# **TITLE PAGE**

| Protocol Number: | 810P301 |
|---|---|
| Title: | A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Molindone Hydrochloride Extended-Release Tablets for the Treatment of Impulsive Aggression in Pediatric Patients with Attention Deficit/Hyperactivity Disorder (ADHD) in Conjunction with Standard ADHD Treatment |
| Sponsor: | Supernus Pharmaceuticals, Inc. |
| IND number: | 106,515 |
| Investigational Medicinal Product: | Molindone Hydrochloride Extended-Release Tablets (SPN-810) |
| Indication: | Treatment of Impulsive Aggression in patients with Attention Deficit/Hyperactivity Disorder (ADHD) in conjunction with standard ADHD treatment |
| Clinical CRO: | |
| Medical Monitor | |
| Phase: | 3 |
| Protocol Version: | 9.0 |

| Release Date: | 01Nov 2018 |
|---|---|
| Good Clinical Practice<br>(GCP) Statement: | This study is to be performed in full compliance with International Conference on Harmonization (ICH) GCP and all applicable local regulations. All required study documentation will be archived as required by regulatory authorities. |

| he undersigned, have rea | d this protocol and agree to condu | ct this trial in accordance with all |
|---|---|---|
| | and in accordance with ICH GCP an | |
| • | | |
| cluding the Declaration of | Helsinki and all its accepted amen | dments to date. |
| Principal Investigator | Signature | Date |



# **SUMMARY OF CHANGES**

This summary table lists all clarifications, administrative changes or amendments to Supernus protocol 810P301. Additions are denoted by bold letters and deletions by strikethrough.

| Section | Page | Description of Change | Rationale |
|---|---|---|---|
| | Changes to 810P301 V5.0 Dated 21 Dec 2015 | | |
| Title Page | 1 | Protocol version and date was updated | Administrative |
| Signature<br>page | 3 | The authorship for revised | For clarification |
| Synopsis | 10 | The following was added: | To understand exposure of metabolites in children |
| Synopsis | 11 | The following was changed: Total subject duration on study: Approximately 13 10 12 weeks Pre-treatment phase: Up to 45 days 4 6 weeks o Screening period: Up to 30 days 2- 4 weeks o Baseline period: At least 15 days 2 weeks | To facilitate study conduct |
| Synopsis | 12 | The following was added: | To understand exposure of metabolites in children |
| Synopsis | 13 | The following was added: | To understand exposure of metabolites in children |

| List of<br>Abbreviations | 19 | List of Abbreviations was updated to include Adverse Event of Special Interest (AESI) | For clarification |
|---|---|---|---|
| 2.3 | 25 | The following was changed: | To understand exposure of metabolites in children |
| 3.2 | 26 | The following was changed: Following screening, eligible subjects will enter a two week flexible baseline period, at which time the IA diary will be issued to the subject's primary caregiver. At the end of the two week baseline period, eligible subjects whose primary caregiver has maintained at least 80% compliance with the IA diary will be randomized 1:1:1 to 18 mg/day SPN-810, 36 mg/day SPN-810, or placebo. | To give caregivers the opportunity to improve diary compliance |
| 3.2.1.1 | 26 | The following was changed: Screening will take place for up to 28 45 days prior to randomization and may be carried out over more than one visit if necessary. | To facilitate study conduct |
| 3.2.1.1 | 26 | The following was added: Staff at study sites are encouraged to complete screening procedures as early as possible to provide more flexibility in the Baseline Period for the caregivers to achieve IA diary compliance (see Section 3.2.1.2). | For clarification |
| 3.2.1.2 | 27 | The following was changed: Subjects who meet study entry requirements will proceed to the two-week flexible 15-day baseline period. At Visit 2 primary and (if assigned) secondary caregivers will receive training on the use of the IA diary. Aan IA diary device (LogPad) will be issued to the primary caregiver. The primary and (if assigned) secondary caregivers will receive training on the use of the IA diary. Every effort will be made to provide adequate caregiver training on the use of the IA diary at Visit 2 and acknowledgement of training will be captured on the device. The caregiver will be instructed to | To give caregivers the opportunity to improve diary compliance |

| | | maintain the diary for two weeks. At the end of this period, | |
|---|---|---|---|
| | | caregiver compliance with the IA diary will be assessed. | |
| | | Following at least 15 days of IA diary use, caregiver | |
| | | compliance with the IA diary will be assessed. Compliance | |
| | | will be calculated as the percentage of days <b>over the past 15</b> | |
| | | days during the baseline period for which an evening diary | |
| | | was completed. Compliance of at least 80% must be | |
| | | demonstrated to continue into the titration period and to be | |
| | | eligible for randomization. Compliance will be measured by | |
| | | the percentage of evening diary entries completed during the | |
| | | baseline period. Subjects whose caregivers demonstrate at | |
| | | least 80% compliance will be eligible for randomization and | |
| | | continue into the titration period. | |
| | | Subjects whose caregivers do not reach 80% compliance | |
| | | during the first 15 days of the Baseline Period may be | |
| | | allowed to continue to use the diary for up to 15 additional | |
| | | days. For these subjects, caregivers will receive remedial | |
| | | training on the use of the IA diary. During this time, | |
| | | caregiver compliance with the IA diary will be monitored | |
| | | daily by study site personnel over the past 15-days as a | |
| | | "rolling window". When the caregivers' performance with | |
| | | the IA diary improves such that the caregivers are able to | |
| | | demonstrate at least 80% compliance over the past 15-day | |
| | | rolling window, the subject will be eligible for | |
| | | randomization and allowed to continue into the titration | |
| | | period. | |
| | | Although there are up to 30 days available for each of the | |
| | | screening and the baseline Period, the total duration of | |
| | | screening and baseline periods may not exceed 45 days. | |
| | | Rescreening | |
| | | As a general rule, rescreening of subjects is not allowed. | |
| | | The only exception to this will be for subjects who had | |
| | | failed screening due to caregiver non-compliance with the | |
| | | IA diary under protocol version 5.0. These subjects may be | |
| | | rescreened to participate in the study under protocol 6.0. | |
| | | These subjects will be assigned a new subject ID number | |
| | | and will complete all study screening procedures. | |
| 3.2.4 | 28 | The following was changed: | For clarification |
| | | Subjects will return to the study site for a final visit, after | |
| | | completing the 1-week Taper/Conversion Period. Those | |
| | L | | l |

| Figure 1 and | 29,<br>30 | subjects who elect to continue in the OLE study will have procedures performed for that study as well. All subjects who discontinue early will return to the study site for a final visit. Any sSubjects who discontinues from the study during the maintenance period will be offered a Taper kit and will return to the study site for a follow-up visit (EOS). Subjects who discontinue during the titration period will not receive a taper kit and will only complete the EOS procedures. These figures were updated with the new visit windows and screening period | Updated as per changes in the protocol |
|---|---|---|---|
| 4.1.1 | 31 | The following was added: 8. α 2- adrenergic agonists (e.g. clonidine and guanfacine) used for any other reason except for monotherapy treatment for ADHD (e.g. aggression or insomnia) must be discontinued at least two weeks prior to Visit 2. | To facilitate study conduct |
| Table 1 | 33,<br>34 | Table 1 was updated with the new visit windows, screening period, baseline period, and footnotes. Due to the addition of a new footnote, this section had to be renumbered | Updated as per changes in the protocol |
| Table 1 | 33,<br>34 | The following new foot note "c" was added for Visit 3 window days: Visit 3 will occur at least 15 days following Visit 2. Footnote "g" was renumbered to "h" and changed as follows: gh Total of 5 PK blood samples will be obtained over one or two visits (Visit 4 and/or Visit 5) to be divided between Visit 4 and Visit 5. Footnote "d" was renumbered to "e" and changed as follows: de Diary compliance must be at least 80% (minimum of 12 days out of 1415) to qualify for randomization. | Updated as per changes in the protocol |
| 4.2.1 | 35 | The following was changed: Subject screening procedures will be performed within 28 45 days prior to Visit 3 and may be done on more than one day. | To facilitate study conduct |

| 4.2.2 | 35 | The following was changed: | To facilitate study conduct |
|---|---|---|---|
| | | Visit 2 will occur at least <b>44 15</b> days prior to Visit 3. | |
| 4.2.2 | 35 | The following was added: | For clarification |
| | | Please note that, per protocol and within the EDC, Visit 1 | |
| | | and Visit 2 may occur on the same day. | |
| 4.2.3 | 35 | The following was changed: | To facilitate study |
| | | Visit 3 will occur at least <b>1415</b> days following Visit 2 according | conduct |
| | | to the Schedule of Visits and Procedures. | |
| 4.2.3 | 36 | The following was changed: | For clarification |
| | | 10. Collect urine samples for urinalysis, <b>urine drug</b> | |
| | | screen (all subjects), and pregnancy test (FOCP only) | |
| 4.2.4 | 36 | The following was changed: | To facilitate study |
| | | Visit 4 will occur 7 (± <b>42</b> ) days following Visit 3 according to | conduct |
| | | the Schedule of Visits and Procedures. | |
| 4.2.5 | 36 | The following was changed: | To facilitate study |
| | | Visit 5 will occur 14 (± <b>12</b> ) days following Visit 3 according to | conduct |
| | | the Schedule of Visits and Procedures. | |
| 4.2.6 | 37 | The following was changed: | To facilitate study |
| | | Visit 6 will occur 21 (±43) days following Visit 5 according to | conduct |
| | | the Schedule of Visits and Procedures. | |
| 4.2.8 | 38 | The following was changed: | To facilitate study |
| | | These will include pre and post-dose samples obtained over | conduct |
| | | one visit (Visit 4 or Visit 5) or can be obtained over two | |
| | | visits (Visit 4 and Visit 5) Blood will be drawn for quantitative | |
| | | PK analysis at Visit 4 and Visit 5. | |
| | | If the subject decides to complete the PK sampling over one | |
| | | visit then he/she will arrive at the clinic in the morning prior to taking the morning dose. | |
| | | A PK sample will be drawn pre-dose; then the dose will be observed in the clinic. Post-dose PK samples will be taken | |
| | | at approximately 1 hour, 2 hours, 4 hours and 6 hours after | |
| | | the time of the observed dose. PK samples should be | |
| | | obtained within 15 minutes of the 1 hour and 2 hour | |

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

| | | timepoints and within 30 minutes of the 4 hour and 6 hour | |
|---|---|---|---|
| | | timepoint. At one of these visits, subjects will arrive at the | |
| | | clinic in the morning, prior to taking their morning dose. A PK | |
| | | sample will be drawn pre-dose; then the dose will be | |
| | | observed in the clinic. Post dose PK samples will be taken at | |
| | | approximately 1 hour and 2 hours after the time of the | |
| | | observed dose. PK samples should be obtained within 15 | |
| | | minutes of the targeted timepoints. | |
| | | If the subject decides to come for the PK sampling over two | |
| | | visits, then on one visit the subject will arrive at the clinic in | |
| | | the morning, prior to taking their morning dose. A PK | |
| | | sample will be drawn pre-dose; then the dose will be | |
| | | observed in the clinic. Post-dose PK samples will be taken | |
| | | at approximately 1 hour and 2 hours after the time of the | |
| | | observed dose. PK samples should be obtained within 15 | |
| | | minutes of the targeted timepoints. | |
| | | 7. ( ) | 5 1 10 11 |
| 4.4 | 41 | The following was added: | For clarification |
| | | 4.4 Prohibited Medications: | |
| | | Subjects may not be on any prohibited medication while on | |
| | | study as indicated in the Inclusion/Exclusion Criteria. These | |
| | | medications include: | |
| | | α 2- adrenergic agonists (e.g. clonidine and) | |
| | | guanfacine) used for any other reason except | |
| | | for monotherapy treatment for ADHD | |
| | | I I I I I I I I I I I I I I I I I I I | |
| | | ., | |
| | | Anti-psychotics including aripiprazole, | |
| | | <ul> <li>Anti-psychotics including aripiprazole,<br/>risperidone, quetiapine, and ziprasidone</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines,</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines,</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity</li> </ul> | |
| | | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known</li> </ul> | |
| 4.5 | 41 | <ul> <li>Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone</li> <li>Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity</li> </ul> | For clarification |
| 4.5 | 41 | Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity Herbal supplements The following was deleted: | For clarification |
| 4.5 | 41 | Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity Herbal supplements The following was deleted: Subjects may not be on any prohibited medication as | For clarification |
| 4.5 | 41 | Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity Herbal supplements The following was deleted: | For clarification |
| 4.5 | 41 | Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity Herbal supplements The following was deleted: Subjects may not be on any prohibited medication as | For clarification For clarification |

| 5.3 | 44 | CGI-I, relative to the condition at baseline Visit 3, will be evaluated by the caregiver and by the Investigator at each post-baseline visit on a 7-point scale with 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse. The following was added: | To understand exposure of metabolites in children |
|---|---|---|---|
| 5.3.2 | 44 | The following was added: | To understand exposure of metabolites in children |
| 5.4.2.1 | 47 | The following was changed: All SAEs must be reported to the Drug Safety Contact within 24 hours of first becoming aware of the SAE. The Investigator must complete an SAE eCRF in EDC Form and include a detailed description of the SAE, as well as other available information pertinent to the case (e.g., hospital records, autopsy reports and other relevant documents). Should the site be unable to access EDC, a paper SAE form must be completed and sent to Drug Safety by email or fax. The investigator will keep a copy of this SAE Report form on file at the study site. Once EDC becomes available, the site must complete the SAE eCRF in EDC. | For Clarification |
| 5.4.2.1 | 48 | The E-mail address for drug safety contact was updated: | Administrative |
| 5.4.2.2. | 48 | The following was added: The Investigator must complete a Pregnancy Outcome Form as a follow up. | For Clarification |
| 5.4.2.2 | 48 | The following was changed: Treatment-emerging EPS (e.g. akathisia, dystonia, Parkinsonism, tardive dyskinesia) and neuroleptic malignant syndrome should be reported to the Drug Safety Contact person(s) by completing the Adverse Event Special Interest (AESI) eCRF in EDC. Should the site be unable to access EDC, | For Clarification |

| | | a paper AESI form must be completed and sent to Safety by email or fax faxing or scanning the appropriate source documentation within 24 hours of first becoming aware of the event. Once EDC becomes available the site must complete AESI eCRF in EDC. EPS incidence will be summarized and shared with study Investigators throughout the trial. | |
|---|---|---|---|
| 5.4.4 | 49 | The following was added: A subject will be excluded if the Screening blood test results indicates > 2 times the upper limit of normal (ULN) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transpeptidase (GGT), and/or serum creatinine. Laboratory tests will not be repeated for these subjects. Any repeat laboratory testing will be conducted under fasting condition. | For Clarification |
| 6.5 | 54 | The following was added: Only one (primary) reason for study discontinuation will be recorded for each subject. | For Clarification |
| | 56 | The following was changed: The secondary endpoints are: | For Clarification |
| 6.9.2 | | <ol> <li>Actual Caregiver CGI-I score at Visit 6</li> <li>Actual Investigator CGI-I score at Visit 6</li> <li>Change from Visit 3 to Visit 6 in Investigator CGI-S score</li> <li>Change from Visit 3 to Visit 6 in CHQ-28 score</li> <li>Change from Visit 3 to Visit 6 in PSI-4-SF scores in: <ul> <li>Parental Distress</li> <li>Parent-Child Dysfunctional Interaction</li> </ul> </li> </ol> | |
| | | a.c. Difficult Child 4. Change from Visit 3 to Visit 6 in Caregiver completed CGI 1 | |

| | | <b>5-6.</b> Change from Visit 3 to Visit 6 in SNAP-IV ADHD | |
|---|---|---|---|
| | | scores in: | |
| | | a. Inattention ratings | |
| | | b. Hyperactivity/Impulsivity ratings | |
| | | c. Combined Scale ratings | |
| 6.13 | 60 | The following was added: | To understand exposure of metabolites in |
| | | | children |
| 7.4.4 | 64 | The following was added: | To understand exposure |
| 7.4.4 | 04 | The following was added. | of metabolites in |
| | | | children |
| | | Changes to 810P301 V6.0 Dated 21 Jul 2016 | |
| | | | <u> </u> |
| Title Page | 1 | Protocol version and date was updated | Administrative |
| Signature | 3 | The signature page was updated | Administrative |
| Page | | | |
| Synopsis | <b>1</b> 5 | | Procedural |
| | | <b>17</b> years (inclusive) will be screened to achieve 291 subjects randomized; 97 per treatment arm | |
| Synopsis | <b>1</b> 5 | Criteria for Inclusion: | Procedural |
| | | Otherwise healthy male or female subjects, age 6 to 12 17 | |
| | | years at the time of screening with a primary diagnosis of ADHD and currently receiving monotherapy treatment with | |
| | | an optimized FDA-approved ADHD medication. IA will be | |
| | | confirmed at screening using R-MOAS and Vitiello Aggression | |
| | | Scale. | |
| List of | 25 | FOCP changed to FOC <b>B</b> P | To Clarify |
| Abbreviation | | | |
| | l | | 1 |

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

| _ | _ | T | Ι |
|---|---|---|---|
| 3.1 | 31 | The present study is designed to evaluate the efficacy, safety, and tolerability of SPN-810 in patients aged 6 to 42 17 years with ADHD and comorbid IA, when taken in conjunction with a standard ADHD treatment. | Procedural |
| 3.2 | 32 | Protocol 810P301 is a randomized, placebo-controlled, double blind, multicenter, parallel group, fixed dose study to demonstrate the efficacy, safety, and tolerability of SPN-810 in the treatment of IA in patients aged 6-12 17 years with ADHD in conjunction with standard ADHD treatment. | Procedural |
| 3.2.1.1 | 32 | The Vitiello Aggression Scale will be used to evaluate subtype of aggression (planned vs. impulsive); only those children <b>and adolescents</b> who score as predominantly impulsive will be included. | Procedural |
| 3.2.1.2 | 33 | These subjects may be rescreened to participate in the study under protocol 6.0 current protocol. | To Clarify |
| 4.1 | 37 | The target population will be male and female subjects aged 6 to 12 17 years with IA and ADHD. | Procedural |
| 4.1.1 | 37 | <ol> <li>Healthy male or female subjects, age 6 to 12 17 years at the time of screening.</li> <li>Weight of at least 20 kg for 6-12 year old subjects.</li> </ol> | Procedural |
| 4.1.2 | 37,38 | <ol> <li>Body Mass Index (BMI) in less than 25th and above 99th percentile or above for 13-17 year old subjects only.</li> <li>Pregnancy or refusal to practice contraception during the study (for female subjects of childbearing potential) and sexually active males).</li> <li>Criminal arrest or report at least 6 months prior to Visit 2.</li> </ol> | |
| Table 1 | 40 | f To be performed for female subjects of childbearing potential prior to administration of first dose of SM and will have to be tested as negative for the subject to continue in the study. | |
| 4.2.1. 4.2.3<br>and 4.2.7 | 41, 42,<br>43 | FOCP changed to FOC <b>B</b> P | To Clarify |
| 4.2.8 | 44 | The following paragraph in Section 4.2.8 was depicted as deleted by a strikethrough in error in the summary of changes; the strikethrough was removed: | Administrative |

| | | <del>,</del> | |
|---|---|---|---|
| | | If the subject decides to complete the PK sampling over one | |
| | | visit then he/she will arrive at the clinic in the morning prior | |
| | | to taking the morning dose. | |
| Table 3 | 56 | FOCP changed to FOC <b>B</b> P | To Clarify |
| | | Changes to 810P301 V7.0 Dated 24 Jul 2017 | |
| Title Page | 1 | Protocol version and date was updated | Administrative |
| Signature<br>Page | 3 | The signature page was updated and revised | Administrative |
| Synopsis | 18 | Number of Subjects: Approximately 378 subjects aged 6-17 | Procedural |
| | | 12 years (inclusive) will be screened to achieve 291 subjects | |
| | | randomized; 97 per treatment arm | |
| Synopsis | 18 | Criteria for Inclusion: | Procedural |
| | | Otherwise healthy male or female subjects, age 6 to 17 12 | |
| | | years at the time of screening with a primary diagnosis of | |
| | | ADHD and currently receiving monotherapy treatment with | |
| | | an optimized FDA-approved ADHD medication. IA will be | |
| | | confirmed at screening using R-MOAS and Vitiello | |
| | | Aggression Scale. | |
| Synopsis | 19 | Primary Efficacy Endpoint | To clarify |
| | | The primary efficacy endpoint is the percent change (PCH <sub>MT</sub> ) | |
| | | in the frequency (unweighted score) of IA behaviors per 7 | |
| | | days in the Maintenance Treatment (Titration and | |
| | | Maintenance) period relative to the Baseline period | |
| | | calculated over the number of days with non-missing IA | |
| | | diary data. | |
| | | The primary efficacy endpoint PCH <sub>MT</sub> will be calculated by | |
| | | PCH <sub>MT</sub> = 100*(MT-B)/B, where MT and B are IA behavior | |
| | | frequencies per 7 days during the maintenance Treatment | |
| | | period and baseline period, respectively. | |
| Synopsis | 20 | Hypotheses: | To clarify |
| | | Let μ₁, μ₂, and μ₃ represent the median percent change in | |
| | | the frequency of IA behaviors per 7 days in the Maintenance | |
| | | Treatment period relative to the Baseline period in the ITT | |
| | | population for subjects treated with Placebo, 18 mg and 36 | |
| | | mg doses of SPN-810, respectively. The null (H <sub>0</sub> ) and the | |
| | | alternative ( $H_a$ ) hypotheses are as in the following. | |
| | | and the fine of the same as an are the following. | |

| Synopsis | 20 | Handling Missing Data: | To clarify |
|---|---|---|---|
| | | For the primary efficacy end point, the frequency of IA behaviors during the maintenance treatment period will be calculated over the number of days with non-missing IA diary data in the maintenance treatment period. | |
| Synopsis | 21 | Statistical Methods: | To clarify |
| | | The primary efficacy analysis will be based on the ITT population. The primary efficacy endpoint is the percent change in the frequency (unweighted score) of IA behaviors per 7 days in the Maintenance Treatment period relative to the Baseline period in the ITT population calculated over the number of days with non-missing IA diary data. | |
| 3.1 | 34 | The present study is designed to evaluate the efficacy, safety, and tolerability of SPN-810 in patients aged 6 to <del>17</del> <b>12</b> years with ADHD and comorbid IA, when taken in conjunction with a standard ADHD treatment. | Procedural |
| 3.2 | 35 | Protocol 810P301 is a randomized, placebo-controlled, double blind, multicenter, parallel group, fixed dose study to demonstrate the efficacy, safety, and tolerability of SPN-810 in the treatment of IA in patients aged 6-17 12 years with ADHD in conjunction with standard ADHD treatment. | Procedural |
| 3.2.1.1 | 35 | The Vitiello Aggression Scale will be used to evaluate subtype of aggression (planned vs. impulsive); only those children and adolescents who score as predominantly impulsive will be included. | Procedural |
| 4.1 | 40 | The target population will be male and female subjects aged 6 to 47 12 years with IA and ADHD. | Procedural |
| 4.1.1 | 40 | <ol> <li>Healthy male or female subjects, age 6 to 47 12 years at the time of screening.</li> <li>Weight of at least 20 kg for 6 12 year old subjects.</li> </ol> | Procedural |
| 4.1.2 | 40,41 | Body Mass Index (BMI) in less than 25th and above 99 <sup>th</sup> percentile or-above for 13-17 year old subjects only. Sign | Procedural |
| 6.2 | 62 | For the primary efficacy end point, the frequency of IA behaviors during the maintenance treatment period will be | To clarify |

| | | calculated over the number of days with non-missing IA diary data in the maintenance treatment period. | |
|---|---|---|---|
| 6.9.1 | 64 | The primary efficacy endpoint is the percent change (PCH <sub>MT</sub> ) in the frequency (unweighted score) of IA behaviors per 7 days in the Maintenance Treatment (Titration and Maintenance) period relative to the Baseline period calculated over the number of days with non-missing IA diary data. | To clarify |
| | | The primary efficacy endpoint PCH <sub>MT</sub> will be calculated by PCH <sub>MT</sub> = 100*( <del>MT</del> -B)/B, where <del>MT</del> and B are IA behavior frequencies per 7 days during the <del>maintenance-Treatment</del> period and baseline period, respectively. | |
| | | Let $\mu_1$ , $\mu_2$ , and $\mu_3$ represent the median percent change in the frequency of IA behaviors per 7 days in the Maintenance Treatment period relative to the Baseline period in the ITT population for subjects treated with Placebo, 18 mg and 36 mg doses of SPN-810, respectively. | |
| 6.11 | 67 | However, the primary endpoint for this study is percent change in the frequency of IA incidence per 7 days in the Maintenance Treatment (Titration and Maintenance) period (PCH <sub>MT</sub> ) relative to the Baseline period in the ITT population calculated over the number of days with nonmissing IA diary data | To clarify |
| | | Changes to 810P301 V8.0 Dated 07 Nov 2017 | |
| Title Page | 1, 2 | Protocol version and date were updated | Administrative |
| Signature<br>Page | 3 | The signature page was updated | Administrative |
| Protocol<br>Synopsis | 19 | Number of Subjects: Approximately <b>426</b> <del>378</del> subjects aged 6-12 years (inclusive) will be screened to achieve <del>291</del> <b>330</b> subjects randomized <del>; 97 per treatment arm</del> | Revised following re-<br>estimation of sample<br>size |
| Protocol<br>Synopsis | 20 | Sample size: Based on results from the Phase 2 study, it is assumed that the average treatment difference between SPN-810 dose groups and placebo is 11.51 15 with a common standard deviation of 27.3. A sample size of 132 77 subjects per arm (264 231 subjects for 3 arms) will yield 90% power to detect | Revised following re-<br>estimation of sample<br>size |

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

| | | a non-zero difference between the median of 18 mg or 36 | |
|---|---|---|---|
| | | mg dose group and the placebo using the Wilcoxon rank- | |
| | | sum test with a 2-sided significance level alpha=0.05. | |
| | | It is assumed that approximately 20% of subjects will | |
| | | dropout before the completion of the study and hence, an | |
| | | adjusted total of <b>330</b> <del>291</del> subjects will be randomized in a | |
| | | 1:1:1 ratio to obtain 264 231 subjects in the ITT population | |
| | | at the completion of the study. | |
| 4.1 | 41 | Approximately <b>330</b> <del>291</del> subjects will be randomized in this | Revised following re- |
| | | clinical investigation. | estimation of sample |
| | | | size |
| 5.2.2 | 53 | ADHD-Combined subscale: the first two subscales items | Clarification |
| | | are combined | |
| | | Each subscale score is the sum average of the scores for the | |
| | | individual items included in the subscale. | |
| 6.10 | 68 | Based on results from the Phase 2 study, it is assumed that | Revised following re- |
| | | the average treatment difference between SPN-810 dose | estimation of sample |
| | | groups and placebo <b>is 11.51 <del>15</del></b> with a common standard | size |
| | | deviation of 27.3. A sample size of <del>77</del> <b>132</b> subjects per arm | |
| | | (231 264 subjects for 3 arms) will yield 90% power to detect | |
| | | a non-zero difference between the median of 18 mg or 36 | |
| | | mg dose group and the placebo using the Wilcoxon rank- | |
| | | sum test with a 2-sided significance level alpha=0.05. | |
| | | It is assumed that approximately 20% <b>of</b> subjects will | |
| | | dropout before the completion of the study and hence, an | |
| | | adjusted total of <del>291</del> 330 subjects will be randomized in a | |
| | | 1:1:1 ratio to obtain 231 264 subjects in the ITT population | |
| | | at the completion of the study. | |
| | | ' ' | |

## **CLINICAL PROTOCOL SYNOPSIS**

| Name of Company: | IND Number: 106,515 |
|------------------------------------------|----------------------------|
| Supernus Pharmaceuticals, Inc. | |
| Name of Product: Molindone Hydrochloride | Name of Active Ingredient: |
| Extended-Release Tablets (SPN-810) | Molindone Hydrochloride |
| Protocol Number: 810P301 | Phase of Development: 3 |

Full Title of Study: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Molindone Hydrochloride Extended-Release Tablets for the Treatment of Impulsive Aggression in Pediatric Patients with Attention Deficit/Hyperactivity Disorder (ADHD) in Conjunction with Standard ADHD Treatment

Investigator(s) / Center(s): Approximately 25 US centers

# Objectives:

#### **Primary**

The primary objective is to assess the efficacy and safety of SPN-810 in reducing the frequency of impulsive aggression (IA) behaviors in pediatric patients with ADHD when taken in conjunction with standard ADHD treatment

## Secondary

The secondary objectives of the study are to assess the following:

- the effect of SPN-810 on the Investigator-rated Clinical Global Impression Improvement Scale (CGI-I)
- the effect of SPN-810 on the Clinical Global Impression Severity Scale (CGI-S)
- the effect of SPN-810 on the child's overall health as measured by the Child Health Questionnaire Parent Form 28-item (CHQ-PF28)
- the effect of treating the child with SPN-810 on the parent-child relationship as measured by the Parenting Stress Index Short Form (PSI-4-SF)
- the effect of SPN-810 on the Caregiver-rated CGI-I
- the effect of SPN-810 on inattention and hyperactivity-impulsivity measured by the SNAP-IV Rating Scale

| • |
|---|

Study Design: Double-blind, placebo-controlled, randomized, parallel group study

**Number of Subjects:** Approximately 426 subjects aged 6-12 years (inclusive) will be screened to achieve 330 subjects randomized

#### Criteria for Inclusion:

Otherwise healthy male or female subjects, age 6 to 12 years at the time of screening with a primary diagnosis of ADHD and currently receiving monotherapy treatment with an optimized FDA-approved ADHD medication. IA will be confirmed at screening using R-MOAS and Vitiello Aggression Scale.

#### Criteria for Exclusion:

Current or lifetime diagnosis of epilepsy, major depressive disorder, bipolar disorder, schizophrenia or related disorder, personality disorder, Tourette's disorder, or psychosis not otherwise specified. Currently meeting DSM criteria for autism spectrum disorder, pervasive developmental disorder, obsessive compulsive disorder, post-traumatic stress disorder, or any other anxiety disorder as primary diagnosis. Known or suspected intelligence quotient (IQ) < 70, suicidality, pregnancy, or substance or alcohol abuse.

# Treatment, Dose, and Mode of Administration:

Molindone hydrochloride extended-release tablet dosage forms of 3mg and 9mg with matching placebo tablets. Treatment to be administered orally twice daily with or without food. Subjects will be force-titrated over a period of 2 weeks to their final randomized dose.

Treatment 1: placeboTreatment 2: 18mgTreatment 3: 36mg

# **Duration of Treatment and Study Duration:**

Total subject duration on study: Approximately 13 weeks

Pre-treatment phase: Up to 45 days

Screening period: Up to 30 days

Baseline period: At least 15 days

Treatment phase: 5 weeks

Titration period: 2 weeksMaintenance period: 3 weeks

Conversion/taper phase: 1 week

## **Endpoints:**

## **Primary Efficacy Endpoint**

The primary efficacy endpoint is the percent change ( $PCH_T$ ) in the frequency (unweighted score) of IA behaviors per 7 days in the Treatment (Titration and Maintenance) period relative to the Baseline period calculated over the number of days with non-missing IA diary data.

The primary efficacy endpoint PCH $_{\rm T}$  will be calculated by PCH $_{\rm T}$ = 100\*(T–B)/B, where T and B are IA behavior frequencies per 7 days during the Treatment period and baseline period, respectively. The IA behavior frequency per 7 days is defined as (SUM/DAY) x 7, where SUM is the total of the IA behaviors reported in the subject IA diary, and DAY is the number of days with non-missing IA score in the subject IA diary during the specified study period.

## Secondary Efficacy Endpoints

- 1. Investigator-rated CGI-I
- 2. CGI-S
- 3. CHQ-PF28
- 4. PSI-4-SF
- 5. Caregiver-rated CGI-I
- 6. SNAP-IV Rating Scale

# Safety and Tolerability Endpoints

- 1. Adverse events (AE)
- 2. Extrapyramidal symptoms (EPS) scales (Simpson-Angus Scale, Barnes Akathisia Scale, Abnormal Involuntary Movement Scale)
- 3. Clinical laboratory tests (Hematology, Chemistry and Urinalysis)
- 4. ECGs
- 5. Vital signs
- 6. Columbia Suicide Severity Rating Scale (C-SSRS)
- 7. Infrequent Behaviors Checklist

#### Sample size:

Based on results from the Phase 2 study, it is assumed that the average treatment difference between SPN-810 dose groups and placebo is 11.51 with a common standard deviation of 27.3. A sample size of 132 subjects per arm (264 subjects for 3 arms) will yield 90% power to detect a non-zero difference between the median of 18 mg or 36 mg dose group and the placebo using the Wilcoxon rank-sum test with a 2-sided significance level alpha=0.05.

It is assumed that approximately 20% of subjects will dropout before the completion of the study and hence, an adjusted total of 330 subjects will be randomized in a 1:1:1 ratio to obtain 264 subjects in the ITT population at the completion of the study.

The sample size was calculated using the nQuery Advisor Software, Version 7.

#### **Analysis Populations:**

Safety Population: will include all randomized subjects who received at least 1 dose of study drug.

<u>Intent-to-Treat (ITT) Population</u>: will include all subjects who received at least 1 dose of study drug and have a baseline and at least 1 valid post-randomization assessment of frequency of IA behaviors based on IA diary entry.

<u>Per-Protocol (PP) Population</u>: will include all of the subjects in the ITT population who completed the treatment period with 80% diary completion compliance and who did not have major protocol deviations.

<u>PK population</u>: will include all subjects in the safety population who had at least one PK sample drawn which had a quantitatable concentration for at least one analyte of interest.

## Hypotheses:

Let  $\mu_1$ ,  $\mu_2$ , and  $\mu_3$  represent the median percent change in the frequency of IA behaviors per 7 days in the Treatment period relative to the Baseline period in the ITT population for subjects treated with Placebo, 18 mg and 36 mg doses of SPN-810, respectively. The null (H<sub>0</sub>) and the alternative (H<sub>a</sub>) hypotheses are as in the following.

- $H_{01}$ :  $\mu_2 = \mu_1$ , (there is no difference between the median of the 18 mg dose SPN-810 and the median of placebo) vs.  $H_{a1}$ :  $\mu_2 \neq \mu_1$ ,(there is a difference between the median of the 18 mg dose SPN-810 and the median of placebo)
- $H_{02}$ :  $\mu_3$ =  $\mu_1$ , (there is no difference between the median of the 36 mg dose SPN-810 and the median of placebo) vs.  $H_{a2}$ :  $\mu_3 \neq \mu_1$ ,(there is a difference between the median of the 36 mg dose SPN-810 and the median of placebo)

# Handling Missing Data:

For the primary efficacy end point, the frequency of IA behaviors during the treatment period will be calculated over the number of days with non-missing IA diary data in the treatment period. No explicit imputation of missing data will be used, but this approach is implicitly equivalent to using the frequency of IA behaviors during the days with non-missing IA diary data to impute the frequency for days after study discontinuation and days with missing IA diary data.

#### Pharmacokinetic Methods:

### Sampling:

5 blood samples divided between 2 visits.

## Bioanalytical Analysis:

| Pharmacokinetic Analysis: |
|---------------------------|

#### Statistical Methods:

Summaries for continuous variables will include the sample size, mean, and standard deviation, median, minimum, and maximum. Summaries for discrete variables will include the tabulation of frequencies and percentages.

The primary efficacy analysis will be based on the ITT population. The primary efficacy endpoint is the percent change in the frequency (unweighted score) of IA behaviors per 7 days in the Treatment period relative to the Baseline period in the ITT population calculated over the number of days with non-missing IA diary data.

The primary efficacy analysis will be performed using the Wilcoxon rank-sum test to compare the medians of each of the two doses of SPN-810 (18 mg and 36 mg) with the median of the Placebo. The Hodges-Lehmann estimate and the associated 95% confidence interval (CI) will be calculated. The robustness of the primary analyses will be checked by performing two sensitivity analyses.

Each one of the six secondary endpoints will be analyzed using the analysis of covariance method based on the ITT population with missing data imputed using the Last Observation Carried Forward (LOCF) method. The model includes treatment and baseline as fixed independent covariates and change from baseline to final maintenance visit as a response variable. The least squares mean of each treatment group, the difference in the least squares mean (18mg dose minus placebo and 36 mg dose minus placebo), and the 2-sided 95% CI for the difference will be obtained.

#### Interim analysis:

A single interim analysis will be performed after approximately 50% of the randomized subjects complete the study. The main purpose of the interim analysis is to re-estimate the sample size.

CONFIDENTIAL Version 9.0


## Safety analysis:

Safety analyses will be based on the safety population. All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized using discrete summaries at the subject and event level by system organ class and preferred term for each treatment group. Similarly, treatment-emergent AEs will be summarized by severity and relationship separately. Vital signs will be summarized using descriptive statistics by treatment groups. The summary includes sample size, mean, and standard deviation, median, minimum, and maximum. Continuous laboratory parameters will be summarized similarly. If applicable, categorical laboratory tests will be summarized using number and percent of subjects by treatment groups. Data on infrequent behaviors will be listed.

# **TABLE OF CONTENTS**

| " | TLE PAGE | | 1 |
|---|---|---|---|
| Sl | JMMARY | OF CHANGES | 4 |
| CI | LINICAL P | ROTOCOL SYNOPSIS | 18 |
| T/ | ABLE OF C | ONTENTS | <b>2</b> 4 |
| LI | ST OF TAI | BLES AND FIGURES | 28 |
| LI | ST OF AB | BREVIATIONS | 29 |
| 1 | INTRO | DUCTION | 31 |
| | 1.1 | Background | 31 |
| | 1.2 | Sponsor's Phase 2a Study | 32 |
| | 1.3 | Sponsor's Phase 2b Study | 33 |
| | 1.4 | Impulsive Aggression Diary (IA Diary) | 34 |
| | 1.5 | Study Rationale | 34 |
| 2 | STLIDY | OBJECTIVES | 3/ |
| _ | | Primary Objective | |
| | | Secondary Objectives | |
| | | Tertiary Objective | |
| , | | FIGATIONAL PLAN | |
| 3 | IIIAAF2 | IIGATIONAL PLAN | |
| _ | 2 1 | | |
| _ | | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of | |
| _ | Measurer | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments | 35 |
| _ | Measurer<br>3.2 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of nents | 35<br>36 |
| | Measurer<br>3.2<br>3.2.1 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments | 35<br>36 |
| _ | 3.2.1<br>3.2.1 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of nents Overall Study Design and Plan Pre-Treatment Phase 1 Screening Period | <b>3</b> 5<br><b>3</b> 6<br>36 |
| | Measurer<br>3.2<br>3.2.1 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments Overall Study Design and Plan Pre-Treatment Phase 1 Screening Period 2 Baseline Period | :<br>36<br>36<br>36 |
| | Measurer<br>3.2<br>3.2.1<br>3.2.1<br>3.2.1. | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of nents Overall Study Design and Plan Pre-Treatment Phase 1 Screening Period 2 Baseline Period. Treatment Phase | 35<br>36<br>36<br>37 |
| | Measurer 3.2 3.2.1 3.2.1 3.2.1 3.2.2 3.2.2 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of nents Overall Study Design and Plan Pre-Treatment Phase 1 Screening Period 2 Baseline Period. Treatment Phase | 35<br>36<br>36<br>37 |
| | Measurer 3.2 3.2.1 3.2.1 3.2.1 3.2.2 3.2.2 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments Overall Study Design and Plan Pre-Treatment Phase 1 Screening Period 2 Baseline Period. Treatment Phase 1 Randomization. 2 Titration Period. | 36<br>36<br>37<br>38<br>38 |
| | Measurer 3.2 3.2.1 3.2.1 3.2.1 3.2.2 3.2.2 3.2.2 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments Overall Study Design and Plan Pre-Treatment Phase 1 Screening Period 2 Baseline Period. Treatment Phase 1 Randomization 2 Titration Period | 36<br>36<br>36<br>37<br>38<br>38 |
| | Measurer 3.2 3.2.1 3.2.1 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of nents Overall Study Design and Plan Pre-Treatment Phase Screening Period Baseline Period Treatment Phase Randomization Titration Period Maintenance Period | 35<br>36<br>36<br>38<br>38<br>38 |
| | Measurer 3.2 3.2.1 3.2.1 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 5.2.3 3.2.4 STUDY | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments Overall Study Design and Plan Pre-Treatment Phase Screening Period Baseline Period Treatment Phase Randomization Titration Period Maintenance Period Conversion/Taper Phase End of Study / Early Termination | 36<br>36<br>36<br>37<br>38 |
| 4 | Measurer 3.2 3.2.1 3.2.1 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 5.2.3 3.2.4 STUDY | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments | 35363638383838383838383838383838 |
| 4 | Measurer 3.2 3.2.1 3.2.1 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 3.2.2 5.2.3 3.2.4 STUDY | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments Overall Study Design and Plan Pre-Treatment Phase Screening Period Baseline Period Treatment Phase Randomization Titration Period Maintenance Period Conversion/Taper Phase End of Study / Early Termination | 35363638383838383838383838383838 |
| 4 | Measurer 3.2 3.2.1 3.2.1 3.2.1 3.2.2 3.2.2 3.2.2 3.2.2 3.2.3 3.2.4 STUDY 4.1 | Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of ments | 36<br>36<br>37<br>38<br>41<br>41 |

| | 4.2.1 | Visit 1 | 45 |
|---|---|---|---|
| | 4.2.2 | Visit 2 | 45 |
| | 4.2.3 | Visit 3 | 45 |
| | 4.2.4 | Visit 4 | 46 |
| | 4.2.5 | Visit 5 | 46 |
| | 4.2.6 | Visit 6 | 47 |
| | 4.2.7 | Visit 7 | 47 |
| | 4.2.8 | Pharmacokinetic Sample Collection | 48 |
| | 4.3 | Treatments | 48 |
| | 4.3.1 | Treatments Administered | 48 |
| | 4.3.2 | Identity of Investigational Product(s) | 48 |
| | 4.3.3 | Study Medication Handling and Accountability | 49 |
| | 4.3.4 | Method of Assigning Subjects to Treatment Groups | 49 |
| | 4.3.5 | Treatment Replacement | |
| | 4.3.6 | Dosing Schedule | |
| | 4.3.7 | Method of Administration | |
| | 4.3.8 | Blinding | 50 |
| | 4.4 | Prohibited Medications: | |
| | 4.5 | Concomitant Medication | 51 |
| | 4.6 | Completion of Study and Discontinuation of Subjects | 52 |
| 5 | ΔΝΑΙ | YSIS VARIABLES | 52 |
| • | 5.1 | Primary Efficacy Variable | |
| | 5.2 | Secondary Efficacy Variables | |
| | 5.2.1 | Clinical Global Impression (CGI) Scales | |
| | 5.2.2 | Swanson, Nolan, Pelham Rating Scale- Revised (SNAP-IV) | |
| | 5.2.3 | Child Health Questionnaire Parent Form 28- Item (CHQ-PF28) | |
| | 5.2.4 | Parenting Stress Index-Short Form (PSI-4-SF) | |
| | 5.2.4 | Pharmacokinetic Measurements | |
| | 5.3.1 | | |
| | 5.3.2<br><b>5.4</b> | Exploratory Pharmacokinetic Variables | |
| | | Cafaty Assassments | |
| | | Safety Assessments | |
| | 5.4.1 | Adverse Events | 55 |
| | <b>5.4.1</b> 5.4.1 | Adverse Events | 55 |
| | <b>5.4.1</b> 5.4.1 5.4.1 | Adverse Events | 55<br>55 |
| | 5.4.1<br>5.4.2<br>5.4.2<br>5.4.2 | Adverse Events | 55<br>55<br>56 |
| | <b>5.4.1</b> 5.4.1 5.4.1 | Adverse Events | 55<br>55<br>56 |
| | 5.4.1<br>5.4.1<br>5.4.1<br>5.4.2 | Adverse Events | 55<br>55<br>56<br>56 |
| | 5.4.1<br>5.4.2<br>5.4.2<br>5.4.2<br>5.4.2 | Adverse Events | |
| | 5.4.1<br>5.4.1<br>5.4.2<br>5.4.2<br>5.4.2<br>5.4.2 | Adverse Events | |

| | - 4 4 | | |
|---|--------|-----------------------------------------------------|----|
| | 5.4.4 | Laboratory Measurements | |
| | 5.4.5 | Vital Sign and Height/Weight Measurements | |
| | 5.4.6 | Medical History | |
| | 5.4.7 | Physical Examinations and Electrocardiograms (ECGs) | |
| | 5.4.8 | Other Special Tests | |
| | 5.4.8. | · · | |
| | 5.4.8. | | |
| | 5.4.8. | | |
| | 5.4.8. | ( , | |
| | 5.4.8. | | |
| | 5.4.8. | | |
| | 5.4.8. | , , , | |
| | 5.4.8. | 8 Infrequent Behaviors Checklist | 62 |
| 6 | STATIS | TICAL METHODS | 62 |
| | 6.1 | Statistical and Analytical Plans | 62 |
| | | Handling Missing Data | |
| | | Analysis Populations | |
| | | Demographic and Baseline Characteristics | |
| | | Subject Disposition | |
| | | Protocol Deviations | |
| | | Study Medication Exposure and Compliance | |
| | | Concomitant Medications | |
| | | Efficacy Analyses | |
| | 6.9.1 | Primary Efficacy Analysis | |
| | 6.9.2 | Secondary Efficacy Analyses | |
| | 6.9.3 | Sensitivity Analysis | |
| | 6.9.3. | 1 Multiple imputation under Missing at Random (MAR) | 67 |
| | 6.9.3. | | |
| | 6.9.3. | | |
| | 6.10 | Sample Size and Power Considerations | 68 |
| | 6.11 | Interim Analysis | 68 |
| | 6.12 | Assessment of MCIC | 68 |
| | 6.13 | Pharmacokinetic Analyses | 70 |
| | 6.14 | Safety Analyses | 70 |
| | 6.14.1 | Adverse Events | 70 |
| | 6.14.2 | Laboratory Values | 71 |
| | 6.14.3 | Vital Signs, Height and Weight | 71 |
| | 6.14.4 | ECG Results | |
| | 6.14.5 | Physical Examinations | |
| | 6.14.6 | Columbia Suicide Severity Rating Scale (C-SSRS) | |
| | 6.14.7 | Infrequent Behaviors Checklist | |
| | | · | |
| | 6.14.8 | Other Special Tests | |

| 7 | DOCU | IMENTATION | 72 |
|---|---|---|---|
| | 7.1 | Adherence to the Protocol | 72 |
| | 7.2 | Changes to the Protocol | 72 |
| | 7.3 | Protocol Deviations | 73 |
| | 7.4 | Data Quality Assurance | 73 |
| | 7.4.1 | Data Collection | 73 |
| | 7.4.2 | Clinical Data Management | 74 |
| | 7.4.3 | Database Quality Assurance | 74 |
| | 7.4.4 | Bioanalytical Data Management and Quality Control | 74 |
| | 7.5 | Retention of Records | 74 |
| | 7.6 | Auditing Procedures | 75 |
| | 7.7 | Publication of Results | 75 |
| | 7.8 | Financing and Insurance | 75 |
| | 7.9 | Disclosure and Confidentiality | 75 |
| | 7.10 | Discontinuation of Study | 76 |
| 8 | FTHIC | S | 76 |
| | 8.1 | Institutional Review Boards / Independent Ethics Committees | |
| | 8.2 | Ethical Conduct of the Study | |
| | 8.3 | Investigators and Study Personnel | |
| | 8.4 | Subject Information and Consent/Assent | |
| 9 | REFER | RENCE LIST | 77 |
| 10 | | PENDICES | |
| | 10.1 | Adaptive Design Plan | |
| | 10.1.1 | | |
| | 10.1.2 | • | |
| | 10.1.3 | • | |
| | 10.1.4 | | |
| | 10.1.5 | , | |
| | 10.1<br>10.1 | .5.1 Responsible Party | |
| | 10.1 | Retrospective Modified Overt Aggression Scale (R-MOAS) | |
| | 10.3 | Clinical Global Impression (CGI) Scale | |
| | 10.4 | Vitiello Scale | |
| | 10.5 | Kiddie-Sads-Present and Lifetime Version (K-SADS-PL) 2013 | |
| | 10.6 | Columbia-Suicide Severity Rating Scales (C-SSRS) | |
| | 10.7 | Swanson, Nolan and Pelham Rating Scale-Revised (SNAP IV) | |
| | 10.7 | Simpson-Angus Rating Scale | |
| | 10.9 | Barnes Akathisia Rating Scale (BARS) | |
| | 10.10 | Abnormal Involuntary Movement Scale (AIMS) | |
| | 10.11 | Child Health Questionnaire Parent Form 28-item (CHQ-PF28) | |

| 810b301 | version 9.0 | |
|---|---|---|
| 10.12 | Parenting Stress Index-Short Form (PSI-4-SF) | 225 |
| LIST OF | TABLES AND FIGURES | |
| Table 1: S | chedule of Visits and Procedures | 43 |
| Table 2: Dosing Schedule (Total Daily Dose) | | |
| Table 3: Clinical Laboratory Tests | | |
| Figure 1: T | reatment Schedule (Conversion) | 39 |
| Figure 2: T | reatment Schedule (Taper) | 40 |

#### LIST OF ABBREVIATIONS

ADHD Attention-Deficit Hyperactivity Disorder

AE Adverse Event

AESI Adverse Event of Special Interest

AIMS Abnormal Involuntary Movement Scale

ASD Autism Spectrum Disorder

BID Twice a Day

CFR Code of Federal Regulations

CGI-S Clinical Global Impression – Severity of Illness
CGI-I Clinical Global Impression – Global Improvement
CHQ-PF 28 Child Health Questionnaire Parent Form 28-item

CL/F Apparent Clearance

CRA Clinical Research Associate

CRO Contract Research Organization

C-SSRS Columbia Suicide Severity Rating Scale

eCRF Electronic Case Report Form
EPS Extrapyramidal Symptoms

FOCBP Females of Childbearing Potential

IA Impulsive Aggression
IAF Informed Assent Form
ICF Informed Consent Form

ICH International Conference on Harmonization

IEC Independent Ethics Committee
IRB Institutional Review Board

ITT Intent to Treat

KBIT-2 Kaufman Brief Intelligence Test, Second Edition

K-SADS-PL 2013 Schedule for Affective Disorders and Schizophrenia for School-aged

Children - Present and Lifetime Versions 2013

LSM Least-square Means MAR Missing at Random

MedDRA Medical Dictionary for Regulatory Activities

MI Multiple Imputation
MNAR Missing Not at Random

ODD Oppositional Defiant Disorder

PK Pharmacokinetic(s)

PSI-4-SF Parenting Stress Index – Short Form

QD Once a Day

R-MOAS Retrospective Modified Overt Aggression Scale

SAE Serious Adverse Event

Supernus® Pharmaceuticals, Inc. CONFIDENTIAL 810P301 Version 9.0 

SAP Statistical Analysis Plan SM Study Medication

SNAP-IV Swanson, Nolan and Pelham Rating Scale - Revised

TDD Total Daily Dose

ULN Upper Limit of Normal

V/F Apparent Volume of Distribution

## 1 INTRODUCTION

## 1.1 Background

Behavior with the immediate intent to cause harm – whether to self, others, objects, or property – constitutes aggression. Aggressive behavior becomes maladaptive when it persists, occurs outside an acceptable social context, and is of an intensity, frequency, severity and/or duration detrimental to the child's interests (Connor 2006; Jensen 2007). Maladaptive aggression is an expression of central nervous system dysfunction and may therefore be amenable to treatments targeting its neurobiologic substrate.

Aggression can be categorized into two broad subtypes based on the aggressor's motivation – 1) reactive or impulsive and 2) proactive or instrumental (Vitiello 1997). Impulsive aggression (IA) is angry, retaliatory aggression arising out of frustration, annoyance, or hostility to real or perceived provocations – stressors that youth of the same age typically experience with equanimity. IA is therefore an unplanned and immediate response reflecting out-of-control emotionality that satisfies immediate emotional pressures, albeit with negative consequences to the aggressor. In contrast, instrumental aggression is consciously planned, goal-oriented behavior with the specific intent of benefiting the aggressor (Jensen 2007).

IA is a common comorbidity in attention-deficit/hyperactivity disorder (ADHD) and is often refractory to primary ADHD therapy. In the Multimodal Treatment of Children with ADHD (MTA) study (MTA 1999), 54% of preadolescent study participants with ADHD Combined subtype displayed clinically significant aggression at baseline. Of these, 44% remained significantly symptomatic in terms of aggressive behavior after 14 months of optimal medication (stimulants) with/without behavioral therapy (Jensen, 2007).

IA amplifies the psychological, academic, emotional, and social problems associated with ADHD (Shelton, 1998), markedly increasing the risk of persistent behavioral problems, conduct disorder, encounters with the justice system, deficits in academic achievement, behavioral and disciplinary problems at school, and substance experimentation/abuse. Early-onset, pervasive and unremitting IA in the context of impulsive thoughts, emotional lability, and impulsive behavior is thought to represent a high-risk profile for progression from childhood ADHD to adult antisocial disorders (McKay, 2001). In the context of ADHD it represents a serious clinical and public health concern and warrants effective and timely intervention.

Since primary ADHD therapy has limited effect on IA, a stepped-care approach has been recommended, with aggression-targeted therapy such as an antipsychotic added to ADHD therapy to manage residual aggressive behaviors (Scotto- Rosato 2012). Risperidone and other "atypical" antipsychotics have historically been at the forefront of treatment recommendations regarding combination therapy for managing comorbid aggression in children with ADHD (Pappadopulos et al. 2003; Pliszka et al. 2006; Pliszka et al. 2007). However, only two double-blind randomized placebo-controlled trials of risperidone as adjunctive therapy in children with ADHD and aggression refractory to stimulants have been published – 1) a pilot study in 25 children that was likely underpowered and did not detect a significant treatment effect (Armenteros 2007; Aman 2014) and 2) the recently completed TOSCA (Treatment of

Severe Childhood Aggression) study (Farmer et al. 2011; Aman 2014; Gadow 2014). The effect size for risperidone's effect on IA was small (0.29), even though the dosage could be adjusted to optimal effect. The TOSCA study provides initial empirical evidence supporting a stepped-care approach in which ADHD children with severe aggression are initially treated with primary ADHD therapy followed by adjunctive antipsychotic therapy targeted to IA. However, the long-term effects of risperidone and similar antipsychotics in terms of metabolic derangements predictive of diabetes and cardiovascular disease, have become cause for considerable concern, especially in the face of very limited evidence of efficacy as aggression-targeted therapy in ADHD. The TOSCA study confirmed that stimulant co-therapy does not attenuate the adverse effects of risperidone or similar agents on body composition, metabolic parameters, prolactin, or sedation (Calarge 2009; Penzner 2009).

Molindone hydrochloride (molindone) is a medium potency antipsychotic, and is currently under development by the Sponsor as an extended-release formulation (SPN-810), for its potential utility in treating IA in children with ADHD.

In an open-label study, molindone improved aggressive behavior in children (N=6, 6-11 years of age) with undersocialized conduct disorder, aggressive type (Greenhill 1981). The optimum dose was 0.5 mg/kg/day. Molindone was also shown to be effective in treating aggressive behavior in a double-blind, 8-week, inpatient study of 31 children, ages 6 to 11, with undersocialized conduct disorder, aggressive type (Greenhill 1985).

Prior to its withdrawal from the US market for commercial reasons, Immediate-Release Molindone (Moban®) was approved for the treatment of schizophrenia in adults and adolescents. Its use was also evaluated in a pediatric population with early-onset schizophrenia and schizoaffective disorder when it was selected as the first-generation antipsychotic on the basis of its more favorable safety profile for comparison with second-generation agents (risperidone, olanzapine) in an NIH-sponsored study (TEOSS, Treatment of Early-Onset Schizophrenia Spectrum Disorders Study) (McClellan 2007). At an average dose of 60 mg/day (range, 10-140 mg/day), molindone was shown to be safe and well-tolerated (Sikich 2008). Molindone (10-140 mg/day) was not associated with significant increases in weight/BMI (in contrast to olanzapine). Molindone was also not associated with more dystonic or parkinsonian symptoms when given with benztropine, although akathisia was reported by more molindone-treated subjects. Results of randomized controlled trials such as TEOSS stimulated interest in the potential usefulness of molindone as a weight- and metabolically-neutral D2-receptor antagonist in children with ADHD and comorbid IA.

#### 1.2 Sponsor's Phase 2a Study

Study 810P201, was a proof-of-concept, multicenter, open-label, parallel-group, randomized, doseranging, safety, and tolerability study of molindone administered as experimental Molindone Immediate Release (IR) capsules in children with ADHD and persistent serious conduct problems (Stocks 2012). Target subjects were healthy male or female children aged 6 to 12 years, inclusive, with a diagnosis of ADHD accompanied by persistent serious conduct problems. A total of 78 subjects (19-20 per treatment group) in ten U.S sites were randomized. The primary objective was to evaluate the safety and tolerability of four weight-based dosages of Molindone IR dosed three times daily in children with ADHD

| and persistent serious conduct problems (<30 kg: |
|---|
| 1.3 Sponsor's Phase 2b Study Sponsor completed a Phase 2b multicenter, randomized, double-blind, placebo-controlled trial in the United States in pediatric subjects 6 to 12 years of age diagnosed with ADHD and IA that was not controlled by optimal stimulant and behavioral therapy (Sponsor Study 810P202). The primary objective of the study was to assess the effect of an extended-release tablet formulation of molindone hydrochloride (SPN-810) (12 to 54 mg/day) in reducing IA as measured by the Retrospective-Modified Overt Aggression Scale (R-MOAS) after at least three weeks of assigned treatment. Secondary endpoints included the rate of remission of IA and measurement of the effectiveness of SPN-810 on Clinical Global Impression (CGI) and ADHD scales as well as evaluation of the safety and tolerability of the drug. Patients who completed the study were offered the opportunity to continue into an open-label phase of six months duration. |
| SPN-810 dose within treatment groups was stratified by weight (below/above 20 kg). Both the medium (24/36 mg) and low (12/18 mg) dose groups showed statistically significant difference from the placebo group in the change from baseline to Visit 10 in R-MOAS but the high (36/54 mg) dose group was not significantly different from the placebo group. Furthermore, both the low dose and medium dose groups were significantly different from the high dose based on pair-wise comparison among the dose groups. |

# 1.4 Impulsive Aggression Diary (IA Diary)

Sponsor has developed and validated a new measurement tool to assess behaviors associated with IA. The impulsive aggression diary (IA diary) is an electronic observer-reported outcome (eObsRO) instrument that comprises an episodic diary (to be reported as soon as possible after the parent or other guardian or observer witnesses the child's IA behavior) and an evening diary (to enable at a minimum, completion of the diary once each day). The IA diary monitors the frequency of occurrence of 15 IA behaviors: Yelling, Screaming, Threatening, Scratching, Throwing, Slamming, Hitting Self, Arguing, Cursing, Name Calling, Shoving, Hair Pulling, Fighting, Hitting Others, Kicking Others. The development process followed FDA's "Guidance for Industry Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims." Through this process, the IA diary was demonstrated to be a psychometrically valid and reliable tool to assess IA in children (Sponsor Study 810P501).

# 1.5 Study Rationale

Additionally, IA severity and improvement will be assessed using Clinical Global Impression (CGI) scales completed by both investigator and caregiver. Subject and caregiver quality of life will also be evaluated.

The effect of molindone on body composition, metabolic parameters, and prolactin will be evaluated. Emergence of extrapyramidal symptoms will be monitored.

# 2 STUDY OBJECTIVES

# 2.1 Primary Objective

The primary objective is to assess the efficacy and safety of SPN-810 in reducing the frequency of IA behaviors in pediatric patients with ADHD when taken in conjunction with standard ADHD treatment.

# 2.2 Secondary Objectives

The secondary objectives of the study are to assess the following:

- the effect of SPN-810 on the Clinical Global Impression Improvement Scale (CGI-I)
- the effect of SPN-810 on the Clinical Global Impression Severity Scale (CGI-S)
- the effect of SPN-810 on the child's overall health as measured by the Child Health Questionnaire Parent Form 28-item (CHQ-PF28)
- the effect of treating the child with SPN-810 on the parent-child relationship as measured by the Parenting Stress Index Short Form version 4 (PSI-4-SF)
- the effect of SPN-810 on the caregiver-completed CGI-I
- the effect of SPN-810 on inattention and hyperactivity-impulsivity measured by the SNAP-IV Rating Scale

# 2.3 Tertiary Objective

#### 3 INVESTIGATIONAL PLAN

# 3.1 Rationale for Study Design, Including Choice of Treatment Groups, Appropriateness of Measurements

The present study is designed to evaluate the efficacy, safety, and tolerability of SPN-810 in patients aged 6 to 12 years with ADHD and comorbid IA, when taken in conjunction with a standard ADHD treatment. In this patient population, IA behaviors persist, despite monotherapy treatment with an FDA-approved ADHD medication, stimulant or non-stimulant, at an FDA-approved optimized dose.

A titration schedule will be followed to ensure a safe escalation to each dose level. The titration rate and dose range under investigation in the present study were demonstrated to be safe, efficacious, and well tolerated in a similar patient population in the previous Phase 2b study. Administration of study medication will be recorded using an electronic dosing diary.

The IA diary will serve as the primary assessment tool for efficacy. The IA diary is a new electronic observer-reported outcome (eObsRO) instrument developed by the Sponsor to record behaviors associated with IA. Secondary measures of efficacy will include the effect of SPN-810 on the Clinical Global Impression – Improvement Scale (CGI-I), the effect of SPN-810 on the Clinical Global Impression – Severity Scale (CGI-S), the effect of SPN-810 on the child's overall health as measured by the Child Health Questionnaire Parent Form 28-item (CHQ-PF28), and the effect of treating the child with SPN-810 on the parent-child relationship as measured by the Parenting Stress Index – Short Form (PSI-4-SF). The child's ADHD symptoms will be measured using the Swanson, Nolan and Pelham Rating Scale - Revised (SNAP-IV).

Safety will be assessed by the monitoring of AEs, concomitant medications, vital signs, clinical laboratory tests, physical examinations, and ECGs, as well as by the Simpson-Angus Scale, the Barnes Akathisia Scale, and the Abnormal Involuntary Movement Scale (AIMS). The scales were chosen to specifically monitor EPS, since youth treated with antipsychotics are at greater risk for EPS side effects than adults (Findling 2005). These scales were utilized in Phase 2 studies and have been used in other clinical studies of atypical antipsychotics in children.

## 3.2 Overall Study Design and Plan

Protocol 810P301 is a randomized, placebo-controlled, double blind, multicenter, parallel group, fixed dose study to demonstrate the efficacy, safety, and tolerability of SPN-810 in the treatment of IA in patients aged 6-12 years with ADHD in conjunction with standard ADHD treatment. The study is presented schematically in Figure 1 and Figure 2. The study is divided into three phases: Pre-Treatment, Treatment, and Conversion/Taper.

Following screening, eligible subjects will enter a flexible baseline period, at which time the IA diary will be issued to the subject's primary caregiver. At the end of the baseline period, eligible subjects whose primary caregiver has maintained at least 80% compliance with the IA diary will be randomized 1:1:1 to 18 mg/day SPN-810, 36 mg/day SPN-810, or placebo. A dose titration schedule will be followed, with dosing in the active treatment groups initiated at 3 mg/day and increased approximately every 3 days until the target dose is reached. After completing the two-week titration period and the three-week maintenance period, subjects will enter the conversion or tapering phase prior to discontinuing SM, at which time subjects will have the option to enter an open label extension (OLE) study. A subject who discontinues during the maintenance period prior to Visit 6 may be allowed to participate in the OLE on a case-by-case basis only after consultation between the Investigator, the Medical Monitor and the Sponsor. The OLE study will be conducted under a separate protocol. Subjects who choose to participate in the OLE will enter that study at a dose of 18 mg/day SPN-810.

#### 3.2.1 Pre-Treatment Phase

#### 3.2.1.1 Screening Period

Screening will take place for up to 45 days prior to randomization and may be carried out over more than one visit if necessary. Prior to conducting any screening procedures, written informed consent/assent must be obtained from the parent or legal representative, and subject (when required). Each screened subject will be assigned a subject number starting from 1001 to 1999 in a sequential manner. Staff at study sites are encouraged to complete screening procedures as early as possible to provide more flexibility in the baseline period for the caregivers to achieve IA diary compliance (see Section 3.2.1.2).

The R-MOAS and CGI-S will be administered to determine entry to the baseline period of the study and also to determine eligibility for randomization to treatment. The Vitiello Aggression Scale will be used to evaluate subtype of aggression (planned vs. impulsive); only those children who score as predominantly
impulsive will be included. The diagnosis of ADHD will be confirmed with the Schedule for Affective Disorders and Schizophrenia for School-aged Children—Present and Lifetime Versions 2013 (K-SADS-PL 2013). The K-SADS-PL 2013 is a semi-structured diagnostic interview designed to diagnose current and past episodes of psychopathology in children and adolescents according to DSM-5 criteria. The Introductory and Screen Interviews will be completed. The Screen Interview will assess the different diagnoses and determine which supplements should be completed. Supplement 4 (Neurodevelopment, Disruptive and Conduct Disorders) must be completed to assess ADHD, ODD, CD, Tic and ASD (Autism Spectrum Disorder). If an exclusionary diagnosis is confirmed, the remainder of the diagnostic will not be completed and the subject will be deemed a screen failure.

#### 3.2.1.2 Baseline Period

Subjects who meet study entry requirements will proceed to the flexible baseline period. At Visit 2 an IA diary device (LogPad) will be issued to the primary caregiver. The primary and (if assigned) secondary caregivers will receive training on the use of the IA diary. Every effort will be made to provide adequate caregiver training on the use of the IA diary at Visit 2 and acknowledgement of training will be captured on the device.

Following at least 15 days of IA diary use, caregiver compliance with the IA diary will be assessed. Compliance will be calculated as the percentage of days over the past 15 days during the baseline period for which an evening diary was completed. Subjects whose caregivers demonstrate at least 80% compliance will be eligible for randomization and continue into the titration period.

Subjects whose caregivers do not reach 80% compliance during the first 15 days of the baseline period may be allowed to continue to use the diary for up to 15 additional days. For these subjects, caregivers will receive remedial training on the use of the IA diary. During this time, caregiver compliance with the IA diary will be monitored daily by study site personnel over the past 15-days as a "rolling window". When the caregivers' performance with the IA diary improves such that the caregivers are able to demonstrate at least 80% compliance over the past 15-day rolling window, the subject will be eligible for randomization and allowed to continue into the titration period.

Although there are up to 30 days available for each of the screening and the baseline period, the total duration of screening and baseline periods may not exceed 45 days.

#### Rescreening

As a general rule, rescreening of subjects is not allowed. The only exception to this will be for subjects who failed screening due to caregiver non-compliance with the IA diary under protocol version 5.0. These subjects may be rescreened to participate in the study under current protocol. These subjects will be assigned a new subject ID number and will complete all study screening procedures.

#### 3.2.2 Treatment Phase

#### 3.2.2.1 Randomization

Inclusion/exclusion criteria will be re-assessed to verify eligibility prior to study randomization at the end of Visit 3 (Randomization). Eligible subjects whose primary caregiver has maintained at least 80% compliance with the IA diary will be randomized. Eligible subjects who complete the baseline period and meet the requirements for the double blind study will be randomized at Visit 3 (Day 1) in a 1:1:1 ratio to receive 18 mg/day, 36 mg/day SPN-810, or placebo and proceed to the titration period, which will be two weeks.

#### 3.2.2.2 Titration Period

Subjects will be titrated to maintenance dose over a period of 2 weeks.

#### 3.2.2.3 Maintenance Period

Following dose titration, subjects on active treatment will be maintained at their designated dose level for 3 weeks.

#### 3.2.3 Conversion/Taper Phase

All subjects who complete the randomized, double blind portion of study 810P301 will have the option to participate in an OLE study (study protocol 810P304) in which all subjects will receive active SM treatment. Subjects choosing to participate will receive blinded conversion medication kits, and their total daily dose for the open label extension will be converted to 18 mg/day (Figure 1). Those subjects who do not elect to participate in this extension will be tapered off SM (Figure 2).

#### 3.2.4 End of Study / Early Termination

Subjects will return to the study site for a final visit, after completing the 1-week Taper/Conversion Period. Those subjects who elect to continue in the OLE study will have procedures performed for that study as well. Subjects who discontinue from the study during the maintenance period will be offered a Taper kit and will return to the study site for a follow-up visit (EOS). Subjects who discontinue during the titration period will not receive a taper kit and will only complete the EOS procedures.

Figure 1: Treatment Schedule (Conversion)



Figure 2: Treatment Schedule (Taper)



#### 4 STUDY METHODS

# 4.1 Selection of Study Population

The target population will be male and female subjects aged 6 to 12 years with IA and ADHD. SM will be administered in conjunction with the subject's standard ADHD treatment. Approximately 330 subjects will be randomized in this clinical investigation.

#### 4.1.1 Inclusion Criteria

- 1. Healthy male or female subjects, age 6 to 12 years at the time of screening.
- Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders-5
  (DSM-5 confirmed by the Schedule for Affective Disorders and Schizophrenia for School-aged
  Children Present and Lifetime Version 2013 (K-SADS-PL 2013).
- Retrospective Modified Overt Aggression Scale (R-MOAS) score of ≥24 at screening.
- 4. CGI-S score of at least moderately ill at both Screening and Randomization.
- 5. Vitiello Aggression Scale score from -2 to -5 at Screening.
- 6. Free of antipsychotic medication for at least two weeks prior to Visit 2.
- Monotherapy treatment with FDA-approved optimized ADHD medication (psychostimulant or non-stimulant) at an FDA-approved dose for at least one month prior to Screening, and willing to maintain that dose throughout the Baseline and Treatment period.
- 8. α 2- adrenergic agonists (e.g. clonidine and guanfacine) used for any other reason except for monotherapy treatment for ADHD (e.g. aggression or insomnia) must be discontinued at least two-weeks prior to Visit 2.
- 9. Medically healthy and with clinically normal laboratory profiles, vital signs, and electrocardiograms (ECGs).
- 10. Weight of at least 20 kg.
- 11. Able and willing to swallow tablets whole and not chewed, cut or crushed.
- 12. Written Informed Consent obtained from the subject's parent or legal representative, and written Informed Assent obtained from the subject if appropriate.
- 13. Measurement of compliance ≥ 80% for completion of IA Diary during Baseline Period.

#### 4.1.2 Exclusion Criteria

- 1. Body Mass Index (BMI) in 99<sup>th</sup> percentile or above.
- Current or lifetime diagnosis of epilepsy, major depressive disorder, bipolar disorder, schizophrenia or related disorder, personality disorder, Tourette's disorder, or psychosis not otherwise specified.
- 3. Currently meeting DSM-5 criteria for autism spectrum disorder, pervasive developmental disorder, obsessive compulsive disorder, post-traumatic stress disorder, or any other anxiety disorder as primary diagnosis.

- Use of anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity within two weeks of Visit 2.
- 5. Use of herbal supplements within one week of Visit 2.
- Known or suspected intelligence quotient (IQ) < 70.</li>
- Unstable endocrinological or neurological conditions which confound the diagnosis or are a contraindication to treatment with antipsychotics.
- 8. Suicidality, defined as either active suicidal plan/intent or active suicidal thoughts in the six months before the Screening Visit or more than one lifetime suicide attempt.
- Pregnancy or refusal to practice contraception during the study (for female subjects of childbearing potential and sexually active males).
- 10. Substance or alcohol use during the last three months.
- 11. Urine drug test at screening that is positive for alcohol or drugs of abuse.
- 12. Known allergy or sensitivity to molindone hydrochloride.
- 13. Any reason which, in the opinion of the Investigator or the Sponsor, would prevent the subject and subject's caregiver from participating in the study or complying with the study procedures.
- 14. Use of an investigational drug or participation in an investigational study within 30 days prior to Visit 2.

#### 4.2 Schedule of Visits and Procedures

All subjects who are randomized and take any SM will be followed according to the protocol regardless of the number of doses of SM taken, unless consent for follow-up is withdrawn. The Sponsor, or the Sponsor's designee, must be notified of all deviations from the protocol visits or procedures, and these procedures, if applicable, will be rescheduled or performed at the nearest possible time to the original schedule. Subjects will be instructed to call study personnel to report any abnormalities during the intervals in between study visits and to come to the study site if medical evaluation is needed and as the urgency of the situation indicates. Unscheduled visits may be conducted at the discretion of the investigator throughout all study periods. The medical monitor must be contacted promptly in the event that any clinically significant findings or information are obtained during the unscheduled visit. This should be captured in the appropriate eCRF. For emergency and other unscheduled visits to a medical facility other than the study site, medical records will be obtained by the Investigator or qualified designee as source data for study follow-up.

Table 1 presents the schedule of visits and procedures for the study.

Table 1: Schedule of Visits and Procedures

| Phase | Pre-treatment | | Treatment | | | | Conversion/ |
|---|---|---|---|---|---|---|---|
| Period | Screening | Baseline | Titration | | Maintenance | | Taper |
| VISIT NUMBER | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| DAY | -45 | -15 | 1 | 8 | 15 | 36 | 43 |
| WINDOW (DAYS) | ≤45d prior to<br>Visit 3 | ≥15d prior to<br>Visit 3 | <b>O</b> c | 7d±2d from<br>Visit 3 | 14d±2d from<br>Visit 3 | 21d±3d from<br>Visit 5 | 7d±1d from<br>Visit 6 |
| Informed Consent/Assent <sup>a</sup> | Хp | | | | | | |
| R-MOAS, K-SADS-PL 2013 & Vitiello<br>Aggression Scale | Х | | | | | | |
| Medical History | Х | | Χq | | | | |
| Demographics | Х | | | | | | |
| Physical Examination | Х | | | | | X | |
| ECG (12-lead) | Х | | | Х | | X | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Randomization | | | X b,e | | | | |
| Urine Drug Screen | X | | X | | | | |
| Urine Pregnancy Test <sup>f</sup> | X | | X | | | | X |
| Diary Training & Distribution or Evaluation | | X | X e | X | X | X | |
| Vital Signs <sup>g</sup> | X | | | | | | X |
| Weight, height, BMI | X | | X | X | X | X | X |
| Hematology/chemistry/Urinalysis | X | | X | | | X | X |
| PK Blood Sampling | | | | Χh | X h | | |
| Columbia Suicide Severity Rating Scale (CSSRS) | Х | | х | х | X | X | х |
| Investigator CGI-S | X | | X | Х | X | X | |
| Caregiver and investigator CGI-I | | | | Х | X | X | |
| Efficacy scales (SNAP-IV, CHQ-PF28, PSI-4-SF) | | | X | | | X | |
| Safety Scales (Simpson-Angus, Barnes, AIMS) | | | X | Х | X | X | Х |
| Infrequent Behaviors Checklist | | | X | Х | X | X | |
| Adverse Events | | | X | Х | X | X | Х |
| Concomitant Medications | Х | X | Х | Х | Х | X | Х |
| Drug Dispensation | | | Хp | | X | Х | |


# 

| Phase | Pre-treatment | | Treatment | | | | Conversion/ |
|---|---|---|---|---|---|---|---|
| Period | Screening | Baseline | Titra | ation | Maintenance | | Taper |
| VISIT NUMBER | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| DAY | -45 | -15 | 1 | 8 | 15 | 36 | 43 |
| WINDOW (DAYS) | ≤45d prior to<br>Visit 3 | ≥15d prior to<br>Visit 3 | <b>0</b> c | 7d±2d from<br>Visit 3 | 14d±2d from<br>Visit 3 | 21d±3d from<br>Visit 5 | 7d±1d from<br>Visit 6 |
| Drug Return and Compliance | | | | | X | X | X |
| Diary Return | | | | | | | X |

- a Written consent must be obtained prior to performing any study-related procedure.
- b Access IWRS.
- c Visit 3 will occur at least 15 days following Visit 2
- d Assess for any clinically significant change in Medical History since screening.
- e Diary compliance must be at least 80% (minimum of 12 days out of 15) to qualify for randomization.
- f To be performed for female subjects of childbearing potential prior to administration of first dose of SM and will have to be tested as negative for the subject to continue in the study.
- g Heart Rate (HR), blood pressure (BP), temperature, and respiratory rate will be measured.
- h Total of 5 PK blood samples will be obtained over one or two visits (Visit 4 and/or Visit 5)

#### 4.2.1 Visit 1

Prior to conducting any screening procedures, written Informed Consent must be obtained from the parent or legal representative, and, if appropriate, Informed Assent from the subject. Subject screening procedures will be performed within 45 days prior to Visit 3 and may be done on more than one day. Abnormal results on screening laboratory tests may be repeated at the discretion of the Investigator.

The following procedures will be performed at Visit 1:

- Obtain written informed consent and assent.
- 2. Obtain demographic information, medical history
- 3. Access Interactive Web Response System (IWRS) for subject number
- 4. Administer K-SADS-PL 2013 for confirmation of ADHD diagnosis
- 5. Administer Vitiello Aggression Scale
- 6. Administer R-MOAS
- 7. Administer Investigator CGI-S
- 8. Perform physical examination
- 9. Record vital signs (HR, BP, temperature, and RR), height, weight and BMI
- 10. Perform 12-lead ECG
- 11. Collect blood samples for hematology and chemistry
- 12. Administer C-SSRS
- 13. Collect urine sample for urinalysis and urine drug screen (all subjects), and pregnancy test (FOCBP only)
- 14. Assess and record concomitant medications
- 15. Assess inclusion/exclusion criteria

#### 4.2.2 Visit 2

Visit 2 will occur at least 15 days prior to Visit 3. Please note that, per protocol and within the EDC, Visit 1 and Visit 2 may occur on the same day.

- 1. Provide training for IA diary and dosing diary module
- 2. Distribute device
- 3. Assess and record concomitant medications

#### 4.2.3 Visit 3

Visit 3 will occur at least 15 days following Visit 2 according to the Schedule of Visits and Procedures.

- 1. Administer efficacy scales (SNAP-IV, CHQ-PF28, PSI-4-SF)
- 2. Assess IA diary compliance / review training as necessary
- 3. Confirm eligibility to randomize to study medication treatment
- 4. Randomize subject via IWRS
- Administer Investigator CGI-S
- 6. Administer Infrequent Behaviors Checklist

- 7. Administer safety scales (Simpson-Angus, Barnes Akathisia, AIMS)
- 8. Record height, weight, and BMI
- Collect blood samples for hematology/chemistry
- Collect urine samples for urinalysis, urine drug screen (all subjects), and pregnancy test (FOCBP only)
- 11. Administer C-SSRS
- 12. Record concomitant medication
- 13. Assess for any clinically significant change in Medical History
- 14. Dispense SM via IWRS.
- 15. Review training on dosing diary module
- 16. Assess adverse events (post-dose)

#### 4.2.4 Visit 4

Visit 4 will occur 7 (±2) days following Visit 3 according to the Schedule of Visits and Procedures.

- 1. Administer Investigator CGI-S
- 2. Administer caregiver and investigator-completed CGI-I
- 3. Administer Infrequent Behaviors Checklist
- 4. Administer safety scales (Simpson-Angus, Barnes Akathisia, AIMS)
- 5. Record height, weight, and BMI
- 6. Perform 12-lead ECG
- 7. Collect blood samples for PK analysis
- 8. Administer C-SSRS
- 9. Record concomitant medication
- 10. Review IA diary compliance and provide training as required
- 11. Collect AEs
- 12. Review dosing diary compliance and provide training as required

#### 4.2.5 Visit 5

Visit 5 will occur 14 (±2) days following Visit 3 according to the Schedule of Visits and Procedures.

- 1. Administer Investigator CGI-S
- 2. Administer caregiver and investigator-completed CGI-I
- 3. Administer Infrequent Behaviors Checklist
- 4. Administer safety scales (Simpson-Angus, Barnes Akathisia, AIMS)
- 5. Record height, weight, and BMI
- 6. Collect blood samples for PK analysis
- 7. Administer C-SSRS
- 8. Record concomitant medication
- 9. Review IA diary compliance and provide training as required
- 10. Collect AEs
- 11. Collect returned SM; assess treatment compliance
- 12. Review dosing diary compliance and provide training as required

#### 13. Dispense SM

#### 4.2.6 Visit 6

Visit 6 will occur 21 (±3) days following Visit 5 according to the Schedule of Visits and Procedures.

- Administer efficacy scales (Investigator CGI-S, caregiver and investigator CGI-I, SNAP-IV, CHQ-PF28, PSI-4-SF)
- 2. Administer Infrequent Behaviors Checklist
- 3. Administer safety scales (Simpson-Angus, Barnes Akathisia, AIMS)
- 4. Record height, weight, and BMI
- 5. Perform 12-lead ECG
- 6. Perform physical examination
- 7. Collect blood samples for hematology/chemistry
- 8. Collect urine sample for urinalysis
- 9. Administer C-SSRS
- 10. Record concomitant medication
- 11. Review IA diary compliance and provide training as required
- 12. Collect AEs
- 13. Collect returned SM; assess treatment compliance
- 14. Review dosing diary compliance and provide training as required
- 15. Determine whether subject wishes to participate in open-label extension
- 16. Dispense SM (either Conversion or Taper based upon subject's decision about participation in open-label extension)

#### 4.2.7 Visit 7

Visit 7 will occur 7 (±1) days following Visit 6 according to the Schedule of Visits and Procedures. These procedures will also be performed for patients who discontinue early. Patients who discontinue early after Visit 5 will be offered a taper kit.

- 1. Administer safety scales (Simpson-Angus, Barnes Akathisia, AIMS)
- 2. Record vital signs (HR, BP, temperature, and RR), height, weight and BMI
- 3. Collect urine sample for pregnancy test (FOCBP only)
- 4. Administer C-SSRS
- 5. Record concomitant medication
- 6. Collect AEs
- 7. Collect SM and assess treatment compliance
- 8. Collect device
- 9. Complete/discontinue subject
- 10. Collect blood samples for hematology/chemistry
- 11. Collect urine sample for urinalysis

#### 4.2.8 Pharmacokinetic Sample Collection

All blood samples for PK analysis will be drawn at the clinical site. A total of 5 blood samples (4 mL each) will be taken for PK analysis over the course of the study. These will include pre- and post-dose samples obtained over one visit (Visit 4 or Visit 5) or over two visits (Visit 4 and Visit 5).

If the subject decides to complete the PK sampling over one visit then he/she will arrive at the clinic in the morning prior to taking the morning dose. A PK sample will be drawn pre-dose; then the dose will be observed in the clinic. Post-dose PK samples will be taken at approximately 1 hour, 2 hours, 4 hours and 6 hours after the time of the observed dose. PK samples should be obtained within 15 minutes of the 1 hour and 2 hour timepoints and within 30 minutes of the 4 hour and 6 hour timepoints.

If the subject decides to come for the PK sampling over two visits, then on one visit the subject will arrive at the clinic in the morning, prior to taking their morning dose. A PK sample will be drawn predose; then the dose will be observed in the clinic. Post-dose PK samples will be taken at approximately 1 hour and 2 hours after the time of the observed dose. PK samples should be obtained within 15 minutes of the targeted timepoints. At the other visit, subjects will arrive at the clinic after taking their morning dose. PK samples will be taken at approximately 4 hours and 6 hours after the time that the morning dose was taken. PK samples should be obtained within 30 minutes of the targeted timepoints.

Blood samples will be collected and processed as per instructions in the Laboratory Manual.

#### 4.3 Treatments

#### 4.3.1 Treatments Administered

Subjects will take molindone hydrochloride extended-release tablet (SPN-810) or placebo twice each day (BID) with or without food, in the morning and in the evening, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if after noon, the evening dose.

Subjects will be randomized to one of three treatments at Visit 3. Subjects will be titrated up to the final randomized total daily dose (TDD).

- Reference treatment
  - Treatment 1: Placebo tablets, PO, BID
- Test treatments
  - o Treatment 2: Molindone extended-release tablets, 18 mg TDD, PO, BID
  - o Treatment 3: Molindone extended-release tablets, 36 mg TDD, PO, BID

#### 4.3.2 Identity of Investigational Product(s)

Test and reference (matching placebo) products are either purple (3mg) or yellow (9mg) round tablets printed on one side with the tablet dose strength (" $\underline{3}$ " or " $\underline{9}$ ") that will be supplied in labeled blister cards by the Sponsor. The Sponsor will package the SM in a double-blind configuration.

Each SM blister card will contain combinations of molindone extended-release and/or placebo tablets, which will supply a subject with 6 (six) to 8 (eight) days of dosing as well as some extras for lost product and/or to account for visit delays associated with patient/site schedules. The SM blister card types include: Titration (two blister cards), Maintenance (three blister cards), Taper (one blister card), and Conversion (one blister card).

A single SM kit contains a total of 7 pre-packaged blister cards (two Titration blister cards, three Maintenance blister cards, one Tapering blister card and one Conversion blister card) and is marked with a unique 4-digit SM kit number.

#### 4.3.3 Study Medication Handling and Accountability

All SM will be supplied to the Investigator by the Sponsor. SM supplies must be kept in an appropriate secure area (e.g., locked cabinet) and stored according to the conditions specified on the SM labels. SM must be stored between  $59^{\circ}F - 86^{\circ}F$  ( $15^{\circ}C - 30^{\circ}C$ ).

Following Sponsor instructions and in compliance with ICH E6 as well as local, state, and federal regulations, the Investigator and study staff will be responsible for the accountability of all clinical supplies (receiving, shipment, dispensing, inventory, and record keeping) in a SM accountability log, a copy of which will be collected by the Sponsor at the end of the study.

Under no circumstances will the Investigator allow the SM to be used other than as directed by this protocol. Clinical supplies will not be dispensed to any individual who is not randomized into the study.

An accurate and timely record of the receipt of all clinical supplies; dispensing of SM to the subject; collection of unused supplies returned by the subject; and subsequent return of unused SM to the Sponsor must be maintained with dates. This SM accountability log includes, but may not be limited to: (a) documentation of receipt of clinical supplies, (b) SM inventory log, (c) SM accountability log, and (d) all shipping service receipts. All forms will be provided by the Sponsor. Any comparable forms that the study site wishes to use must be approved by the Sponsor.

The supplies and inventory records must be made available, upon request, for inspection by the designated representative of the Sponsor, a representative of the FDA, or a representative of a non-US health authority. The assigned Clinical Research Associate (CRA) will review these documents along with all other study conduct documents at each and every visit to the study site once SM has been received by the study site. All used, partly used, and unused clinical supplies, including empty containers, are to be returned to the Investigator by the subject and ultimately to the Sponsor at the conclusion of the study, unless provision is made by the Sponsor for destruction of supplies and containers at the study site. Upon completion of SM accountability and reconciliation procedures by study site personnel and documentation procedures by Sponsor personnel, SM is to be returned to the Sponsor with a copy of the completed SM disposition form as outlined in the Study Medication Manual.

#### 4.3.4 Method of Assigning Subjects to Treatment Groups

Allocation of study drug will be completed centrally through the use of an interactive web response system (IWRS) that will determine which kit to assign to the subject. The randomization schedules will

be created by a designated unmasked statistician using SAS (SAS Institute, Cary, North Carolina, Version 9.2 or higher). Separate schedules for subject randomization and drug list will be created. The randomization scheme assigns treatment to each randomization number in a 1:1:1.

Upon admission to the study, subjects will be assigned site (01-99) and subject numbers (1001-1999), in the sequence that they are entered. Subjects who complete the Baseline Period and continue to meet all eligibility criteria will be assigned kit numbers, according to the randomization schedule, by using the IWRS.

#### 4.3.5 Treatment Replacement

In the event that a subject's original kit is lost, damaged, or consumed prior to the end of treatment, the Investigator will use the IWRS which will specify a new Kit Number to be dispensed to that subject from the supplies already available at the site. Separate reserve supplies will not be provided to the Investigators.

#### 4.3.6 Dosing Schedule

During Visit 3, subjects will be randomized to Treatments 1, 2, or 3 and start dosing. Table 2 below presents the details of the dosing schedule for each active treatment group throughout the 6-week treatment phase for this study. Dose reduction will not be permitted in the study.

Table 2: Dosing Schedule (Total Daily Dose)

| Treatment | Final Dose | | Study Days | | | | | |
|---|---|---|---|---|---|---|---|---|
| Arm | rillal Dose | | 1-2 | 3-5 | 6-8 | 9-11 | 12-14 | 15+ |
| | | Period* | Т | Т | Т | T | T | М |
| 1 | Placebo | | РВО | PBO | РВО | PBO | РВО | РВО |
| 2 | 18 mg | | | | | | | |
| 3 | 36 mg | | | | | | | |

<sup>\*</sup> T = titration period; M = maintenance period; PBO=Placebo

#### 4.3.7 Method of Administration

The SM must be swallowed whole. SM must not be crushed, chewed or cut. The SM must be taken with or without food in the morning and in the evening, preferably within 12 hours.

#### 4.3.8 Blinding

The subject and all personnel involved with the conduct and the interpretation of the study, including the Investigators, study site personnel, and the Sponsor and CRO clinical staff, will be blinded to the medication codes. A limited number of Supernus personnel will perform and interpret the plasma assays for the population PK analysis and will be aware of these plasma data during the study. These personnel will not have access to the randomization schedule, are not associated with the clinical

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

conduct of the study, and will not reveal to any clinical personnel involved in the study the treatment to which a subject is assigned. Randomization schedule data will be kept strictly confidential, filed securely by the IWRS vendor, and accessible only to authorized persons until the time of unblinding.

The test tablets have matching placebo tablets. The blind is maintained primarily through the IWRS. The blind will be maintained through the end of the Conversion/Taper period.

The Investigator must try to avoid breaking the blind. The decoding information will not be viewed unless an actual medical or medication safety emergency occurs. The Investigator can access the subject's randomized treatment information via IWRS only if knowledge of the treatment regimen will influence or assist with medical management of the subject in an acute emergency. Before breaking the blind, every effort must be made to contact the Medical Monitor to ascertain the necessity of breaking the code. If the Investigator is unsuccessful in contacting the Medical Monitor, he/she will contact the backup Medical Monitor (or other appropriate designee if the backup Medical Monitor is unavailable). If it is not possible to contact the Medical Monitor or the backup Medical Monitor (or designee), and the situation is an emergency, the Investigator may break the blind and contact the Medical Monitor as soon as possible. The Investigator is to make a careful note of the date and time of decoding, the reason that necessitated breaking the code, and the signature of the person who broke the code. Upon breaking the randomization code, the subject should be withdrawn from the study but should be followed up for safety purposes.

#### 4.4 Prohibited Medications:

Subjects may not be on any prohibited medication while on study as indicated in the Inclusion/Exclusion Criteria. These medications include:

- α 2- adrenergic agonists (e.g. clonidine and guanfacine) used for any other reason except for monotherapy treatment for ADHD
- Anti-psychotics including aripiprazole, risperidone, quetiapine, and ziprasidone
- Anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors or any drug known to inhibit CYP2D6 activity
- Herbal supplements

# 4.5 Concomitant Medication

The dose of the ongoing ADHD medication will not be adjusted during the study, starting at Visit 1. No additional concomitant medications are allowed during the study, with the following exceptions:

- Chronic medication for conditions not related to ADHD or IA that are allowed by Investigator at Screening
- Nutritional supplements (e.g. multivitamins, fish oil)
- Emla or other numbing cream for PK venipuncture
- Benztropine is permitted for the treatment of emerging EPS at a starting dose of 0.5mg BID up to a range of 1 to 4mg/day. Lorazepam (1 to 2 mg per dose not to exceed three times daily) and

- clonazepam (0.25 to 1 mg per dose not to exceed twice daily) will also be permitted to treat emerging EPS.
- Common over-the-counter (OTC) therapies for minor transient ailments (e.g. acetaminophen for headache, ibuprofen for fever) will be allowed without exception.
- Treatment for AEs other than EPS or minor transient ailments is only permitted in consultation with the Medical Monitor.

All concomitant medications will be recorded in the eCRF.

# 4.6 Completion of Study and Discontinuation of Subjects

Subjects will be considered to have completed the study if they complete all visits up to and including Visit 6. All subjects who discontinue early will complete Visit 7. Any subject who discontinues from the study after Visit 5 will be offered a Taper kit.

The Investigator(s) or subjects themselves may stop SM treatment at any time for safety or personal reasons. A subject is free to withdraw from the study at any time for any reason without prejudice to their future medical care by the physician or at the institution. The Investigator or Sponsor may also withdraw the subject at any time in the interest of subject safety. The withdrawal of a subject from the study should be discussed where possible with the Medical Monitor and/or CRA before the subject stops SM. Subjects removed from the study for any reason will not be replaced.

Reasons for withdrawal may include but are not limited to subject withdrawal of consent, occurrence of unmanageable AEs, or if it is in the best interest of the subject as per Investigator's discretion.

The primary reason for withdrawal must be recorded in the subject's medical record and on the eCRF. If a subject is withdrawn for more than one reason, each reason should be documented in the source document and the most medically significant reason should be entered on the eCRF.

#### 5 ANALYSIS VARIABLES

#### 5.1 Primary Efficacy Variable

The primary efficacy endpoint will be based on a checklist of 15 IA behaviors collected in an electronic IA diary. The IA diary comprises two parts: 1) An episodic diary that will be used by the primary caregiver (or alternate) to enter events as soon as possible after they are observed; and 2) an evening diary that will prompt the caregiver to review events for the day and to enter any events that were not previously captured. Events can be directly observed by the caregiver or could be reported to the caregiver by another observer such as a teacher. Each event will be characterized by a checklist of 15 observed behaviors: Yelling, Screaming, Threatening, Scratching, Throwing, Slamming, Hitting Self, Arguing, Cursing, Name Calling, Shoving, Hair Pulling, Fighting, Hitting Others, Kicking Others. The checklist will indicate whether each behavior was observed (coded 1) or was not observed (coded 0) during the incidence of an event. Each day can have multiple events. A day can have no event, as can be attested

in the evening diary. In this case, if no event is reported during a day, and the evening diary confirms this, the daily event score for that subject will be 0. Behaviors not on this list will not be captured.

# 5.2 **Secondary Efficacy Variables**

The following efficacy scales will be administered at visits designated in the Schedule of Visits and Procedures (Table 1).

#### 5.2.1 Clinical Global Impression (CGI) Scales

The CGI scale was developed to provide a brief, stand-alone assessment of the clinician's view of a subject's global functioning prior to and after administration of a SM (Guy 1976). Severity of illness (CGI-S) and global improvement (CGI-I) are both rated on a scale of 1 to 7 with 7 being "extremely ill" or "very much worse", respectively. Successful therapy is indicated by a lower overall score in subsequent testing. Investigators should consider their total clinical experience with children who have IA comorbid with ADHD and rate how severe the subject's condition is at the time.

- CGI-S will be evaluated by the Investigator at each visit on a 7-point scale with 1=Normal,
   2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill.
- CGI-I, relative to the condition at Visit 3, will be evaluated by the caregiver and by the
  Investigator at each post-baseline visit on a 7-point scale with 1=Very much improved, 2=Much
  improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very
  much worse.

CGI-S will be assessed by the Investigator at Visit 1, Visit 3, Visit 4, Visit 5 and Visit 6. CGI-I will be assessed by the caregiver and the Investigator at Visit 4, Visit 5 and Visit 6.

#### 5.2.2 Swanson, Nolan, Pelham Rating Scale- Revised (SNAP-IV)

The SNAP-IV rating scale includes 18 ADHD and 8 oppositional defiant disorder (ODD) symptoms as specified in the DSM-IV-TR and International Statistical Classification of Diseases and Health Related Problems 10th Revision (ICD-10) Classification of Mental and Behavioral Disorders. The symptoms are scored by assigning a severity estimate for each symptom on a 4-point scale (Swanson 2001). The SNAP-IV rating should be performed by the same parent or legal representative at each visit when possible.

The ratings from the SNAP-IV scale are grouped into the following 4 subscales:

- ADHD-Inattention (items #1-9),
- ADHD-Hyperactivity/Impulsivity (items #10-18)
- ODD (items #19-26)
- ADHD-Combined subscale: the first two subscale items are combined

Each subscale score is the average of the scores included in the subscale.

The SNAP-IV rating scale will be administered at Visit 3 and Visit 6.

#### 5.2.3 Child Health Questionnaire Parent Form 28- Item (CHQ-PF28)

The Child Health Questionnaire Parent Form 28-item (CHQ-PF28) is a short generic measure of health status and health related quality of life (Landgraf 1996). CHQ-PF28 items have four, five, or six response options, divided over eight multi-item scales (physical functioning, general behavior, mental health, self-esteem, general health perceptions, parental impact: emotional, parental impact: time, and family activities) and five single item concepts (role functioning: emotional/behavior, role functioning: physical, bodily pain, family cohesion, and change in health). The CHQ-PF28 should be performed by the primary caregiver when possible.

The CHQ-PF28 will be administered at Visit 3 and Visit 6.

# 5.2.4 Parenting Stress Index-Short Form (PSI-4-SF)

Reduction in stress is considered important for parents of children with disruptive behavior problems, developmental disabilities, and chronic illness (Haskett 2006). The Parenting Stress Index – Short Form (PSI-4-SF) is a 36-item self-report measure of parenting stress (Abidin 1995). Three subscales (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child) consist of 12 items each. Parents use a 5-point scale to indicate the degree to which they agree with each statement.

The PSI-4-SF will be administered at Visit 3 and Visit 6.

| 5.3 | Pharmacokinetic Measurements |
|-----|------------------------------|

#### 5.3.1 Pharmacokinetic Variables

The pharmacokinetic variables are:

- Apparent clearance (CL/F) of molindone in the pediatric population
- Apparent volume of distribution (V/F) of molindone in pediatric population
- Effect on molindone apparent clearance (CL/F) of co-administration of amphetamines, methylphenidate, clonidine, guanfacine and atomoxetine

# 5.3.2 Exploratory Pharmacokinetic Variables

| • |
|---|
| • |
| - |

# 5.4 Safety Assessments

Safety assessments will consist of monitoring of and recording of all concomitant medications and AEs, clinical laboratory tests, measurement of vital signs and 12-lead ECGs, suicidality monitoring, and the performance of physical examinations at visits designated in the Schedule of Visits and Procedures (Table 1).

Assessment of possible neurological side effects and EPS will be performed using the Simpson-Angus scale, the Barnes Akathisia scale and the AIMS. A positive rating or finding on the safety scale will be captured as an AE at the discretion of the Investigator.

#### 5.4.1 Adverse Events

As defined by the ICH Guideline for GCP, an adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with treatment.

#### An AE can be:

- Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
- Any new disease, intercurrent injuries, or exacerbation of an existing disease.
- Any deterioration in a laboratory value or other clinical test (e.g., ECG) that results in symptoms, a change in treatment, or discontinuation from SM.
- Recurrence of an intermittent medical condition (e.g., headache) not present at baseline.

Surgical procedures are not AEs; they are therapeutic measures for conditions that require surgery. The condition for which the surgery is required is an AE, if it occurs or is detected during the study period.

#### **5.4.1.1** *Causality*

AEs may be categorized as either Adverse Drug Reactions or Suspected Adverse Drug Reactions based on their relationship to SM and the degree of certainty about causality.

Suspected adverse drug reactions (SADRs) are a subset of adverse events for which there is evidence to suggest a causal relationship between the drug and the AE, i.e., there is a reasonable possibility that the drug caused the adverse event.

**Adverse drug reactions** (ADRs) are a subset of all SADRs for which there is reason to conclude that the drug caused the event.

#### 5.4.1.2 Recording and Evaluation of Adverse Events

All subjects who are enrolled (starting at Visit 3) will be questioned regarding the occurrence of AEs. At each contact with the subject, the investigator must seek information on AEs by specific questioning and, as appropriate, by examination. Information on all AEs should be recorded immediately in the source document, and also in the appropriate adverse event module of the eCRF. All clearly related

signs, symptoms, and abnormal diagnostic procedures results should be recorded in the source document, though they may be grouped under one diagnosis. For example, fever, elevated WBC, cough, abnormal chest X-ray, etc., can all be reported as "pneumonia".

All AEs occurring after enrollment and throughout the study period must be recorded. A treatmentemergent adverse event (TEAE) is defined as an AE with a start date on or after the first dose of study drug, or that worsened following first administration of study drug. For subjects who receive SM, TEAEs will be collected starting from the first dose of SM. The clinical course of each AE should be followed until resolution or until, in the medical judgment of the Investigator, the event has stabilized or is assessed as chronic.

An increase in the CSSRS, Simpson Angus Scale, Barnes Akathisia Scale, or the AIMS will not necessarily be rated as an AE unless the event meets AE criteria.

The Investigator is responsible for evaluating AEs and determining the following:

- Serious vs. Non-serious: Is the event a Serious Adverse Event (SAE)?
- Causality: Was AE related or possibly related to the SM?
- Severity: How pronounced is the incapacity/discomfort caused by an AE?

#### 5.4.1.3 Criteria for Assessing Severity

The Investigator will evaluate the comments of the subject and the response to treatment in order that he or she may judge the true nature and severity of the AE. Severity refers to the accumulated intensity of discomfort/impairment of health since the last recording of AEs and will be assessed according to the following criteria:

- Mild: Awareness of sign, symptom, or event, but easily tolerated
- Moderate: Discomfort enough to interfere with usual activity and may warrant intervention
- Severe: Incapacitating with inability to do usual activities or significantly affects clinical status and warrants intervention

The criteria for assessing severity are different from those used for seriousness.

#### 5.4.1.4 Criteria for Assessing Causality

The Investigator is responsible for determining the relationship between the administration of SM and the occurrence of an AE as **not suspected** or as a **suspected** reaction to SM. These are defined as follows:

<u>Not suspected</u>: The temporal relationship of the AE to SM administration makes a **causal relationship unlikely**, or other drugs, therapeutic interventions, or underlying conditions provide a sufficient explanation for the observed event.

• Not related: Temporal relationship to SM administration is missing or implausible, or there is an evident other cause.

• Unlikely related: Temporal relationship to SM administration makes a causal relationship improbable; and other drugs, chemicals, or underlying disease provide plausible explanations.

<u>Suspected</u>: The temporal relationship of the AE to SM administration makes a causal relationship possible, and other drugs, therapeutic interventions, or underlying conditions do not provide a sufficient explanation for the observed event.

- Possibly related: Temporal relationship to SM administration is plausible, but concurrent disease or other drugs or chemicals could also explain event. Information on drug withdrawal may be lacking or unclear. This will be reported as a Suspected Adverse Drug Reaction (SADR).
- Definitely related: Temporal relationship to SM administration is plausible, and concurrent
  disease or other drugs or chemicals cannot explain event. The response to withdrawal of the
  medication (dechallenge) should be clinically plausible. The event must be definitive
  pharmacologically or phenomenologically, using a satisfactory rechallenge procedure if
  necessary. This will be reported as an Adverse Drug Reaction (ADR).

#### 5.4.2 Serious Adverse Events (SAE)

AEs are classified as serious or non-serious. An AE or ADR is considered "serious" if, in the view of either the investigator or Sponsor, it results in one of the following outcomes:

- death
- life-threatening AE (i.e., the subject was at immediate risk of death from the AE as it occurred. This does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death.)
- in-patient hospitalization or prolongation of existing hospitalization
- persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions
- a congenital anomaly or birth defect
- an important medical event

Important medical events are those that may not be immediately life threatening or result in death or hospitalization, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above. For example, drug dependence or abuse, blood dyscrasias, a seizure that did not result in in-patient hospitalization, or intensive treatment for allergic bronchospasm in an emergency department would typically be considered serious.

#### 5.4.2.1 Investigator Responsibilities for Reporting SAEs

The Investigator must immediately report to the Sponsor all SAEs, regardless of whether the Investigator believes they are drug related.

All SAEs must be reported to the Drug Safety Contact within 24 hours of first becoming aware of the SAE. The Investigator must complete an SAE eCRF in EDC and include a detailed description of the SAE,

as well as other available information pertinent to the case (e.g., hospital records, autopsy reports and other relevant documents). Should the site be unable to access EDC, a paper SAE form must be completed and sent to prug Safety by email or fax. The investigator will keep a copy of this SAE Report form on file at the study site. Once EDC becomes available, the site must complete the SAE eCRF in EDC.

The Investigator or study physician, after thorough consideration of all facts that are available, must include an assessment of causality of an AE to SM in the report to the Sponsor.

Follow-up information, or new information available after the initial report, should be actively sought and reported to the Sponsor as it becomes available using the SAE Report Form.

The Drug Safety Contact for SAE reporting is:



#### 5.4.2.2 Other Events Requiring Immediate Reporting

The Investigator must report a pregnancy that occurs in a subject during a clinical study to the Drug Safety Contact within 24 hours of first becoming aware of the event. Pregnancy should be reported on a Pregnancy Report Form. The Investigator should discuss the case with the Medical Monitor; the Investigator must follow any pregnant subject for 3 months after the child is born. The Investigator must complete a Pregnancy Outcome Form as a follow up. Any AEs concerning the pregnancy of the subject during pregnancy or the child after birth must be documented and reported to the Sponsor.

Treatment-emerging EPS (e.g. akathisia, dystonia, Parkinsonism, tardive dyskinesia) and neuroleptic malignant syndrome should be reported to the Drug Safety Contact person(s) by completing the Adverse Event of Special Interest (AESI) eCRF in EDC. Should the site be unable to access EDC, a paper AESI form must be completed and sent to Drug Safety by email or fax within 24 hours of first becoming aware of the event. Once EDC becomes available the site must complete AESI eCRF in EDC. EPS incidence will be summarized and shared with study Investigators throughout the trial.

Overdosage of molindone presumably may be manifested by severe EPS and sedation. Coma with respiratory depression and severe hypotension resulting in a shock-like syndrome could occur. In the event of a suspected overdose, the parent or legal representative should be instructed to call 911 or their local poison control center at

Symptomatic, supportive therapy should be the rule. Gastric lavage is indicated for the reduction of absorption of molindone which is freely soluble in water. Since the adsorption of molindone by activated charcoal has not been determined, the use of this antidote must be considered of theoretical value.

Emesis in a comatose patient is contraindicated. Additionally, while the emetic effect of apomorphine is blocked by molindone in animals, this blocking effect has not been determined in humans.

#### 5.4.2.3 Sponsor Responsibilities for Expedited Reporting of SAEs

The Sponsor will inform Investigators and regulatory authorities of reportable events, in compliance with applicable regulatory requirements, on an expedited basis (i.e., within specific timeframes). For this reason, it is imperative that study sites submit SAE information to the Sponsor in the manner described above.

Investigators must comply with the applicable regulatory requirements related to the reporting of SAEs to the IRB/IEC. Investigators must also submit the safety information provided by the Sponsor to the IRB/IEC unless the country legal regulation requires that the Sponsor should be responsible for the safety reporting to the IRB/IEC.

It is the responsibility of the Sponsor to notify all participating investigators, in a written IND safety report, of any SADR that is both serious and unexpected. The Sponsor will also notify participating investigators of any findings from other sources (other studies, animal and in vitro testing, etc.) that suggest a significant risk for human subjects. Such findings will typically lead to safety-related changes in the study protocol, Informed Consent, and/or Investigator's Brochure.

#### 5.4.3 Management of Treatment-Emerging EPS

If a subject experiences treatment-emerging EPS (including akathisia, dystonia, Parkinsonism, or tardive dyskinesia), benztropine will be permitted at a starting dose of 0.5 mg BID up to a range of 1 to 4 mg/day. Lorazepam (1 to 2 mg per dose not to exceed three times daily) and clonazepam (0.25 to 1 mg per dose not to exceed twice daily) will also be permitted to treat emerging EPS.

A positive finding on an EPS safety assessment scale (Barnes Akathisia, Simpson-Angus, AIMS) does not necessarily equate to an EPS event. Investigators should evaluate positive findings on the EPS safety assessment scales and integrate them into a global clinical observation to determine if an AE of EPS should be recorded.

#### 5.4.4 Laboratory Measurements

With the exception of urine pregnancy test, clinical laboratory tests will be performed by a central laboratory as specified in the reference binder.

Details for collecting, handling, and shipping samples (including shipment addresses) will be detailed in a separate laboratory manual. The Schedule of Visits and Procedures (Table 1) shows the time points at which urine samples will be collected for urinalysis and blood samples will be collected for clinical laboratory tests and plasma concentration levels.

Table 3 presents the clinical laboratory tests to be performed. Metabolic parameters (including insulin, glucose, triglycerides, and cholesterol) and prolactin will be measured. A subject will be excluded if the Screening blood test results indicates > 2 times the upper limit of normal (ULN) of alanine

aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transpeptidase (GGT), and/or serum creatinine. Laboratory tests will not be repeated for these subjects.

All laboratory tests will be reviewed in a timely manner by qualified site personnel to ensure safety. Abnormal lab findings may be confirmed if necessary by one repeated testing at the discretion of the Investigator. Any repeat laboratory testing will be conducted under **fasting condition**. Any laboratory abnormality may qualify as an AE in the Investigator's judgment.

A total of approximately 42 mL of blood per subject will be drawn during the study: 22 mL is for clinical laboratory tests and 20 mL is for PK sampling.

**Table 3: Clinical Laboratory Tests** 

| Category | Parameters |
|---|---|
| Hematology | RBC, WBC, Hgb, HCT, MCH, MCHC, MCV, platelet count, and WBC with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils, large unstained cells) |
| Chemistry | Electrolytes: Na+, K+, chloride, bicarbonate |
| | <b>Liver function tests:</b> alkaline phosphatase, AST, ALT, total bilirubin, direct bilirubin ,indirect bilirubin |
| | Renal function parameters: BUN, creatinine |
| | Other: glucose, Ca <sup>+2</sup> , albumin, phosphorus, lactate dehydrogenase, total protein, CK/CPK, globulin, uric acid, triglycerides, insulin, prolactin, cholesterol – total, HDL and LDL Amylase, gammaGT (GGT), Iron, Lipase, Magnesium |
| Urine | Urinalysis |
| Office | Urine Drug Screen Urine pregnancy test (FOCBP only) |

#### 5.4.5 Vital Sign and Height/Weight Measurements

Vital sign measurements (e.g., blood pressure, heart rate, temperature, and respiratory rate) and height, weight and BMI will be obtained at visits designated on the Schedule of Visits and Procedures (Table 1). Blood pressure and heart rate will be measured after the subject has been sitting for 5 minutes. Vital signs may be taken at any other time, as deemed necessary by the Investigator.

#### 5.4.6 Medical History

Medical history will be collected at visits designated on the Schedule of Visits and Procedures (Table 1).

#### 5.4.7 Physical Examinations and Electrocardiograms (ECGs)

A physical examination and a 12-lead ECG will be obtained at visits designated on the Schedule of Visits and Procedures (Table 1). Additional ECGs may be performed at other times if deemed necessary by the Investigator.

The ECG will be recorded while the subject is resting in a supine position. The ECG will electronically measure the PR, QRS, QT, and QTc intervals, and heart rate.

All ECG tracings will be reviewed within 24 hours by the Investigator or qualified Sub-Investigator. PR intervals will be determined for each of these ECGs from a single reading. Invalid measurements will be repeated. QTc will be reported as QTcF (QT corrected using Fridericia's method).

### 5.4.8 Other Special Tests

The following special tests will be administered in the clinic at visits designated in the Schedule of Visits and Procedures (Table 1).

#### 5.4.8.1 K-SADS-PL 2013 Diagnostic Interview

The K-SADS-PL 2013 is a semi-structured diagnostic interview designed to diagnose current and past episodes of psychopathology in children and adolescents according to DSM-5 criteria (Kaufman 1997). We will use a version of K-SADS 2013 that was revised to be compatible to the DSM-5 criteria. It includes the parent and child DSM-5 cross-cutting symptoms measures (DSM-5 CC-SM); an unstructured Introductory Interview; the Diagnostic Screening Interview; the Supplement Completion Checklist; the Diagnostic Supplements and the Summary Lifetime Diagnostic Checklist. The K-SADS-PL 2013 will be used at screening to confirm the diagnosis of ADHD, as well as to rule out exclusionary diagnoses. The Screen Interview will assess the different diagnoses and determine which supplements should be completed. Supplement 4 (Neurodevelopment, Disruptive and Conduct Disorders) must be completed to assess ADHD, ODD, CD Tic and ASD. If an exclusionary diagnosis is confirmed, the remainder of the diagnostic will not be completed. This assessment will be administered at Visit 1.

#### 5.4.8.2 Simpson-Angus Scale

The Simpson-Angus scale is a 10-item rating scale that is widely used for assessment of neuroleptic-induced Parkinsonism (Simpson 1970). It consists of 1 item measuring gait, 6 items measuring rigidity, and three items measuring glabella tap, tremor and salivation, respectively. This assessment will be administered at Visit 3 and all subsequent visits.

#### 5.4.8.3 Barnes Akathisia Scale

The Barnes Akathisia scale is a rating scale for drug-induced akathisia and includes components for rating the observable, restless movements characteristic of akathisia, the awareness of restlessness, and any distress associated with the condition (Barnes 1989). This assessment will be administered at Visit 3 and all subsequent visits.

#### 5.4.8.4 Abnormal Involuntary Movement Scale (AIMS)

The AIMS test is a rating scale used to measure tardive dyskinesia (Munetz 1988). There are 12 items that rate involuntary movements of various areas of the subject's body. This assessment will be administered at Visit 3 and all subsequent visits.

#### 5.4.8.5 Vitiello Aggression Scale

The Vitiello Aggression Scale is a 10-item rating scale that uses a cluster analysis to categorize aggression into two subtypes, predatory (or planned) and affective (or impulsive) (Vitiello 1990). This assessment will be administered at Visit 1.

#### 5.4.8.6 Retrospective-Modified Overt Aggression Scale (R-MOAS)

The Retrospective-Modified Overt Aggression Scale (R-MOAS) was developed to gauge the severity of aggressive behavior (Blader 2010). Parents rate the frequency over the past week of 16 aggressive behaviors in four areas: verbal aggression; physical aggression toward others; aggression toward oneself; and destruction or hostile misuse of property. Numeric weighting amplifies the seriousness of more harmful behaviors in the total score. This assessment will be administered at Visit 1.

#### 5.4.8.7 Columbia Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a questionnaire that prospectively assesses suicidal ideation and behavior using a semistructured interview to probe patient responses (Posner 2011). The C-SSRS versions applicable to the current study are the Baseline version and the Since Last Visit version.

The Baseline version of the scale assesses lifetime suicidal ideation and behavior. This version is suitable as part of a subject's first interview and will be used at Visit 1 to identify volunteers who must not participate in the trial due to their suicidal tendencies.

The Since Last Visit version of the scale assesses any suicidal thoughts or behaviors the subjects may have had since the last administration of the C-SSRS. This version will be used for the other study visits.

#### 5.4.8.8 Infrequent Behaviors Checklist

The infrequent behaviors checklist is a checklist of 15 behaviors that (along with the 15 IA Diary behaviors) were qualitatively linked to IA during the development of the IA diary. These behaviors include teasing, spitting, biting, weapons, ripping, breaking, vandalizing, destroying, fire setting, hitting animal, kicking self, kicking animal, severe injury self, severe injury others, severe injury animal. Caregivers will be asked which, if any, of these behaviors have been observed since the patient's last visit. This assessment will be administered at Visit 3, Visit 4, Visit 5, and Visit 6.

#### **6 STATISTICAL METHODS**

### 6.1 Statistical and Analytical Plans

Tabular summaries of the data collected during the study will be presented to provide a general description of the subjects studied and an overview of the Efficacy, PK and safety results. Data from all sites will be combined in the computation of these summaries and summaries will be presented by treatment group. Continuous variables will be summarized using descriptive statistics (number of subjects, mean, standard deviation [SD], median, and minimum and maximum values). Categorical (nominal) variables will be summarized using frequency tables (number and percentage of subjects in each category).

In addition to tabular summaries, subject data listings, as specified in Sections 16.2 and 16.4 of ICH Guidance E3, will be provided. Additional subject data listings to be provided for this study are listed under the relevant subsections below. All data analyses will be performed by the CRO after the study is completed and the database is released. Statistical programming and analyses will be performed using SAS° and/or other validated statistical software as required.

Complete details of the statistical analysis will be provided in a separate statistical analysis plan (SAP), which will be written, finalized, and approved prior to database lock and will be included in the Clinical Study Report (CSR) for this protocol. The statistical analysis plan will supersede the statistical analysis methods described in this clinical protocol. Any deviation from the statistical plan will be documented and described in the final report. If changes to principal features stated in the protocol are required, these will be documented in a protocol amendment. The final SAP will take into account any amendment to the protocol.

In general, the baseline value for a variable is defined as the last observation prior to the first dose of double-blind study medication, ideally Visit 3, but including the screening value, if necessary.

# 6.2 Handling Missing Data

For the primary efficacy end point, the frequency of IA behaviors during the treatment period will be calculated over the number of days with non-missing IA diary data in the treatment period. No explicit imputation of missing data will be used, but this approach is implicitly equivalent to using the frequency of IA behaviors during the days with non-missing IA diary data to impute the frequency for days after study discontinuation and days with missing IA diary data.

#### 6.3 Analysis Populations

The population of "all enrolled subjects" consists of all those screened subjects who meet the requirements for study participation and are entered in the Baseline period of the study. The population of "all randomized subjects" consists of all those enrolled subjects who complete the Baseline Period, meet the inclusion/exclusion criteria and are randomized.

Safety Population: will include all randomized subjects who received at least 1 dose of study drug.

<u>Intent-to-Treat (ITT) Population</u>: will include all subjects who received at least 1 dose of study drug and have a baseline and at least 1 valid post-randomization assessment of frequency of IA behaviors based on IA diary entry.

<u>Per-Protocol (PP) Population</u>: will include all of the subjects in the ITT population who completed the treatment period with 80% diary completion compliance and who did not have major protocol deviations.

<u>PK population</u>: will include all subjects in the safety population who had at least one PK sample drawn which had a quantifiable concentration for at least one analyte of interest.

The safety, ITT, PP, and PK populations are based on randomized treatment received.

# 6.4 Demographic and Baseline Characteristics

Demographic/baseline variables include age, sex, ethnicity, race, and height at screening, weight at screening and baseline, and medical history. Tabular summaries of the demographic/baseline variables will be presented for the safety, ITT, and PP populations, except for medical history, which will be summarized for the safety population only.

# 6.5 Subject Disposition

A disposition of subjects will include the number and percentage of subjects in each of the following categories:

- Subjects in the randomized population
- Subjects in the ITT population
- Subjects treated (safety population)
- Subjects in the PP study population

Within each of the previous categories, the number and percentage of subjects who completed and discontinued from the study will be summarized. The reasons for study discontinuation will also be summarized. The reason for discontinuation may include any of the following:

- Subject withdrew consent
- Lost to follow-up
- Administrative reason
- Adverse event
- Investigator decision
- Failure to follow required study procedures
- Other

Only one (primary) reason for study discontinuation will be recorded for each subject.

#### 6.6 Protocol Deviations

Protocol deviations will be presented in listings. If applicable, the number and percent of subjects within each type of protocol deviation will be presented using discrete summary statistics. Protocol deviations will include, but are not limited to:

- Non-compliance with any scheduled study visit
- · Non-compliance with study treatment
- Disallowed concomitant medications
- Non-compliance with study inclusion or exclusion criteria
- Non-compliance with study assessment procedures

# 6.7 Study Medication Exposure and Compliance

Duration of exposure is defined as the total number of days a subject is exposed to any study treatment. This will be calculated for each subject by taking the difference between the date of last dose *minus* the date of the first dose, *plus* 1 (date of last dose – date of first dose +1).

Duration of Treatment exposure will also be summarized using descriptive statistics (n, mean, SD, median, minimum, and maximum).

Percent of study drug compliance is defined as  $\{(\text{number of tablets dispensed} - \text{number of tablets returned}) / 2*(date of last dose - date of first dose + 1)}* 100%.$ 

For each treatment, SM compliance will be summarized by compliance category (<80%, 80-120%, and >120%) and number of subjects in each compliance category. Study medication compliance will also be summarized as a continuous variable using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) for each treatment.

Summaries of treatment compliance and exposure will be presented separately for the Titration Period, Maintenance Period, and combined Titration and Maintenance Periods.

#### 6.8 Concomitant Medications

Concomitant medications will be assigned an 11-digit code using the World Health Organization Drug Dictionary (WHO DD) drug codes. Concomitant medications will be further coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating therapeutic classification. A tabular summary of concomitant medications by drug class will be presented for the safety population.

# 6.9 Efficacy Analyses

#### 6.9.1 Primary Efficacy Analysis

The primary efficacy endpoint is the percent change ( $PCH_T$ ) in the frequency (unweighted score) of IA behaviors per 7 days in the Treatment (Titration and Maintenance) period relative to the Baseline period calculated over the number of days with non-missing IA diary data. The frequency of IA behaviors per 7 days is the sum of scores for all events in a given period of sequential days, adjusted to 7 days.

The primary efficacy endpoint PCH $_T$  will be calculated by PCH $_T$ = 100\*(T–B)/B, where T and B are IA behavior frequencies per 7 days during the Treatment period and baseline period, respectively. The IA behavior frequency per 7 days is defined as (SUM/DAY) x 7, where SUM is the sum of the IA behaviors reported in the subject IA diary, and DAY is the number of days with non-missing IA frequency data in the subject IA diary during the specified study period.

Let  $\mu_1$ ,  $\mu_2$ , and  $\mu_3$  represent the median percent change in the frequency of IA behaviors per 7 days in the Treatment period relative to the Baseline period in the ITT population for subjects treated with Placebo, 18 mg and 36 mg doses of SPN-810, respectively. The null (H<sub>0</sub>) and the alternative (H<sub>a</sub>) hypotheses are as in the following.

- $H_{01}$ :  $\mu_2 = \mu_1$ , (there is no difference between the median of the 18 mg dose SPN-810 and the median of placebo) vs.  $H_{a1}$ :  $\mu_2 \neq \mu_1$ , (there is a difference between the median of the 18 mg dose SPN-810 and the median of placebo)
- $H_{02}$ :  $\mu_3 = \mu_1$ , (there is no difference between the median of the 36 mg dose SPN-810 and the median of placebo) vs.  $H_{a2}$ :  $\mu_3 \neq \mu_1$ , (there is a difference between the median of the 36 mg dose SPN-810 and the median of placebo)

The primary efficacy analysis will be performed using the Wilcoxon rank-sum test to compare the medians of each of the two doses of SPN-810 (18 mg and 36 mg) with the median of the Placebo. The Hodges-Lehmann estimate and the associated 95% confidence interval (CI) will be calculated. To preserve the overall Type I error-rate at 0.050 for the primary efficacy endpoint, multiplicity adjustment due to interim analysis and two comparisons of SPN-810 dose group (18 mg and 36 mg) with the Placebo will be performed as described in Section 10.1.4.

### 6.9.2 Secondary Efficacy Analyses

The secondary endpoints are:

- 1. Actual Caregiver CGI-I score at Visit 6
- 2. Actual Investigator CGI-I score at Visit 6
- 3. Change from Visit 3 to Visit 6 in Investigator CGI-S score
- 4. Change from Visit 3 to Visit 6 in CHQ-28 score
- 5. Change from Visit 3 to Visit 6 in PSI-4-SF scores in:
  - a. Parental Distress
  - b. Parent-Child Dysfunctional Interaction
  - c. Difficult Child
- 6. Change from Visit 3 to Visit 6 in SNAP-IV ADHD scores in:
  - a. Inattention ratings
  - b. Hyperactivity/Impulsivity ratings
  - c. Combined Scale ratings

Each one of the six secondary endpoints will be analyzed using the analysis of covariance method based on the ITT population with missing data imputed using the Last Observation Carried Forward (LOCF) method. The model includes treatment and baseline as fixed independent covariates and change from baseline to final maintenance visit as a response variable. The least squares mean of each treatment group, the difference in the least squares mean (18mg dose minus placebo and 36 mg dose minus placebo), and the 2-sided 95% CI for the difference will be obtained.

To preserve the overall type I error rate at 0.05 for the secondary endpoints, a sequential testing procedure will be used with the following features. First only dose or doses that are significantly different from placebo for the primary endpoint will be tested for secondary endpoints. The first of the secondary endpoints will be compared to placebo using the Hochberg step up procedure but only using those doses retained as a result of testing the primary endpoint (Hochberg 1988). The second secondary endpoint will be tested in the same manner but only using those doses that were retained from the

primary and the first secondary endpoint and so forth. As the endpoints are gone through in the predefined order doses will only be retained if significant for all endpoints tested so far and at the given stage the Hochberg step-up procedure will be applied.

The ordering of the 6 secondary endpoints from first to be tested to sixth is: Investigator Clinical Global Impression – Improvement Scale (CGI-I)(Endpoint 1), Clinical Global Impression – Severity Scale (CGI-S) (Endpoint 2), Child Health Questionnaire (CHQ-28) (Endpoint 3), Parenting Stress Index (PSI-4-SF) (Endpoint 4), Caregiver-completed CGI-I (Endpoint 5) and SNAP-IV Rating Scale (Endpoint 6).

#### 6.9.3 Sensitivity Analysis

In the presence of a high drop-out rate, performance of sensitivity analysis is crucial. The purpose of sensitivity analysis is to see whether different methods of handling missing data provide consistent and similar results for the primary efficacy analysis. To this end, the three sensitivity analyses will be performed:

- 1. Multiple imputation under MAR using available data on the primary endpoint
- 2. Placebo- based imputation under MNAR
- 3. Per Protocol Analysis

#### 6.9.3.1 Multiple imputation under Missing at Random (MAR)

The multiple imputation (MI) method assumes that the missing data are missing at random (MAR), that is, the probability that an observation is missing may depend on the observed values but not the missing values. For example, if a subject's Diary values are available on Day 1 and Day 2 but missing on Day 3, then the missing value on Day 3 is related to the non-missing value on Day 1 and Day 2.

MI is implemented using the following three steps.

- 1) SAS PROC MI is applied with input dataset containing some missing values for all days during the titration and maintenance period to create 100 datasets. The data sets will include separate columns for the frequency of incidences during each day starting from baseline. The Markov Chain Monte Carlo (MCMC) method will be used to complete the missingness pattern to a monotone pattern separately by treatment arm. The monotone patterns will be achieved by applying sequential imputation based on Bayesian regression with the treatment arm included as a covariate. All copies contain identical values of the non-missing data items, but different values imputed for missing values.
- 2) For each of these MI data sets, the percent change will be computed as in the observed data set and the primary analysis based on the Wilcoxon rank-sum test will be conducted and asymptotic 95% confidence intervals will be constructed.
- 3) To produce a single confidence interval for each dose placebo comparison (e.g., Dose 1 versus placebo), PROC MIANALYZE will be used and Rubin's combination rules will be applied to the treatment effect estimates and associated asymptotic standard errors from the MI data sets.

The treatment effect estimates will be defined as the midpoints of the asymptotic confidence intervals and the standard errors will be defined as the asymptotic standard errors (based on the width of the associated 95% confidence intervals) from the Hodges-Lehmann estimate of the individual datasets (Rubin 1987).

#### 6.9.3.2 Multiple imputation under Missing Not at Random (MNAR)

This approach can be labeled "worst-case" sensitivity analyses as it assumes that after discontinuation subjects from the dosing arms would adopt the outcome model estimated from the placebo arm. To generate missing values from this "placebo-based" imputation model, PROC MI with the MNAR statement (available in SAS 9.3 and later versions) will be used or, alternatively, SAS macros available at the DIA Missing Data Working Group site (Ratitch et al., 2013; Ayele et al., 2014) can be used.

#### 6.9.3.3 Per Protocol Analysis

This analysis will be conducted by repeating the primary analysis on the per protocol population.

# 6.10 Sample Size and Power Considerations

Based on results from the Phase 2 study, it is assumed that the average treatment difference between SPN-810 dose groups and placebo is 11.51 with a common standard deviation of 27.3. A sample size of 132 subjects per arm (264 subjects for 3 arms) will yield 90% power to detect a non-zero difference between the median of 18 mg or 36 mg dose group and the placebo using the Wilcoxon rank-sum test with a 2-sided significance level alpha=0.05.

It is assumed that approximately 20% of subjects will dropout before the completion of the study and hence, an adjusted total of 330 subjects will be randomized in a 1:1:1 ratio to obtain 264 subjects in the ITT population at the completion of the study.

The sample size was calculated using the nQuery Advisor Software, Version 7.

#### 6.11 Interim Analysis

The main purpose of the interim analysis is to re-estimate the sample size. The sample size estimate described in the sample size Section 6.10 is based on effect size assumptions from the Phase 2 data in which the primary endpoint was the change from baseline to endpoint in R-MOAS ratings. However, the primary endpoint for this study is percent change in the frequency of IA incidence per 7 days in the Treatment (Titration and Maintenance) period (PCH<sub>T</sub>) relative to the Baseline period in the ITT population calculated over the number of days with non-missing IA diary data. Hence, there is uncertainty as to what magnitude of alternative hypothesis treatment difference and between-subject variability is appropriate to pre-specify. To this end, a single interim analysis is planned after approximately 50% of subjects complete the study. The adaptive design plan for the interim analysis plan is presented in the Appendix 10.1.

#### 6.12 Assessment of MCIC

Based on unblinded data available at study close, the ability of a percent change (PCH) endpoint to detect change will be evaluated using three anchor-based minimal clinically important change (MCIC)

estimates obtained from two global impression of change (CGI-I) variables and one global impression of severity (CGI-S) variable. Consistent with the recommendations of Hays (Hays et al., 2005), the assessment of detection of clinically meaningful change will emphasize unstandardized anchor-based estimates "so that users of the measure will be able to interpret differences in the raw metric."

The anchor-based MCIC values will be obtained by estimating the average PCH for minimal improvement groups defined by ratings from two raters for two concepts. Investigators and caregivers will each rate global impression of change. These will be known as Investigator-rated CGI-I and Caregiver-rated CGI-I, respectively. However, only investigators will rate global impression of severity (CGI-S). These CGI-I/CGI-S measures will be obtained at multiple site visits (Visit 3, Visit 4, Visit 5, and Visit 6) throughout the study period to reduce recall error and quantify incremental change over time. Investigator-rated CGI-I and Caregiver-rated CGI-I will be assessed on a 7-point scale with 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse. CGIS will be evaluated on a 7-point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill. Minimal improvement groups (rating of 3) for a fixed assessment contrast (e.g. Visit 3 vs. Visit 4, Visit 3 vs. Visit 5, and Visit 3 vs. Visit 6) define the MCIC anchor on Investigator-rated CGI-I and Caregiver-rated CGI-I. To define an MCIC anchor on CGI-S, the difference in severity ratings across assessment interval (e.g. Visit 4 minus Visit 3, Visit 5 minus Visit 3, and Visit 6 minus Visit 3) will be calculated with those exhibiting minimal improvement in severity across intervals used to define the MCIC anchor. Minimal improvement on CGI-S is calculated as a one category change of improvement, e.g. changing from a value of mildly ill at baseline to borderline ill at titration or markedly ill at baseline to moderately ill at maintenance.

To calculate MCIC for each of the CGI-I/CGI-S anchors defined above, PCH scores will be calculated by visit: Visit 4, Visit 5, and Visit 6. With three visits at which MCIC will be calculated, the three PCH variables may be expressed as  $PCH_{3,4} = 100 * \left(\frac{V4-B}{B}\right)$ ,  $PCH_{3,5} = 100 * \left(\frac{V5-B}{B}\right)$ , and  $PCH_{3,6} = 100 * \left(\frac{V6-B}{B}\right)$ , where V4-B, V5-B, and V6-B are the difference in unweighted scores adjusted to 7 days between Visit 4 and baseline, Visit 5 and baseline, and Visit 6 and baseline, respectively. The MCIC values will be obtained from an ANOVA estimated using SAS' GLM procedure with PCH as outcome and the anchors: Investigator-rated CGI-I, Caregiver-rated CGI-I, and change in CGI-S scores as fixed independent classification variables. With three assessment occasions (Visit 4, Visit 5 and Visit 6) for which PCH will be calculated and three anchors (Investigator-rated CGI-I, Caregiver-rated CGI-I, and CGI-S) at each occasion there will be a total of 9 PCH and anchor combinations. A Separate one-way ANOVA will be fit for each of the 9 PCH and anchor combinations. Within a given PCH and anchor combination, the average PCH value for each level of the anchor will be estimated, with the MCIC estimate corresponding to the average PCH value for the minimal improvement group. Consistent with current best practice for MCIC reporting, (Hays et al., 2005) the ANOVA estimated 95% confidence interval for the MCIC estimates will also be provided. MCIC estimates will be triangulated in an attempt to establish the ability of the IA diary score to detect clinically meaningful change.

In addition, the cumulative distribution functions (CDFs) for PCH from baseline to each visit will be explored graphically. The CDFs for each anchor category stratum will be plotted for each assessment

combination (visit 3 vs. 4, visit 3 vs. 5, and visit 3 vs. 6), and within each assessment combination three anchor-specific CDF plots will be generated. Given that the CGI-I and CGI-S each have seven categories, CDFs for the CGI-I and CGI-S measures will display seven total CDFs. Given that the CGI-S has seven categories but the anchor will be converted to one-category change values for MCIC estimation, an additional CGI-S plot will be produced displaying six CDFs, one for each one-category change value (1 to 2, 2 to 3, . . . , 6 to 7) at each assessment combination in order to assess the uniformity of PCH across each possible one-point change combination. In addition, the CDFs for each treatment arm will be plotted. To augment the interpretation of the IA diary's ability to detect meaningful change, the MCIC estimates will be demarcated in the treatment-stratified CDF plots and the treatment-arm specific proportions achieving the MCIC estimates will be reported and compared.

# 6.13 Pharmacokinetic Analyses

#### 6.14 Safety Analyses

Evaluation of safety will be performed for the safety population. Safety data that will be evaluated include concomitant medications, AEs, clinical laboratory results, vital signs, ECGs, and findings from the physical examinations. The occurrence of neurological side effects will be assessed by looking at any worsening in scores from Visit 3 to each subsequent visit for each of the Simpson-Angus scale, Barnes Akathisia scale, and AIMS. Suicidal ideation and suicidal behavior will be measured by C-SSRS.

All summary tables related to safety analyses will use the safety population.

#### 6.14.1 Adverse Events

AEs will be classified into standardized medical terminology from the verbatim description (Investigator term) using the Medical Dictionary for Regulatory Activities (MedDRA). AEs will be summarized using discrete summaries at the subject and event level by system organ class and preferred term for each treatment group. Similarly, treatment-emergent AEs will be summarized by severity and relationship separately. Verbatim description and all MedDRA level terms, including the lower level terms, for all AEs will be contained in the subject data listings.

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

All AEs occurring after randomization and throughout the study period will be recorded. For subjects who receive SM, treatment-emergent AEs (TEAEs) will be collected starting after the first dose of SM (Visit 3) to the end of the study. These AEs include those that emerge during treatment or worsen in severity during treatment. These AEs will be tabulated, listed and analyzed.

Separate TEAE incidence tables will be presented for the three treatment groups. The incidence rates for all SADRs will also be summarized as described for all TEAEs.

In addition, these same tables will be presented by treatment period (Titration, Maintenance, and combined Titration and Maintenance). For the combined Titration and Maintenance Periods, the incidence of TEAEs will also be presented by highest severity reported and the dose of SM at first occurrence.

Listings (and tabular summaries, if warranted) of deaths, other SAEs, and other significant TEAEs, including TEAEs resulting in treatment discontinuation, will be provided.

#### 6.14.2 Laboratory Values

Clinical laboratory values will be summarized by visit by treatment group using descriptive statistics for hematology and biochemistry. For quantitative laboratory parameters, both actual values and change from baseline values will be summarized.

Laboratory test results will be assigned a low, normal, high (LNH) classification according to whether the values were below (L), within (N), or above (H) the laboratory parameters' reference ranges provided by the central laboratory. Within-treatment comparisons will be based on three by three tables (shift tables) that, for a particular laboratory test, compare the LNH classification at baseline to the LNH classification at visit. By subject-listings of all abnormal laboratory values, i.e., those with L or H classification will be provided.

#### 6.14.3 Vital Signs, Height and Weight

Vital signs will be summarized by visit by treatment group using descriptive statistics. Both actual values changes from baseline to visit will be summarized. Descriptive summary statistics (mean, SD, median, and range) for vital sign data, height, weight and BMI will be evaluated by treatment group.

#### 6.14.4 ECG Results

By-visit tabular summaries of the quantitative ECG parameters and the overall ECG findings (normal, abnormal not clinically significant, or abnormal clinically significant) will be presented. The QT will be corrected using Fridericia's method.

ECG results will be summarized by visit by treatment group using descriptive statistics (for quantitative ECG parameters) and frequency tables (for qualitative ECG parameters, including the overall ECG finding). For quantitative ECG parameters, both actual values and change from screening values will be summarized.

#### 6.14.5 Physical Examinations

Findings from the physical examinations will be listed for each system or area examined.

#### 6.14.6 Columbia Suicide Severity Rating Scale (C-SSRS)

C-SSRS outcomes will be summarized using number and percent of subjects by categories for suicidal ideation only, suicidal behavior only and suicidality (ideation and behavior combined). The summary will be presented by treatment groups. The proportion of subjects in each treatment group will be compared with the proportion of subjects in the placebo group using Fisher's exact test or Chi-square test as applicable if appropriate.

#### 6.14.7 Infrequent Behaviors Checklist

Infrequent behaviors will be listed for each subject by treatment group.

#### 6.14.8 Other Special Tests

The occurrence of neurological side effects will be assessed by looking at the changes in scores from baseline to post-baseline visits for each of the Simpson-Angus scale, Barnes Akathisia scale, and AIMS. For each item on each of these scales, the number (and percentage) of subjects with a worse score at any post-baseline visit, compared to baseline, will be presented. A listing of these subjects will also be provided.

#### 7 DOCUMENTATION

#### 7.1 Adherence to the Protocol

The Investigator agrees, when signing the protocol, to adhere to the instructions and procedures described in the protocol and to adhere to the principles of ICH GCP to which the protocol conforms as well as all governing local regulations and principles for medical research.

The protocol, ICF, and appropriate related documents must be reviewed and approved by an IRB constituted and functioning in accordance with ICH E6 and any local regulations. Documentation of IRB compliance with the ICH and any local regulations regarding constitution and review conduct will be provided to the Sponsor.

A signed letter of study approval from the IRB Chairman must be sent to the Investigator with a copy to the Sponsor prior to study start and the release of any SM to the site by the Sponsor or its designee. If the IRB decides to suspend or terminate the study, the Investigator will immediately send the notice of study suspension or termination by the IRB to the Sponsor.

Study progress is to be reported to IRB annually (or as required) by the Investigator or Sponsor, depending on local regulatory obligations. If the Investigator is required to report to the IRB, he/she will forward a copy to the Sponsor at the time of each periodic report.

#### 7.2 Changes to the Protocol

There are to be no changes to the protocol without written approval from the Sponsor.
Any change to the protocol requires a written protocol amendment or administrative change that must be approved by the Sponsor before implementation. Amendments specifically affecting the safety of subjects, the scope of the investigation, or the scientific quality of the study require additional approval by the applicable IRBs and, in some countries, by the regulatory authority. These requirements should in no way prevent any immediate action from being taken by the Investigator, or by the Sponsor, in the interest of preserving the safety of all subjects included in the study. If an immediate change to the protocol is warranted as per the Investigator, for safety reasons, the Medical Monitor and IRB must be notified promptly.

Changes affecting only administrative aspects of the study do not require formal protocol amendments or IRB approval, but the IRB must be kept informed of such changes. In these cases, the Sponsor will send a letter to the IRB detailing such changes.

#### 7.3 Protocol Deviations

There are to be no Investigator-initiated deviations from the protocol. Any subject whose treatment deviates from the protocol or who is not qualified for study participation may be ineligible for analysis and may compromise the study. The date of and reason for deviations must be documented in all cases. Significant or major protocol deviations impacting the safety of the subject or the integrity of the study must be reported by the Investigator to the IRB immediately. Reporting of all other protocol deviations must adhere to the requirements of the governing IRB. Protocol assessments will continue until the end of the study, unless the protocol deviations put the subject at risk or the subject's condition requires that he/she be discontinued from the study.

#### 7.4 Data Quality Assurance

This study will be organized, performed, and reported in compliance with the protocol, standard operating procedures (SOPs), working practice documents, and applicable regulations and guidelines. Site visit audits may be made periodically by the Sponsor's Quality Assurance team or qualified designee, which is an independent function from the study conduct team.

#### 7.4.1 Data Collection

The primary source document will be the subject's medical record. If separate research records are maintained by the Investigator(s), both the medical record and the research record will be considered the source documents for the purposes of monitoring and auditing the study.

Electronic data collection techniques will be used to collect data directly from the study sites using eCRFs. The electronic data will be stored centrally in a fully validated clinical database.

| /programs. |
|------------|

Data recorded on source documents will be transcribed into the eCRFs in accordance with the eCRF Completion Instructions that are provided to the study sites. The Investigator is responsible for ensuring that all sections of each eCRF are completed correctly, and that entries can be verified against source documents. The eCRFs will be monitored for completeness and accuracy against the source documents by the CRA(s) on a regular basis. Inconsistencies between the eCRFs and source documents will be resolved in accordance with the principles of GCP.

Completed eCRFs will be extracted from the clinical database, stored as PDF files on a CD-ROM and sent to the respective study site for archiving. A CD-ROM containing all eCRFs will be kept by the Sponsor in the Sponsor's Trial Master File.

#### 7.4.2 Clinical Data Management

Data from eCRFs and other external data (e.g., laboratory data) will be entered into or merged with a clinical database as specified in the data management plan. Quality control and data validation procedures will be applied to ensure the validity and accuracy of the clinical database.

#### 7.4.3 Database Quality Assurance

In accordance with the vendor's procedures, the clinical database will be reviewed and checked for omissions, apparent errors, and values requiring further clarification using computerized and manual procedures. Data queries requiring clarification will be documented and returned to the study site for resolution. Only authorized personnel will make corrections to the clinical database, and all corrections will be documented in an audit trail.

# 7.4.4 Bioanalytical Data Management and Quality Control

#### 7.5 Retention of Records

The Investigator has the responsibility to retain all study "essential documents", as described in ICH E6. Essential documents include but not limited to the protocol, copies of paper CRFs or eCRFs, source documents, laboratory test results, SM inventory records, Investigator's Brochure, regulatory agency registration documents (e.g., FDA form 1572, ICFs, and IRB/IEC correspondence). The investigator should take measures to prevent accidental or premature destruction of these documents. Study essential documents should be retained until at least two years after the last approval of a marketing application or after formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by an agreement with the Sponsor. The Investigator must obtain written permission from the Sponsor prior to the destruction of any study document.

It is requested that at the completion of the required retention period, or should the Investigator retire or relocate, the Investigator contact the Sponsor, allowing the Sponsor the option of permanently retaining the study records.

These records must be made available at reasonable times for inspection and duplication, if required, by a properly authorized representative of the US FDA in accordance with the US 21 CFR 312.68 or other national or foreign regulatory authorities in accordance with regulatory requirements.

#### 7.6 Auditing Procedures

In addition to the routine monitoring procedures, the Sponsor's Corporate Quality Assurance department or qualified designee may conduct audits of clinical research activities in accordance with the Sponsor's written SOPs to evaluate compliance with the principles of ICH GCP and all applicable local regulations. A government regulatory authority may also wish to conduct an inspection (during the study or after its completion). If an inspection is requested by a regulatory authority, the Investigator must inform the Sponsor and the CRO immediately that this request has been made.

These records must be made available at reasonable times for inspection and duplication, if required, by a properly authorized representative of the US FDA in accordance with the US 21 CFR 312.68 or other national or foreign regulatory authorities in accordance with regulatory requirements.

#### 7.7 Publication of Results

Any presentation or publication of data collected as a direct or indirect result of this trial will be considered as a joint publication by the Investigator(s) and the appropriate personnel at the Sponsor's site. Authorship will be determined by mutual agreement. All manuscripts, abstracts or other modes of presentation arising from the results of the study must be reviewed and approved in writing by the Sponsor, prior to submission for publication or presentation. No publication or presentation with respect to the study shall be made until any Sponsor comments on the proposed publication or presentation have been addressed to the Sponsor's satisfaction.

The detailed obligations regarding the publication of any data, material results, or other information, generated or created in relation to the study shall be outlined in the agreement between each Investigator and the Sponsor or designee.

#### 7.8 Financing and Insurance

Financing and Insurance information will be set forth in a separate document between the Investigator and Sponsor (provided by the Sponsor or designee).

#### 7.9 Disclosure and Confidentiality

The contents of this protocol and any amendments and results obtained during the course of this study will be kept confidential by the Investigator, the Investigator's staff, and IRB and will not be disclosed in whole or in part to others or used for any purpose other than reviewing or performing the study without the written consent of the Sponsor. No data collected as part of this study will appear in any written work, including publications, without the written consent of Sponsor.

All persons assisting in the performance of this study must be bound by the obligations of confidentiality and non-use set forth in the Confidentiality Agreement between the Investigator and Sponsor.

#### 7.10 Discontinuation of Study

The Sponsor reserves the right to discontinue the study for medical or administrative reasons at any time. The Investigator will be reimbursed for reasonable expenses covering subjects, use of live-in facilities, laboratory tests, and other professional fees. The Investigator will refund the excess of payments made in advance.

The Investigator reserves the right to discontinue the study should his/her judgment so dictate. The Investigator will notify the IRB in case of study discontinuation. Study records must be retained as noted above.

#### 8 ETHICS

#### 8.1 Institutional Review Boards / Independent Ethics Committees

A list of the Institutional Review Board(s) (IRB) and/or Independent Ethics Committee(s) (IEC) that approved this study and the approval letters will be included in the clinical study report for this protocol.

The protocol, any protocol amendments, and the informed consent form (ICF) will be reviewed and approved by the appropriate IRB before subjects are screened for entry. Verification of the IRB unconditional approval of the protocol will be transmitted to the Sponsor prior to the shipment of study medication to the investigational site. The Investigators or Sponsor will submit, depending on local regulations, periodic reports and inform the IRB of any reportable adverse events (AEs) per International Conference on Harmonization (ICH) guidelines and local IRB standards of practice.

#### 8.2 Ethical Conduct of the Study

This study will be conducted in accordance with standard operating procedures (SOPs) of the Sponsor and the Contract Research Organizations (CRO) that will conduct the study. These SOPs are designed to ensure adherence to Good Clinical Practice (GCP) guidelines as required by:

- Declaration of Helsinki, 1964 ("Recommendations Guiding Physicians in Biomedical Research Involving Human Patients"), and all its accepted amendments to date concerning medical research in humans.
- ICH Guideline for GCP (Committee for Proprietary Medicinal Products/ICH/135/95) of the European Agency for the Evaluation of Medicinal Products, Committee for Proprietary Medicinal Products, ICH of Pharmaceuticals for Human Use.
- United States (US) Code of Federal Regulations (CFR) dealing with clinical studies (21 CFR, including parts 50 and 56 concerning Patient Informed Consent and IRB regulations).
- Local, national legal guidelines.

#### 8.3 Investigators and Study Personnel

This study will be conducted by qualified Investigators under the Sponsorship of Supernus Pharmaceuticals, Inc. (Sponsor) at approximately 25 study sites in the US.

Contact persons at the Sponsor and the CROs are listed in the reference binder provided to each investigational site. The study will be monitored by qualified personnel from the designated CRO by visiting the study sites. The Sponsor will oversee and review the monitoring activities of the monitors. Medical writing, data management, and statistical analyses will be performed by the CROs. Laboratory tests will be conducted by a central laboratory as designated in the reference binder.

#### 8.4 Subject Information and Consent/Assent

The Investigator (or designee) will inform the subject and their parent(s), or legal representative, of all aspects pertaining to the subject's participation in the study and will provide oral and written information describing the nature and duration of the study, the procedures involved, the expected duration, the potential risks and benefits involved, and any potential discomfort.

The process for obtaining informed consent/assent will be in accordance with all applicable regulatory requirements. The Investigator (or designee) and the parent (or legal representative) must sign and date the Informed Consent Form (ICF)/Informed Assent Form (IAF) before the subject can participate in the study. The parent or legal representative and the subject will be given a copy of the signed and dated consent/assent form and the original will be retained in the investigational site study records.

The decision regarding subject participation in the study is entirely voluntary. The Investigator (or designee) must emphasize to the subject and their parent(s) or legal representative that consent regarding study participation may be withdrawn at any time without penalty or loss of benefits to which the subject is otherwise entitled.

The ICF/IAF should be given by means of a standard written statement, written in non-technical language. The subject should understand the statement before signing and dating it. If written consent is not possible, oral consent may be obtained if witnessed by at least one person not involved in the study. The verbal consent will be documented and signed by the Investigator and the witness(es). No subject can enter the study before his/her ICF has been obtained.

If the ICF/IAF is amended during the study, the Investigator must follow all applicable regulatory requirements pertaining to approval of the amended ICF by the IRB and use the amended informed consent form (including ongoing subjects).

#### 9 REFERENCE LIST

Abidin RR. Parenting Stress Index. (3rd ed.) Odessa, FL: Psychological Assessment Resosurces, Inc., 1995.

Aman MG, Bukstein OG, Gadow KD et al. What does risperidone add to parent training and stimulant for severe aggression in child attention-deficit/hyperactivity disorder? J Am Acad Child Adolesc Psychiatry 2014; 53:47-60 e1.

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

Armenteros JL, Lewis JE, Davalos M. Risperidone augmentation for treatment-resistant aggression in attention-deficit/hyperactivity disorder: A placebo-controlled pilot study. J Am Acad Child Adolesc Psychiatry 2007; 46:558-65.

Ayele BT, Lipkovich I, Molenberghs, G, Mallinckrodt, CH. A multiple imputation based approach to sensitivity analyses and effectiveness assessments in longitudinal clinical trials. Journal of Biopharmaceutical Statistics 2014; 24, 211-228.

Barnes TRE. A rating scale for drug-induced akathisia. Br. J. Psychiatry 1989; 154:672-676.

Blader JC, Pliszka SR, Jensen PS, Schooler NR, Kafantaris V. Pediatrics 2010;126(4):e796-806.

Calarge CA, Acion L, Kuperman S et al. Weight gain and metabolic abnormalities during extended risperidone treatment in children and adolescents. J Child Adolesc Psychopharm 2009; 19:101-9.

Chen YH, DeMets DL, Lan KKG. Increasing the sample size when the unblinded interim result is promising. Statistics in Medicine 2004; 23: 1023-1038.

Connor DF, Mc Laughlin TJ. Aggression and diagnosis in pychiatrically referred children. Child Psychiatry Hum. Dev. 2006; 37(1):1-14.

Farmer CA, Arnold LE, Bukstein OG, Findling RL, Gadow KD, Li X, Butter EM, Aman MG. The treatment of severe child aggression (TOSCA) study: Design challenges. Child and Adolescent Psychiatry and Mental Health 2011; 5:36.

Findling RL, Steiner H, Weller EB. Use of antipsychotics in children and adolescents. J. Clin. Psychiatry 2005; 66:29-40.

Gadow KD, Arnold LE, Molina BS et al. Risperidone added to parent training and stimulant medication: Effects on attention-deficit/hyperactivity disorder, oppositional defiant disorder, conduct disorder, and peer aggression. J Am Acad Child Adolesc Psychiatry 2014; 53:948-59.

Greenhill LL, Barmack JE, Spalten D, Anderson M, Halpern F. Molindone hydrocholoride in the treatment of aggressive, hospitalized children. Psychopharmacol. Bull. 1981; 1:125-127.

Greenhill LL, Solomon M, Pleak R, Ambrosini P. Molindone hydrochloride treatment of hospitalized children with conduct disorder. J. Clin. Psychiatry 1985; 46:20-25.

Guy W. Clinical global impressions. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD. U.S. National Institute of Health, Psychopharmacology Research Branch 1976; 217-222.

Haskett ME, Ahern LS, Ward CS, Allaire JC. Factor structure and validity of the parenting stress index-short from. J. Clin. Child Adolesc. Psychol. 2006; 35(2):302-312.

Hays RD, Farivar SS, Liu H. Approaches and recommendations for estimating minimally important differences for health related quality of life measures. COPD 2005; 2(1): 63–67.

Hochberg Y. A sharper Bonferroni procedure for multiple significance testing. Biometrika 1988; 75(4):800-802.

Jensen PS, Youngstrom EA, Steiner H, Findling RL, Meyer RE, Malone RP, Carlson GA, Coccaro EF, Aman MG, Blair J, Dougherty D, Ferris C, Flynn L, Green E, Hoagwood K, Hutchinson J, Laughren T, Leve LD, Novins DK, Vitiello B. Consensus Report on Impulsive Aggression as a Symptom Across Diagnostic Categories in Child Psychiatry: Implications for Medication Studies. J. Am. Acad. Child Adolesc. Psychiatry 2007; 46 (3):309-322.

Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, et al. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry 1997; 36(7):980-8.

Kaufman, AS, Lichtenberger, E. Assessing Adolescent and Adult Intelligence. 3rd Edition; 2005.

Landgraf JM, Abetz L, Ware JE. The CHQ User's Manual. Boston. First Edition Boston, MA: The Health Institute, New England Medical Center 1996.

McClellan J, Sikich L, Findling RL, Frazier JA, Vitiello B, Hlastala SA, et al. Treatment of early-onset schizophrenia spectrum disorders (TEOSS): Rationale, design, and methods. J. Am. Acad. Child Adolesc. Psychiatry 2007; 46:969-978.

McKay KE, Halperin JM. ADHD, aggression, and antisocial behavior across the lifespan. Ann NY Acad Sci 2001; 931:84-96.

Mehta CR, Pocock SJ. Adaptive increase in sample size when interim results are promising: a practical guide with examples. Statistics in Medicine 2000; 00:1-6.

The MTA Cooperative Group. A 14-month randomized clinical trial of treatment strategies for attention-deficit/hyperactivity disorder. The MTA Cooperative Group. Multimodal Treatment Study of Children with ADHD. Arch Gen Psychiatry 1999; 56:1073-86.

Munetz MR, Benjamin S. How to examine patients using the abnormal involuntary movement scale. Hosp. Commun. Psychiatry 1988; 39:1172-1177.

Pappadopulos E, Macintyre II JC, Crismon ML et al. Treatment recommendations for the use of antipsychotics for aggressive youth (TRAAY). Part II. J Am Acad Child Adolesc Psychiatry 2003; 42:145-61.

Penzner JB, Dudas M, Saito E et al. Lack of effect of stimulant combination with second-generation antipsychotics on weight gain, metabolic changes, prolactin levels, and sedation in youth with clinically relevant aggression or oppositionality. J Child Adolesc Psychopharm 2009; 19:563-73.

Pliszka S, AACAP Work Group on Quality Issues. Practice parameter for the assessment and treatment of children and adolescents with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry 2007; 46:894-921.

Pliszka SR, Crismon ML, Hughes CW et al. The Texas Children's Medication Algorithm Project: Revision of the algorithm for pharmacotherapy of attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry 2006; 45:642-57.

Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity rating scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry 2011; 68: 1266-1277.

Ratitch B, O'Kelly, M, Tosiello, R. Missing data in clinical trials: from clinical assumptions to statistical analysis using pattern mixture models. Pharmaceutical Statistics, 2013; 12, 337-347.

Rubin D.B. Multiple Imputation for Nonresponse in Surveys, New York, Wiley; 1987.

Scotto Rosato N, Correll CU, Pappadopulos E et al. Treatment of maladaptive aggression in youth: Cert guidelines ii. Treatments and ongoing management. Pediatrics 2012; 129:e1577-86.

Shelton TL, Barkley RA, Crosswait C et al. Psychiatric and psychological morbidity as a function of adaptive disability in preschool children with aggressive and hyperactive-impulsive-inattentive behavior. J Abnorm Child Psychology 1998; 26:475-94.

Sikich L, Frazier JA, McClellan J et al. Double-blind comparison of first- and second-generation antipsychotics in early-onset schizophrenia and schizo-affective disorder: Findings from the treatment of early-onset schizophrenia spectrum disorders (TEOSS) study. Am J Psychiatry 2008; 165:1420-31.

Simpson GM, Angus JWS. A rating scale for extrapyramidal side effects. Acta Psychiatr. Scand. Suppl. 1970; 212:11-19

Stocks JD, Taneja BK, Baroldi P et al. A phase 2a randomized, parallel group, dose-ranging study of molindone in children with attention-deficit/hyperactivity disorder and persistent, serious conduct problems. J Child Adolesc Psychopharm 2012; 22:102-11.

Swanson JM, Kraemer HC, Hinshaw SP, Arnold LE, Conners CK, Abikoff HB, et al. Clinical relevance of the primary findings of the MTA: Success rates based on severity of ADHD and ODD symptoms at the end of treatment. J. Amer. Acad. Child Adolesc. Psychiatry 2001; 40:168-179.

Supernus Pharmaceuticals, Inc. Single-Center, Single-Dose, Open-Label, Randomized, Incomplete Crossover Pilot Study to Evaluate the Single Dose Pharmacokinetics of Controlled and Immediate Release Formulations of Molindone Hydrochloride in Healthy Adult Volunteers Under Fed and Fasted Conditions 2010.

Supernus Pharmaceuticals, Inc Study 810P202. A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of Molindone Hydrochloride Extended-Release Tablets as Adjunctive Therapy in Children with Impulsive Aggression Comorbid with Attention-Deficit/Hyperactivity Disorder (ADHD) 2013.

Supernus Pharmaceuticals, Inc Study 810P501. Psychometric Testing of an Electronic Observer-Reported Outcome Measure of Impulsive Aggression of Children with Attention Deficit Hyperactivity Disorder 2015.

Vitiello B, Behar D, Hunt, J, Stoff, D, Riccuiti, A. Subtyping Aggression in Children and Adolescents. J. Neuropsychiatry Clin. Neurosciences 1990; 2:189-192.

Vitiello B, Stoff DM. Subtypes of aggression and their relevance to child psychiatry. J. Am. Acad. Child Psychiatry 1997; 36(3):307-315.

#### 10 APPENDICES

#### 10.1 Adaptive Design Plan

#### 10.1.1 Introduction

The document defines the key elements of the adaptive design for Protocol 810P301 (A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Molindone Hydrochloride Extended-Release Tablets for the Treatment of Impulsive Aggression in Pediatric Subjects with Attention Deficit/Hyperactivity Disorder (ADHD) in Conjunction with Standard ADHD Treatment).

#### 10.1.2 Trial Design

The trial will be designed to evaluate the efficacy and safety profiles of two doses of SPN-810 compared to placebo. For compactness, the doses will be denoted by Dose 1 (18 mg) and Dose 2 (36 mg).

A two-stage design with a single interim analysis and final analysis (FA) will be utilized in this trial:

- Stage 1 will include subjects who complete the trial prior to the Interim Analysis.
- Stage 2 will include subjects who complete the trial after the Interim Analysis.

The Interim Analysis data will be reviewed in an unblinded manner to potentially increase the number of subjects in Stage 2. The sample sizes in each stage of the trial will be denoted as follows:

- Let  $n_1$  denote the total number of subjects who complete the trial prior to Interim Analysis (in other words, this will be the total sample size in Stage 1). The number of subjects allocated to Dose 1, Dose 2 and Placebo in Stage 1 will be denoted by  $n_{11}$ ,  $n_{12}$  and  $n_{13}$ , respectively. Note that  $n_{11} + n_{12} + n_{13} = n_1$
- Let  $n_2$  denote the total number of subjects in Stage 2 without sample size adjustment at Interim Analysis. The number of subjects allocated to Dose 1, Dose 2 and Placebo in Stage 2 will be denoted by  $n_{21}$ ,  $n_{22}$  and  $n_{23}$ , respectively. Note that some of these sample sizes will be set to 0 if a decision to drop a dosing arm is made at IA and  $n_{21} + n_{22} + n_{23} = n_2$ .

#### 10.1.3 Decision Rules at Interim Analysis

As indicated above, Interim Analysis will be conducted mainly to support a decision to increase the number of subjects in Stage 2 if the observed treatment difference for the primary endpoint is less than anticipated. It is important to note that subject enrollment will not be terminated in either dosing arm at Interim Analysis due to overwhelming efficacy and, as a consequence, no  $\alpha$  will be spent at Interim Analysis. However, subject enrollment may be terminated due to futility as explained below.

Interim Analysis will be performed after a pre-defined fraction the total number of subjects complete the trial, i.e., approximately 50% of subjects complete the final visit.

The following sample size reassessment rule will be applied at Interim Analysis. Let CP define the dose-specific conditional power at Interim Analysis, i.e., the probability of establishing a significant treatment effect on the primary endpoint conditional upon the primary endpoint data available at Interim Analysis under the original sample size assumptions. In particular, CP1 is defined as conditional power based on the comparison of Dose 1 to placebo at Interim Analysis and CP2 is defined as conditional power based on the comparison of Dose 2 to placebo at Interim Analysis.

The trial's design will be modified at Interim Analysis using the following thresholds (CP refers to either CP1 or CP2):

- If CP < 0.1, discontinue subject enrollment in this particular dosing arm (e.g., subjects will be allocated to Dose 2 or placebo in Stage 2 if CP1 < 0.1 and CP2 ≥ 0.1).</li>
- If  $CP \ge 0.1$  and  $CP \le 0.36$ , retain the original sample size in the dosing arm.
- If CP ≥ 0.36 and CP ≤ 0.8, increase the sample size in the dosing arm.
- If CP > 0.8, retain the original sample size in the dosing arm.

The sample size will be increased in a dosing arm to achieve the nominal power of 80% before the multiplicity adjustment or the sample size will be doubled, whichever is smaller.

The following rules will be applied to compute the sample sizes across the treatment arms in Stage 2:

- If a decision to discontinue subject enrollment is made for a particular dosing arm at Interim
  Analysis, subjects who were planned to be enrolled in that arm after Interim Analysis will be redistributed to the remaining treatment arms. For example, if Dose 1 is dropped and Dose 2 is
  retained, the sample sizes for the three treatment arms in Stage 2 will be defined as follows:
  - o Dose 1: 0.
  - $\circ$  Dose 2:  $n_{22} + n_{12}/2$ .
  - o Placebo:  $n_{23} + n_{12}/2$ .
- If a decision is made to increase the sample size in at least one dosing arm, the modified sample size in the placebo arm will be equal to the larger modified sample size in the two dosing arms. For example, if the modified sample sizes in the two dosing arms in Stage 2 are n<sub>31</sub> and n<sub>32</sub>, respectively, the modified sample size in the placebo arm in Stage 2 will be set to max(n<sub>31</sub>, n<sub>32</sub>). However, if the sample size is increased in one dosing arm, the sample size in the other dosing arm will not be automatically increased.

#### 10.1.4 Adaptive Design

This section defines the mathematical approach used in the proposed adaptive design with two stages and data-driven decision rules (e.g., sample size modification at Interim Analysis). The derivation of the adaptive design is based on the combination function approach applied in conjunction with the closure principle, see, for example, Wang et al. (2001), Brannath et al. (2002) and Hommel (2005). This general approach is commonly used to construct adaptive designs in confirmatory trials and guarantees that the overall Type I error rate is protected in the trial at the nominal level (two-sided  $\alpha$ = 0.05) regardless of the type of design modifications at an Interim Analysis, including decisions to drop a treatment arm or adjust the sample size in one or more arms.

Let  $H_1$  and  $H_2$  denote the null hypotheses of no treatment effect for the two dose-placebo comparisons (Dose 1 versus placebo and Dose 2 versus placebo). According to the combination function approach, the amount of evidence to reject these null hypotheses will be evaluated separately in each individual stage of the trial and the inferences at FA will be performed by combining the evidence across the two stages. Further, the rejection rules for  $H_1$  and  $H_2$  will be chosen to achieve consistency with the Hochberg procedure (Dmitrienko and D'Agostino, 2013) that was pre-defined as multiplicity adjustment tool in this trial. To achieve this consistency, the Hochberg procedure will be applied within each stage (Hochberg, 1988).

Let  $p_i$  and  $q_i$  denote the p-values for testing the null hypothesis  $H_i$ , i=1,2, based on the data in Stages 1 and 2, respectively. The Stage 2 p-values are computed from the samples obtained after Interim Analysis, i.e., the sample size in a dosing arm may be adjusted. Further,  $p_{(1)} < p_{(2)}$  will denote the ordered treatment effect p-values in Stage 1 and similarly  $q_{(1)} < q_{(2)}$  will denote the ordered treatment effect p-values in Stage 2. These p-values will be used to construct a closure-based representation of the Hochberg procedure in each of the two stages. To define the closure-based representation, a closed family of intersection hypotheses that includes all possible non-empty intersections of the two null hypotheses will be set up. Table 1 and Table 2 display the intersection hypotheses in the closed family and associated intersection p-values that define the Hochberg procedure in Stage 1 and Stage 2 respectively.

Table 1: Intersection hypothesis and Hochberg intersection p-values in Stage 1.

| Intersection hypothesis | Hochberg intersection p-value |
|-------------------------|--------------------------------------|
| $H_1 \cap H_2$ | $p_{12} = \min (2 p_{(1)}, p_{(2)})$ |
| H <sub>1</sub> | <i>p</i> <sub>1</sub> |
| H <sub>2</sub> | <i>p</i> <sub>2</sub> |

Table 2: Intersection hypothesis and Hochberg intersection p-values in Stage 2.

| Intersection hypothesis | Hochberg intersection p-value |
|-------------------------|----------------------------------------|
| $H_1 \cap H_2$ | $q_{12} = \min (2 \ q_{(1)}, q_{(2)})$ |
| H <sub>1</sub> | $q_1$ |
| H <sub>2</sub> | $q_2$ |

Note that, if a certain dose is dropped due to futility at Interim Analysis, the corresponding p-values in Stage 2 is automatically set to 1 to remove the dosing arm from consideration. This guarantees that a null hypothesis cannot be rejected at FA if the corresponding dose was dropped due to futility at Interim Analysis. Further, the p-values computed at Interim Analysis (Stage 1 p-values) are not used for inferential purposes and therefore no  $\alpha$  will be spent at Interim Analysis to stop the trial early due to overwhelming efficacy.

As an illustration, if Dose 1 is dropped at Interim Analysis, the corresponding treatment effect p-value in Stage 2 ( $q_1$ ) will be set to 1. As a result, the intersection p-values will be defined in Stage 2 as shown in Table 3 (note that the smaller ordered p-value will be equal to  $q_2$  and the larger ordered p-value will be equal to 1).

Table 3: Intersection hypotheses and Hochberg intersection p-values in Stage 2 if dose 1 is dropped at Interim Analysis.

| Intersection hypothesis | Hochberg intersection p-value |
|-------------------------|-------------------------------|
| $H_1 \cap H_2$ | $q_{12} = \min(2 q_2, 1)$ |
| H <sub>1</sub> | 1 |
| H <sub>2</sub> | $q_2$ |

The inferences for the two null hypotheses will be performed at FA using the composite treatment effect p-values that will be defined as follows. Let  $w_1$  and  $w_2$  define the stage weights that are prospectively defined based on the expected amount of information at Interim Analysis. Since Interim Analysis is planned to be taken after 50% of the subjects have completed the trial,

 $n_1$  (total sample size in Stage 1) =  $n_2$  (total sample size in Stage 2 before sample size adjustment), and thus the pre-specified stage weights are given by

$$w_1 = \frac{n_1}{n_1 + n_2} = 0.5$$
,  $w_2 = \frac{n_2}{n_1 + n_3} = 0.5$ .

Using the stage weights, the combination function to be used at FA will be defined as follows:

$$c(x_1, x_2) = 1 - \Phi \left[ \sqrt{w_1 \Phi^{-1} (1 - x_1)} + \sqrt{w_2 \Phi^{-1} (1 - x_2)} \right],$$

where  $\Phi(x)$  is the cumulative distribution function of the standard normal distribution.

This combination function will be applied to compute composite intersection p-values for each intersection hypothesis in the closed family. The resulting composite intersection p-values are denoted by  $r_{12}$ ,  $r_1$ ,  $r_2$ , and are defined in Table 4.

Table 4: Intersection hypothesis and composite intersection p-values at FA.

| Intersection hypothesis | Composite intersection p-value |
|-------------------------|--------------------------------|
| $H_1 \cap H_2$ | $r_{12} = c(p_{12}, q_{12})$ |
| H <sub>1</sub> | $r_1=c(p_1,q_1)$ |
| H <sub>2</sub> | $r_2=c(p_2,q_2)$ |

After that, the null hypothesis  $H_1$  will be rejected at FA (which implies a statistically significant treatment effect at Dose 1) if the composite p-values for all intersection hypotheses in the closed family that contain  $H_1$  are significant at  $\alpha = 0.05$  (two-sided), i.e.,

$$r_{12} \le \alpha$$
 and  $r_1 \le \alpha$ .

Similarly, the null hypothesis  $H_2$  will be rejected at FA (and a statistically significant treatment effect will be established at Dose 2) if the composite p-values for all intersection hypotheses in the closed family that contain  $H_2$  are significant at  $\alpha = 0.05$ , i.e.,

$$r_{12} \le \alpha$$
 and  $r_2 \le \alpha$ .

As indicated above, the resulting approach accounts for two sources of multiplicity in this clinical trial (multiple data looks and multiple dose-placebo comparisons) and guarantees Type I error rate control at  $\alpha = 0.05$ . The  $\alpha$  control is retained even if the sample size is adjusted in or more treatment arms at Interim Analysis. In addition, it needs to be emphasized that a null hypothesis cannot be rejected at FA if the corresponding dose was dropped due to futility at Interim Analysis.

#### 10.1.5 Important Interim Analysis Considerations

#### 10.1.5.1 Responsible Party

The Interim Analysis will be performed by an independent unblinded statistician who is not affiliated to the trial sponsor, trial management, data cleaning, and analysis.

The Head of Clinical Research and Director of Biostatistics at Supernus (sponsor) will receive recommendation letter from the independent unblinded statistician. They will make the final decision for the sample size adjustment.

#### 10.1.5.2 Confidentiality

The independent statistician will sign the confidentiality agreement. He/she will not reveal any unblinded data/information to any persons within his/her own organization or to the sponsor, with the exception of sending recommendation as described in Section 10.1.5.1 above.

#### References

Brannath W, Posch M, Bauer P. Recursive combination tests. Journal of the American Statistical Association. 2002; 97: 236-244.

Dmitrienko, A., D'Agostino, R.B. Tutorial in Biostatistics: Traditional multiplicity adjustment methods in clinical trials. Statistics in Medicine. 2013; 32:5172-5218.

Hommel, G. Adaptive modifications of hypotheses after an interim analysis. Biometrical Journal. 2005; 5: 581-589.

Wang, SJ, Hung HMJ, Tsong Y, Cui L. Group sequential test strategies for superiority and non-inferiority hypotheses in active controlled clinical trials. Statistics in Medicine. 2001; 20: 1903-1912.

#### 10.2 Retrospective Modified Overt Aggression Scale (R-MOAS)

| A. Child's First Name: B. Child's Last Name | | Staff Entries | roject Participant |
|---|---|---|---|
| | | 1 1 1 1 1 1 | i II I I I I |
| C. Your First Name: D. Your Last Name: | | Visit Type V | isit # |
| | | | 100 |
| E. Your Relationship to Child: | | Month De | av {ear |
| Mother O Father O Grandmother O Grandfather | er Other | 1 1 1/1 | <u>run ta</u> |
| Retrospective Modified Overt | Aggressi | on Scale | (R-MOAS) |
| nstructions: These questions focus on difficulties indicate how many times each of the | | | |
| /erbal Incidents: | <u>0 - 1 times</u> | 2 - 4 times | 5 or more time |
| . How many times did your child shout angrily, curse, or insult people but then stopped quickly? | | 0 | |
| . How many times did your child shout angrily, curse, or insult people in a repetitive, out-of-control way durin episodes that lasted less than five minutes? | | _0_ | |
| . How many times did your child shout angrily, curse, or insult people in a repetitive, out-of-control way durin episodes that lasted more than five minutes? | | 0 | |
| . How many times did your child threaten to hurt someon | ne?O | O | O |
| Other verbal incidents (Please describe): | | | |
| ncidents Toward Other People: Nor How many times did your child act like he/she | ne <u>1 - 2 times</u> | 3 - 4 times | 5 or more time |
| was about to hit somebody or took a swing at someone without actually hitting another person? | 0 | 0 | O |
| . How many times did your child hit someone with hands or an object, kick, push, scretch or | | | |
| pull hair, without causing real injury? | )0 | 0_ | |
| How many times did your child do any of the things in Item 2 and caused some mild injury (bruises, sprains, welts, etc.)? | | _0_ | |

| | | (/Ei-/) | | |
|---|---|---|---|---|
| ncidents Involving Property: | None | 1 - 2 times | 3 - 4 times | 5 or more times |
| How many times did your child slam a door or<br>cabinet, rip clothing, or knock something<br>over in anger? | 0_ | | | |
| t. How many times did your child throw things<br>down, kick furniture, or otherwise misuse<br>things angrily but did not break them? | | 0 | 0 | -0 |
| How many times did your child break things, smash windows, or damage or deface property on purpose? | | 0 | 0 | 0 |
| How many times did your child set a fire or<br>throw things at people in order to hurt them? | - | _0_ | 0 | 0 |
| Other incidents involving property (Please descri | ibe): | | | |
| ncidents Directed Toward Self: How many times did your child pick at or scratch his or her skin, pull out hair, or hit himself or herself while upset or angry? | None | 1 - 2 times | 3 - 4 times | 5 or more time |
| | O_ | O | _0_ | 0 |
| or throw himself or herself on the floor? | O- | 0 | 0 | |
| <ol> <li>How many times did your child cut, bruise,<br/>or burn himself or herself on purpose?</li> </ol> | | o | 0 | |
| How many times did your child severely<br>injure himself or herself, or try to kill<br>himself or herself? | | 0 | 0 | 0 |
| 5. Other incidents in which your child acted harmful | lly toward | himself or herse | elf (Please des | cribe): |
| | | | Staff Use: | |
| | | | | H |
| | | | | R |
| | | | Si | |
| | | | Total | |

#### 10.3 Clinical Global Impression (CGI) Scale

| (1) NOT DONE | | |
|---|---|---|
| appropriate numbered be | ate only one response for the quest<br>ox. | ion by placing a cross (x) in the |
| | | cular population ( <i>impulsive aggression</i> ition at this time? |
| (0) NOT ASSESSED | (1) Normal, not at all ill | (4) Moderately ill |
| | (2) Borderline mentally ill | (5) Markedly ill |
| | (3) Mildly ill | (6) Severely ill |
| | | $\square$ (7) Among the most extremely ill patient |
| | ent. Compared to his/her conditi | hether or not, in your judgment, it is due<br>ion at Visit 1/Baseline, how much has the |
| (0) NOT ASSESSED | (1) Very much improved | (4) No change |
| (0) NOT ASSESSED | (1) Very much improved (2) Much improved | (4) No change (5) Minimally worse |
| (0) NOT ASSESSED | | |

#### 10.4 Vitiello Scale

#### Predatory-Affective Aggression Scale

| Patie | nt | - | |
|---|---|---|---|
| Rater | | Date | _ |
| Chec | k if any these behaviors is usual for this patient (i.e., it in): | has occurred at leas | at 3 times during the last |
| | | YES | NO |
| 1. | Non profitable damaging of own property | 1 | 0 |
| 2. | Hides aggressive acts | 1 | 0 |
| 3. | Exposes self to physical harm when aggressive | 1 | 0 |
| 4. | Is aggressive without a purpose | 1 | 0 |
| 5. | Can control own behavior when aggressive | 1 | 0 |
| 6. | Aggression is unplanned, out of the blue | 1 | 0 |
| 7. | Very careful to protect self when aggressive | 1 | 0 |
| 8. | Completely out of control when aggressive | 1 | 0 |
| 9. | Plans aggressive acts | 1 | 0 |
| 10. | Steals | 1 | 0 |

#### Scoring:

Predatory score: sum of items 2, 5, 7, 9, and 10 Affective score: sum of items 1, 3, 4, 6, and 8 Total score: difference of Predatory score minus Affective score/

Possible range of total score: from 5 (completely predatory) to -5 (completely affective)

#### Reference:

B. Vitiello et al. (1990), J. Neuropsychiatry Clin. Neurosciences 2:189-192.

#### 10.5 Kiddie-Sads-Present and Lifetime Version (K-SADS-PL) 2013

# K-SADS-PL 2013

#### Includes:

- A. Screen Interview
- **B. Supplements** 
  - I. Depressive and Bipolar Related Disorders Supplement
  - II. Schizophrenia Spectrum and Other Psychotic Disorders Supplement
  - III. Anxiety, Obsessive-Compulsive, and Trauma-Related Disorders Supplement
  - IV. Neurodevelopmental, Disruptive, and Conduct Disorders Supplement
  - V. Eating Disorders and Substance-Related Disorders Supplement

Advanced Center for Intervention and Services Research (ACISR)

for Early Onset Mood and Anxiety Disorders

Western Psychiatric Institute and Clinic

Child and Adolescent Research and Education (CARE)

Program, Yale University

| Subject | | | |
|---------|-----|-------------|-----|
| Date / | 2 0 | Interviewer | Fr. |



#### **ACKNOWLEDGEMENTS**



The authors extend appreciation to the many consultants who contributed to this instrument including Oscar Bukstein MD, John Campo MD, Carrie Christopher Fascetti, MSW, Andrew Gilbert MD, Benjamin Goldstein MD, Tina Goldstein PhD, Diane Goudreau, PhD, Megan Muir Grivas, MA, Ben Handen MD, Ami Klin, PhD, David Kolko PhD, Walter Kaye, MD, Rolf, Loeber, PhD, Catherine Lord, PhD, Martin Lubetsky MD, William Pelham, PhD, David Rosenberg, MD, Rita Scholle BA, Eunice Torres, MS, and John Walkup, MD. Special thanks are given to Denise Carter-Jackson and Jason Lyons, MA for the extensive reformatting of earlier version of this instrument.

The authors of the KSADS-PL 2013 acknowledge the prior authors and earlier versions of this instrument which laid the foundation of the current KSADS-PL: the K-SADS-P (Present Episode Version), which was developed by William Chambers, MD and Joaquim Puig-Antich, MD, and later revised by Joaquim Puig-Antich, MD and Neal Ryan, MD; the K-SADS-E by Helen Orvaschel, PhD and Joaquim Puig-Antich, MD, the K-SADS-PL by Joan Kaufman, PhD, Boris Birmaher, MD, David Brent, MD, Uma Rao, MD, and Neal Ryan, MD, and the KSADS-PL-2009 Working. Draft was developed by David Axelson MD, Boris Birmaher MD, Jamie Belazny RN,

MPH, Joan Kaufman PhD, and Mary Kay Gill MSN with support provided by the Advanced Center for Intervention and Services Research (ACISR, MH66371) Pt. David Brent MD. The current instrument is also greatly indebted to several other existing structured and semi-structured psychiatric instruments including the SADS-L (Spitzer and Endicott), the SCID (Spitzer, Williams, Gibbon, and First), the DIS (Robins and Helzer), the ISC (Kovacs), the DICA (Reich, Shayka, and Taibleson), and the DUSI (Tarter, Laird, Bukstein, and Kaminer). Guidelines for the introductory interview at the beginning of this instrument were initially provided by Michael Rutter, M.D. and Philip Graham, M.D., and refined with subsequent renditions of the KSADS.

| - | 1 1 1 1 | |
|---------|---------|------------|
| Subject | | المريو الم |
| | | n Com |



## TABLE OF CONTENTS Screen Interview









#### Schedule for Affective Disorders and Schizophrenia for School Aged Children (6-18 Years)

page I of xiv

#### Kiddie-SADS - Lifetime Version (K-SADS-PL 2013

The K-SADS-PL 2013 combines dimensional and categorical assessment approaches to diagnose current and past episodes of psychopathology in children and adolescents according to DSM-5 criteria. Prior to administering the interview portion of the K-SADS-PL, parents and children are to complete the DSM-5 cross-cutting 25-item symptom rating scales. Responses on these dimensional rating scales are then taken into account in completing the interview portion of the assessment. The primary diagnoses assessed with the K-SADS-PL 2013 include: Major Depression, Persistent Depression, Mania, Hypomania, Cyclothymia, Bipolar Disorders, Disruptive Mood Dysregulation Disorder, Schizoaffective Disorders, Schizophrenia, Schizophreniform Disorder, Brief Psychiotic Disorder, Panic Disorder, Agoraphobia, Separation Anxiety Disorder, Simple Phobia, Social Anxiety Disorder, Selective Mutism, Generalized Anxiety, Obsessive Compulsive Disorder, Attention Deficit Hyperactivity Disorder, Conduct Disorder, Oppositional Defiant Disorder, Enuresis, Encopresis, Anorexia Nervosa, Bulimia, Binge Eating Disorder, Transient Tic Disorder, Tourette's Disorder, Chronic Motor or Vocal Tic Disorder, Alcohol Use Disorder, Substance Use Disorder, Post-Traumatic Stress Disorder, Adjustment Disorders, and Autism Spectrum Disorder.

The K-SADS-PL 2013 is a semi-structured interview. The probes that are included in the interview do not have to be, and should <u>not</u> be recited verbatim. Rather, they are provided to illustrate ways to elicit the information necessary to score each item. The interviewer should feel free to adjust the probes to the developmental level of the child, and use language supplied by the parent and child when querying about specific symptoms.

After reviewing parent and child responses on the DSM-5 cross-cutting rating scales, the K-SADS-PL 2013 is administered by interviewing the parent(s), the child, and finally achieving summary ratings which include all sources of information (parent, child, school, chart, and other). In general, when administering the instrument to pre-adolescents, conduct the parent interview first. In general, when working with adolescents, begin with them. There may be clinical reasons to alter the order of administration.

When there are discrepancies between different sources of information, the rater will have to use his/her best clinical judgment. In the case of discrepancies between parents' and child's reports, the most frequent disagreements occur in the items dealing with subjective phenomena where the parent does not know, but the child is very definite about the presence or absence of certain symptoms. This is particularly true for items like guilt, hopelessness, interrupted sleep, hallucinations, and suicidal ideation. If the disagreements relate to observable behavior (e.g. truancy, fire setting, or a compulsive ritual), as appropriate, the examiner should query the parent(s) and child about the discrepant information. Ultimately the interviewer will have to use his/her best clinical judgment in assigning the summary ratings.



2013

## KSADS-PL SCREEN INTERVIEW:

page ii of xiv



The following guidelines should be used in coding symptoms:

- 1) Current Diagnoses: In coding current episodes (CE) of disorders, symptoms should be rated for the time period when they were the most severe during the episode. Note in the margins if and when particular symptoms (e.g. insomnia) improved or resolved. Patients typically present when symptoms are at the worst. In follow-up research assessments, symptoms may be in partial remission.
- 2) Disorders Targeted with Medication. In coding disorders treated with medication (e.g. ADHD), use the ratings to describe the most intense severity of symptoms experienced prior to initiation of medication, when medications wear off, or during 'drug holidays'. Note in margins symptoms targeted effectively with medication.
- 3) Past Diagnoses: In order for an episode to be considered 'resolved' or 'past', the child should have had a minimum of two months free from the symptoms associated with the disorder. Episodes rated in the past disorders section should represent the most severe past (MSP) episode experienced of that given disorder.
- 4) Time Line: For children with a history of recurrent or episodic disorders, it is recommended that a time line be generated to chart lifetime course of disorder and facilitate scoring of symptoms associated with each episode of illness.

In the process of completing the full interview, diagnoses initially believed to be 'past' may turn out to be current diagnoses in partial remission. Corrections in the coding of current and past severity ratings can be made after completion of the interview.

Administration of the K-SADS-PL 2013 requires the completion of; 1) the parent and child DSM-5 cross-cutting symptoms measures (DSM-5 CC-SM); 2) an unstructured Introductory Interview; 3) a Diagnostic Screening Interview; 4) the Supplement Completion Checklist; 5) the appropriate Diagnostic Supplements; andd6) the Summary

Lifetime Diagnostic Checklist. The K-SADS-PL is initially completed with each informant separately. If there is no suggestion of current or past psychopathology, no assessments beyond the Screen Interview will be necessary. The Summary Lifetime Diagnostic Checklist is completed after synthesizing all the data and resolving discrepancies in informants' reports. Each of the phases of the KSADS-PL interview is discussed briefly below.

- 1) The DSM-5 Cross-Cutting Symptom Measures (DSM-5 CC-SM). The DSM-5 CC-SM are designed to be self-report measures completed independently by the parent and child before beginning the KSADS interview. Scores on these self-report scales should be reviewed and recorded in the spaced provided before beginning the interview portion of the KSADS. The DSM-5 CC-SM include 25-items that assess symptom severity over the past two weeks. The parent and child DSM-5 CC-SM are included at the end of the KSADS. The American Psychiatric Association recommends specific follow-up measures that can be completed if threshold scores are obtained on the 25-item DSM-5 CC-SM, and several disorder specific severity scales. These additional scales can be accessed at: http://www.psychiatry.org/practice/dsm/dsm5/online-assessment-measures#Level1, but do not need to be completed as part of the KSADS diagnostic assessment.
- 2) The Unstructured Introductory Interview. This section of the K-SADS-PL 2013 takes approximately 10 to 15 minutes to complete. In this section, the parent provides information about health, presenting complaint and prior psychiatric treatment data, and both the parent and the child are surveyed about the child's school functioning, hobbies, and peer and family relations. Discussion of these latter topics is extremely important, as it provides a context for eliciting mood symptoms (depression and irritability), and obtaining information to evaluate functional impairment. This section of the K-SADS-PL should be used to establish rapport with the parent(s) and the child, and should never be omitted.
- 3) The Screen Interview. The Screen Interview surveys the primary symptoms of the different diagnoses assessed in the K-SADS-PL 2013. Specific probes and scoring criteria are provided to assess each symptom. The rater is not obliged to recite the probes verbatim, or use all the probes provided, just as many as is necessary to score each item. Probing should be as neutral as possible, and leading questions should be avoided (e.g. "You don't feel sad, do you?") Symptoms rated in the screen interview are surveyed for current (CE) and most severe past (MSP) episodes simultaneously. Begin by asking if the child has ever experienced the symptom. If the answer is no, rate the symptom negative for current and past episodes and proceed to the next question. If the answer is yes, find out when the symptom was present. If the symptom is endorsed for one time frame (e.g. currently), inquire if it was ever present at another time (e.g. past).

| Subject | | | 500 |
|---------|-------|------|-----|
| | _ _ | <br> | |

2013



#### KSADS-PL SCREEN INTERVIEW: Introduction

page iii of xiv



The diagnoses assessed with the screen interview do not have to be surveyed in order. The interviewer may begin inquiring about relevant diagnoses suggested by the presenting complaint information obtained during the unstructured interview. All sections of the Screen Interview must be completed, however, and most people find it easiest to proceed from start to finish.

Skip Out Criteria. After the primary symptoms associated with each diagnosis are surveyed in the Screen Interview, skip out criteria are delineated for current and past episodes of the disorder. A space is provided to indicate if the child met the skip out criteria, or if the child has clinical manifestations of the primary symptoms associated with the specific diagnosis. If the child failed to meet the skip out criteria for some diagnoses, the appropriate supplements should be administered after the Screen Interview is completed in its entirety.

Scoring. While interviewers are free to utilize latitude in the manner in which symptoms are queried, the scoring criteria are to be applied rigidly. The majority of the items in the K-SADS-2013 are scored using a 0–3 point rating scale. Scores of 0 indicate no information is available, scores of 1 suggest the symptom is not present, scores of 2 indicate subthreshold levels of symptomatology, and scores of 3 represent threshold criteria. The remaining items are rated on a 0-2 point rating scale on which 0 implies no information, 1 implies the symptom is not present, and 2 implies the symptom is present. When determining whether a symptom meets threshold vs subthreshold level criteria, it is important to assess the severity, frequency, and duration of the symptom, as well as impairment from the symptom. It is often helpful to ask for examples of specific behaviors or symptoms. To attain a threshold score of 3, the child must meet or exceed the threshold scoring criteria. If his symptom severity falls between the threshold and subthreshold criteria, the symptom would be rated subthreshold; a score of 2.

Subthreshold Symptoms While subthreshold manifestations of symptoms are not sufficient to count toward the diagnosis of a disorder, further inquiry may be warranted in certain cases. Subthreshold scores of psychotic symptoms or clusters of other symptoms associated with a given diagnosis should be brought to the attention of the attending physician or research supervisor. If subthreshold scores are attained on multiple items within a given diagnostic section of the Screen Interview, the supplement for that section can be completed to further assess relevant clinical symptomatology.

- 4) Supplement Completion Checklist. The Supplement Completion Checklist is on the last page of this Screen Interview. It should be torn off before starting the interview. Supplements requiring completion should be noted in the spaces provided, together with the dates of possible current and past episodes of disorder.
- 5) Diagnostic Supplements. There are five Diagnostic Supplements included with the K-SADS-PL: Supplement #1: Depressive and Bipolar Related Disorders; Supplement #2: Schizophrenia Spectrum and Other Psychotic Disorders; Supplement #3: Anxiety, Obsessive Compulsive, and Trauma-Related Disorders; Supplement #4: Neurodevelopmental. Disruptive, and Conduct Disorders; Supplement #5: Eating Disorders and Substance-Related Disorders. The format of the KSADS with its Screen Interview and five Diagnostic Supplements is designed to facilitate differential diagnoses, with the Screen Interview providing a good overview of potentially relevant diagnostic categories before surveying symptoms associated with the different disorders in detail.

The diagnoses surveyed in each of these supplements are outlined in the Supplement Completion Checklist, and in the Table of Contents at the beginning of each supplement. The skip out criteria in the Screening Interview specify which supplements, if any, should be completed. Like in the Screen Interview, each supplement has a list of symptoms, probes, and criteria to assess current (CE) and most severe past (MSP) episodes of disorder.

Supplements should be administered in the order that symptoms for the different diagnoses appeared. For example, if the child had evidence of Attention Deficit Hyperactivity Disorder (ADHD) beginning at age 5, and possible Major Depression (MDD) beginning at age 9, the Supplement for ADHD should be completed before the supplement for MDD. If the child had a history of attention difficulties associated with ADHD, when inquiring about concentration difficulties in assessing MDD, it is important to find out if the onset of depressive symptoms was associated with a worsening of the long standing concentration difficulties. If there was no change in attention problems with the onset of the depressive symptoms, the symptom concentration difficulties should not be rated positively in the MDD supplement.

When the time course of disorders overlap, supplements for disorders that may influence the course of other disorders should be completed first. For example, if there is evidence of substance use and possible Mania or Psychosis, the substance abuse supplement should be completed first, and care should be taken to assess the relationship between substance use and possible manic and/or psychotic symptoms.

2013 KSADS-PL SCREEN INTERVIEW:

Introduction page iv of xiv

6) The Summary Lifetime Diagnostic Checklist is a template that was designed to record basic lifetime and current diagnostic information. Clinicians / Investigators may wish to record additional, more specific information (e.g., dates of onset/offset or duration of additional episodes). The Follow-up Summary Diagnostic Checklist is a template designed to record longitudinal course of illness. These template checklists are included at the end of the supplements of the KSADS.

Using the K-SADS in Longitudinal Studies. When the KSADS is used to monitor subjects longitudinally, it is important to be sure that the symptoms and diagnoses are being scored since the last interview. The timeframe for the Current ratings needs to be defined, based on the aims of the study. For example, the Current period could be the month prior to the interview (or 2 weeks, or 2 months, etc.). Then symptoms and diagnoses are rated for the most symptomatic time during the current period. Past symptoms and diagnoses are rated based on the most severe symptomatology between the last interview and whatever time is defined as the Current rating period. These rules are more relevant for episodic disorders such as depression and mania/hypomania. It is recommended that each study define a priori the timeframes to be used in administering the KSADS for longitudinal assessments. Results from the follow-up interviews can then be recorded on the Longitudinal Summary Diagnostic Checklist. The longitudinal summary diagnostic checklist may require some modifications by Investigators to accommodate the aims, methodology, and outcome definitions (e.g., remission, recovery, remission, recurrence) utilized in each study.

As depicted below, the KSADS can be used to characterize subject's longitudinal course of illness. The space between the first two lines on the left side of each diagram below depicts the course of illness since the last assessment up to the "current episode" timeframe, and the space on the right side of each diagram depicts the characterization of the current (e.g., last two months) symptomatology.



Legend. A) Figure A depicts a child with a chronic course of illness from the last interview; B) Figure B depicts a child who met full criteria during the last interview and continued to meet criteria during his most severe past episode during the follow-up interval, then met partial remission criteria during the "current" time frame assessed at follow-up; C) Figure C depicts a child who was in partial remission but never went into full remission during the "past" or "current" follow-up intervals, and is currently in partial remission: D) Figure D depicts a child who had no diagnosis at the initial interview, and then had an onset of a full diagnosis during the follow-up, but met for partial remission during the "current" follow-up interval.

Guidelines for the Administration of the Introductory Unstructured Interview

The unstructured interview should take at least 15 minutes to administer. The aim of the unstructured interview is to establish rapport, obtain information about presenting complaints, prior psychiatric problems, and the child's global functioning. It is helpful to spend a few minutes in general conversation in order to make the child and parent feel at ease.

The interview opens with questions about basic demographics. This is a very easy thing for most people to talk about, and the information helps to orient the interviewer to the child's life circumstances. Health and developmental history data should also be obtained from the parent, as this information may be helpful in making differential diagnoses. The child does not need to be queried about these things.

| - | Subject |
|-------|---------|
| (4.4) | |

2013



CUR ITOT INCODMATION

#### KSADS-PL SCREEN INTERVIEW: Subject Information

page v of xiv



In discussing onset and course of symptoms, many children will be unable to provide reliable time data. This is developmentally normal. If the child does not provide such data in the first questioning, s/he will probably not provide it at all.

In interviewing the parent, modify the questions to refer to the child.

In the introductory interview and throughout the K-SADS, interviewers are encouraged to use language generated by the child and/or parent when asking about symptoms (e.g., "For how long did you feel bummed?")

After surveying the reason for referral, obtain information about treatment history. Then ask about the child's school adaptation and social relations.

In interviewing children, it is not necessary — and usually not productive to try to complete all of the introductory interview. Review basic demographics (e.g. age, grade, family constitution, siblings' names and ages), presenting complaints (likely in less detail than with the parent), and family, school adaptation, and peer relations information. The discussion of these latter topics are extremely *important*, as it provides a context for eliciting mood symptoms (depression and irritability) from children, generate hypotehese about possible relevant diagostic areas, and obtain preliminary information to evaluate functional impairment.

| irst Name: | Las | t Name: | |
|---|---|---|---|
| Date of Birth: | | | |
| Gender: O Ma | le O Female | | |
| thnicity: O Hi | spanic or Latino O Not Hispanic or Latino | | |
| ace (Mark all | O Black or African American | O Native Hawaiian or Pacific | c Islander |
| nat apply): | O Asian | O Native American or Alask | an Native |
| | O White or Caucasian | | |
| | O Other Specify: | | |
| Vith whom is s | ubject currently living (choose one)? | | |
| | O Both biological parents | O Biological father only | O Group home |
| | | ACCESS TO A THEORY OF THE | |
| | O Both biological parents, but joint custody | O Stepmother only | O Residential institution |
| | O Both biological parents, but joint custody O Biological mother and stepfather | O Stepfather only | O Residential institution O Boarding home |
| | 가게 하게 되지 않아 많아 되는 것 같아. 이렇게 하다. | | |
| | O Biological mother and stepfather | O Stepfather only | O Boarding home |
| | O Biological mother and stepfather O Biological father and stepmother | O Stepfather only O Grandparent | O Boarding home O Runaway |

| | | | KSAE | | | | | | 200 | EW: | | | | | F | page | e v. c | of xiv | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| TICIPATIO | N: | | | | | | | | | | | | | | | | | | | |
| nant/repor | ter for | this i | ntervi | ew? | | | | | | | | | | | | | | | | |
| ogical pare | nts | | | ( | O Ad | optive | moth | er | | | | OG | rand | pare | ent | | | | | |
| mother | | | | ( | O Ad | optive | fathe | F | | | | 00 | ther | rela | tive | | | | | |
| father | | | | ( | O Ste | ep-mo | ther | | | | | 00 | ther | | | | | | | |
| ptive parer | its | | | ( | O Ste | ep-fath | ner | | | | | | | | | | | | | |
| ease specif | y: | | | | | | | | | | | | | Ü | | | | | | |
| | | | e) | | | Last | Nam | e: | | | | | | | | | | | | |
| | | 4 | | _ | | | | | 1 | | | | | | | | | | | |
| O Step | pted Mo | other | O S | dpte | ed Fa | ther C | Gra | ndmo | ther | | Gra | andfa | ather | | | | | | | |
| O Ado | CAREC | SIVER | O A | Ī | | Last | Nam | <b>9</b> : | | | | | | | | | | | | Ī |
| O Ado | CAREC | SIVER | O A | Ī | | Last | | <b>9</b> : | | | | | ather | er e | | | | | | |
| O Ado | CAREC | SIVER | O A | о Ма | other | Last | Nam | e:<br>r Fati | her | 0 | Fos | ter M | | | 0 | ther | Sp | ecify | | |
| O Ado | CAREC | GIVER<br>licable | O A | o Mo | other | Last | Nam- | e:<br>r Fati | her | O I | Fos | ter M | Nothe | 0 | 0 | tther | Sp | ecify | | |
| O Ado | CAREC | GIVER<br>licable | O A | o Mo | other | Last O | Nam- | e:<br>r Fati | her | O I | Fos | ter M | /othe | 0 | 0 | ther | Sp | ecify | | |
| O Ado | CAREC | GIVER<br>licable | O A | o Mo | other | Last O O other C | Nam- | r Fati | her | O I | Fos | ter M | /othe | 0 | 0 | ther | Sp | ecify | | |
| O Ado | CAREC | GIVER<br>licable | O A | o Mo | other | Last O O other C | Name<br>Foste<br>Uncl | r Fati | her | O I | Fos | ter M | /othe | 0 | 0 | ther | Sp | ecify | | |
| | mant/repor<br>ogical pare<br>mother<br>father<br>ptive paren<br>wase specif | ogical parents I mother I father ptive parents pase specify: MARY CAREGIVE ps with subject, if applications O Biological M | mant/reporter for this in agical parents in mother in father potive parents wase specify; MARY CAREGIVER's as with subject, if applicable is: O Biological Mother | mant/reporter for this intervi- pgical parents I mother I father ptive parents pase specify: MARY CAREGIVER's ps with subject, if applicable) St. O Biological Mother O B | pricipation: mant/reporter for this interview? pricipal parents mother father prive parents mase specify: MARY CAREGIVER's prive swith subject, if applicable) Six O Biological Mother O Bio Father materials of the subject of the s | pricipation: mant/reporter for this interview? pricipal parents O Add mother O Add father O Ste prive parents O Ste prive pare | pricipation: nant/reporter for this interview? pricipal parents O Adoptive I mother O Step-mo prive parents O Step-fath prive parents O Step-fath prive parents D Step-fath pr | pricipation: mant/reporter for this interview? pricipal parents | pricipation: mant/reporter for this interview? pricipal parents | mant/reporter for this interview? ogical parents O Adoptive mother on Manther O Step-mother optive parents O Step-father observed by: MARY CAREGIVER's os with subject, if applicable) Last Name: or O Biological Mother O Bio Father O Foster Mother | pricipation: mant/reporter for this interview? pricipal parents | ricipation: nant/reporter for this interview? original parents | price parents O Adoptive mother O G Adoptive parents O Step-mother O Step-father Prive parents O Step- | pricipation: mant/reporter for this interview? program of parents | pricipation: mant/reporter for this interview? pricipal parents | Pricipation: nant/reporter for this interview? pigical parents O Adoptive mother O Grandparent mother O Adoptive father O Other relative father O Step-mother O Other prive parents O Step-father pase specify: MARY CAREGIVER'S ps with subject, if applicable) Last Name: Step O Biological Mother O Bio Father O Foster Mother O Foster Father | Inant/reporter for this interview? Ogical parents O Adoptive mother O Grandparent I mother O Adoptive father O Other relative I father O Step-mother O Other Optive parents O Step-father Passe specify: MARY CAREGIVER's Os with subject, if applicable) Last Name: Sign O Biological Mother O Bio Father O Foster Mother O Foster Father | Inant/reporter for this interview? Inant/reporter for this interview. Inant/reporter for this interv | Inant/reporter for this interview? Ogical parents O Adoptive mother O Grandparent I mother O Adoptive father O Other relative I father O Step-mother O Other Optive parents O Step-father O Step-father Dase specify: MARY CAREGIVER's Os with subject, if applicable) Last Name: C O Biological Mother O Bio Father O Foster Mother O Foster Father | Inant/reporter for this interview? Ogical parents O Adoptive mother O Grandparent I mother O Adoptive father O Other relative I father O Step-mother O Step-father O Step-father Dase specify: MARY CAREGIVER's Oswith subject, if applicable) Last Name: C O Biological Mother O Bio Father O Foster Mother O Foster Father |

| O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS First Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Full sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Excellent | 2013 | | | SCREEN INTERV / Sibling Information | - Tare 2 - 2 | page vii | of xiv |
|---|---|---|---|---|---|---|---|
| Does child live with biological mother: | BIOLOGICAL FA | THER | | | | | |
| fino, describe nature of contact/relationship: O Mother deceased O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS First Name: Last Name: Quality of Relationship: O Excellent O Good O Fair O Poor O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive, sporadic contact C Mother alive, regular visitation O Mother alive, regular visitation O Mother alive, regular visitation O Mother alive, regular visitation O Excellent O Good O Fair O Poor O Foor O | First Name: | | | Last Name: | | | |
| fino, describe nature of contact/relationship: O Mother deceased O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS First Name: Last Name: Quality of Relationship: O Excellent O Good O Fair O Poor O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive, sporadic contact O Mother alive, regular visitation O Excellent O Good O Fair O Poor O Foor O Poor O Excellent O Good O Fair O Poor O Poor O Excellent O Good O Fair O Poor O Poor O Excellent O Good O Fair O Poor O Poor O Excellent O Good O Fair O Poor O Poor O Excellent O Good O Fair O Poor O | | 100000 | | | | | |
| f no, describe nature of contact/relationship: O Mother deceased O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS First Name: Last Name: Quality of Relationship: O Excellent O Good O Fair O Poor O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive, sporadic contact O Mother alive, regular visitation O Excellent O Good O Fair O Poor O Foor O Poor O Foor O Foo | | | | * A. | | | |
| Quality of Relationship: O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS irst Name: Age: O Half sibling O Full sibling | oes child live w | ith biological mo | ther: O Yes | O No | | | |
| O Mother alive, regular visitation O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS irst Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling Age: O Half sibling O Full sibling O Excellent O Good O Fair O Poor Cuality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Poor Cuality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Poor O Excellent O Good O Fair | | | elationship: | E | 20 | | |
| O Mother alive, sporadic contact O Mother alive but no contact SUBJECT'S SIBLINGS irst Name: Age: O Half sibling O Full sibling O Excellent O Good O Fair O Potential O Good O Fair O Fotential O Good O Fair | | | tion | Quality of R | elationship: | | |
| O Mother alive but no contact SUBJECT'S SIBLINGS irst Name: Age: O Half sibling O Full sibling Age: O Half sibling O Full sibling Quality of Relationship between Sibling and Subject: East Name: Last Name: Quality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Potential Sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Full sibling O Excellent O Good O Fair O Potential Sibling O Excellent O Good O Fair | and the state of t | | | O Excellent | O Good | O Fair | O Poor |
| Age: O Half sibling O Full sibling | | | | | | | |
| Age: O Half sibling O Full sibling Age: O Half sibling O Full sibling Age: O Half sibling O Full sibling Age: O Half sibling O Full sibling Age: O Half sibling O Full sibling Quality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Political Polit | SUBJECT'S SIBL | INGS | | | | 0=0=0=0 | - |
| O Half sibling O Full sibling O Excellent O Good O Fair O Police Inst Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Police Inst Name: Last Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Police Age: O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibling O Full sibling O Full sibling O Excellent O Good O Fair O Police O Half sibling O Full sibli | irst Name: | | | Last Name: | | | |
| O Half sibling O Full sibling O Excellent O Good O Fair O Politicate Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Politicate Name: Last Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Politicate O Good O Fair O Politicate O Half sibling O Full sibling O Excellent O Good O Fair O Politicate O Good O Fair O Po | | | | | | | |
| irst Name: Age: O Half sibling O Full sibling Quality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Potential Sibling O Excellent O Good O Fair O Potentiate Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Potentiate Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Potentiate Name: | Age: | | | Quality of Relationsh | nip between Sibl | ing and Subject | ct: |
| Age: O Half sibling O Full sibling Last Name: Quality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Po Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Po | | O Half sibling | | | | 하게 없었는 나무하다 | O Poor |
| Age: O Half sibling O Full sibling Last Name: Quality of Relationship between Sibling and Subject: O Excellent O Good O Fair O Po Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Po | | | | | عاملوند | | |
| O Half sibling O Full sibling D Excellent O Good O Fair O Politicat Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Excellent O Good O Fair O Politicationship Detween Sibling and Subject: O Half sibling O Excellent O Good O Fair O Politicationship Detween Sibling and Subject: O Half sibling | irst Name: | | | Last Name: | | | |
| O Half sibling O Full sibling O Excellent O Good O Fair O Politicate Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Politicationship of State O | | | | | | | |
| irst Name: Last Name: Quality of Relationship between Sibling and Subject: O Half sibling O Full sibling O Excellent O Good O Fair O Po | Age: | | | Quality of Relationsh | nip between Sibl | ing and Subject | et: |
| Age: O Half sibling O Full sibling O Excellent O Good O Fair O Po | | O Half sibling | O Full sibling | O Excellent | O Good | O Fair | O Poor |
| Age: O Half sibling O Full sibling O Excellent O Good O Fair O Po | | | | | | | |
| O Half sibling O Full sibling O Excellent O Good O Fair O Po | irst Name: | | | Last Name: | | | |
| O Half sibling O Full sibling O Excellent O Good O Fair O Po | | 4 11 11 11 11 11 | | | | | |
| O Excellent O Good O Pail O Po | Age: | San San San | | Quality of Relationsh | nip between Sibl | ing and Subject | ct; |
| | | O Half sibling | O Full sibling | O Excellent | O Good | O Fair | O Poor |
| | 1-1- | | | | | | 5 |
| if the people in your family, or among the people you live with, who would you say you are closet to? | f the people in ve | virtamily or amor | on the people you live | a with who would you | reav vou are clos | ot to? | |
| The people in your family, or althoughte people you live with, who would you say you are closer to? | the people in ye | our fairlily, or airlor | ig the people you live | e with, who would you | a say you are clos | et to: | |
| | | Subject | | | | 170 | |

| 2013 | KSADS-I | Health Sc | N INTERVII | EVV: | | pa | age vili d | of xiv | ı |
|---|---|---|---|---|---|---|---|---|---|
| CHILD AND ADOLESCE | NT HEALTH SCR | REEN | | | | | | | |
| PREGNANCY AND BIRTH | <b>l</b> : | T-T | _ | | | | | | |
| <ol> <li>Mother's age at birth of chi</li> </ol> | ld | | | | | | | | |
| <ol><li>Did mother have any illness<br/>pregnancy?</li></ol> | s or injury during | O Yes | O No | | | | | | |
| <ol> <li>Did she take any medication vitamins and iron?</li> </ol> | ons other than | O Yes | O No | | | | | | |
| 4. Did mother drink or use eli | | | O No | | | | | | |
| 5. Did mother smoke during p | orgnancy? | O Yes | O No | | | | | | Ť |
| 6. Was the baby premature? | | | O No | | | | | | Î |
| 7. What was the birth weight? | | | lbs. | | | | | | |
| 8. Did the baby have any trou | ble at birth? | O Yes | O No | | | | | | |
| <ol> <li>Did the baby have any other<br/>(Jaundice, infections, other</li> </ol> | | O Yes | O No | | | | | | Ì |
| 0. How many days did the ba | | after | days | | | | | | |
| 10. How many days did the babirth? | aby stay in the hospital | after | | | | -0-2- | | | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA | aby stay in the hospital | | days Weight: | | ].[ | lbs | | - | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA 11. Current height: | L HISTORY: | | | | ].[ | ibs | | | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA 11. Current height: fe 12. Where does your child go care? | L HISTORY: eet inches | | | | ].[] | lbs | | | |
| O. How many days did the bibirth? MEDICAL AND SURGICA Ourrent height: Where does your child go care? Date of last medical exam | L HISTORY: eet inches for medical c reactions to any | | Weight. | | | lbs | | | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA 11. Current height: 12. Where does your child go care? 13. Date of last medical examination of the company of th | L HISTORY: eet inches for medical c reactions to any | s<br> | Weight. | | | ibs | | | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA 11. Current height: 12. Where does your child go care? 13. Date of last medical examinations? If YES, please Allergic research. | L HISTORY: eet inches for medical c reactions to any ase specify: | o Yes | Weight. | | | lbs | | | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA 11. Current height: 12. Where does your child go care? 13. Date of last medical examinations? If YES, please Allergic reaction | L HISTORY: eet inches for medical c reactions to any ase specify: eactions to foods? ns to insect bites? | O Yes | Weight: | | | lbs. | | | |
| 10. How many days did the bibirth? MEDICAL AND SURGICA 11. Current height: 12. Where does your child go care? 13. Date of last medical examinations? If YES please. | L HISTORY: eet inches for medical c reactions to any ase specify: eactions to foods? ns to insect bites? nunizations? | O Yes O Yes O Yes | Weight: O No O No O No O No O No O No O No O N | | | lbs. | | | |

| | L SCREE<br>I / Developr | | | | | pag | e ix of xiv | , |
|---|---|---|---|---|---|---|---|---|
| MEDICAL AND SURGICAL HISTORY cont: | | | | | | | | |
| 7. Any hospitalizations? If <u>YES</u> , for what? | O Yes | O No | | | | | | |
| | | Ť | | | | | 11 | |
| | | Ł | ++ | $\pm$ | + | | + | |
| | | Ĺ | | | 111111 | | Ш | |
| 8. Any serious injuries? If <u>YES</u> , what kind? | O Yes | O No | | | | | T | |
| | | Ī | | | + | | | + |
| | | Ļ | | | 1 | | | |
| | | L | | | | | | |
| | | | -11-1 | | li l | | | |
| Any head injuries? (Indicate if your child lost | | | | 1 1 | | | | 1 1 |
| consciousness): | O Yes | O No | | | | | | |
| 0. Any other current or past significant medical | O Yes | O No | TT | П | Ť | | 1.1 | |
| health problems? If <u>YES</u> , please specify: | 0 103 | C 140 | ++ | - | + | | ++ | |
| | | L | | | 144 | 11.11 | 117 | |
| | | | | | 1111 | | | |
| | | Ī | 111 | | Til | | Ħ | H |
| | | | | | | 2-2- | | |
| EVELOPMENTAL HISTORY: | | | | | | | | |
| Problems with social relatedness during infancy as | nd early child | dhood: | C | Yes | O No | | | |
| If no, explain: | | | | | | | | |
| | | | | | 5.7 | | | |
| Developmental milestones within normal limits: | | | C | Yes | O No | | | |
| If no, explain: | | | | | | | | |
| Subject | | | | | | | - | |

| 2013 | KSADS-PL SCREEN INTERVIEW: <u>Presenting Complaint</u> | page x of xiv |
|---|---|---|
| | Clinician | |
| - | Supervising Physician/Supervising Researcher | - |
| | Date | |
| resenting Complaint: | | |
| | | _ |
| ;= | | |

#### CONFIDENTIAL Version 9.0


| 1 | KSADS-PL SCREEN INTERVIEW | |
|------|-----------------------------------------|----------------|
| 2013 | Family History for Biological Relatives | page xi of xiv |

Probe: Have you or anyone else in the family had psychiatric treatment before? For what sorts of problems?

Criteria:

0 = No Information 1 = Not Present 2 = Probable 3 = Definite

| | | Ma | ther | | | Fa | ther | | 1 | Sit | ling | - | - F | talf: | Siblin | 19 | G | tand | ipare | nt | 1 | \unit | Urid | 0 | | 100 | her | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Payonatric Tx | 0 | 1 | 2 | 3 | 0 | 1 | 5 | 3 | Ü. | T | 2 | 8 | 0 | 1 | - 2 | 3 | 0 | 3 | 2 | 3 | D | 1 | 2 | 3 | 0 | 1 | 2 | 2 |
| Depression | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 7 | 2 | 3 | 0 | 1 | 2 | 3 | - 0 | 1 | 2 | 3 | 0 | 1 | .2 | 3 |
| Mania | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 9 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0. | t | 2 | 3 |
| ADHD | 0 | 1 | 2 | 3 | C | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | T | 2 | 3 |
| Conduct/Antisocial | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | - 27 |
| Schizophrenia | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0. | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | -1 | 2 | - 3 |
| Other Psychosis | Ō | 1 | 2 | 3 | Ô | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 4 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 4 | 2 | 3 | 0 | -1 | 2 | - 3 |
| Alcohol Use Dinorder | Ö | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | В | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | - 0 | 1 | 2 | 3 | 0 | 1 | 2 | - 3 |
| Substance Use De. | - 0 | 1 | 2 | 3 | u | 1 | 2 | -9 | 0 | 1 | 2 | 3 | 0 | 1 | .2 | 3 | 0 | 9 | 2 | 3 | | 1 | 2 | 3 | - 0 | -1 | 3 | - 2 |
| Autism Spectrum | 0 | 1 | 2 | 3. | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | -1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | -1 | 2 | 3 | 0 | -1 | 2 | - 3 |
| Suicide Attempt | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | U | 1 | 2 | 3 . | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | . 3 | . 0 | 1 | 2 | 3 |
| Suicide Completion | 0 | 1 | 2 | 3 | Û | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 3 | 2 | 3 | . 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 |
| Other | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0. | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 1 | 2 | 3 | 0 | 4 | 2 | 3 | 0 | 1 | -2 | - 3 |

| 201 | 3 | | | UN | | | DS-PL | | | | | | | | | page | xii of | xiv | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| LIF | ETIME | TREA | ATME | NT HI | STO | RY | | | | | | | | | | | first tx | ionths) | |
| | Outpa | atient Ti | eatme | nt | | | | | | O No | o info | O No | 0 | Yes | | | | | |
| | Psych | niatric H | losptial | ization | 1 | | | | | O No | o info | O No | 0 | Yes | Ē | | Ī | | |
| | Partia | Il Hospi | talizatio | on | | | | | | O No | o info | O No | 0 | Yes | | | | | |
| | Resid | ential T | reatme | ent Fac | ility | | ***** | | | O No | o info | O No | 0 | Yes | | | | | |
| | In-Ho<br>Based | me Ser | vices T | x (e.g., | , Wra | p Arour | nd/Family | <i>r</i> | | O No | o info | O No | 0 | Yes | | | į | | |
| | Ducc | | | | | | | | | | | | | | | | | | |
| | | per of P | sychiat | ric Hos | pitaliz | zations | | | | ***** | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | <b>Y OF</b> □ Po | or | |
| Med | | per of P | | ric Hos | pitaliz | zations | Pacti | Curren | | | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | 7 | - | |
| Med | Numb | per of P | | ric Hos | pitaliz | zations | Past/<br>O | Curren | t 7 | | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | 7 | Past/ | |
| Med | Numb | per of P | | ric Hos | pitaliz | zations | | | t 7 2 | | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | 7 | Past/ | ( |
| Med | Numb | per of P | | ric Hos | pitaliz | zations | | 0 | 7 | | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | 7 | Past/<br>O | ( |
| Med | Numb | per of P | | ric Hos | pitaliz | zations | | 0 | 7<br>8<br>8 | | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | 7 | Past/<br>O | ( |
| Med | Numb | per of P | | ric Hos | pitaliz | zations | | 0 0 | 7 8 9 9 E | | | 9 | OVERA<br>NFORI | LL R | ELIA<br>ON: | - | 7 | Past/<br>O | 0 |

| 2013 | KSADS-PL SCREEN INTERVIEW: School Information page xiii of xiv |
|---|---|
| chool Information | |
| Current Grade (or highes | st grade completed): Any Repeated Grades? List: |
| Current School Setting | O Regular Public School O Specialized School for Youth with Emotional/Behavioral Problems O Regular Private School O Vocational-TechnicalSchool O Not in School O Other, specify: |
| Specialized Services: | O Full-time Emotional Support Classroom O Special Education for specific subjects (partially mainstreamed) O Full-time Learning Support Classroom O Part-time Aide O Resource Room O Tutoring Support O Other, specify: |
| Recent Grades - Acade | emic Classes: Best: O A O B O C O D O F Average: O A O B O C O D O F Worst: O A O B O C O D O F |
| Strengths. | |
| Subject<br>Weaknesses: | |
| Concerns from teacher Detentions (past | Fights in school |

| 013 | | | | | KSA | Pee | | | | | | ER\<br>ation | | V: | | | | | pag | e xiv | of x | ív | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| er Relations | | | | | | | | | | | | | | | | | | | | | | | |
| Best friend(s)? | | | | | | | Оує | s | Оп | 10 | | | | | | | | | | | | | |
| Relations with p | eers at | scho | ol: | | | | O E | xcell | ent | 0 | Go | od | | | | | | +->-> | | | | | |
| Relations with p | eers in | the n | neigh | borh | ood: | | 0 E | xcell | ent | 0 | Go | od | OF | air | 0 | Poo | | | •••• | | | | |
| Bullied by other | s? | | | | | | | | | | | a pr | | | | | | | | | prob | | |
| ther Activities / In | | | ify) | | - | | - | | | | | | | | | | | | | | | | |
| O Hobbies | | | | | | | | | | | | 2 | | | | | | | | | | I | |
| | | | | **** | | | | | | teke | | | *** | *** | | 9999 | *** | | | | | | |
| O Preferred<br>Activies during 1<br>free-time | | | | | | | | | | | | 3 | | | 1 | | | | | | | | |
| 2 | | | | | | | | | | | 1 | 4 | | | 1 | | | | 1 | | | | |
| O Sports | | 1 | 1 | T | | ***** | 7777 | **** | 777 | | | 3 | | T | 7 | ,,,,,, | | 1 | 1 | | | 1 | |
| | Н | | | - | | | | | | | = | Ē | | T | 1 | ÷ | + | Ť | + | $\pm$ | + | Ť | + |
| 2 | Ш | | _ | _ | | | _ | | | | | 4 | 1 | J | 1 | 1 | 1 | | _ | | | | |
| O Organizations | | | | | | | I | | | | | 2 | | T | Ì | | | Ì | | Ĭ | | Ī | |
| | | | | | - | - | | - | | | . 5 4 | | - | | | | | | | | | | = 10 |

| Parent Rating: Child Rating: () () () 2 - Subthreshold: Depressed mood at least 2-3 days/ week, for much of the day. | P C S | DSM-5 DR# 6; Felt down, depressed: | | Depression | <u>P</u> () | | | |
|---|---|---|---|---|---|---|---|---|
| DSM-5 DR# 6: Felt down, depressed: Parent Rating: Child Rating: | DSM-5 DR8 6: Felt down, depressed: DSM-5 DR8 6: Felt down, depressed: Dam-5 DR8 6: Felt down, depressed: Parent Rating: | DSM-5 DR# 6: Felt down, depressed: | | | () | | | 0 - No information. |
| DSM-5 DR# 6: Felt down, depressed: Parent Rating: Child Rating: | DSM-5 DR# 6: Felt down, depressed: Parent Rating: Child R | DSM-5 DR# 6: Felt down, depressed: | | | - | () | () | 0 - No information. |
| Parent Rating: Child Rating: () () () 2 - Subthreshold: Depressed mood at least 2-3 days/ week, for much of the day. Have you ever felt sad, blue, down, or empty? Did you feel like crying? When was that. Do you feel now Was there ever another time you felt Did you have a bad feeling all the time that you couldn't get rid of Did you cry or were you tearful? Did you feel ( ) all the time, some o the time? (Percent of awake time: summation of % of all labels if they do not occur simultaneously). (Assessment of dlurnal variation can secondarily clarify daily duration of depressive mood) Did it come and go How often? Every day? How long did it last? What do you think brought it on? Could other people tell that you were sad? Duration of Depressed Mood: Duration of Depressed Mood: | Parent Rating: Child Rating: | | | | (1) | | | a seem to the second |
| Have you ever felt sad, blue, down, or empty? Did you feel like crying? When was that Do you feel now Was there ever another time you felt Did you have any other bad feelings Did you have a bad feeling all the time that you couldn't get rid of Did you cry or were you tearful? Did you feel all the time, some o the time? (Percent of awake time: summation of % of all labels if they do not occur simultaneously). (Assessment of diurnal variation can secondarily clarify daily duration of depressive mood) Did it come and go How often? Every day? How long did it last? What do you think brought it on? Could other people tell that you were sad? Duration of Depressed Mood: Duration of Depressed Mood: | Have you ever felt sad, blue, down, or empty? Did you feel like crying? When was that Do you feel now Was there ever another time you felt Did you have any other bad feelings Did you have a had feeling all the time that you couldn't get rid of Did you cry or were you tearful? Did you feel () all the time, some o the time? (Percent of awake time: summation of % of all labels if they do not occur simultaneously). (Assessment of diurnal variation can secondarily clarify daily duration of depressive mood) Did it come and go How often? Every day? How long did it last? Could other people tell that you were sad? NOTE: SOMETIMES THE CHILD WILL INITIALLY GIVE A NEGATIVE ANSWER AT THE START OF THE INTERVIEW GOES ON, THEN THESE OULESTIONS SHOULD BE REPEATED ELICITING THE PRESENT MOOD AND USING IT AS AN EXAMPLE TO DETERMINE ITS PREGUENCY. SIMILARLY, IF THE MOTHER'S OPPINS ITS THAT ECHILD SHOULD BE CONFRONTED WITH THE MOTHER'S OPPINS ITS THAT CHILD SHOULD BE CONFRONTED WITH THE MOTHER'S OPPINS ITS THAT CHILD SHOULD BE CONFRONTED WITH THE MOTHER'S OPPINS ITS THAT CHEILD SHOULD BE CONFRONTED WITH THE MOTHER'S OPPINS ITS THAT CHEILD SHOULD BE CONFRONTED WITH THE MOTHER'S OPPINS OF NING HAND SHOULD BE | Parent Rating: Child Rating: | | | 1.3 | () | () | 1 - Not present. Not at all or less than once a wee |
| Have you ever telt sad, blue, down, or empty? Did you feel like crying? When was that Do you feel now Was there ever another time you felt Did you have any other bad feelings Did you have a bad feeling sll the time that you couldn't get rid of Did you cry or were you tearful? Did you feel () all the time, some o the time? (Percent of awake time: summation of % of all labels if they do not occur simultaneously). (Assessment of diurnal variation can secondarily clarify daily duration of depressive mood) Did it come and go How offer? Every day? How long did it last? What do you think brought it on? Could other people tell that you were sad? Duration of Depressed Mood: Duration of Depressed Mood: | Note: Sometimes the Child Will Initially Give a Negative Anegative Answer and the Stand To you were people left that you were sad? Note: Sometimes the Child Will Initially Give a Negative Anegative Answer and Should Be repeated Eliciting The Interview But will be Gow and Should Be governed and Should Be governed and Should Be governed And Sh | | | | () | () | () | |
| Was there ever another time you felt | Was there ever another time you felt | Did you feel like crying? When was that | | | () | () | 0 | (4-7 days/week), most of the day (at least |
| | ANSWER AT THE START OF THE INTERVIEW BUT WILL BECOME OBVIOUSLY SAD AS THE INTERVIEW GOES ON, THEN THESE QUESTIONS SHOULD BE REPEATED ELICITING THE PRESENT MOOD AND USING IT AS AN EXAMPLE TO DETERMINE ITS FREQUENCY. SIMILARLY, IF THE MOTHER'S REPORT IS THAT THE CHILD IS SAD MOST OF THE TIME AND THE CHILD DENIES IT, THE CHILD SHOULD BE CONFRONTED WITH THE MOTHER'S OPINION AND THEN ASKED WHY HE | Was there ever another time you felt | ) all the time, .<br>If all labels if th | ney do not | | | | PAST: P C S Duration of Depressed Mood: (current) Duration of Depressed Mood: |
| 013 | | KS | ADS-PL SCREEN INT<br>Depression | ERV | IEW: | |
|---|---|---|---|---|---|---|
| | | | <u>P</u> | c | <u>s</u> | |
| Irritability and Anger | | | () | () | () | 0 - No information |
| DSM- | 5 DR# 7: Felt me | ore imtated than usual: | () | () | () | 1 - Not present. Not at all or less than once a wee |
| | Rating: | Child Rating: | () | () | () | <ol> <li>Subthreshold; Feels definitely more angry or<br/>irritable than called for by the situation at least<br/>(2-3 days/week), for much of the day.</li> </ol> |
| things Did yi Are y What Were How More What Did yi With Your Who At so What Did a How All of Lots o | s? ou ever have a ou ever have a ou like that now kinds of things you feeling ma angry? than before? kinds of things ou sometimes fi his happen ofter ou lose your ten your family? friends? else? hool? ridd you do? nybody say any much of the time? of the time? | time when you lost your temper? Was there ever another time made you? do another time and you did was a feel angry? The seel angry and/or irritable and/or proper? | a lot? When was that? ( ) you felt? "It show it)? cranky and didn't know | () | () | 3 - Threshold: Feels irritable/angry, more days than (4-7 days/week), most of the day (at least 50 of awake time.). PAST: P C S Duration of Irritable Mood (current) |
| Just now and then? None of the time? When you got mad, what did you think about? Did you think about killing others or hurting yourself? Or about hurting them or torturing them? Whom? Did you have a plan? How? | | | | | | Duration of Irritable Mood (most severe past) |
| | | Y MAY BE DUE TO OTHER I | | | | |

| 2013 KSADS-PL SCREEN Depression | 0.000 | RVI | EW: | |
|---|---|---|---|---|
| | P | <u>c</u> | <u>s</u> | |
| Anhedonia, Lack of interest, Apathy, Low Motivation, or Boredom | () | () | () | 0 - No information |
| DSM-5 DR# 5; Has less fun doing things: | () | () | () | 1 - Not present. |
| Parent Rating: Child Rating: | () | () | () | 2 - Subthreshold: Several activities definitely less |
| Boredom is a term all children understand and which frequently refers to loss of ability to enjoy (anhedonia) or to loss of interest or both. Loss of pleasure and loss of interest are not mutually exclusive and may coexist. | | | | pleasurable or interesting. Or bored or<br>apathetic at least 3 times a week during<br>activities. |
| What are the things you do for fun? Enjoy? (Get examples: nintendo, sports, friends, favorite games, school subjects, outings, family activities, favorite TV programs, computer or video games, music, dancing, playing alone, reading, going out, etc.). | () | () | () | 3 - Threshold: Most activities much less<br>pleasurable or interesting. Or bored or<br>apathetic daily, or almost daily, at least 50%<br>the time. |
| Has there ever been a time you felt bored a lot of the time? When Do you feel bored a lot now Was there another time you felt bored a lot Did you feel bored when you thought about doing the things you usually like to do for fun? (Give examples mentioned above). Did this stop you from doing those things Did you (also) feel bored while you were doing things you used to enjoy | | | | PAST: P C S |
| Anhedonia refers to partial or complete (pervasive) loss of ability to get pleasure, enjoy, have fun during participation in activities which have been attractive to the child like the ones listed above, it also refers to basic pleasures like those resulting from eating favorite foods and, in adolescents, sexual activities. | | | | Duration of Anhedonia:<br>(current) |
| Did you look forward to doing the things you used to enjoy? (Give examples) Did you try to get into them Did you have to push yourself to do your favorite activities Did they interest you Did you get excited or enthusiastic about doing them? Why not Did you have as much fun doing them as you used to before you began feeling (sad, etc.) If less fun, did you enjoy them a little less? Much less? Not at all Did you have as much fun as your friends How many things are less fun now than they used to be (use concrete examples provided earlier by child) How many were as much fun? More fun Did you do less than you used to? How much less | | | | Duration of Anhedonia:<br>(past) |
| In adolescents: (if sexually active) Do you enjoy sex as much as you used to? Are you less sexually active than you used to be | | | | |
| This item does not refer to inability to engage in activities (loss of ability to concentrate on reading, games, TV, or school subjects) | | | | |
| Two comparisons should be made in each assessment: Enjoyment as compared to that of peers and/or enjoyment as compared to that of child when not depressed. The second is not possible in episodes of long duration because normally children's preferences change with age. Severity is determined by the number of activities which are less enjoyable to the child, and by the degree of loss of ability to enjoy. | | | | |
| Do not confuse with lack of opportunity to do things which may be due to excessive parental restrictions. | | | | |
| Subject | | | | |

| 2013 | KSADS-PL SCREEI<br>Suicide | | | | |
|---|---|---|---|---|---|
| | | P | С | <u>s</u> | |
| 4a. Recurrent Thought | s of Death | () | () | () | 0 - No information. |
| Sometimes children w | tho get upset or feel bad, wish they were dead or feel | () | () | () | 1 - Not present. |
| they'd be better off de<br>Have you ever had th<br>Do you feel that way | ead.<br>ese type of thoughts? When?<br>now? | () | () | () | Subthreshold: Infrequent thoughts of death (e. less than once per month, vague, |
| Was there ever anoth | er time you felt that way? | () | () | () | non-specific). 3 - Threshold: Recurrent thoughts of death, "I would be better off dead" or "I wish I were dead." |
| | | | | | PAST: P C S |
| | | P | <u>c</u> | <u>s</u> | |
| 4b. Suicidal Ideation | | () | () | () | 0 - No information |
| potts pougs | | () | () | () | 1 - Not at all. |
| Parent Rating: | hts of committing suicide Child Rating: | () | () | () | <ul> <li>2 - Subthreshold: Infrequent or vague thoughts of<br/>suicide (e.g., less than once per month).</li> </ul> |
| Sometimes children w | tho get upset or feel bad think about dying or even | () | () | () | 3 - Threshold: Recurrent thoughts of suicide. |
| Have you ever had si<br>How would you do it?<br>Did you have a plan? | 2.1 1 2 2 2 2 2 2. | | | | PAST: P C S |
| | | <u>P</u> | <u>c</u> | <u>s</u> | |
| 4c. Suicidal Acts - Inte | <u>nt</u> | () | () | () | 0 - No information. |
| DSM-5 DR# 25: Ever tri | ed to kill self | () | () | () | 1 - No attempt. |
| | Child Rating: d to kill yourself? When? | O | () | () | 2 - Subthreshold, Preparations with no actual inter<br>to die (e.g., held pills in hand) or planned<br>attempt but did not follow through or engage is<br>self harming behavior. |
| What did you do?<br>Any other things?<br>Did you really want to<br>How close did you co<br>Was anybody in the r | | () | () | () | <ol> <li>Threshold: Self injurious behavior with ANY<br/>suicidal intent. (If subject endorses even a 1%<br/>intent to die, code as threshold here).</li> </ol> |
| Did you tell them in ac<br>How were you found!<br>Did you ask for any h | Did you really want to die? | | | | PAST: P C S |
| | HARMING BEHAVIOR WITH NO INTENT TO DIE AS<br>F-INJURIOUS BEHAVIOR - NOT AS SUICIDAL | | Eve | r atter | mpted suicide: O Yes O No |
| | | | | | of lifetime attempts<br>hreshold of (3): |

| 20 | 13 KSADS-PL SCREE<br>Suicid | 10-110-6- | KVI | EVV: | |
|---|---|---|---|---|---|
| | | P | <u>c</u> | s | |
| 4d. | Suicidal Acts - Medical Lethality | () | () | 0 | 0 - No information. |
| | Actual medical threat to life or physical condition following the most serious suicidal act. Take into account the method, impaired consciousness at time of being rescued, seriousness of physical injury, toxicity of ingested material, | () | () | () | <ol> <li>No attempt or engaged in behavior with no inte<br/>to die (e.g., held pills in hand). No medical<br/>damage.</li> </ol> |
| | reversibility, amount of time needed for complete recovery and how much<br>medical treatment needed. | () | () | () | 2 - Subthreshold: superficial cuts, scratch to wristook a couple of extra pills. |
| | How close were you to dying after your (most serious suicidal act)?<br>What did you do when you tried to kill yourself?<br>What happened to you after you tried to kill yourself? | () | () | () | Threshold: Medical intervention occurred or<br>was indicated, or significant cut with bleedin<br>or took more than a couple of pills. |
| | NOTE: CODE SELF-HARMING BEHAVIOR WITH NO INTENT TO DIE<br>AS NON-SUICIDAL, SELF-INJURIOUS BEHAVIOR - NOT AS SUICIDAL<br>BEHAVIOR. | | | | PAST: P C S |
| | | P | <u>c</u> | <u>s</u> | |
| 4e. | Non-suicidal, Self-Injurious Behavior | () | () | () | 0 - No information |
| | Refers to intentional self-inflicted damage to the surface of the body, of a | | 0 | () | 1 - Not present. |
| | sort likely to induce bleeding or pain for purposes that are not socially sanctioned AND done without intent of killing himself, with the expectation that the injury will lead to only minor or moderate physical harm. | () | () | 0 | 2 - Subthreshold: Once. Has engaged in the<br>behavior on 1-4 occasions. Has never<br>caused serious injury to self. |
| | Did you ever try to hurt yourself? Have you ever burned yourself with matches/candles? Or sorratched yourself with needles/ a knife? Your nails? Or put hot pennies on your skin? Anything else? Why did you do it? How often? Use you have many accidents? What kind? How often? | () | () | () | 3 - Threshold: Repetitive. Has engaged in the behavior more than 5 times and/or has engaged in the behavior with significant injur to self (e.g., burn left scar, out required stitches). PAST: PC S |
| | Some kids do these types of things because they want to kill themselves,<br>and other kids do them because it makes them feel a little better afterwards.<br>Why do you do these things? | | | | |
| 3 | IF RECEIVED A SCORE OF 3 ON <u>CURRENT</u> RATING OF <u>ANY</u> ODEPRESSIVE/DYSTHYMIC DISORDERS (CURRENT) SECTION DISORDERS SUPPLEMENT, AFTER FINISHING THE SCREEN I | OF THE | DEPR | | |
| _ | IF RECEIVED A SCORE OF 3 ON <u>PAST</u> RATING OF <u>ANY</u> OF THE DEPRESSIVE/DYSTHYMIC DISORDERS (PAST) SECTION OF DISORDERS, AFTER FINISHING THE SCREEN INTERVIEW. | | | | |
| | NO EVIDENCE OF DEPRESSIVE/DYSTHYMIC DISORDER. | | | | |
| - | | | | | |

| 2013 | | KSADS-PL SCREEN<br>Mania / Hypo | | RVI | EW: | |
|---|---|---|---|---|---|---|
| | | | P | <u>c</u> | <u>s</u> | |
| 1. Eleva | ited, Elated, or Expans | ive Mood | () | () | () | 0 - No information. |
| ⊟ev | ated mood and/or excessiv | vely optimistic attitude which is out of | () | () | () | 1 - Not present. |
| child<br>nom<br>mild<br>goin<br>child | iren of the same age or sal<br>mal mood in chronically<br>I elation is reported in si<br>ng to amusement parks,<br>dren very excited. | id above and beyond what is expected in me developmental level. Differentiate from depressed subjects. Do not rate positive if tuations like Christmas, birthdays, which normally overstimulate and make | O | () | () | 2 - Definitely elevated and optimistic outlook that<br>somewhat out of proportion to the<br>circumstances (above and beyond what is<br>expected in a child of the subject's age). Oo<br>less than 4 hours in a day and/or for fewer to<br>3 separate days. |
| PSY | CHIATRIC OR MEDICAL | GS, MEDICATIONS, OR ANY OTHER | () | () | () | <ul> <li>Mood and outlook are clearly out of proportion<br/>circumstances. Noticeable to others and<br/>perceived as odd or exaggerated. Occurs for</li> </ul> |
| work Did I Have ever Were Did I drug Did S Have silly | d? Way more than your n<br>the super-happy feeling se<br>e there been times when y<br>yone else around you?<br>e you laughing about thing<br>it feel like you couldn't stop<br>it seem like you were drun<br>is or alcohol?<br>offer people notice?<br>e your friends ever said at<br>or too high? | ormal happy feeling? wen to come out of the blue? ou were super silly, much more silly than s that normally you would not find funny? laughing? k or high, even though you weren't taking nything to you about being way too happy, too | | | | least 4 hours out of a day for at least 2 consecutive days or on at least 3 separate within one week. PAST: P C S |
| Did y the v Did y reas Can How Wou Did y Ask his/h | you have the feeling that e<br>way you wanted;<br>you feel really excited or it,<br>on to feel this way?<br>you give me some examp,<br>long did this feeling usual<br>it come and go through<br>you ever have problems or<br>Parent/Caregiver: Was | ly last? | | | | |
| | | | P | C | S | |
| Evol | oriva Irritability / Ango | | () | () | () | K - W - |
| Explosive Irritability / Anger | | | | | 0 - No information. | |
| DSN | M-5 DR# 8: Felt angry or lost | your temper; | () | () | () | 1 - Not present. |
| Parent Rating: Child Rating: Was there ever a time you were so irritable and angry that you exploded? When you are feeling really mad, do you throw things or break things. Tear your room apart. Have you ever punched a hole in the wall when you were angry. | | () | () | () | 2 - Subthreshold: Definite periods of excessive<br>irritable/angry mood. Anger / Irritability is of<br>proportion for the situation and occurs for<br>much of the day or intensely for a brief per<br>(< 1 hour). | |
| Whe<br>a tea<br>Wha<br>Have | en you got really angry, dia<br>acher? What about other<br>at was going on at the lime<br>e there been times when y<br>little things that you norm | you ever threaten or actually hurt a parent or<br>kids or pets<br>when this happened? What set you off?<br>ou got super angry without knowing why or<br>ally would not get upset about? | () | () | () | 3 - Threshold: Episodes of explosive irritability<br>anger that are far out of proportion to any<br>stressor or stimuli - has associated aggres<br>behavior (e.g. threats, property destruction<br>physical aggression). Occurs on at least 2<br>consecutive days or on at least 3 separate<br>days within one week. |
| | <ul> <li>Univ rate irritiability ar</li> </ul> | nd explosiveness in this item that occurs<br>represents a change from baseline. Do | | | | PAST: |

| | | SADS-PL SCREEN INTERVIEW:<br>Mania / Hypomania | | EW: | page 7 of 5 <b>2</b> |
|---|---|---|---|---|---|
| | | Р | c | s | |
| sed Energy or Activ | ity | O | () | () | 0 - No information. |
| | | () | () | () | 1 - Not present. |
| DR #9: Starting lots n | nore projects | 17. | | | 2 - Subthreshold: Brief period(s) of increased |
| ere ever been a time w | here you had much more energy than us | ual, | ., | ., | energy, or mild intensification from baseline<br>(cr) likely caused by environmental stimulus<br>questionable clinical significance. |
| hen that happened? | | | () | () | 3 - Threshold: Definite episodes of clear increas |
| eem like you were doin<br>ng did that feeling last?<br>different than other pec<br>thing seem to cause the<br>ere anything else differ | g too many things or were super hyper? Did other people notice it? nple around you? nat feeling? ent about you during the time of high ene | | ,,- | | energy or activity, well beyond baseline or far excess of same age peers in the same situation. PAST: |
| ETIC AT BASELINE,<br>CT PERIOD OF SUBS<br>The (hypo)manic sy | ONLY RATE POSITIVE IF THIS IS A STANTIAL INCREASE IN ENERGY, imptom of increased energy should or | | | | |
| eased Need for Slee | ep | <u>P</u> | <u>c</u> | <u>s</u> | |
| 5 DR 3: PProblems fai | lling asleep, staying asleep, or waking ea | arly. | | | 0 - No information. |
| l Rating: | Child Rating:: | | | | 1 - Not present. |
| 5 DR 10: Sleeping les: | s than usual, still have energy: | () | () | () | 2 - At least 1 1/2 hours less than usual without<br>feeling tired, for at least 2 consecutive days<br>at least 3 separate days. |
| Reting: | Child Rating::: | () | () | () | 3 - At least 3 hours less than usual because he/s |
| leep than usual yet still<br>less sleep). | feels rested (average for several days wh | en | | | felt energetic or high and did not feel tired.<br>Occurs for at least 2 consecutive days, or on<br>least 3 separate days within one week. |
| ich sleep do you ordina<br>ich had you been sleep<br>stay up because you f<br>or by yourself? Had you<br>ne did you wake up? | rily need?<br>ing?<br>elt especially high or energetic? Were you<br>u taken any drugs? Were you up busy doi | ng | | | PAST: C S |
| TRIGGERED BY SOC<br>TMENTS OR DRUG L | ISE, OR REFLECTIVE OF TYPICAL | | | | |
| | DR #9: Starting lots in it Rating: are ever been a time with energy that it felt like then that happened? If the interest in | sed Energy or Activity DR #9: Starting lots more projects It Rating:: Child Rating:: the ever been a time where you had much more energy than us the energy that it felt like too much? What kinds of things were you hen that happened? The energy that it felt like too much? What kinds of things were you hen that happened? The energy that it felt like too much? What kinds of things were you hen that happened? The energy that it felt like too much? What kinds of things were you had the feling? The gean like you were doing too many things or were super hyper? The gean like you were doing too many things or were super hyper? The gean like you were doing too many things were were super hyper? The gean like you glos different about you during the time of high energed of talking, thinking, any thing else? The CHILD HAS ADHD OR IS VERY ACTIVE AND settle AT BASELINE, ONLY RATE POSITIVE IF THIS IS A CT PERIOD OF SUBSTANTIAL INCREASE IN ENERGY. The (hypo)manic symptom of increased energy should on ability). If the symptom is only questionably associated with the symptom is only question | sed Energy or Activity (1) DR #9: Startling lots more projects It Rating:; Child Rating:: | seed Energy or Activity () () () () () () () () () () () () () () () () () () () () ( | sed Energy or Activity (1) (2) (3) (2) (3) (3) (3) (4) (5) (4) (5) (7) (5) (7) (7) (8) (6) (8) Starling lots more projects (7) (8) (9) (9) (10) (10) (8) Rating: |

| 2013 | KSADS-PL SCREEN<br>Mania / Hypo | | RVI | EW: | |
|---|---|---|---|---|---|
| 5. Hypersexuality | | P | c | s | |
| | High Risk Pleasurable Activities] | () | () | () | 0 - No information. |
| | IN THE ABSENCE OF SEXUAL ABUSE OR | () | () | () | 1 - Not present. |
| SYMPTOM FAIRLY SPECIF<br>SEPARATE DSM-5 DIAGNO<br>IT CAN POTENTIALLY FUL | RE TO SEXUAL BEHAVIOR OR MEDIA IS A IC TO MANIC/HYPOMANIA. IT IS NOT A OSTIC CRITERION. BUT WHEN PRESENT. FILL EITHER BOTH THE INCREASED Y AND THE RISKY, PLEASURE-SEEKING | () | () | () | <ol> <li>Isolated, brief incidents of mildly inappropriat<br/>sexual behavior, of questionable clinical<br/>significance.</li> </ol> |
| BEHAVIOR B CRITERION. | AND THE RISKT. PLEASURE-SEEKING | () | () | () | 3 - Definite episodes of clearly inappropriate |
| nudity, his/her private parts or<br>Did your child show an unusu<br>or dressing in an inappropriat<br>Would your child kiss or toucl | your child was excessively focused on sex, touching others' private parts? laid increase in touching their privates in public e or sexual manner? I you in a sexual way or be way too sual way of showing affection? luring these times? | | | | PAST: C S |
| than usual or that your sex dr<br>Did you do anything differentl<br>way, talk about sex a lot or as<br>you)? | y when this happened (dress in a revealing<br>sk other people to be intimate / have sex with<br>were driven to have sex much more than usual | | | | |
| | TIVE, NEED TO RULE OUT SEXUAL ABUSE<br>ISURE TO SEXUAL MATERIAL OR | | | | |
| CURRENT MANIA/HYPO<br>SUPPLEMENT. IF RECEIVED A SCORE | OF 3 ON THE <u>CURRENT</u> RATINGS FOR DMANIA SECTION OF <u>THE</u> DEPRESSIVE OF 3 ON THE <u>PAST</u> RATINGS FOR ANY CTION OF THE DEPRESSIVE AND BIPOLEDO MANIA | OF THE | POLA | R RE | LATED DISORDERS S ITEMS, COMPLETE THE PAST |
| | OF POSSIBLE CURRENT AND PAST HY | POMAN | IA OF | RMAN | NIA). |
| Subject | | | | | K |

| 201 | 3 | KSADS-PL SCREE<br>Disruptive Mood Dysre | 55 377 25 | = (4,7) | 22.5 | |
|---|---|---|---|---|---|---|
| | | | Р | С | <u>s</u> | |
| 1. Irri | itability | | () | () | () | 0 - No information. |
| | Do you often feel cranky, irritable, | or angry? Have you had these | () | () | () | 1 - Not present |
| fe<br>ir<br>ti<br>kc<br>V | eelings in the past few weeks at a<br>n the past year? (if not) How often<br>here been a period of time when y<br>ong as a couple of months at a tin<br>Vinen you are feeling cranky or an | IP Have you felt this way most days<br>do you have these feelings? Has<br>ou didn't have those feelings for as<br>le? | () | () | () | 2 - Subthreshold: Irritable mood present less than half the day or less than most days in the past 12 months, or not severe enough to be noticeable to other people |
| 0 | | e, at school, or when you are with<br>tice the way you feel? What do your<br>out how you are feeling? | () | () | () | Threshold: Irritable and/or angry mood present<br>at least half the day most days for at least 12<br>months. Severity is sufficient to be noticeable to<br>other people (parents, teachers, peers). |
| | IOTE: IN THIS SECTION CODE<br>RRITABILITY OF ONE YEAR DU | | | | | PAST: P C S |
| | | | P | <u>c</u> | <u>s</u> | |
| 2. Re | current Temper Outbursts | | () | () | () | 0 - No information. |
| | Is it pretty easy or common for you to become irritable, angry, or to explode? When you are feeling very angry, do you yell or scream? Do | | | () | () | 1 - Not present. |
| d<br>p | explode? Wrien you are reeing very angry, do you yell or scream? Do you swear a lot, call people names or put them down? Do you throw or destroy things? Have you ever threatened or actually hurt another person? Did you punch, kick, or beat anyone? What was going on at the time when this happened? What set you off? | | | | () | 2 - Subthreshold: Verbal or physical outbursts had<br>not occurred as often as 3 times a week or have n<br>persisted for as long as 12 months. |
| H | | y for so long that you exploded at least | () | () | () | 3 - Threshold: Subject has verbal rages, and/or displays aggressive behaviors toward people or property. Such events occur, on average, at least times a week and have been consistently preserover the past 12months. |
| | | | | | | PAST: C S |
| E | DYSRUPTIVE MOOD DYSRI | 3 ON THE <u>CURRENT</u> RATINGS ON DEGULATION DISORDER (CURRENT) PLEMENT AFTER FINISHING THE S | SECTIO | N OF | THE | DEPRESSIVE AND BIPOLAR |
| | DYSRUPTIVE MOOD DYSRI | 3 ON THE <u>PAST</u> RATINGS ON <u>EITH</u><br>EGULATION DISORDER (PAST) SEC<br>PLEMENT AFTER FINISHING THE S | TION OF | THE | DEPR | ESSIVE AND BIPOLAR |
| _ | NO EVIDENCE OF DYSRU | PTIVE MOOD DYSREGULATION DIS | ORDER | | | |
| NOT | ES: (RECORD DATES OF | POSSIBLE CURRENT AND PAST DY | SRUPTI | VE MO | OOD D | YSREGULATION DISORDER) |
| | | Subject | | | | |
| | | | _ | | | |

| 2013 | KSAL | OS-PL SCREEN INTE<br><u>Psychosis</u> | RVI | EVV: | |
|---|---|---|---|---|---|
| | | P | c | s | |
| 1. Hallucinations | | () | () | () | 0 - No information. |
| DSM-5 DR# 14: Heard \ | laiser | () | () | () | 1 - Not present. |
| Parent Rating: | Child Rating: | () | () | () | 2 - Subthreshold: Suspected or likely. |
| Parent Raung. | Child Rating. | () | () | () | 3 - Threshold: Definitely present. |
| DSM-5 DR# 15: Had visi | ons: | | | | PAST: |
| Parent Rating: | Child Rating: | | | | |
| Sometimes children mig<br>other people cannot her | ime when your mind played tricks<br>ht hear voices or see things, or sn<br>ir, see or smell.<br>I to you? Tell me about it. | | | | P C S |
| | ime when you heard voices that o | other people could | | | |
| | at kind of things did you hear?<br>which other people could not? | | | | |
| other people could not<br>What did you see? How | time when you saw things like peo<br>see? If yes can you tell me abou<br>v often did it happen? When did it I<br>night while you were trying to slee | ut it<br>happen | | | |
| Has there ever been a<br>smell or felt things that | time when you smelled things that<br>weren't there? | other people can't | | | |
| What did you think it wa<br>Did you think it was you<br>Did you think it was rea | | | | | |
| These voices you hear when you were awake Did they happen when was dark? Did they hap Were you sick with feve Have you ever been drugs when it happened | nking beer, wine, liquor? Or taking | ream<br>p? Only when it.<br>g any | | | |
| | ATIONS POSSIBLY PRESENT. R<br>NS WITH THE PROBES BELOW | | l. ASS | ESS T | HE SUBJECT'S CONVICTION OF THE REALIT |
| | TIONS ARE PRESENT. CAREFU<br>OOD SYMPTOMS. THIS WILL F | | | | IN RELATION TO MOOD SYMPTOMS OR |
| NOTE: DO NOT RAT<br>TWICE, | E AS POSITIVE IF ONLY ENDOR | RSES HAVING HEARD SOMEO | NE C | ALLING | THEIR NAME OCCURRING ONLY ONCE OR |
| frequently occur due t | | ness, noisy locale) or inattention and | | | sory slimuli which is momentarily transformed. The<br>diately corrected when attention is focused on the |
| NOTE: TAKE INTO | ACCOUNT CULTURAL BACKG | ROUND OF THE SUBJECT. | | | |
| | | S ACTING ON HALLUCINATION | | | |

| any ideas about things that you didn't tell anyone because a might not understand? The property of the proper | P () () () () | <u>c</u> () | <u>s</u> () () () () | O - No information. 1 - Not present 2 - Subthreshold, Suspected or likely delusional 3 - Threshold: Definite delusions. PAST: PCS |
|---|---|---|---|---|
| In might not understand? In might not understand? In a time you felt that someone was out to hurt you or that ving you or spying an you? Who? Why? In a time you felt that someone was out to hurt you or that ving you or spying an you? Who? Why? In your mind or body (like a robot)? You were an important or great person? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time then you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was coming to an end? In a time you or that the world was coming to an end? In a time you or that the world was coming to an end? In a time you or that the world was coming to an end? In a time you or that you | () | () | () | Not present. Subthreshold, Suspected or likely delusional Threshold: Definite delusions. PAST: |
| In might not understand? In might not understand? In a time you felt that someone was out to hurt you or that ving you or spying an you? Who? Why? In a time you felt that someone was out to hurt you or that ving you or spying an you? Who? Why? In your mind or body (like a robot)? You were an important or great person? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time then you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was happening to your body? In a time you felt something was coming to an end? In a time you or that the world was coming to an end? In a time you or that the world was coming to an end? In a time you or that the world was coming to an end? In a time you or that you | () | () | () | Subthreshold. Suspected or likely delusions Threshold: Definite delusions. PAST: |
| the delusions surveyed below: In a time you felt that someone was out to hurt you or that ving you or spying on you? Who? Why? Of your mind or body (like a robot)? Ou were an important or great person? secial powers? secople you do not know, do you think that they are me when you felt something was happening to your body? rotting from the inside, or that something was very wrong invinced that the world was coming to an end? SINS ARE PRESENT, CAREFULLY ASSESS THE ERMINE IF IN RELATION TO MOOD SYMPTOMS OR | | | | 3 - Threshold: Definite delusions. PAST: |
| the delusions surveyed below: In a time you felt that someone was out to hurt you or that wing you or spying on you? Who? Why? In a time you felt that someone was out to hurt you or that wing you or spying on you? Who? Why? In a time you felt that someone was out to hurt you or that wing you or spying on you? Who? Why? In a time you felt that someon? In when you felt something was happening to your body? In word from the inside, or that something was very wrong winvinced that the world was coming to an end? In same PRESENT, CAREFULLY ASSESS THE ERMINE IF IN RELATION TO MOOD SYMPTOMS OR | () | O | () | PAST: |
| n a time you felt that someone was out to hurt you or that wing you or spying an you? Who? Why? of your mind or body (like a robot)? ou were an important or great person? eacial powers? people you do not know, do you think that they are me when you felt something was happening to your body? rotting from the inside, or that something was very wrong invinced that the world was coming to an end? hink about? | | | | |
| n a time you felt that someone was out to hurt you or that wing you or spying an you? Who? Why? of your mind or body (like a robot)? ou were an important or great person? eacial powers? people you do not know, do you think that they are me when you felt something was happening to your body? rotting from the inside, or that something was very wrong invinced that the world was coming to an end? hink about? | | | | P C S |
| NG THE SCREEN INTERVIEW.<br>SCORE OF 3 ON THE <u>PAST</u> RATINGS ON <u>EITHE</u><br>IE SCHIZOPHRENIA SPECTRUM AND OTHER PS | OTHER | PSY | CHOT | OUS ITEMS. COMPLETE THE PAST |
| OF PSYCHOSIS. | | | | |
| DATES OF POSSIBLE CURRENT AND PAST HAL | LUCINA | ATION | is an | D DELUSIONS). |
| 14 5 | ION OF THE SCHIZOPHRENIA SPECTRUM AND<br>G THE SCREEN INTERVIEW. SCORE OF 3 ON THE <u>PAST</u> RATINGS ON <u>EITHE</u> E SCHIZOPHRENIA SPECTRUM AND OTHER PS SCREEN INTERVIEW. IF PSYCHOSIS. | ION OF THE SCHIZOPHRENIA SPECTRUM AND OTHER G THE SCREEN INTERVIEW. SCORE OF 3 ON THE PAST RATINGS ON EITHER OF THE SCHIZOPHRENIA SPECTRUM AND OTHER PSYCHOT SCREEN INTERVIEW. OF PSYCHOSIS. ATES OF POSSIBLE CURRENT AND PAST HALLUCINA | ION OF THE SCHIZOPHRENIA SPECTRUM AND OTHER PSY G THE SCREEN INTERVIEW. SCORE OF 3 ON THE PAST RATINGS ON EITHER OF THE PE E SCHIZOPHRENIA SPECTRUM AND OTHER PSYCHOTIC DI SCREEN INTERVIEW. OF PSYCHOSIS. ATES OF POSSIBLE CURRENT AND PAST HALLUCINATION | ION OF THE SCHIZOPHRENIA SPECTRUM AND OTHER PSYCHOL G THE SCREEN INTERVIEW. SCORE OF 3 ON THE PAST RATINGS ON EITHER OF THE PREVIOUS E SCHIZOPHRENIA SPECTRUM AND OTHER PSYCHOTIC DISORE SCREEN INTERVIEW. OF PSYCHOSIS. ATES OF POSSIBLE CURRENT AND PAST HALLUCINATIONS AN |

| | | KSADS-PL SCREE<br>Panic Disc | | RVI | EW: | |
|---|---|---|---|---|---|---|
| | | | P | c | s | |
| 1. Panic A | Attacks | | () | () | () | 0 - No information. |
| 100 | | | () | () | () | 1 - Not present. |
| DSM-5 | 5 DR# 11: Felt nervous, a | anxious, or scared: | 100 | | | |
| Have | you ever had a time wh | Child Rating:<br>nen, all of a sudden, out of the blue, for no | () | () | () | Subthreshold: Occasional unanticipated attactor less than 4 of the associated symptoms |
| about i | it. | elt anxious, nervous, or frightened? Tell me<br>nck like this, what did you think brought it on?<br>t of the blue? | () | () | () | Threshold: Recurrent unexpected attacks without or more associated symptoms. |
| How lo | was it like?<br>ong did it last?<br>he first time this happe | ned, did you worry about it happening again? | | | | PAGE |
| If spec | cific symptoms are no | ot elicited spontaneously when describing the following symptoms: | | | | PAST: |
| | lated Symptoms: | | | | | P C S |
| | art palpitations, | | | | | Note: DSM-V does not have threshold criteria |
| 2. swe | | | | | | the minimum number of attacks. |
| | mbling or shaking. | | | | | |
| 4, sen | sations of shortness of | breath, or smothering sensations, | | | | |
| | elings of choking. | | | | | |
| | est pains, | | | | | |
| | usea or abdominal distr | ress, | | | | |
| | ziness or lightheadedne | | | | | |
| | at sensations or chills. | | | | | |
| | imbing of hands or feet<br>epersonalization or der | | | | | |
| 12. fe | ar of losing control. | | | | | |
| 13. fe | ear of dying, | | | | | |
| IFAS | CORE OF 3 ON CL | ASTS ALL DAY OR DIRECTLY CAUSED BY D | ЕМ, СОМ | PLET | E THE | E PANIC DISORDER (CURRENT) |
| | | ETY, OBSESSIVE COMPULSIVE, AND TR<br>SCREEN INTERVIEW. | RAUMA-F | RELAT | rED [ | DISORDERS SUPPLEMENT |
| - SECTI | ION OF THE ANXIE | AST RATING OF PANIC ATTACK ITEM, (<br>ETY, OBSESSIVE COMPULSIVE, AND TR<br>SCREEN INTERVIEW. | | | | |
| | VIDENCE OF PANI | C DISORDER. | | | | |
| - NO EV | CONTRACTOR AND ADDRESS OF | OF POSSIBLE CURRENT AND PAST PA | NIC DICC | RDF | 3) | |

| 2013 KSADS-PL SCI | REEN INTE<br>raphobia | RVI | EW: | |
|---|---|---|---|---|
| | <u>P</u> | c | <u>s</u> | |
| I. Agoraphobia | () | () | () | 0 - No information. |
| Marked fear or anxiety about at least one situation from two or more | () | () | () | 1 - Not present. |
| of the following five groups: 1) being outside home or alone in other situations; 2) standing in line or being in a crowd; 3) being in closed spaces (e.g., shops, theaters or cinemas); 4) open spaces (e.g., parking lots, marketplaces, bridges); 5) using public transportation. | | () | () | <ul> <li>Subthreshold: Fear limited to one situation or<br/>fear only mild or transient, but more severe than a<br/>typical child his/her age.</li> </ul> |
| Have you ever gone through a period when you did not want to leave your home? Have you ever been really afraid of being in a crowded place or going outside in public? Were you bothered by standing in lines? Were you ever afraid to go to the mall, movie theatres, or any other places? Did being in open spaces bother you? Have you ever avoided public transportation including buses or subways? Did these feelings last for several months or longer? | () | () | () | 3 - Threshold: Fears two mor more situations and<br>fears have persisted and are are clearly out of<br>proportion to the circumstances. |
| NOTE: RATE POSITIVELY ONLY IF BEHAVIOR IS ABOVE AND BEYOND WHAT WOULD BE EXPECTED IN CHILDREN OF SAME AGE AND DEVELOPMENTAL LEVEL. | | | | PAST: P C S |
| Do not rate positively if exclusively accounted for by other psychlatr disorders (i.e. psychosis, depression) separation anxiety, social | lc | | | |
| anxiety or medical problems. | <u>P</u> | <u>C</u> | <u>s</u> | |
| Distress / Avoidance How scared did make you? Did it make your stomach upset or your heart race? How long did last? Are you more scared of than any of your friends? Has there ever been a time when your fear of kept you from doing anything? Did you try to avoid? | | () | () | 0 - No information. |
| | | 0 | () | 1 - Not present. |
| | | () | () | <ol> <li>Subthreshold: Associated with only mild<br/>transient symptoms of distress. Minimal or<br/>inconsistent avoidance.</li> </ol> |
| Were there times you could? If someone was with you, could you? | () | () | () | 3 - Threshold: Feared stimuli or situations associal<br>with moderate to severe symptoms of distre-<br>Stimuli or situations consistently avoided or<br>requires presence of companion/support |
| | | | | PAST: P C S |
| IF RECEIVED A SCORE OF 3 ON THE <u>CURRENT</u> RATINGS AGORAPHOBIA (CURRENT) SECTION OF THE ANXIETY, DISORDERS SUPPLEMENT AFTER FINISHING THE SCRE | OBSESSIVE C | OMP | | EVIOUS ITEMS, COMPLETE THE |
| IF RECEIVED A SCORE OF 3 ON THE PAST RATINGS ON AGORAPHOBIA (PAST) SECTION OF THE ANXIETY, OBSI DISORDERS SUPPLEMENT AFTER FINISHING THE SCRE | ESSIVE COMP | ULSI | | |
| NO EVIDENCE OF AGORAPHOBIA. | | | | |
| IOTES: (RECORD DATES OF POSSIBLE CURRENT AND PAS | T AGORAPHO | (BIA) | | |
| Subject | | | | |
| Date / / 2 0 | | | ntervi | |

KSADS-PL SCREEN INTERVIEW: 2013  Separation Anxiety NOTE: KEEP IN MIND THE DEVELOPMENTAL LEVEL OF THE CHILD. RATE POSITIVELY ONLY IF SYMPTOM IS ABOVE AND BEYOND WHAT WOULD BE EXPECTED IN A CHILD OF THE SAME AGE AND DEVELOPMENTAL LEVEL. C S () () () 0 - No information. 1. Fears Calamitous Event that will Cause Separation () () () 1 - Not present. Did you ever worry that something bad might happen to you where you would never see your parents again? Like getting lost, kidnapped, killed, or getting into an accident? () () () 2 - Subthreshold: Occasionally worries. Worries How much do you worry about this? more severely and more often than a typical child his/her age. () () 3 - Threshold: Frequently worries in separation situations. Persistent and excessive worry that an untoward event will lead to separation from major attachment figure PAST: C S P C S () () () 0 - No information. 2. Fears Harm Befalling Attachment Figure () () () 1 - Not present. Has there ever been a time when you worried about something bad happening to your parents? Like what? Were you afraid of them being in an accident or getting killed? () () () 2 - Subthreshold: Occasionally worries. Worries Were you afraid that they would leave you and not come back? more severely and more often than a typical child his/her age. How much did you worry about this? () () () 3 - Threshold: Frequently worries in separation situations. Persistent and excessive worry about losing, or about possible harm befalling major attachment figure PAST: P S C P C S () () 0 - No information 3. School Reluctance/Refusal Was there ever a time when you had to be forced to go to school? () () () 1 - Not present. Did you have worries about going to school? Tell me about those feelings. () () What were you afraid of? 2 - Subthreshold: Frequently somewhat resistant Had you been going to school? about going to school but usually can be How often did you miss school or did you leave school early? persuaded to go, missed no more than 1 day in 2 weeks. NOTE; ONLY COUNT IF SCHOOL AVOIDED IN ORDER TO STAY WITH () () ATTACHMENT FIGURE 3 - Threshold: Protests intensely about going to school, or sent home or refuses to go at least 1 day per week. Persistent reluctance or refusal to go to school. PAST: P C

| 2013 | | KSADS-PL SCREE<br>Separation | | KVI | EVV: | |
|---|---|---|---|---|---|---|
| | | | P | <u>c</u> | <u>s</u> | |
| 4. Fears | Sleeping Away From Ho | ne/Sleeping Alone | () | () | () | 0 - No information. |
| | | e age of four, when you were afraid of | () | () | () | 1 - Not present, |
| Did y<br>parei<br>Do y | oing alone?<br>You get scary feelings if you ha<br>Ints being with you?<br>You move to your parent's bed<br>Yo you need your parent to slee | | () | () | () | <ul> <li>2 - Subthreshold: Occasionally fearful. Fears of<br/>sleeping away or alone more severe and more<br/>frequent than a typical child his/her age.</li> </ul> |
| Do y | ou avoid sieepovers? | p iii you bediesiii. | () | () | () | 3 - Threshold: Frequently fearful, some avoidance<br>sleeping alone or away from home. Persistent<br>refusal to go to sleep without being near a maj<br>attachment figure or to sleep away from home |
| | | | | | | PAST: P C S |
| | | | P | c | <u>s</u> | |
| 5. Fears | Being Alone at Home | | () | () | () | 0 - No information. |
| | | e of 4, when you used to follow your | () | () | () | 1 - Not present. |
| Did y<br>Did y<br>Did y | er wherever she went?<br>ou get upset if she was not in<br>ou cling to your mother?<br>ou check up on your mother a<br>ou always want to know wher | lot? | () | () | () | Subthreshold: Occasionally fearful. Fears of<br>being alone more severe and more frequent<br>than a typical child his/her age. |
| | afraid were you?<br>often did this happen? | | () | () | () | 3 - Threshold: Clings to mother; fearful, some<br>avoidance of being alone. Persistent and<br>excessively fearful or reluctant to be alone or<br>without major attachment fugures at home. |
| | | | | | | PAST: P C S |
| SEP | ARATION ANXIETY DISC | ON THE <u>CURRENT</u> RATINGS OF <u>A</u><br>ORDER (CURRENT) SECTION IN TH<br>BERS SUPPLEMENT AFTER FINISH | E ANXIE | TY, O | BSES | SIVE COMPULSIVE, AND |
| SEP | ARATION ANXIETY DISC | ON THE <u>PAST</u> RATINGS OF <u>ANY</u> OP ORDER (PAST) SECTION IN THE AND PLEMENT AFTER FINISHING THE S | XIETY, C | BSE | SSIVE | COMPULSIVE, AND TRAUMA- |
| NO E | EVIDENCE OF SEPARAT | ION ANXIETY DISORDER. | | | | |
| NOTE: ( | RECORD DATES OF PO | SSIBLE CURRENT AND PAST SEP | ARATION | KAN A | JETY | DISORDER) |


| 1. Fear of Social Situations Are you a very shy person? Have you ever felt nervous, self-conscious or shy around people that you didn't know very well? Is it difficult for you to be with other kids - even kids you know? What kind of situations make you feel uncomfortable? | () | <u>c</u> | <u>s</u> | |
|---|---|---|---|---|
| Are you a very shy person? Have you ever felt nervous, self-conscious or shy around people that you didn't know very well? Is it difficult for you to be with other kids - even kids you know? | () | | | |
| Have you ever felt nervous, self-conscious or shy around people that you didn't know very well?<br>Is it difficult for you to be with other kids - even kids you know? | () | 4.7 | () | 0 - No information. |
| Have you ever felt nervous, self-conscious or shy around people that you<br>didn't know very well?<br>Is it difficult for you to be with other kids - even kids you know? | 0.7 | () | () | 1 - Not present. |
| is it difficult for you to be with other kids - even kids you know? | 2.4 | 100 | | |
| Speaking in front of others (e.g. answering questions in class, giving ora<br>reports, show & tell? | ()<br>al | () | () | 2 - Subthreshold: Clearly self-conscious and<br>uncomfortable in social performance<br>situations; avoids only 1 or 2 activities that<br>not critical to the child's well being (e.g.<br>avoiding large parties where child knows no<br>one). |
| Eating in front of others (e.g. school cafeteria, fast food | () | () | () | 3 - Threshold: Considerable self-consciousness |
| restaurant)? Writing in front of others (e.g., at chalkboard, taking tests)? Using public bathrooms when others are around? Performance situations (e.g., gym class, recess, sports activities)? Changing clothes when others are present (e.g., in gym/pool locker room)? Going to parties or social events? How old were you when you first started to feel this way? For how long have you been feeling this way? NOTE: SHYNESS AND FEAR OF SOCIAL SITUATIONS MUST BE SIGNIFICANTLY AFFECTING THE CHILD, DO NOT RATE POSITIVELY IF EXCLUSIVELY ACCOUNTED FOR BY ANOTHER PSYCHIATRIC DISORDER (i.e., AUTISM SPECTRUM DISORDER) How old were you when you first started to feel this way? For how long have you been feeling this way? | | | | that makes the child uncomfortable in seve social settings; at least 1 activity is avoider (e.g., repeatedly and persistently refusing answer questions in class, avoiding gatherings where child does not know everyone). A marked and persistent fear of social performance situations - fears actin a way (or showing anxiety symptoms) that will be humiliating or embarrassing. DO NC CODE AS THRESHOLD IF THE CHILD'S ONLY FEAR IS GIVING ORAL PRESENTATIONS AT SCHOOL. PAST: P C S |
| 2. Failure to Speak in Specific Social Situations | () | () | () | 0 - No information. |
| Have you ever felt like you couldn't talk in school or other situations? Have you ever felt so shy that you just couldn't say anything? Even to | | ( | | ) 1 - Not present 2 - Subthreshold: Child unable to speak in nov |
| another kid?<br>Are there certain situations that you just can't talk in? | 1 | , , | ) ( | situations, including the start of school year |
| | χ) | r | ) ( | <ul> <li>but symptom does not persist.</li> <li>3 - Threshold: Consistent failure to speak in social situations when expected to speak.</li> </ul> |
| | | | | PAST: |
| | | | | P C S |
| IF RECEIVED A SCORE OF 3 ON THE CURRENT RATINGS O ANXIETY DISORDER/SELECTIVE MUTISM (CURRENT) SECT AND TRAUMA-RELATED DISORDERS SUPPLEMENT AFTER IF RECEIVED A SCORE OF 3 ON THE PAST RATINGS OF EI DISORDER/SELECTIVE MUTISM (PAST) SECTION IN THEAN RELATED DISORDERS SUPPLEMENT AFTER COMPLETING NO EVIDENCE OF SOCIAL ANXIETY DISORDER | TON IN THE<br>COMPLETING<br>THER ITEM,<br>XXIETY, OBS | ON<br>ESSI | ETY,<br>HE SO<br>IPLE<br>VE C | OBSESSIVE COMPULSIVE,<br>CREEN INTERVIEW.<br>TE THE SOCIAL ANXIETY<br>COMPULSIVE, AND TRAUMA- |
| NOTES: (RECORD DATES OF POSSIBLE CURRENT AND PAST | SOCIAL AN | XIET | Y OR | R SELECTIVE MUTISM DISORDER) |

| Only rate most intense phobia. 1. Specific Phobias Are you very, very afraid of anything? Like really, really scared to death of spiders, other insects, dogs, horses, heights, elevators, the subway, or the dark? What about crowds, being outside alone, being on a bridge or traveling in a bus, train or automobile? (ask about all situations listed). Were you afraid of any other things? | ()<br>()<br>() | ()<br>()<br>() | <u>s</u> () () () | O - No information. 1 - Not present. 2 - Subthreshold: Fear of stimuli or situation more severe than a typical child his/her age. |
|---|---|---|---|---|
| Are you very, very afraid of anything? Like really, really scared to death of spiders, other insects, dogs, horses, heights, elevators, the subway, or the dark? What about crowds, being outside alone, being on a bridge or traveling in a bus, train or automobile? (ask about all situations listed). | () | () | () | Not present. 2 - Subthreshold: Fear of stimuli or situation more severe than a typical child his/her age. |
| Like really, really scared to death of spiders, other insects, dogs,<br>horses, heights, elevators, the subway, or the dark?<br>What about crowds, being outside alone, being on a bridge or traveling in<br>a bus, train or automobile? (ask about all situations listed). | () | () | () | 2 - Subthreshold: Fear of stimuli or situation more severe than a typical child his/her age. |
| horses, heights, elevators, the subway, or the dark? What about crowds, being outside alone, being on a bridge or traveling in a bus, train or automobile? (ask about all situations listed). | | 100<br>100 | | severe than a typical child his/her age. |
| | () | () | () | w. weeks the second of a constraint of the second of the s |
| | | | | 3 - Threshold: Marked and persistent fear that is<br>excessive and unreasonable, cued by the<br>presence or anticipation of a specific object<br>or situation. |
| | | | | PAST: P C S |
| | P | С | S | |
| 2. Distress/Avoidance | () | () | () | 0 - No information. |
| How scared did make you? | () | () | () | 1 - Not present. |
| Did it make your stomach upset or your heart race? How long did last? Are you more scared of than any of your friends? Has there ever been a time when your fear of kept you from doing | () | () | () | Subthreshold: Associated with only mild transis<br>symptoms of distress. Minimal or inconsister<br>avoidance. |
| anything? Did you try to avoid? Were there times you could? If someone was with you, could you? | () | () | () | 3 - Threshold: Fear of stimuli or situation associat<br>with moderate to severe symptoms of distres<br>Feared stimuli or situation consistently avoide |
| | | | | PAST: P C S |
| Specify most intense phobia: | - | 1 | 7 | |
| | | | _ | |
| Specify other phobias: | | | | |
| | | | 7 | |
| | Ŧ | $\pm$ | = | |
| | | | 1 | |

| 013 KSADS-PL SCRE<br>Generalized An | | | | |
|---|---|---|---|---|
| | P | c | <u>s</u> | |
| Excessive worries | () | () | () | 0 - No information. |
| DSM-5 DR# 12: Not been able to stop worrying: | () | () | () | 1 - Not present. |
| Parent Rating: Child Rating: | () | () | () | 2 - Subthreshold: Frequently worries somewhat |
| Paralle Raing, Gilla Raing, | | | | excessively (at least 3 times per week) about anticipated events or current behavior. |
| Are you a worrier? Do you worry too much?<br>Do you worry more than other kids your age? Have people said | () | 0 | Ó | 3 - Threshold: Most days of the week is excessive |
| you worry too much? Has there ever been a time when you worried about things | | | ., | worried about at least two different life |
| before they happened?<br>Can you give me some examples? | | | | circumstances or anticipated events or curr<br>behavior. |
| NOTE: IF THE ONLY WORRIES THE CHILD BRINGS UP RELATE TO | | | | PAST: |
| THE ATTACHMENT FIGURE OR A SIMPLE PHOBIA, DO NOT SCORE HERE. ONLY RATE POSITIVELY IF THE CHILD WORRIES ABOUT MULTIPLE THINGS. | | | | PCS |
| In order to rate positively, child must worry above and beyond other children | | | | |
| of the same age. Worries must be exaggerated and out of context: | | | | |
| | Р | c | S | |
| Somatic Complaints | () | () | () | 0 - No information. |
| Projectory C. H. and Colored St. Colored S | () | () | () | 1 - Not present. |
| DSM-5 DR# 1: Bothered by stomachaches, etc.: | () | () | () | 2 - Subthreshold: occasional worries |
| Parent Rating: Child Reting: DSM-5 DR# 2: Worried about getting sick: | | 3.5 | | /complaints. Symptoms/complaints more severe and more often than experienced by typical child his/her age. |
| Parent Rating: Child Rating: | () | () | () | 3 - Threshold: Frequent worries /complaints. |
| | 7.1 | | | Worres about health preoccupy child and cause distress. |
| Do you worry a lot about your health? Do you get a lot of headaches? Stomachaches? | | | | |
| Have a lot of aches and pains? Do you worry that you might have a serious illness? | | | | P C S |
| NOTE: DO NOT COUNT IF SYMPTOMS ARE KNOWN TO BE CAUSED B | V A DEAL N | EDIC | AT II TA | iece. |
| NOTE, DO NOT GOOD IN STANFORD ARE KNOWN TO BE SAUGED E | / HINERE II | LUIO | L ILLI | |
| | | | | _ |
| | | _ | | |
| Subject | | | | |

| 013 | KSADS-PL SCREEN INTE<br>Generalized Anxiety Diso | |
|---|---|---|
| THE GENERALIZED A | E OF <u>3</u> ON THE CURRENT RATINGS OF <u>EITHER</u> (<br>NXIETY DISORDER (CURRENT) SECTION IN THE<br>D DISORDERS SUPPLEMENT AFTER FINISHING T | ANXIETY, OBSESSIVE COMPULSIVE, |
| GENERALIZED ANXIET | OF 3 ON THE PAST RATINGS OF EITHER OF THE Y DISORDER (PAST) SECTION IN THE ANXIETY, O SUPPLEMENT AFTER FINISHING THE SCREEN IN | BSESSIVE COMPULSIVE, AND TRA |
| NO EVIDENCE OF GEN | ERALIZED ANXIETY DISORDER. | |
| OTES: RECORD DATES | OF POSSIBLE CURRENT AND PAST GENERALIZE | D ANXIETY DISORDER). |

#### KSADS-PL SCREEN INTERVIEW: Obsessive-Compulsive Disorder




| | | P | <u>c</u> | S | |
|---|---|---|---|---|---|
| Obsessions | | () | () | () | 0 - No information. |
| DSM-5 DR# 16: Recurr | rent thoughts that you would do something bad or | () | () | () | 1 - Not present. |
| something bad would ha | appen to you or someone else: | () | () | () | 2 - Subthreshold: Suspected or likely. |
| Parent Rating: | Child Rating: | | | 77 | |
| | | () | () | () | <ul> <li>Threshold: Definite obsessions, causes som<br/>effect on functioning or distress.</li> </ul> |
| DSM-5 DR# 18; Wome | d a lot that things you touch were dirty, etc. | | | | PAST: |
| Parent Rating: | Child Rating. | | | | |
| | which is a second of the second | | | | P C S |
| | e thoughts, impulses, or images that, are distressing<br>er which the person has little control. | | | | |
| | a time when thoughts popped into your mind over and | d | | | |
| over and you couldn't<br>Has there ever been a | get rid of them<br>a time when you were bothered by thoughts, "picture. | s" | | | |
| | oming into your head for no reason and that yo | | | | |
| couldn't stop or get rio<br>Did you ever worry a | or<br>lot about having dirt or germs on your hands, or worr | ý | | | |
| that you might get ill fr | | | | | |
| or arranging things in | out doing things perfectly or about making things eve<br>a certain way | en | | | |
| What about thoughts | that something bad might happen, or that you did | | | | |
| | en though you knew it wasn't true<br>oughts that kept running around your mind | | | | |
| | ints, words, or numbers which wouldn't go away | | | | |
| How often did you thin | | | | | |
| again | ip that won't go away, just kept coming again and | | | | |
| re these thoughts an | | | | | |
| | make anv sense | | | | |
| Did they not seem to | t in your way or stop you from doing things | | | | |

NOTE: DO NOT SCORE OBSESSIONS TEMS POSITIVELY IF IDEAS /THOUGHTS ARE DELUSIONAL, OR ARE EXCLUSIVELY DUE TO ANOTHER AXIS I DISORDER (e.g. thoughts of food in the presence of an eating disorder; thoughts that parents will get harmed in the presence of a separation anxiety disorder; increased worries from GAD). DO NOT RATE POSITIVELY IF SAYS, "I cannot stop thinking about boy/girlfriend or music."

| | V |
|----------|-----|
| Subject | Po- |
| 2.447.44 | 1.7 |

| 2013 | KSADS-PL SCREE Obsessive-Comput | | 22, 2, 2, 5 | 7.7.7. | |
|---|---|---|---|---|---|
| | | <u>P</u> | c | <u>s</u> | |
| 2. Compulsions | | () | () | () | 0 - No information, |
| DSM-5 DR# 17: Felt the n | reed to check thinkgs over and over again, etc. | () | () | () | 1 - Not present |
| Parent Rating: | Child Rating: | () | () | () | 2 - Subthreshold: Suspected or likely. |
| DOM 5 DD# 10: Eath you | nad to do things in a certain way, like counting, etc | () | () | () | <ul> <li>Threshold: Definite compulsions, causes seeffect on functioning or distress.</li> </ul> |
| | Child Rating: | | | | |
| Parent Rating: | Critic Raung | | | | PAST: |
| to an obsession, accordi | titive, purposeful behaviors performed in response<br>ng to certain rules, or in stereotyped fashion that are<br>ng and over which the person has little control. | | | | P C S |
| seemed silly over and o | ime when you found yourself having to do things that<br>ver, or things which you could not resist repeating<br>ounting or washing your hands many times, or<br>things? | | | | |
| | urself having to repeat certain actions over and | | | | |
| | y control over them? Did these things bother you?<br>Iways felt you had to do exactly the same way or in | | | | |
| read parts of an assignr<br>re-writing your homewor | le making it to school on time because it takes too | | | | |
| | n your school work, did you have to start at the | | | | |
| What about when you w<br>several times before you | | | | | |
| | nge things in your room in a particular way?<br>commented about these habits? | | | | |
| NOTE: DO NOT RATE | POSITIVELY IF BEHAVIOR IS EXCLUSIVELY ACC | OUNTED | FOR E | BY ANG | OTHER DISORDER (e.g., PDD, Asperger's, tic |
| OBSESSIVE COMP | ORE OF <u>3</u> ON <u>CURRENT</u> RATINGS OF <u>EITHE</u><br>ULSIVE DISORDER (CURRENT) SECTION IN<br>DISORDERS SUPPLEMENT AFTER FINISH | THE AN | XIET | Y, OBS | SESSIVE COMPULSIVE, AND |
| OBSESSIVE COMP | ORE OF <u>3</u> ON <u>PAST</u> RATINGS OF <u>EITHER</u> O<br>ULSIVE DISORDER (PAST) SECTION IN THE<br>ERS SUPPLEMENT AFTER FINISHING SCRE | ANXIET | Y, OE | SESS | TO 이 급하게 되고 있다면서 이번 등에 생물을 하게 있다면서 하면 없을까지 않는 것입니다. |
| NO EVIDENCE OF | OBSESSIVE COMPULSIVE DISORDER. | | | | |

| 2013 | KSADS-PL SCREEI<br>Enures | | :RVI | EW: | |
|---|---|---|---|---|---|
| | Lituies | 13 | | | page 22 01 02 — |
| . Repeated Voiding | | | | | |
| A lot of kids sometimes have acc<br>at night. Has there ever been a ti<br>Did you ever have accidents duri | | | | | |
| What about if you laughed or sne | | P | C | S | |
| a. Night time | | () | () | () | 0 - No information. |
| How often did this happen a | t night? | () | () | () | 1 - Not present. |
| | | () | () | () | 2 - At least one to four times a month for three of more months. |
| | | () | () | () | 3 - At least two times a week for three consecutive months. |
| | | | | | PAST: |
| | | P | C | <u>s</u> | P C S |
| b. Daytime | | () | () | () | 0 - No information. |
| How often did this happen of | luring the day? | () | () | () | 1 - Not present. |
| | | () | () | () | At least one to four times a month for three o more months. |
| | | () | () | () | At least two times a week for three consecution months. |
| | | | | | PAST: |
| | | P | C | s | P C S |
| c. Total | | () | () | () | 0 - No information. |
| Estimate frequency of c | ombined nighttime and | () | () | () | 1 - Not present. |
| daytime accidents. | STATE OF THE STATE | () | () | () | At least one to four times a month for three of more months. |
| NOTE: Do not rate positiv | rely if enuresis due to | () | () | () | At least two times a week for three consecution months. |
| medical condition. | | | | | PAST: |
| | | | | | P C S |
| IF RECEIVED A SCORE OF<br>THE QUESTIONS ON THE | 3 OR ABOVE ON THE <u>CURRENT</u> RA<br>FOLLOWING PAGE. | TINGS | OF AN | IY OF | THE PREVIOUS ITEMS, COMPLETE |
| IF RECEIVED A SCORE OF QUESTIONS ON THE FOL | | GS OF A | NY O | F THE | PREVIOUS ITEMS, COMPLETE THE |
| IF NO EVIDENCE OF ENU | RESIS, GO TO ENCOPRESIS SECTIO | N ON P | AGE 2 | 24. | |
| | Subject | | | | |
| | Guijest | | | | |

| 013 | | KSADS-PL SCREEN INTERVIEW:<br>Enuresis | |
|---|---|---|---|
| Dist | tress | | |
| | | when you had an accident? Did you tell your mom? Your teacher? What mes had accidents? How much did it bother you when you had an accider | |
| Imp | airment: (home, sch | ool, peers) | |
| Dura | ation: (specify) | | |
| DSM<br>A. R.<br>B. T | he behavior is clinically si<br>significant distress or in | e into bed or clothes, whether involuntary or intentional;<br>gnificant as manifested by either a frequency of twice a week for at least three consecutive r<br>mpairment in social, academic (occupational), or other important areas of functioning; | months, or the presence of clinically |
| DSM<br>A. R<br>B. T | M-5 Criteria Repeated voiding of urining the behavior is clinically significant distress or in Chronological age is at l | gnificant as manifested by either a frequency of twice a week for at least three consecutive r<br>mpairment in social, academic (occupational), or other important areas of functioning;<br>east 5 years (or equivalent developmental level);<br>outable physiological effect of a substance (e.g., a diuretic, an antipsychotic medication) | |
| A R B T C. C. D. 1 | N-5 Criteria Repeated voiding of urining the behavior is clinically significant distress or inchronological age is at Inthe behavior is not attribudiabetes, spina bifida, | gnificant as manifested by either a frequency of twice a week for at least three consecutive of mpairment in social, academic (occupational), or other important areas of functioning; east 5 years (or equivalent developmental level); outable physiological effect of a substance (e.g., a diuretic, an antipsychotic medication) a seizure disorder). A FOR ENURESIS (CURRENT), (Scored 3 plus impairment). | |
| DSM<br>A. R.<br>B. T<br>C. C.<br>D. 1 | W-5 Criteria Repeated voiding of urining the behavior is clinically significant distress or in chronological age is at I the behavior is not attributed abetes, spina bifida. TS DSM-5 CRITERIAL SITES IN CRITERIAL SITES IN COLUMN IN CRITERIAL SITES IN CRITERIA | gnificant as manifested by either a frequency of twice a week for at least three consecutive of maximment in social, academic (occupational), or other important areas of functioning; east 5 years (or equivalent developmental level); outable physiological effect of a substance (e.g., a diuretic, an antipsychotic medication), a seizure disorder). A FOR ENURESIS (CURRENT), (Scored 3 plus impairment). Diurnal Only: Nocturnal and Diurnal; | |
| A R B T C C D T | Repeated voiding of urinche behavior is clinically si significant distress or in Chronological age is at I The behavior is not attrib diabetes, spina bifida. TS DSM-5 CRITERIA (If): TS DSM-5 CRITERIA (IT): TS DSM-5 CRITERIA (IT): TS DSM-5 CRITERIA (IT): TS DSM-5 CRITERIA (IT): | gnificant as manifested by either a frequency of twice a week for at least three consecutive of manifested by either a frequency of twice a week for at least three consecutive of manifested in social, academic (occupational), or other important areas of functioning; east 5 years (or equivalent developmental level); autable physiological effect of a substance (e.g., a diuretic, an antipsychotic medication) a seizure disorder). A FOR ENURESIS (CURRENT). (Scored 3 plus impairment). Diumal Only: Nocturnal and Diumal; | |
| A R B T C C D T | Repeated voiding of urinche behavior is clinically si significant distress or in Chronological age is at I The behavior is not attrib diabetes, spina bifida. TS DSM-5 CRITERIA (If): TS DSM-5 CRITERIA (IT): TS DSM-5 CRITERIA (IT): TS DSM-5 CRITERIA (IT): TS DSM-5 CRITERIA (IT): | gnificant as manifested by either a frequency of twice a week for at least three consecutive of maximment in social, academic (occupational), or other important areas of functioning; east 5 years (or equivalent developmental level); outable physiological effect of a substance (e.g., a diuretic, an antipsychotic medication), a seizure disorder). A FOR ENURESIS (CURRENT), (Scored 3 plus impairment). Diurnal Only: Nocturnal and Diurnal; | |

| 201 | 3 | KSADS-PL SCREE<br>Encopre | | RVI | EW: | |
|---|---|---|---|---|---|---|
| 1. R | epeated Passage of Fece | 25 | | | | |
| 1 | his ever happen to you?<br>Has there ever been a time w<br>bathroom in your pants during | eally scared, or for some reason couldn't get to<br>I to? | | | | |
| | NOTE: ONLY RATE POSITI | VELY IF THERE ARE STOOLS IN THE | | | | |
| | | | <u>P</u> | <u>c</u> | <u>s</u> | |
| 3 | a. Night time | | () | () | () | 0 - No information, |
| | How often did this happe | en at night? | () | () | () | 1 - Not present. |
| | | | () | () | () | 2 - Subthreshold: Less than 1 time a month. |
| | | | () | () | () | 3 - Threshold: 1 or more times a month for at least<br>3 months. |
| | | | | | | PAST: P C S |
| | | | <u>P</u> | C | <u>s</u> | |
| | b. Daytime | | () | () | () | 0 - No information. |
| | How often did this happe | en during the day? | () | () | () | 1 - Not present. |
| | | | () | () | () | 2 - Subthreshold; Less than 1 time a month. |
| | | | () | () | () | 3 - Threshold: 1 or more times a month for at leas<br>3 months. |
| | | | | | | PAST: |
| | | | <u>P</u> | <u>c</u> | <u>s</u> | P C S |
| 2 | c. Total | | () | () | () | 0 - No information. |
| | Estimate total number of | nighttime and daytime accidents. | () | () | () | 1 - Not present. |
| | | | () | () | () | 2 - Subthreshold: Less than 1 time a month. |
| | | | () | () | () | 3 - Threshold: 1 or more times a month for at leas 3 months. |
| | | | | | | PAST: P C S |
| | | OF <u>3</u> OR ABOVE ON THE <u>CURRENT</u> RA | ATINGS ( | OF AN | Y OF | THE PREVIOUS ITEMS, COMPLETE |
| | F RECEIVED A SCORE | OF 3 OR ABOVE ON THE PAST RATING | GS OF A | NY OF | THE | PREVIOUS ITEMS, COMPLETE THE |
| | F NO EVIDENCE OF EN | COPRESIS, GO TO ANOREXIA NERVO | SA SECT | ION | ON PA | AGE 26. |

| Distress What did you usually do when you had an accident? Did you tell your mom? Your teacher? What did they do? Did the kids school know you sometimes had accidents? How much did it bother you when you had an accident? Impairment: (home, school, peers) Duration: (specify) |
|---|
| school know you sometimes had accidents? How much did it bother you when you had an accident? Impairment: (home, school, peers) |
| Duration: (specify) |
| Duration: (specify) |
| DSM-5 Criteria A. Repeated passage of feces into inappropriate places (e.g. clothing or floor) whether involuntary or intentional; B. At least one such event occurs each month for at least 3 months; C. Chronological age is at least 4 years (or equivalent developmental level); D. The behavior is not attributable to the physiological effect of a substance (e.g., laxatives) or another medical condition except through a |
| DSM-5 Criteria A. Repeated passage of feces into inappropriate places (e.g. clothing or floor) whether involuntary or intentional; B. At least one such event occurs each month for at least 3 months; C. Chronological age is at least 4 years (or equivalent developmental level); |
| DSM-5 Criteria A. Repeated passage of feces into inappropriate places (e.g. clothing or floor) whether involuntary or intentional; B. At least one such event occurs each month for at least 3 months; C. Chronological age is at least 4 years (or equivalent developmental level); D. The behavior is not attributable to the physiological effect of a substance (e.g., laxatives) or another medical condition except through a |
| A. Repeated passage of feces into inappropriate places (e.g. clothing or floor) whether involuntary or intentional; B. At least one such event occurs each month for at least 3 months; C. Chronological age is at least 4 years (or equivalent developmental level). D. The behavior is not attributable to the physiological effect of a substance (e.g., laxatives) or another medical condition except through a mechanism involving constipation. MEETS DSM-5 CRITERIA FOR ENCOPRESIS (CURRENT). |
| A. Repeated passage of feces into inappropriate places (e.g. clothing or floor) whether involuntary or intentional; B. At least one such event occurs each month for at least 3 months; C. Chronological age is at least 4 years (or equivalent developmental level); D. The behavior is not attributable to the physiological effect of a substance (e.g., laxatives) or another medical condition except through a mechanism involving constipation. MEETS DSM-5 CRITERIA FOR ENCOPRESIS (CURRENT). Specify: With constipation and overflow incontinenece or Without constipation and overflow incontinenece MEETS DSM-5 CRITERIA FOR ENCOPRESIS (PAST). |

KSADS-PL SCREEN INTERVIEW: 2013  **Eating Disorders** Begin this section with a brief (2-3 minute) semi-structured interview to obtain information about eating habits: Are you happy with your weight? Do you eat regular meals? Are you a dieter? Has there ever been a time when you weighed a lot more or a lot less? What was your weight? What did you want your weight to be? P C S () 0 - No information. () () 1. Fear of Becoming Obese () () () Has there ever been a time when you were afraid of getting fat? 1 - Not present Did you believe you were fat? () () () 2 - Subthreshold: Intense and persistent fear of Have you ever been really overweight? Did you watch what you ate and think about what you ate all the time? becoming fat, which defies prior weight history Were you afraid of eating certain foods because you were afraid they'd and/or present weight, reassurance, etc. Fears make you fat? What foods? have only moderate impact on behavior and/or How much time did you spend thinking about food and worrying about functioning (e.g., weight loss methods utilized at least once a month, but less than once a getting fat? week). If you saw that you had gained a pound or two, did you change your eating habits? Fast for a day or do anything else? () () 3 - Threshold: Intense and persistent fear of becoming fat, that has severe impact on NOTE: KEEP IN MIND DIFFERENTIAL DIAGNOSES OF ANXIETY behavior and/or functioning (e.g., constantly DISORDER, OCD, AND PSYCHOSIS. pre-occupied with weight concerns; or use of weight loss methods 1 time a week or more). PAST: P C S P C S () () () 2. Emaciation 0 - No information. () () () Weight is proportionally lower than ideal weight for height. 1 - Not present. () () 2 - Subthreshold: Weight below 90% of ideal If, by observation, there is any suspicion of emaciation, you must weigh the child, and look at the table (see attached). If in doubt do not ask, just weigh the child. () () 3 - Threshold: Weight below 85% of ideal. NOTE: DO NOT RATE POSITIVELY IF WEIGHT LOSS IS DUE TO A MEDICAL CONDITION, MOOD DISORDER, OR FOOD SCARCITY PAST: RELATED TO POVERTY.

#### KSADS-PL SCREEN INTERVIEW: Eating Disorders




#### 3. Weight Loss Methods

Have you ever used diet pills to control your weight?
How about laxatives, or water pills to lose weight?
Did you sometimes make yourself throw up?
Did you exercise a lot, more than was usual for you, in order to lose weight? How much? How many hours a day?
Did you have periods of at least 1 week during which you had nothing but liquids with no calories (teas, diet sodas, coffee, water)?

| 1 2 | ia No Information Not present Less than one time a week One or more times a week | | 10 | rent | | | 2. 40 | rent<br>SP | | | | ild<br>E | | | - | nild<br>SP | | s | um<br>C | | У | s | um<br>M: | ma<br>SP | гу |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| a. | using diet pills | 0 | 1 | 2 | 3 () | 0 | 1 | 2 | 3 () | 0 | 1 | 2 | 3 () | 0 | 1 | 2 | 3 () | 0 () | 1 () | 2 | 3 | 0 () | 1 | 2 | 3 |
| b. | taking laxatives | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () |
| c. | taking water pills | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | ( |
| d. | throwing up | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | ( |
| e. | exercising a lot | () | () | () | () | () | () | () | () | () | () | () | () | (.) | () | () | () | () | () | () | () | () | () | () | ( |
| f. | taking only non-caloric fluids for<br>a week or more; restricting<br>energy (e.g., food) intake | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | ( |
| g. | combined frequency weight loss<br>methods | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | ( |

| Subject | | | |
|---------|-----|-------------|-------|
| Date / | 120 | Interviewer | ו רבל |

| 2013 | KSADS-PL SCREET | | RVI | EW: | |
|---|---|---|---|---|---|
| | | P | c | <u>s</u> | |
| 4. Eating Binges or Attacks | | () | () | () | 0 - No information |
| Binge eating episode associated with three | or more of the following: | () | () | () | 1 - Not present |
| Eating much more rapidly than normal. Eating until feeling uncomfortably full. Eating large amounts of food when not personal. | physically hungry. | () | () | () | Subthreshold: Eating binges that occur less<br>than once a week or have fewer than three<br>associated features. |
| <ol> <li>Eating alone because of being embarras</li> <li>Feelng disgusted, depressed, or very gu</li> </ol> | | () | () | () | Threshold: Eating binges once a week or mo |
| Has there ever been a time when you had What's the most you ever ate at one time? Have there ever been times you ate so mu happen? (ascertain all details in definition) What did you usually eat when you binged? What did you usually eat when you binged? What was the most food you have eaten do Did you ever make yourself throw up after thow did you feel after you binged? Did you usually binge alone or with other people know you binged? NOTE: ONLY RATE EATING BINGES THAID HINGE THOUGHT TO NOTE SATING ORGIES (e.g., outlings with friends) | ch you felt sick? How often did it ouring a binge? a binge? a binge? apple? AT ARE PATHOLOGICAL (e.g., followed by depressed mood, AATE TYPICAL ADOLESCENT | | | | PAST: P C S |
| IF RECEIVED A SCORE OF 3 ON C<br>COMPLETE THE EATING DISORDI<br>DISORDERS SUPPLEMENT AFTER | ERS SECTION IN THE EATING | DISOR | DERS | | |
| IF RECEIVED A SCORE OF 3 ON P<br>COMPLETE THE EATING DISORDE<br>DISORDERS SUPPLEMENT AFTER | ERS SECTION IN THE EATING | DISORE | DERS | | |
| NO EVIDENCE OF AN EATING DIS | SORDER. | | | | |
| | | | 2.5 | 201 | |
| NOTE: (RECORD DATES OF POSSIBL | E CURRENT AND PAST EATI | NG DISC | RDE | <u> </u> | |



### KSADS-PL SCREEN INTERVIEW: **Attention Deficit Hyperactivity**




Compared to other children/adolescents this age, how would parent/adult rate this child/adolescent. Also ask if teachers or others have

| urrent rating to describe the symptom's most intense severity over the p<br>rior episode of symptomatology was followed by a period of six months | ast year | Scor | e sym | |
|---|---|---|---|---|
| f the symptoms are episodic, consider the presence of a mood disorder of | or other | cause | s (e.g. | , alcohol, drugs or medical problems). |
| Probe: For how long has been a problem? Has it been a problem<br>earlier? Note: According to the DSM-5, onset of ADHD symptoms can appear | | | arten? | First grade? Did the problem start even |
| | <u>P</u> | <u>c</u> | <u>s</u> | ************ |
| Difficulty Sustaining Attention on Tasks or Play Activities | () | () | () | 0 - No information. |
| DSM-5 DR# 4: Not able to pay attention: | 0 | 0 | () | 1 - Not present. |
| Parent Rating: Child Rating: | () | () | () | <ol> <li>Subthreshold: Occasionally has difficulty<br/>sustaining attention on tasks or play activities.<br/>Problem has only minimal effect on<br/>functioning.</li> </ol> |
| Has there ever been a time when you had trouble paying attention in<br>school? Did it affect your school work.<br>Did you get into trouble because of this<br>When you were working on your homework, did your mind wander<br>What about when you were playing games? Did you forget to go when it | () | () | 0 | <ol> <li>Threshold: Often (4-7 days/week) has difficulty<br/>sustaining attention. Problem has significant<br/>effect on functioning.</li> </ol> |
| was your turn<br>Did teachers complain | | | | PAST: |
| NOTE: RATE BASED ON DATA REPORTED BY INFORMANT (e.g., parent or teacher) OR OBSERVATIONAL DATA | | | | P C S |
| NOTE: DO NOT RATE POSITIVELY IF OCCURS ONLY DURING MOOD EPISODE, PSYCHOSIS, EPISODES OF DRUG USE, OR SECONDARY TO A MEDICAL CONDITION., | | | | |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| 2 Easily Distracted | () | () | () | 0 - No information. |
| Was there ever a time when little distractions would make it very hard for<br>you to keep your mind on what you were doing? | () | () | () | 1 - Not present. |
| Like if another kid in class asked the teacher a question while the class was<br>working quietly, was it hard for you to keep your mind on your work? | () | () | () | <ul> <li>2 - Subthreshold: Occasionally distractible. Proble<br/>has only minimal effect on functioning.</li> </ul> |
| When there was an interruption, like when the phone rang, was it hard to get back to what you were doing before the interruption? Were there times when you could keep your mind on what you were doing, and little noises and things didn't bother you? How often were they a problem? | () | () | () | <ul> <li>Threshold: Attention often (4-7 days/week)<br/>disrupted by minor distractions other kids wou<br/>be able to ignore. Problem has significant lefter<br/>on functioning.</li> </ul> |
| Did teachers complain? NOTE: RATE BASED ON DATA REPORTED BY INFORMANT OR OBSERVATIONAL DATA. | | | | PAST: P C S |
| NOTE: DO NOT RATE POSITIVELY IF OCCURS ONLY DURING MOOD EPISODE, PSYCHOSIS, EPISODES OF DRUG USE, OR SECONDARY TO A MEDICAL CONDITION | | | | |

| 0.000 | |
|---------|------|
| Subject | D. 1 |

| 20 | 12 | S-PL SCREEN INTE | 333 | | |
|---|---|---|---|---|---|
| | | <u>P</u> | <u>c</u> | <u>s</u> | |
| 3. C | Difficulty Remaining Seated | () | () | () | 0 - No information |
| | Was there ever a time when you got out of your seat a lot | at school? () | () | () | 1 - Not present. |
| | Did you get into trouble for this?<br>Was it hard to stay in your seat at school? What about din | 11 | () | () | Subthreshold: Occasionally has difficulty remaining seated when required to do so. |
| | Parents: When your child was young, were you able to ta<br>church? Restaurants? | ke him/her to | | | Problem has only minimal effect on function |
| | Were these difficulties beyond what you would expect for age? | a child his/her () | () | () | <ul> <li>Threshold: Often (4-7 days/week) has difficultied remaining seated when required to do so.</li> <li>Problem has significant effect on functioning</li> </ul> |
| | NOTE: RATE BASED ON DATA REPORTED BY INFOR<br>OBSERVATIONAL DATA. | MANT OR | | | PAST: |
| | Take into account that these symptoms tend to impro<br>Carefully check if this symptom was present when the<br>younger. | | | | P C S |
| | | <u>P</u> | <u>c</u> | <u>s</u> | |
| l. Ir | mpulsivity | () | () | () | 0 - No information. |
| | Do you act before you think, or think before you act?<br>Has there ever been a time when these kinds of behaviors<br>trouble? Give some examples. | The state of the s | () | () | 1 - Not present. |
| | | () | () | () | <ul> <li>2 - Subthreshold: Occasionally impulsive.</li> <li>Problem has only minimal effect on function</li> </ul> |
| | (THIS ITEM IS NOT A DSM-5 CRITERION - DO NOT IN<br>SYMPTOM COUNT) | () | () | () | <ol> <li>Threshold: Often (4-7 days/week) impulsive.</li> <li>Problem has significant effect on functionin</li> </ol> |
| | | | | | PAST: P C S |
| , | IF RECEIVED A SCORE OF 3 ON THE CURREL<br>ATTENTION DEFICIT HYPERACTIVITY DISOR<br>DISRUPTIVE, AND CONDUCT DISORDERS SU | DER (CURRENT) SECTION | INT | HEN | EURODEVELOPMENTAL, |
| | IF RECEIVED A SCORE OF 3 ON THE PAST R<br>DEFICIT HYPERACTIVITY DISORDER (PAST)<br>DISORDERS SUPPLEMENT AFTER COMPLET | SECTION IN THE NEURO | DEVE | LOPN | |
| 3 | NO EVIDENCE OF ATTENTION DEFICIT DISO | RDER. | | | |
| | | | | | PERACTIVITY DISORDER). |



### KSADS-PL SCREEN INTERVIEW: Oppositional Defiant Disorder




The essential feature of this disorder is a recurrent pattern of negativistic, defiant, disobedient, and hostile behavior toward authority figures that persists for at least 6 months and occurs more frequently than is typically observed in individuals of comparable age and developmental level.

Keep in mind differential diagnoses of depressive disorder, bipolar disorder, anxiety disorders, ADHD, psychosis, substance use disorders or medical illness. Also consider environmental issues.

While the DSM-5 is not clear regarding this issue, consider making this diagnosis if symptoms are present in more than one setting (i.e., home and school) consider diagnosis of Parent-Child Relational Problem if symptoms occur ONLY at home

| | P | C | S | |
|---|---|---|---|---|
| Loses Temper | () | | () | 0 - No information. |
| LOSES TOTIFIED | - | | | |
| DSM-5 DR# 8: Felt angry or lost your temper. | () | () | () | 1 - Not present. |
| Parent Rating: Child Rating: | () | () | () | <ol> <li>Subthreshold; Occasional severe temper outburs<br/>(less than 1 time weekly).</li> </ol> |
| Has there ever been a time when you would get upset easily and lose your temper? Did it take much to get you mad? How often did you get really mad or annoyed and lose your temper? | () | () | () | Threshold: Less severe outbursts daily or severe temper outbursts at least once a week Outbursts more severe and more often than a typical child his/her age; cause impairment. PAST: P. C. S. |
| In order to be sure this is a temper outburst, ask: Where do you lose your temper? What do you do when you have a temper tantrum | | | | P C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| Argues A Lot With Adults/Authority Figures | () | () | () | 0 - No information, |
| Was there ever a time when you would argue, talk back, "smart mouth" a lot | () | () | () | 1 - Not present. |
| with adults? Your parents or teachers?<br>What kinds of things did you argue with them about?<br>Did you argue with them a lot?<br>How bad did the fights get? | () | () | () | 2 - Subthreshold: Occasionally argues with parents and/or teachers; less than once per week. |
| NOTE: ARGUING INCLUDES AN UNWILLINGNESS TO COMPROMISE, GIVE IN, OR NEGOTIATE WITH ADULTS OR PEERS. | () | () | () | 3 - Threshold: Often argues with parents and/or<br>teachers (at least one time per week).<br>Arguments more severe and more often<br>than a typical child his/her age. |
| | | | | PAST: P C S |
| Subject | | | | |

| | 13 KSADS-PL SCREEN Oppositional Defia | | | | |
|---|---|---|---|---|---|
| | | P | <u>c</u> | <u>s</u> | |
| 3. [ | Disobeys Rules A Lot/Defies or refuses to comply with adult | () | () | () | 0 - No information. |
| | requests | () | () | () | 1 - Not present. |
| | Do you ever deliberately defy or disobey the rules at home? School? How often? Do you think that your parents/teachers ask you to do things that you shouldn't have to do? Like what? | () | () | () | <ul> <li>2 - Subthreshold: Occasionally actively defies or<br/>refuses adult requests or rules; less than one<br/>time per week.</li> </ul> |
| | In addition ask the following for adolescents:<br>How often to you get away with things without getting into trouble or without<br>getting caught? Does this get you into trouble? | () | () | () | Threshold: Often actively defies or refuses adult requests or rules (at least once a week). Disobedient more often than a typical child his/her. |
| | | | | | PAST: C S |
| - | IF RECEIVED A SCORE OF 3 ON THE CURRENT RATINGS OF A OPPOSITIONAL DEFIANT DISORDER (CURRENT) SECTION OF CONDUCT DISORDERS SUPPLEMENT AFTER FINISHING THE | THE NE | URO | DEVE | LOPMENTAL, DISRUPTIVE, AND |
| 3 | IF RECEIVED A SCORE OF 3 ON THE PAST RATINGS OF ANY OPPOSITIONAL DEFIANT DISORDER (PAST) SECTION OF THE CONDUCT DISORDERS SUPPLEMENT AFTER FINISHING THE STATE OF | NEURO | DEV | ELOPI | MENTAL, DISRUPTIVE, AND |
| | NO EVIDENCE OF OPPOSITIONAL DEFIANT DISORDER. | | | | |
| NO | TE: (REGORD DATES OF POSSIBLE CURRENT AND PAST OPPO | SITION | IAL D | EFIAN | NT DISORDER). |

KSADS-PL SCREEN INTERVIEW: 2013  Conduct Disorder The essential feature of Conduct Disorder is a repetitive and persistent pattern of behavior in which the basic rights of others or major age appropriate societal rules are violated. Three behaviors must have been present during the past 12 months with at least one present in the past 6 months. Keep in mind differential diagnoses of mood disorders, ADHD, psychosis, substance abuse. If symptoms occur only during manic episode, consider NOT giving both diagnoses. P C S () () 0 - No information. 1. Lies () () () 1 - Not present. Everybody lies. Some kids tell lies to exaggerate, some kids tell lies to get out of trouble, while others tell lies to con/cheat others. () () () 2 - Subthreshold: Occasionally lies. Lies more often Do you ever tell lies? than a typical child his/her age. What type of lies do you tell? () () 3 - Threshold: Lies often, multiple times per week Who do you lie to? or more (to con or cheat). Have people ever called you a liar? What's the worst lie you ever told? PAST: Did you lie to get other people to do things for you? Did you lie to get out of paying people back money or some favor you owe them? P C S Has anyone ever called you a con? Complained that you broke promises a lot? How often did you lie? NOTE: ONLY RATE POSITIVE EVIDENCE OF LYING TO CHEAT OR "CON." P C S () () () 2. Truant 0 - No information. () () () 1 - Not present. Has there ever been a time when you skipped a whole day of school when your parents didn't know about it? Did you ever go to school and leave early when you were not really supposed to? How about going in late? () () () 2 - Subthreshold: Truent on one isolated incident. Did you sometimes miss or skip classes in the morning? () () 3 - Threshold: Truant on numerous occasions Did you get into trouble? How aften? (e.g. 2 or more days or numerous partial days) For adolescents: How old were you when you first started to play hooky? PAST: NOTE: ONLY RATE POSITIVE INCIDENTS OF TRUANCY BEGINNING BEFORE THE AGE OF 13. IN ADDITION, TRUANCY IS ACTIVELY MISSING PART OR ALL OF A SCHOOL DAY REGARDLESS OF P C S PARENT ABILITY TO ENFORCE ATTENDANCE. Subject

Interviewer

| | sorder | :RVI | EW: | |
|---|---|---|---|---|
| | P | <u>c</u> | <u>s</u> | |
| Initiates Physical Fights | () | () | () | 0 - No information. |
| Has there ever been a time when you got into many fist fights? | () | () | () | 1 - Not present. |
| Who usually started the fights? What's the worst fight you ever got into? What happened? Did anyone get hurt? Who did you usually fight with? | () | () | () | Subthreshold: Fights with peers only. No fight<br>has resulted in serious injury to peer (e.g. no<br>medical intervention required, stitches, etc.). |
| Have you ever hit a teacher? One of your parents? Another adult? How often did you fight? Have you ever tried or wanted to kill someone? NOTE: TAKE INTO ACCOUNT CULTURE, BACKGROUND, AND NEIGHBORHOOD. | O | () | () | 3 - Threshold: Reports at least one physical fight<br>involving an adult (e.g. teacher, parent) OR<br>reports starting frequent fights, with one or<br>more fights resulting in serious injury to a per<br>or frequent fights not resulting in injury (at lea |
| INQUIRE ABOUT BOTH OF THE FOLLOWING: | | | | 1-2 times per month). PAST: |
| Gang Involvement. Are you or any of your friends in a gang? The Crips? Bloods? Another gang? | | | | P C S |
| O Check here if evidence of gang involvement. | | | | |
| 2 - Homicidal Intent. Have you ever thought about wanting to kill someone | or a group | of | | |
| people? Do you have a gun or any other weapons? O Check here if evidence of homicidal intent. | | | | |
| Dulles Thomas on Law Marketon Office | <u>P</u> | <u>c</u> | <u>s</u> | 0 - No information. |
| Bulles, Inreatens or Intimidates Others | | | | |
| Bullies, Threatens, or Intimidates Others Do you ever try to bully kids or threaten kids to get them to do something | () | () | () | 1 - Not present. |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? | () | () | () | 2 - Subthreshold: Occasionally bullies, threatens, |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things: call names or make fun of other kids | () | () | () | Subthreshold: Occasionally bullies, threatens, intimidates. |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things: call names or make fun of other kids threaten to hurt other kids push trip | | | | 2 - Subthreshold: Occasionally bullies, threatens, |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things: call names or make fun of other kids threaten to hurt other kids push | () | () | () | Subthreshold: Occasionally bullies, threatens, intimidates. Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things: call names or make fun of other kids threaten to hurt other kids push trip come up from behind and slap or knock kids down knock items out of kids hands | () | () | () | 2 - Subthreshold: Occasionally bullies, threatens, intimidates. 3 - Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost daily, or at least several times per week. |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things:cell names or make fun of other kids _ threaten to hurt other kids _ push _ trip _ come up from behind and slap or knock kids down _ knock items out of kids hands _ make other kids do things for you | () | () | () | 2 - Subthreshold: Occasionally bullies, threatens, intimidates. 3 - Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost daily, or at least several times per week. PAST: |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things:cell names or make fun of other kids _ threaten to hurt other kids _ push _ trip _ come up from behind and slap or knock kids down _ knock items out of kids hands _ make other kids do things for you | () | () | () | 2 - Subthreshold: Occasionally bullies, threatens, intimidates. 3 - Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost daily, or at least several times per week. PAST: |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things:call names or make fun of other kidsthreaten to hurt other kidspushtripcome up from behind and stap or knock kids downknock items out of kids handsmake other kids do things for you | () | () | () | 2 - Subthreshold: Occasionally bullies, threatens, intimidates. 3 - Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost daily, or at least several times per week. PAST: |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things:call names or make fun of other kidsthreaten to hurt other kidspushtripcome up from behind and stap or knock kids downknock items out of kids handsmake other kids do things for you | () | () | () | 2 - Subthreshold: Occasionally bullies, threatens, intimidates. 3 - Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost daily, or at least several times per week. PAST: |
| Do you ever try to bully kids or threaten kids to get them to do something you want them to do? How often did you do these things:call names or make fun of other kidsthreaten to hurt other kidspushtripcome up from behind and stap or knock kids downknock items out of kids handsmake other kids do things for you | () | () | () | Subthreshold: Occasionally bullies, threatens, intimidates. Threshold: Bullies, threatens, or intimidates others on multiple occasions, daily, almost daily, or at least several times per week. PAST: |


| 2013 | KSADS-PL SCREE<br>Conduct Di | | RVI | EW: | |
|---|---|---|---|---|---|
| | | <u>P</u> | <u>c</u> | <u>s</u> | |
| 5. Nonaggressive Stealing | | () | () | () | 0 - No information. |
| In the past year, have you stolen anythin | | () | () | () | 1 - Not present. |
| What is the most expensive thing you sto<br>What other things have you stolen? From<br>Have you stolen a toy from a store? Mor | n whom? From which stores? | () | () | () | 2 - Subthreshold. Has stolen without confrontati<br>of victim on only one occasion. |
| How often have you stolen things? | N TOWAL VALUE (s. c. \$20.00 av | () | () | () | <ul> <li>Threshold: Has stolen without confrontation victim on 2 or more occasions.</li> </ul> |
| NOTE: ONLY COUNT THEFTS OF NO<br>more) . EXCEPTION: MULTIPLE THEF<br>TRIVIAL VALUE. | TS OUTSIDE THE HOME OF | | | | PAST: |
| | | | | | P C S |
| - IF RECEIVED A SCORE OF 3 ON<br>CONDUCT DISORDER (CURREN<br>DISORDERS SUPPLEMENT AFT | NT) SECTION IN THE NEURODE | EVELOP | MENT | AL, D | |
| CONDUCT DISORDER (CURREN<br>DISORDERS SUPPLEMENT AFT | NT) SECTION IN THE NEURODE<br>TER FINISHING THE SCREENIN<br>IN THE <u>PAST</u> RATINGS OF <u>ANY</u><br>IN THE NEURODEVELOPMENTA | OF THE | MENT<br>RVIEW | AL, D | SITEMS, COMPLETE THE CONDUCT |
| CONDUCT DISORDER (CURREN<br>DISORDERS SUPPLEMENT AFT<br>IF RECEIVED A SCORE OF 3 ON<br>DISORDERS (PAST) SECTION II | NT) SECTION IN THE NEURODE<br>TER FINISHING THE SCREENIN<br>IN THE <u>PAST</u> RATINGS OF <u>ANY</u><br>IN THE NEURODEVELOPMENTA<br>IN THE SCREENING INTERVIEW | OF THE | MENT<br>RVIEW | AL, D | SITEMS, COMPLETE THE CONDUCT |
| CONDUCT DISORDER (CURREN<br>DISORDERS SUPPLEMENT AFT<br>IF RECEIVED A SCORE OF 3 ON<br>DISORDERS (PAST) SECTION IN<br>SUPPLEMENT AFTER FINISHING | NT) SECTION IN THE NEURODE<br>TER FINISHING THE SCREENING THE SCREENING IN THE PAST RATINGS OF ANY IN THE NEURODEVELOPMENTAGE THE SCREENING INTERVIEW ISORDER. | EVELOPI<br>IG INTER<br>OF THE<br>AL, DISR<br>W. | PRE'S | AL, D | SITEMS, COMPLETE THE CONDUCT<br>ND CONDUCT DISORDERS |

| 2013 KSADS-PL SCREEN<br>Tic Disord | | RVI | EW: | |
|---|---|---|---|---|
| | P | <u>c</u> | <u>s</u> | |
| Motor Tics | () | () | 0 | 0 - No information. |
| Has there ever been a time when you noticed your muscles moved in a way | () | () | () | 1 - Not present. |
| that you did not want them to, or that you didn't expect?<br>Like raising your eyebrows (demonstrate), blinking a whole lot<br>(demonstrate), scrunching up your nose (demonstrate), shrugging your<br>shoulders (demonstrate), or moving your head like this (demonstrate)? | () | () | () | Subthreshold: Specific tic behaviors present<br>Tics have not persisted for a full year. |
| Ever blink a whole lot or real hard and not be able to stop? About how often did this happen? | () | () | () | Threshold: Specific tic behaviors are present The frequency may wax and wane, but tics |
| NOTE: RATE BASED ON REPORT AND OBSERVATION. | | | | have been present for at least a year. |
| Do not rate positively if due to compulsions of OCD or stereotypic movements of PDD. | | | | PAST: P C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| Phonic Ties | () | () | () | 0 - No information. |
| Has there ever been a time when you made noises that you didn't want to | () | () | () | 1 - Not present. |
| make, repeated sounds or words that you don't want to say?<br>Like sniffing, coughing, or clearing your throat when you didn't have a cold?<br>Making animal sounds or grunting sounds, or even repeating things that you<br>or other people said? | () | () | () | 2 - Subthreshold: Specific tic behaviors present<br>Tics have not persisted for a full year. |
| NOTE: RATE BASED ON REPORT AND OBSERVATION. | () | () | O | 3 - Threshold: Specific tic behaviors are present The frequency may wax and wane, but tics have been present for at least a year. PAST: P C S. |
| IF RECEIVED SCORE OF 3 ON <u>CURRENT</u> RATINGS OF MOTOR DISORDERS (CURRENT) SECTION IN THE NEURODEVELOPME DISORDERS SUPPLEMENT AFTER FINISHING THE SCREEN IN IF RECEIVED SCORE OF 3 ON <u>PAST</u> RATINGS OF MOTOR <u>OR</u> F | NTAL, I | DISRU<br>W. | JPTIVI | E, AND CONDUCT |
| (PAST) SECTION IN THE NEURODEVELOPMENTAL, DISRUPTIVE FINISHING THE SCREEN INTERVIEW. | | | | |
| NO EVIDENCE OF TIC DISORDER. | | | | |
| OTE: (RECORD DATES OF POSSIBLE CURRENT AND PAST TIC D | ISORDE | RS). | | |

## CONFIDENTIAL Version 9.0


2013



# KSADS-PL SCREEN INTERVIEW:

Autism Spectrum Disorders




Autism Spectrum Disorders are characterized by severe and pervasive impairment in several areas of development: reciprocal social interaction skills, communication skills, and the presence of stereotyped behavior, interests, and activities. The qualitative impairments that define these conditions are distinctly deviant relative to the individual's developmental level or mental age.

- These disorders are usually evident early in life. For each item below, remember to assess the duration of the symptom and whether it has been present
  by preschool or before. Also, for each item, please remember to synthesize your clinical observation of behavior observed during the interview into the
  Summary rating.
- Summary rating.

  2) If the child denies it, but parents report and/or you also observe symptom while interviewing the child, give more weight to parents and/or your observation than the child's report because s/he may not be aware of his/her problem.
- 3) For all symptoms below, take into account whether they are better accounted by other psychiatric disorder (mainly OCD, ADHD, psychosis, mental retardation, severe social anxiety), or medical or neurological conditions. Also, take into account the developmental stage of the child, normal behaviors and reproduces before or pedical, and the publical background of the family and the child.

| Oces your child have any unusual motor mannerisms like hand flapping, mead weaving, body rocking, or body spinning? What about a preoccupation with wiggling his/her fingers? Does your child repeat what you say? Parrot your speech or the speech of others? Repeatedly use idio syncratic phrases? Any other repetitive habits? Maybe an unusual or odd use of a toy or household object? Child: Do you like to watch your hands while you wiggle your fingers? Does rocking back and forth calm you when you are upset? Do people ever tell you to stay still and stop spinning? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND BEHAVIORAL OBSERVATION. |
|---|
| Lobes your child repeat what you say? Parrot your speech or the speech of others? Repeatedly use idiosyncratic phrases? Any other repetitive habits? Maybe an unusual or odd use of a toy or household object? Child: Do you like to watch your hands while you wiggle your fingers? Does rocking back and forth calm you when you are upset? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |
| What about a preoccupation with wiggling his/her fingers? Does your child repeat what you say? Parrot your speech or the speech of others? Repeatedly use idiosyncratic phrases? Any other repetitive habits? Maybe an unusual or odd use of a toy or household object? Child: Do you like to watch your hands while you wiggle your fingers? Does rocking back and forth calm you when you are upset? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |
| Does your child repeat what you say? Parrot your speech or the speech of others? Repeatedly use idiosyncratic phrases? Any other repetitive habits? Maybe an unusual or odd use of a toy or household object? Child: Do you like to watch your hands while you wiggle your fingers? Does rocking back and forth calm you when you are upset? Do people ever tell you to stay still and stop spinning? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |
| Any other repetitive habits? Maybe an unusual or odd use of a toy or household object? Child: Do you like to watch your hands while you wiggle your fingers? Does rocking back and forth calm you when you are upset? Do people ever tell you to stay still and stop spinning? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |
| Child: Do you like to watch your hands while you wiggle your fingers? Does rocking back and forth calm you when you are upset? Do people ever tell you to stay still and stop spinning? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |
| Does rocking back and forth calm you when you are upset? Do people ever tell you to stay still and stop spinning? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |
| Does rocking back and forth calm you when you are upset? Do people ever tell you to stay still and stop spinning? NOTE: RATE BASED ON PARENT AND CHILD REPORT AND |

This document is confidential. It contains proprietary information of Supernus® Pharmaceuticals, Inc. Any viewing or disclosure of such information that is not authorized in writing by the Sponsor is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.
| 2 Insistence on sameness, infloxible adherence to routines. Ritualized for patterns of verbal or nonverbal behavior Is you rehist rigid and unable to tolerate small changes in plans or routines that you would not expect to cause a problem (like driving to school a different way, point glown the goods) process plan askins a different router, on the positive process plan askins a different router, on the positive process plans askins a different router, on the positive process plans askins a different router. The process plans askins a different router, on the positive process plans askins a different router. The process plans askins a continue of the process plans askins a plan askins a ball to reject descend at a certain threat and is unable to do so for some particular reason, does your child outgrows his her clothes, the set of the read a delay in the state of soften way than usual. Child: Do you get ready upset when there is an unexpected change in your phase or the way you usually do things, like if there is a delay in the start of soften way than usual. Child: Do you get ready upset when there is an unexpected change in your phase or the way you usually do things, like if there is a delay in the start of soften and way than usual. Child: Do you get ready upset when there is an unexpected change in your phase or the way you usually do things, like if there is a delay in the start of soften and way than usual. Child: Do you get ready upset when there is an unexpected plan and the soften have a get interest that are altituded in the start of soften and ask and activities are pursued with great interest, and activities are pursu | 1 | 20 | KSADS-PL SCREEN Autism Spectrum | | | EW: | |
|---|---|---|---|---|---|---|---|
| 2. Insistence on sameness, inflexible adherence to routines. Ritualized () | | | | Р | C | S | |
| to your child rigid and unable to tolar ale small changes in plans or routines that you would not expect to cause a problem (like driving to school a development of the family count floar and the strength of the family count floar artificial of calling a print on the family count floar artificial of calling at the habble? Do you work keel hard to avoid changes in schedule as to not upset your child? Has he or she been that way since before knidergarden? For example, when your child outgrows his her cicties, does he resist wearing new clicities? Does your child hale changes in routine, like if he riche usually takes a bath or yet dressed at a certain time and is unable to do so for some particular reason, does your child get very upset? Child: Do you get really upset when there is an unexpected change in your plans or the way you usually do things, like if there is a deality in the start of school, if families is all the earlier than usual; or if you have to chive home a different way than usual? I highly restricted, fixated interests that are abnormal in intensity or focus Often these are primarily manifest in the development of encompassing precoupledors about a circumscribed topic or interest, about which the individue loan amass a great deal of facts and information. These interests and achities are pursued with greal intensity often to the exclusion of other children histories are primarily manifest in the development of encompassing precoupledors about a circumscribed topic or interest, about which the individue clause of the start of the shart precoupled or the start of facts that precouply finance has table? Parent: Does your child have interests that are not typical for other children children. Parent: Does your child have interests that are not typical for other children. Note: Rate This As Positive if it is in Appropriate for its that precoupled with one or more sterectyped and restricted patterns of interest that is shormatic albert in intensity or focus about it. Note: Rate This As Positi | | 2. [ | Insistence on sameness, inflexible adherence to routines, Ritualize | df | | | 0 No information |
| that you would not expect to cause a problem (the driving to school a different way, going down the grocery store asses in a different roler, or shawing a price, or the family come flow instead or easing at the table? Ob you work heal hard to avoid changes in schoolube as to not upset your bits as the cor she been that way since before kindergarten? For example, when your child outgrows his/her clothes, does he resist weaning new clothes? Does your child hate changes in schoolube as to not upset your passes. Child: Do you get really upset when there is an unexpected change in your plans or the way you usually do things, like if there is a delay in the stat of school if dinner is a little earlier than usual? Highly restricted, fixated interests that are abnormal in intensity or focus Offer these are primally manifest in the development of encompassing precoupled rose of the state of the exhibition and only a state of the state of the exhibition of the exhibitions and children and the procoupled or facts and informatic houses of the exhibition of the exhibitions and achildren are provided with greal intensity often to the exhibitions. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children his/her age, the an interest in ceiling fans or radiators? Has he or she memorated unusual facts like bus schedules, history facts, or other sorts of facts that procupy him or her daily? Does your child have one specific schily that her/she is focused on? Doe you think the/she is focused on? Does your child have one specific schily that her/she is focused on? Child: Is there a comething special you are interested in that you really like to that allow of the schilles. PAST: I have a comething special you are interested in that you really like to that allow of the schilles. Past: Does of the fact that proceduly the child of his/her age? Child: Is there a comething special you are interested in that you really like to that allow of the children and the children a | | 1 | patterns of verbal or nonverbal behavior | | -00 | | 3 15/00/2019 |
| different way, going down the grocery store asks in a different order, or having a pricinc on the family room floor instead of eating at the table? Do you work real hard to avoid change in schedule as to not upset your child? Has he or she been that way since before kindergarten? For example, when your child outgrows his his clidhes, does he resist wearing new clidhes? Does your child that changes in routine, like if the rish usually takes a bath or get dressed at a certain time and is unable to do so for some particular reason, does your child get very upset? Child: Do you get really upset when there is an inexpected change in your plans or the way you usually do things, like if there is a delay in the start of school, if dinner is a little earlier than usual, or if you have to drive home a different way than usual? A Highly restricted, fixated interests that are abnormal in intensity or focus Often these are primarily manifest in the development of encompassing precocupidicins about a circumscribed topic or interest, about which the individual can amiss a great deal of facts and information. These intensity and activities are purisued with greal intensity often to the exclusion of other activities. Rate tools and/or intensity. Parent. Does your child have intensests that are not typical for other children his/her egg, like an interest in challing from cradiators? Parent. Does your child have intensests that are not typical for other children his/her egg, like an interest in challing from cradiators? Parent. Does your child have intensests that are not typical for other children his/her egg, like an interest is too obsessed with craftan activities or interests beyond what you would expect for a child of his/her age? Child: Is there something special you are interested in that your really like to lask about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND Clittures of the child. And the crafts activities or interests beyond what you would expec | | | | | | | |
| Do you work real hard to avoid changes in schedule as to not upset your child? Has he or she been that way since before kindergaten? For example, when your child outgrows his her clothes, does he resist wearing new clothes? Does your child hale changes in routine, like if he Jeho usually takes a bath or get dressed at a certain time and is unable to do so for some particular reason, does your child get very upset? Child: Do you get really upset when there is an unexpected change in your plans or the way you usually do timps, like if there is a delay in the start of school, if direms is a like earlier than usual, or if you have to drive home a different way than usual? Step the search primarily manifest in the development of encompassing preoccupations about a circumscribed topic or interest, shoult which the individual can amass a great deal of facts and information. These interests and activities are pursued with great intensity often to the exclusion of other activities. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children his/her age, like an interect in ceiling fans or radiators? Parent: Does your child have interests that are not typical for other children his/her age, like an interect in ceiling fans or radiators? Parent: Does your child have interests that are not typical for other children his/her age, like an interect in ceiling fans or radiators? Child: It here something special you are witherested in that you really like to laik about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED, DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER CAMES HERE. Do not rate positively if behavior related to cither diagnosis such as OCD or a | | 9 | different way, going down the gracery store aisles in a different order, or | () | () | () | |
| ## C S ## Company of the search of the sear | | | Do you work real hard to avoid changes in schedule as to not upset your | () | () | () | |
| Does your child hate changes in routine, fike if he /she usually takes a bath or get dressed at a certain time and is unable to do so for some particular reason, does your child yet very upset? Child: Do you get really upset when there is an unexpected change in your plans or the way you usually do things, like if there is a delay in the state of school, if driner is a life earlier than usual, or if you have to drive home a different way than usual? PC S Highly restricted, fixated interests that are abnormal in intensity or focus Often these are primarily manifest in the development of encompassing precocupations about a circumscribed topic or interest, about which the individual can amass a great dead of facts and information. These interests and activities are pursued with great intensity often to the exclusion of other activities. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children his/her age, like an interest in celling fans or radiators? Has he or she memorize du musual facts like bus schedules, history facts, or other sorts of facts that preoccupy him or her daily? Child: Is there something special you are interested in that you really like to talk about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD. AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER CAMES. Do not rate positively if behavior related to other diagnosis such as OCD or a | | | | | | | distress when interrupted. Pattern of behavior |
| Does your child halte changes in routine, like if he /she usually takes a bath or get dressed at a certain time and is unable to do so for some particular reason, does your child get very upset? Child: Do you get really upset when there is an unexpected change in your plans or the way you usually do things, like if there is a delay in the start of school, if drimer is a like artier than usual, or if you have to drive home a different way than usual? P C S Highly restricted, fixated interests that are abnormal in intensity or focus Often these are primarily manifest in the development of encompassing preoccupations about a circumscribed topic or interest, about which the individual can amass a great deal of fatas an interest and activities are pursued with great intensity often to the exclusion of other activities. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children hisher age, like an interest in ceiling fans or radiators? Has he or she memorate durinsual facts like bus schedules, history facts, or other sorts of facts that preoccupy him or her daily? Does your child have expect for a child by that he/she is focused on? Do you think that he/she is 'too obsessed' with certain activities or interests beyond what you would expect for a child his three specific activity that he/she is focused on? Do you think that he/she is 'too obsessed' with certain activities or interests beyond what you would expect for a child his three specific activity that he/she is focused on? Do you think that he/she is 'too obsessed' with certain activities or interests beyond what you would expect for a child of hisher age? Child: Is there something special you are interested in that you really like to talk about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER. Do not rate positively if behavior related to other diagn | | | | | | | |
| Jelian or the way you usually do things, like if there is a delay in the start of school, if dimme is a little earlier than usual, or if you have to drive home a different way than usual? Highly restricted, fixated interests that are abnormal in intensity or focus | | - 3 | or get dressed at a certain time and is unable to do so for some particular | | | | |
| 3. Highly restricted, fixated interests that are abnormal in intensity or focus Often these are primarily manifest in the development of encompassing preoccupations about a circumscribed topic or interest, about which the individual can amass a great deal of facts and information. These interests and activities are pursued with great intensity often to the exclusion of other activities. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children his/her age, like an interest in ceiling fans or radiators? Has he or she memorized unusual facts like bus schedules, history facts, or other sorts of facts that preoccupy him or her daily? Does your child have one specific activity that he/she is focused on? Do you think that he/she is "too obsessed" with certain activities or interests beyond what you would expect for a child of his/her age? Child: Is there something special you are interested in that you really like to talk about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER GAMES HERE. Do not rate positively if behavior related to other diagnosis such as OCD or a | | 3 | plans or the way you usually do things, like if there is a delay in the start of<br>school, if dinner is a little earlier than usual, or if you have to drive home a | | | | |
| and activities are pursued with great intensity often to the exclusion of other activities. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children his/her age, like an interest in ceiling fans or radiators? Has he or she memorized unusual facts like bus schedules, history facts, or other sorts of facts that preoccupy him or her daily? Does your child have one specific activity that he/she is focused on? Do you think that he/she is "too obsessed" with certain activities or interests beyond what you would expect for a child of his/her age? Child: Is there something special you are interested in that you really like to talk about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER GAMES HERE. Do not rate positively if behavior related to other diagnosis such as OCD or a | 3 | | intensity or focus Often these are primarily manifest in the development of encompassing preoccupations about a circumscribed topic or interest, about which the | () | () | () | Not present. Subthreshold: Unusual preoccupations that do |
| other sorts of facts that preoccupy him or her daily? Does your child have one specific activity that he/she is focused on? Do you think that he/she is "too obsessed" with certain activities or interests beyond what you would expect for a child of his/her age? Child: Is there something special you are interested in that you really like to talk about, read about, or do? Tell me about it. NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER GAMES HERE. Do not rate positively if behavior related to other diagnosis such as OCD or a | | 3 0 00 | and activities are pursued with great intensity often to the exclusion of other activities. Rate focus and/or intensity. Parent: Does your child have interests that are not typical for other children his/her age, like an interest in ceiling fans or radiators? | O | () | () | Threshold: Definitely preoccupied with one or more stereotyped and restricted patterns of interest that is abnormal either in intensity or |
| NOTE: RATE THIS AS POSITIVE IF IT IS INAPPROPRIATE FOR THE AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER GAMES HERE. Do not rate positively if behavior related to other diagnosis such as OCD or a | | | other sorts of facts that preoccupy him or her daily? Does your child have one specific activity that he/she is focused on? Do you think that he/she is "too obsessed" with certain activities or interests | | | | functioning or limits participation in other activities. |
| AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER GAMES HERE. Do not rate positively if behavior related to other diagnosis such as OCD or a | | | | | | | PCS |
| | | | AGE AND CULTURE OF THE CHILD, AND IT IS EXAGGERATED. DO NOT SCORE PREOCCUPATION WITH VIDEOGAMES OR COMPUTER | | | | |
| | | | Subject | | | | Ø. 1 = |

| Autism Spectrum | N INTE | 2000 | EVV: | |
|---|---|---|---|---|
| | P | <u>c</u> | <u>s</u> | |
| Deficits in nonverbal communicative behaviors used for social interaction | () | () | () | 0 - No information. |
| Eye to Eye Gaze: Do you frequently have to remind your child to look at you | () | () | () | 1 - Not present. No problems in any of these area |
| or the person s/he is talking to? Facial Expressions: Does your child show the typical range of facial expressions? | () | () | () | Subthreshold; Subtle problems in one or more<br>area, which is evident to family members and |
| Can you see joy on his/her face when /she is happy? Does s/he pout when s/he is sad? | 4.0 | 4.0 | | professionals but not to teachers or classme |
| Does s/he show less common facial expressions like surprise, interest,<br>and guilt? Gestures: As a loddler or preschooler, did your child use common gestures | () | () | () | 3 - Threshold: Problems with one or more aspect<br>of non-verbal behaviors cause functional<br>impairment. |
| like pointing to show interest, clapping when happy, and nodding to<br>indicate 'yes'? | | | | PAST: |
| For school age children and adolescents: Does he /she use gestures to<br>help show how something works or while they are explaining something? | | | | P C S |
| Indicate problematic areas of non-verbal behavior: | | | | |
| O Gaze O Expressions O Gestures | | | | |
| IF RECEIVED A SCORE OF 3 ON <u>CURRENT</u> RATING OF <u>ANY</u> OF SPECTRUM DISORDERS (CURRENT) SECTION IN THE NEURO DISORDERS SUPPLEMENT AFTER FINISHING THE SCREEN IN | DEVELO | PME | | |
| SPECTRUM DISORDERS (CURRENT) SECTION IN THE NEURO | PREVI | OPME<br>W.<br>OUS I | NTAL, | DISRUPTIVE, AND CONDUCT GOMPLETE THE AUTISM |
| SPECTRUM DISORDERS (CURRENT) SECTION IN THE NEUROI DISORDERS SUPPLEMENT AFTER FINISHING THE SCREEN IN IF RECEIVED A SCORE OF 3 ON PAST RATING OF ANY OF THE SPECTRUM DISORDERS (PAST) SECTION IN THE NEURODEVE | PREVI | OPME<br>W.<br>OUS I | NTAL, | DISRUPTIVE, AND CONDUCT GOMPLETE THE AUTISM |
| SPECTRUM DISORDERS (CURRENT) SECTION IN THE NEUROI DISORDERS SUPPLEMENT AFTER FINISHING THE SCREEN IN IF RECEIVED A SCORE OF 3 ON PAST RATING OF ANY OF THE SPECTRUM DISORDERS (PAST) SECTION IN THE NEURODEVE DISORDERS SUPPLEMENT AFTER FINISHING THE SCREEN INTO | DEVELC<br>TERVIE<br>PREVI<br>LOPME<br>TERVIEV | OPME<br>W.<br>OUS I<br>NTAL<br>V. | TEMS | DISRUPTIVE, AND CONDUCT COMPLETE THE AUTISM RUPTIVE, AND CONDUCT |

| 2013 | EEN INTERVIEW<br>co Use | | | | | pag | e 40 | of 52 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Codes for the Following Items: 0 = N | No Information 1 = N | lo | 2 | = Yes | 5 | | | | | |
| | | F | arer | ıt | | Chile | 1 | Su | mma | ary |
| 1. Use | *************************************** | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| A. Ever smoked | | () | () | () | () | () | () | () | () | ( |
| B. Ever chewed tobacco | | () | () | () | () | () | () | () | () | ( |
| C. Ever smoked (or chewed) tobacco daily for 1 month or more | - | () | () | () | () | () | () | () | () | ( |
| DSM-5 DR# 21; Smoked? Parent Rating: Child Rating: IF EVER USED TOBACCO, COMPLETE QUESTIONS BELOW | v. | | | | | | | | | |
| IF NO EVIDENCE OF TOBACCO USE, GO TO ALCOHOL US | E SECTION ON THE | | LOW | 7 | | Chile | d | Su | mma | ary |
| 2. Quantity of Tobacco Use | | Г | T | | Г | T | | | T | |
| A. Current Use (cigarettes/day or "dips" of chew/day) | | L | 1 | | L | | | L | 1 | |
| B. Greatest amount of Use (cigarettes/day or "dips" of chew/day Age (years): | ) | | | | | | | | I | |
| 3. Have you ever smoked or "dipped" chew at least once a day for a month or more? | | 0 | 1 () | 2 | 0 | 1 | 2 | 0 () | 1 | 2 |
| (1 cigarette or 1 "dip" of chew a day or more for at least 30 days) | | | | | | | | | | |
| Age of first regular use (in months): | | L | | | | | | | | |
| | | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| 4. Ever attempt to quit | | () | () | () | () | () | () | () | () | ( |
| 5. Ever quit | | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| If yes, report longest number of months: | | Ī | | | ĺ | | | | | |
| Notes: | | | | | | | | | | |
| | | | | | | | | | | _ |

| 2013 | | | SCREEN INTER | VIEW: | | | | page | e 41 c | of 52 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Codes for Remaining Items: | 0 = No Information | 1 = No | 2 | = Yes | | | | | | |
| Probes: h<br>usually drir<br>drink than | low old were y<br>nk alone? Whe<br>others? Schoo | rith a brief (2-3 minute) semi-structur<br>rou when you had your first drink? What's you<br>ere do you usually drink? At home? Parties? A<br>Il dances or other parties?How old were you w<br>ne week in which you had at least two drinks? | ur favorite thing to drinkDo<br>friend's house? The stree<br>hen you started to drink reg | you have a gr<br>t? Bars? Are t | oup of<br>here s | friends<br>pecial t | you u | sually<br>then yo | drink v | more | likely t | 0 |
| DSM-5 DR | # 20: Alcoholic | Beverage: | | | | | | | | | | |
| Parent Rati | ing: | Child Rating: | | | | | | | | | | |
| | | | | 11.1 | arer | nt | 1 19 | Child | 1 | Su | mma | iry |
| 1. Use | | | | | | | | | | 1 | | |
| (6 | | ks in one week four or more times<br>uivalent to a 12oz bottle of beer, 5oz glass of<br>or) | wine, or 1.5oz shot of | 0 | () | () | () | () | () | () | 1 () | () |
| B. Ag | e above (at | first regular use - years) | | | I | | | 1 | | | 1 | |
| C. Cu | irrent freque | ncy of use (days per month) | | | I | | | Ī | | | 1 | ] |
| D. Ha | ave you ever | r had 3 or more drinks in a single day? | | 0 () | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| 2. Probler | ms related to | o alcohol | | 0 | 1 () | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| school | Mork? With yo | used you any problems at home? With your p<br>uur teachers? With your friends? With a job?<br>n in trouble while drinking? | arents? With your | 1,7 | () | ,, | ., | 1,7 | 3.2 | ., | 1.7 | ,, |
| 3. Receive | ed treatment | t for alcohol problems. | | 0 () | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| Notes: | | | | | | | | | | | | |
| | - T 12 | | | | | | | 7.1 | - | | | |
| PAGE | E. | SCORE OF <u>2</u> ON ANY OF THE PREVI | | | | | | | | NIWC | <u>IG</u> | |
| _ IF NO | EVIDENCE | OF CURRENT OR PAST ALCOHOL | USE, GO TO SUBSTA | ANCE USE | SECT | ON C | N PA | GE 4 | 3. | | | |
| | | | 1 | | | | | | | | | |

| 2013 KSADS-PL SCREEN Alcohol Use Di | | | _ vv . | |
|---|---|---|---|---|
| | P | <u>c</u> | <u>s</u> | |
| 1. Quantity | () | () | () | 0 - No information. |
| A. How many drinks do you usually have when you sit down to | () | () | () | 1 - 1 - 2 drinks. |
| drink? | () | () | () | 2 - 3 or more drinks. |
| | | | | PAST: P C S |
| | P | <u>c</u> | S | |
| B. What's the most you ever drank in a single day? When was that? | () | () | () | 0 - No information. |
| How about in the last six months? What's the most you drank in a day? | () | () | () | 1 - 1 - 2 drinks. |
| | () | () | () | 2 - 3 or more drinks. |
| | | | | PAST: P C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| 2. Frequency | () | () | () | 0 - No information. |
| What's the most number of days in a given week that you had something to | () | () | () | 1 - 1 - 2 days. |
| drink? Do you usually drink Friday and Saturday night? Midweek too? | () | () | () | PAST: C S |
| | P | <u>c</u> | <u>s</u> | |
| 3. Concern from Others about Drinking | () | () | () | 0 - No information. |
| Has anyone ever complained about your drinking? Friends? Parents? | () | () | () | 1 - No. |
| Teachers?<br>Have you ever been worried about it at all? | () | () | () | 2 - Yes. |
| | | | | PAST: P C S |
| — IF RECEIVED A SCORE OF 2 ON THE <u>CURRENT</u> RATINGS OF ∆ USE DISORDER (CURRENT) SECTION IN THE EATING DISORDE SUPPLEMENT AFTER COMPLETING THE SCREEN INTERVIEW. | ERS AN | | | |
| IF RECEIVED A SCORE OF 2 ON THE PAST RATINGS OF ANY OUSE DISORDER (PAST) SECTION IN THE EATING DISORDERS A SUPPLEMENT AFTER COMPLETING THE SCREEN INTERVIEW. | AND SU | | | |
| NO EVIDENCE OF ALCOHOL USE DISORDER. | | | | |
| NOTE: (RECORD DATE OF POSSIBLE CURRENT AND PAST ALCOH | OL USE | DISC | ORDE | RS). |

ON PAGE 46.

Subject

| 2013 KSADS-PL SCREE Substance | | VIEW: | | | | page | e 43 c | of 52 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Codes for Remaining Items: 0 = No | nformation | 1 = No | 2 | = Yes | 6 | | | | | |
| Prior to beginning this section, give the subject the list of drugs in about the confidential nature of the interview prior to beginning pr 1. Drug Use Let me know if you have used any of the drugs on this list before, | obes (if ap | propriate). | | | | | | | | |
| DSM-5 DR# 22: Marijuana, cocaine, etc: DSM-5 DR# 23: Use medications with | thout MD preso | cription: | | | | | | | | |
| Parent: Child: Parent: Child Rating: | | _ 1 | Parer | | | Child | | | mm:<br>Eve | |
| a. Cannabis<br><i>Marijuana, pot, hash, THC</i> | | 0 () | 1 | 2 | 0 | 1 | 2 | 0 | 1 () | 2 |
| b. Stimulants<br>Speed, uppers, amphetamines, dexedrine, diet pills, crystal meth | | () | () | () | () | () | () | () | () | ( |
| <ul> <li>c. Sedatives/Hypnotics/Anxiolytics Barbiturates (sedatives, downers), Benzodiazepine, quaalude (ludes), val<br/>xanax </li> </ul> | | () | () | () | () | () | () | () | () | () |
| d. Cocaine<br>Coke, crack | | () | () | () | () | () | () | () | () | () |
| e. Opioids<br>Heroin, morphine, codeine, methadone, demerol, percodan, oxycontin | | () | () | () | () | () | () | () | () | () |
| f. PCP<br>Angel dust | | () | () | () | () | () | () | () | () | ( ) |
| g. Hallucinogens Psychedelics, LSD, mescaline, peyote | | () | () | () | () | () | () | () | () | () |
| h. Solvents/Inhalants Glue, gasoline, chloroform, ether, paint | | () | () | () | () | () | () | () | () | () |
| i. Other Prescription drugs, nitrous oxide, ecstasy, MDA, etc. | | () | () | () | () | () | () | () | () | ( |
| Specify: | | | | | | | | | | |
| | 112222111 | | | | | | | | | |
| <ul> <li>j. Polysubstance<br/>(Assess for combined use of all listed substances)</li> </ul> | | () | () | () | () | () | () | () | () | ( |
| Notes: | | - 1 | | | | | | | | |

IF NO EVIDENCE OF CURRENT OR PAST SUBSTANCE USE, GO TO POST-TRAUMATIC STRESS DISORDER SECTION

| () ( | MSP 3 0 1 2 3 () | | Summary MSP 0 1 2 3 () |
|---|---|---|---|
| CE 2 3 0 1 2 () | MSP 3 0 1 2 3 () | CE 0 1 2 3 0 0 0 0 0 | () ( |
| | 0 0000 | | 000 |
| | 0 0000 | 00000 | () () () |
| 00000 | 0 0000 | 0000 | () () () |
| 00000 | | | ********* |
| | () () () () () | 0000 | () () () |
| 0000 | *** | | |
| | () () () () () | ()()()() | () () () |
| 0000 | () () () () () | () () () () | () () () |
| () () () () | () () () () | () () () () | ()()() |
| 0000 | 0 0000 | 0000 | 000 |
| 0000 | () () () () () | () () () () | () () () |
| | 000 | 00 0000 0000 | |

| | | Co | des for R | emainin | g I | tems: | 0 = No Ir | nformation | 1 = No | 2 = | Yes | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | F | arer | nt | - 3 | Child | | Su | mma | ary |
| | ems related t | | | | | 6000 | | 2 | 0 () | 1 | 2 | 0 | 1 | 2 | 0 () | 1 | 3 |
| | your use of<br>oolwork? With to | | | | | ? With you | ur parents? V | Vith your | | | | | | | | | |
| lotes: | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | n as | | | | | | |
| - IF | RECEIVED | ASCORE | OF 3 ON | THE CUI | RRENI | FREQU | JENCY ITE | M FOR AN | Y DRUG | CON | <b>IPLE</b> | re th | HE SU | BST | ANCE | | |
| | RECEIVED / | | | | | | | | | | | | | BST | ANCE | | |
| A | RECEIVED A | ENT) SEC | TION IN | THE EAT | TING D | ISORDE | | | | | | | | BST | ANCE | | |
| A | BUSE (CURR | ENT) SEC | TION IN | THE EAT | TING D | ISORDE | | | | | | | | BSTA | ANCE | | |
| SI | BUSE (CURR<br>JPPLEMENT | ENT) SEC<br>AFTER F | TION IN<br>INISHING | THE EAT | TING D | ISORDE<br>RVIEW. | RS AND S | UBSTANC | E-RELAT | ED D | ISOR | DERS | S | | | | |
| Al SI | BUSE (CURR | AFTER F | TION IN<br>INISHING<br>OF <u>3</u> ON | THE EAT | TING D<br>N INTE | RVIEW. | RS AND S | UBSTANC | E-RELAT | ED D | ISOR | DERS | S | | | | |
| - IF | BUSE (CURR<br>IPPLEMENT<br>RECEIVED | AFTER F | TION IN INITION IN INITION IN INITION IN INITION IN THE | THE EAT SCREE THE PAS EATING | TING D<br>IN INTE | RVIEW. | RS AND S | UBSTANC | E-RELAT | ED D | ISOR | DERS | S | | | | |
| - IF | BUSE (CURR<br>IPPLEMENT<br>RECEIVED A<br>BUSE (PAST | AFTER F | TION IN INITION IN INITION IN INITION IN INITION IN THE | THE EAT SCREE THE PAS EATING | TING D<br>IN INTE | RVIEW. | RS AND S | UBSTANC | E-RELAT | ED D | ISOR | DERS | S | | | | |
| Al<br>SU<br>IF<br>Al<br>SU | BUSE (CURR<br>IPPLEMENT<br>RECEIVED A<br>BUSE (PAST | AFTER F A SCORE SECTION AFTER F | TION IN<br>INISHING<br>OF 3 ON<br>I IN THE<br>INISHING | THE EAT<br>SCREE<br>THE PAS<br>EATING<br>SCREE | TING D<br>IN INTE<br>SI FRE<br>DISOR<br>IN INTE | EQUENC<br>ROLERS A<br>ROLERS A<br>ROLERS A | RS AND S | UBSTANC | E-RELAT | ED D | ISOR | DERS | S | | | | |
| Al<br>SU<br>IF<br>Al<br>SU | BUSE (CURR JPPLEMENT RECEIVED A BUSE (PAST JPPLEMENT | AFTER F A SCORE SECTION AFTER F | TION IN<br>INISHING<br>OF 3 ON<br>I IN THE<br>INISHING | THE EAT<br>SCREE<br>THE PAS<br>EATING<br>SCREE | TING D<br>IN INTE<br>SI FRE<br>DISOR<br>IN INTE | EQUENC<br>ROLERS A<br>ROLERS A<br>ROLERS A | RS AND S | UBSTANC | E-RELAT | ED D | ISOR | DERS | S | | | | |
| AI SI AI SI SI NO | BUSE (CURR IPPLEMENT RECEIVED / BUSE (PAST IPPLEMENT EVIDENCE | A SCORE SECTION AFTER F A SCORE SECTION AFTER F OF SUBS | TION IN<br>INISHING<br>OF 3 ON<br>I IN THE<br>INISHING<br>TANCE U | THE EAT<br>SCREE<br>THE PAS<br>EATING<br>SCREE<br>USE DISC | TING DEN INTE | EQUENC<br>RVIEW.<br>EQUENC<br>RDERS A<br>RVIEW. | RS AND S | UBSTANC<br>DR ANY DR<br>TANCE-RE | E-RELAT | ED D | ISOR | DERS | S | | | | |
| AI SI AI SI NO | BUSE (CURR JPPLEMENT RECEIVED A BUSE (PAST JPPLEMENT | A SCORE SECTION AFTER F A SCORE SECTION AFTER F OF SUBS | TION IN<br>INISHING<br>OF 3 ON<br>I IN THE<br>INISHING<br>TANCE U | THE EAT<br>SCREE<br>THE PAS<br>EATING<br>SCREE<br>USE DISC | TING DEN INTE | EQUENC<br>RVIEW.<br>EQUENC<br>RDERS A<br>RVIEW. | RS AND S | UBSTANC<br>DR ANY DR<br>TANCE-RE | E-RELAT | ED D | ISOR | DERS | S | | | | |

KSADS-PL SCREEN INTERVIEW: 2013  Post Traumatic Stress Disorder Codes for the Following Items: 0 = No Information 2 = Yes 1. Traumatic Events Probe:

I am going to ask you about a number of bad things that sometimes happen to children your age, and I want you to tell me if any of these things have ever happened, even if they only happened one time. have ever happened to you. Be sure to tell me if any of these things have ever happened, even if they only happened one time. Parent Child Summary Criteria Ever Ever A. Car Accident () Have you ever been in a bad car accident? Significant car accident in which child or other individual in car was injured and What happened? required medical intervention. Were you hurt? Was anyone else in the car hurt? B. Other Accident 2 0 () () () 0 0 0 0 0 0 Have you ever been in any other type of Significant accident in which child was bad accidents? injured and required medical intervention What about a biking accident? Other accidents? What happened? Were you hurt? C. Fire 1 2 0 1 2 0 () Were you ever in a serious fire? Child close witness to fire that caused significant property damage or moderate to Did your house or school ever catch on severe physical injuries. Did you ever start a fire that got out of control? What happened? Did anyone get hurt? Was there a lot of damage? D. Witness of a Disaster 2 0 2 0 () Child witness to natural disaster that Have you ever been in a really bad storm, like a tornado or a hurricane? caused significant devastation. Have you ever been caught in floods with waters that were deep enough to swim in? Subject

KSADS-PL SCREEN INTERVIEW: 2013  Post Traumatic Stress Disorder Codes for the Following Items: 0 = No Information 2 = Yes 1. Traumatic Events (cont') Probe:

I am going to ask you about a number of bad things that sometimes happen to children your age, and I want you to tell me if any of these things have ever happened even if they only happened one time. have ever happened to you. Be sure to tell me if any of these things have ever happened, even if they only happened one time Parent Child Summary Criteria Ever Ever E. Witness of a Violent Crime 0 () Did you ever see someone rob someone or Child close witness to threatening or violent shoot them? crime. Steal from a store or jump someone? Take someone hostage? What happened? Where were you when this happened? Was anyone hurt? F. Victim of Violent Crime 2 0 2 0 1 1 0 2 () Child victim of seriously threatening or Did anyone ever mug you or attack you in some other way? What happened? violent crime. Were you hurt? G. Confronted with Traumatic News () Learned about sudden, unexpected death Have you ever gotten some really bad news unexpectedly? Like found out of a loved one, or that loved one has life-threatening disease. someone you loved just died or was sick and would never get better? H. Terrorism Related Trauma 2 1 2 0 1 0 () Were you affected by the events of Boston Loved one missing for extended period of Marathon bombing or any other terrorist time or seriously injured or killed by terrorist attack? attack. Subject

| Codes for the Folia Traumatic Events (cont') Obe: I am going to ask you about a number of bad things ever happened to you. Be sure to tell me if any of the | owing Items: 0 = No Information | 1 = No | 2 | = Yes | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| obe:<br>I am going to ask you about a number of bad things | | | | - 9.55 | | | | | |
| I am going to ask you about a number of bad things | | | | | | | | | |
| | | | | | | y of th | ese th | nings h | ave |
| | Criteria | , | Paren<br>Ever | | | Child<br>Ever | | | mm:<br>Ever |
| I, War Zone Trauma Have you ever lived in a war zone? | Lived in war zone. Witnessed death a | 0<br>() | 1 | 2 | 0 | 1 () | 2 | 0 () | 1 |
| Had your home attacked? Witnessed the killing or rape of others? Seen everything around you set on fire? | mass destruction. | | | | | | | | |
| Protective Services: Has your family ever re | eceived services from CYS/DCF? C | O Curren | t | O P | astt | | | | |
| J. Witness to Domestic Violence | | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 |
| Some kids' parents have a lot of nasty fights. They call each other bad names, throw things, threaten to do bad things to each other, or sometimes really hurt each | Child witness to explosive argument involving threatened or actual harm to parent. | | () | () | () | () | () | () | () |
| other. Did your parents (or does your mother and her boyfriend) ever get in really bad fights? Tell me about the worst fight you remember your parents having. What happened? | | | | | | | | | |
| K. Physical Abuse | | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 |
| When your parents got mad at you, did<br>they hit you?<br>Have you ever been hit so that you had<br>bruises or marks on your body, or were<br>hurt in some way? What happened? | Bruises sustained on more than one occasion, or more serious injury sustain | е | () | () | () | () | O | () | () |


| 2013 | | ADS-PL SCF<br>Post Traumati | c Stress | Disor | der | 250 | | | | page | 9 49 | of 52 | 2 | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 77-11-7-11-1-1 | Codes for the Follo | wing Items: 0 = | No Inforn | nation | 1= | No | 2 | = Yes | | | | | | |
| . Traumatic Events (con | nt') | | | | | | | | | | | | | |
| Probe:<br>I am going to ask you ab | oout a number of bad things t | hat sometimes hann | en to childre | n vour s | ige an | d I want | vou te | tell m | e if ar | v of th | ese th | inas I | nave | |
| | Be sure to tell me if any of the | | | | | y happe | ned o | ne time | 9. | | | | | |
| | | | Criteria | | | 1 | Ever | | | Child | | S | Ever | - |
| L. Sexual Abuse | | | | | | () | () | () | 0 | 1 | () | () | () | ( |
| parts when they sh<br>happened?<br>Has someone ever<br>that made you feel<br>Has anyone who si<br>you undress, touch<br>make you get in be<br>you play with his pr | houldn't have ever made<br>n you between the legs,<br>nd with him/her, or make | Isolated or rep<br>fondling, ora<br>i | | | | Lesso | | | | | | | | |
| that was really bad, | lse that happened to you<br>or something else you | Record incident | below. | | | 0 () | 1 () | 2 () | 0 () | 1 () | 2 () | 0 () | 1 () | |
| saw that was really<br>tell me about? | scary, that you want to | | Hi | | | | | - | 1 | | | | T | - |
| neglect known or<br>ever been a time<br>went on a drug bin<br>siblings alone for a<br>you worried they | stance abuse and/or<br>suspected: Has there<br>when your mom or dad<br>ge and left you and your<br>a day or longer? Were<br>wouldn't come home or<br>d happened to them? | Incident | | | | | | | | | | | | |
| QUESTIONS ON THE | AST TRAUMA (A SCORI<br>E FOLLOWING PAGE.<br>F PAST TRAUMA, END<br>APPROPRIATE SUPPLE | THE SCREENING | | | | | | | | | | | | |

| | | | Pos | t Tra | uma | tic S | tress | Dis | orde | r | | | | page | 50 c | of 52 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Codes for the | Follo | wing | Iten | ns: ( | ) = N | o Info | rmatio | on | 1 = 1 | lo | 2 : | Yes | | | | | | |
| NOTE: If more than one traumatic event was e | ndors | ed, in | quire : | about | symp | tom p | resend | e in n | elatio | n to A | NY of | the tra | aumas | | | | | |
| NOTE: IN DISCUSSING TRAUMATIC EVENTS you think about when he stuck his pee-pee up | | | | | IMPO | RTAN | тто | USE T | HEIR | LANC | SUAG | E IN Y | OUR I | DIALC | GUE. | (e.g. l | Oo. | |
| | 1 | Parer | nt | | aren<br>MSP | | | Child | | | Child<br>MSP | | Su | m ma | iry | | mma<br>MSP | |
| Recurrent Memories, Thoughts, or Images | 0 | 1 () | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| Has there ever been a time when you kept seeing again and again? How often did this happen? Did what happen keep coming into your mind? Did you think about it a lot? | 6226 | | ==== | L | ,,,,,, | | L ===== | | , - b - s | | | | | | | | | |
| 2. Feelings of Detachment | 0 | 1 | 2 | 0 | 1 () | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| Is it hard for you to trust other people? Do you feel like being alone more often than before? Like you just don't feel like being around people now that you used to like being around before? Do you feel alone even when you are with other people? | | | | | | | | | | | | | | | | | | |
| 3. Efforts to Avoid Activities or Situations<br>that Remind you of the Trauma | 0 () | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 () | 0 | 1 () | 2 | 0 | 1 () | 2 |
| Are there places or thigs that remind you of? Do you try to avoid them? You said before that sometimes reminds you of what happened. Dio you try to avoid? | L | | | L | | | | | | | | | | | | de e e e | | |
| 4. Nightmares | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| | 10 | () | | () | () | () | () | () | () | () | () | () | () | () | | () | () | C |
| Has there ever been a time when you had a lot of nightmares? Did you ever dream about? How often? Do you have other scary dreams? | | | | | | | | | | | | | | | | | | |

| | | KSADS-PL SCREEN INTERVIEW: | 2042 | |
|----|---------------|----------------------------|------|------|
| 52 | | Past Traumatic Events | | 2013 |
| | page 51 of | Past Traumatic Events | | |

| Codes for the | e Following | Items: | 0 = No | Infor | matic | n 1 | = N | 0 | 2 : | Yes | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Paren<br>CE | t | Parent | | | Child<br>CE | 1 | | Child<br>MSP | | Su | mma<br>CE | iry | | mma<br>MSP | гу |
| 5. Hypervigilance Since happened, are you more careful? Do you feel like you always have to watch what's going on around you? Do you double check the doors or windows to make sure they are locked? | 0 1 | 750 | <b>0 1</b> | <b>2</b><br>() | <b>0</b> () | 1 () | 2 | 0 () | <b>1</b> () | <b>2</b> () | <b>0</b> () | 1 () | <b>2</b> () | 0 () | 1 () | ( |
| IF RECEIVED A SCORE OF 2 ON <u>CU</u><br>- AND PAST POST-TRAUMATIC STRE | | | | | | | | | | | | | | | | |

- NO EVIDENCE OF POST-TRAUMATIC STRESS DISORDER .

NOTE: (RECORD DATES OF POSSIBLE CURRENT AND PAST POST-TRAUMATIC STRESS DISORDER).

| T. | 1 1 1 | |
|---------|-------|-----|
| Subject | | 170 |

2013



#### KSADS-PL SCREEN INTERVIEW: Supplement Completion Checklist




**DIRECTIONS:** Check the sections to be completed in each supplement. Note dates and/or ages of onset for each current and past possible disorder.

| Supplement #1: Depressive and Bipolar Related Disorders | Supplement #4: Neuro developmental, Disruptive, and Conduct Disorders |
|---|---|
| Depressive Disorders - Current | |
| Depressive Disorders - Past | ADHD - Current |
| Mania - Current | ADHD - Past |
| Mania - Past | Oppositional Disorder - Current |
| Disruptive Mood Dysregulation Disorder - Current | |
| Disruptive Mood Dysregulation Disorder - Past | Conduct Disorder - Current |
| | Conduct Disorder – Past |
| | Tic Disorders - Current |
| Supplement #2: Schizophrenia Spectrum and Other | Tic Disorders – Past |
| Psychotic Disorders | Autism Spectrum Disorders - Current |
| 22.7 Many Procession | Autism Spectrum Disorders - Past |
| Psychosis - Current | |
| Psychosis - Past | |
| Supplement #3: Anxiety, Obsessive Compulsive, and Trauma-Related Disorders | Supplement #5: Eating Disorders and Substance-Related Disorders |
| | Eating Disorders - Current |
| Panic Disorders - Current | Eating Disorders - Past |
| Panic Disorders - Past | Alcohol Use Disorder - Current |
| Agoraphobia - Current | Alcohol Use Disorder - Past |
| Agoraphobia - Past | Substance Use Disorders - Current |
| Separation Disorders - Current | Substance Use Disorders - Past |
| Separation Disorders – Past | dubalance dae biadiuera - 1 dat |
| Social Anxiety/Selective Mulism - Current | |
| Social Anxiety/Selective Mutism – Past | |
| Specific Phobias - Current | |
| Spedfic Phoblas - Past | |
| Generalized Disorders - Current | |
| Generalized Disorders - Past | |
| Obsessive Compulsive Disorder -Current | |
| Obsessive Compulsive Disorder - Past | |
| Posttraumatic Stress Disorder - Current | |
| Posttraumatic Stress Disorder - Past | |

### **KSADS-PL 2013:**

### SUPPLEMENT # 4: NEURODEVELOPMENTAL, DISRUPTIVE, AND CONDUCT DISORDERS SUPPLEMENT

| TABLE OF CONTENTS |
|------------------------------------------|
| Attention Deficit Hyperactivity Disorder |
| Oppositional Defiant Disorder 8 |
| Conduct Disorder |
| Tic Disorders |
| Autism Spectrum Disorders 23 |

| Subject | 44114 | | 17-167 |
|---------|-------|-------------|--------|
| Date / | 20 | Interviewer | |

Subject

Neurodevelopmental, Disruptive, and Conduct Disorders Supplement 2013 Attention Deficit Hyperactivity Disorder  (If child is on medication for ADHD, rate behavior when not on medication) NOTE: DO NOT RATE SYMPTOMS POSITIVELY IF THEY ARE EXCLUSIVELY ACCOUNTED FOR BY MDE. BIPOLAR DISORDER, DYSTHYMIA, AN ANXIETY DISORDER, SUBSTANCE ABUSE, PSYCHOSIS, OR ASD. P C S 1. Makes a lot of Careless Mistakes () () 0 - No Information () () () Do you make a lot of careless mistakes at school? 1 - Not Present Do you often get problems wrong on tests because you didn't read the () () () 2 - Subthreshold: Occasionally makes careless instructions right? mistakes. Problem has only minimal effect on Do you often leave some questions blank by accident? functioning Forget to do the problems on both sides of a handout? How often do these types of things happen? () () () 3 - Threshold: Often (4-7 days/week) makes Has your teacher ever said you should pay more attention to detail? careless mistakes. Problem has significant effect on functioning. PAST: C P C S 2. Doesn't Listen () () () 0 - No Information. () () () 1 - Not Present is it hard for you to remember what your parents and teachers say? Do your parents or teachers complain that you don't listen to them when () () 2 - Subthreshold: Occasionally doesn't listen. they talk to you? Problem has only minimal effect on Do you "tune people out"? functioning. Do you get into trouble for not listening? 3 - Threshold: Often (4-7 days/week) doesn't listen. () () Rate based on data reported by informant or observational data. Problem has significant effect on functioning. PAST. S 3 P C 3. Difficulty Following Instructions () () () 0 - No Information () () () 1 - Not Present Do your teachers complain that you don't follow instructions? When your parents or your teacher tell you to do something, is it sometimes () () 2 - Subthreshold: Occasionally has difficulty hard to remember what they said to do? following instructions. Problem has only Does it get you into trouble? minimal effect on functioning Do you lose points on your assigments for not following directions or not completing the work? () () 3 - Threshold: Often (4-7 days/week) has difficulty Do you forget to do your homework or forget to turn it in? following instructions. Problem has significant Do you get in to trouble at home for not finishing your chores or other things effect on functioning. your parents ask you to do? How often? PAST: S

| Attention Deficit Hypera | activity | Disc | order | |
|---|---|---|---|---|
| | | 12 | 2 | |
| Call to the control of the call to the cal | P | <u>C</u> | <u>s</u> | |
| 4. Difficulty Organizing Tasks | () | () | () | 0 - No Information. |
| is your desk or locker at school a mess? | () | () | () | 1 - Not Present |
| Does it make it hard for you to find the things you need? Does your teacher complain that your assignments are messy or disorganized? | | () | () | <ol> <li>Subthreshold: Occasionally disorganized.</li> <li>Problem has only minimal effect on functionin</li> </ol> |
| When you do your worksheets, do you usually start at the beginning and do<br>all the problems in order, or do you like to skip around?<br>Do you often miss problems? | () | () | () | 3 - Threshold: Often (4-7 days/week) disorganized<br>Problem has significant effect on functioning. |
| Do you have a hard time getting ready for school in the morning? | | | | PAST: C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| 5. Dislikes/Avoids Tasks Requiring Attention | () | () | () | 0 - No Information. |
| Do you hate or dislike doing things that require a lot of concentration/effort? | () | () | () | 1 - Not Present. |
| Like certain assignments, homework or reading a book? Are there some kinds of school work you hate doing more than others? Which ones? Why? Do you try to get out of doing your assignments? About how many times a week do you not do your homework? | () | () | () | <ul> <li>Subthreshold: Occasionally avoids tasks that<br/>require sustained attention, and/or expresses<br/>mild dislike for these tasks. Problem has only<br/>minimal effect on functioning.</li> </ul> |
| NOTE: IN CHILDREN/TEENS WITH ADHD, ABILITY TO SUSTAIN<br>ATTENTION TO VERY REWARDING ACTIVITES LIKE COMPUTER OR<br>VIDEO GAMES MAY NOT BE IMPAIRED. | () | () | () | 3 - Threshold: Often (4-7 days/week) avoids tasks<br>that require sustained attention, and/or<br>expresses moderate dislike for these tasks.<br>Problem has significant effect on functioning. |
| | | | | PAST: P C S |
| 6. Loses Things | <u>P</u> | <u>C</u> | <u>S</u> | Martin Maria Sancia |
| D. Loses Hings | () | () | () | 0 - No Information. |
| Do you lose things a lot? Your pencils at school? Homework assignments?<br>Things around home?<br>About how often does this happen? | () | () | () | Not Present. Subthreshold: Occasionally loses things. Problem has only minimal effect on functionin. |
| | () | () | () | 3 - Threshold: Often loses things (e.g. once a wee<br>or more). Problem has significant effect on<br>functioning. |
| | | | | PAST: P C S |
| Subject Subject | | | | |

| | activity | Dis | order | |
|---|---|---|---|---|
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| . Forgetful in Daily Activities | () | () | () | 0 - No Information. |
| Do you often leave your homework at home, or your books or coats on the | () | () | () | 1 - Not Present. |
| bus? Do you leave your things outside by accident? How often do these things happen? | () | () | () | Subthreshold: Occasionally forgetful. Problem<br>has only minimal effect on functioning. |
| Has anyone ever complained that you are too forgetful? | () | () | () | 3 - Threshold: Often (4-7 days/week) forgetful.<br>Problem has significant effect on functioning |
| | | | | PAST: P C S |
| works to | P | C | S | |
| Fidgets | () | () | () | 0 - No Information. |
| Consider restlessness, tapping fingers, chewing things, squirming, "ants in pants", etc. | () | () | () | 1 - Not Present. |
| Do people often tell you to sit still, to stop moving, or stop squirming in your | () | () | () | 2 - Subthreshold: Occasionally fidgets with hand |
| seat? Your teachers? Parents?<br>Do you sometimes get into trouble for squirming in your seat or playing with | | | 3// | or feet or squirms in seat. Problem has only minimal effect on functioning. |
| little things at your desk? Do you have a hard time keeping your arms and legs still? How often? For parents about children: When you take your child to church or to a | () | () | () | 3 - Threshold: Often (4-7 days/week) fidgets with<br>hands or feet or squirms in seat. Problem h<br>significant effect on functioning. |
| restaurant, do you have to bring a lot of games or loys? About adolescents: When your child was younger, were you able to take him/her to church? Restaurants? Were these difficulties beyond what you would expect for a child his/her age? | | | | PAST: P C S |
| Take into account that these symptoms tend to improve with age. Careful NOTE: RATE BASED ON DATA REPORTED BY INFORMANT OR OBSERVA | | | | tom was present when the child was younger. |
| Pour as Clinks Successively | <u>P</u> | <u>c</u> | <u>s</u> | |
| Runs or Climbs Excessively | <u>P</u> | () | () | 0 - No information |
| Do you get into trouble for running down the hall in school? | 0 | () | () | 1 - Not Present. |
| | - | () | () | |
| Do you get into trouble for running down the hall in school? Does your mom often have to remind you to walk instead of run when you are out together? Do your parents or your teacher complain about you climbing things you shouldn't? What kinds of things? How often does this happen? Adolescents: Do you feel restless a lot? Feel like you have to move around, or that it is very hard to stay in one place? | 0 | () | () | Not Present. Subthreshold: Occasionally runs about or climbs excessively. Problem has only minim effect on functioning. (In addescents, may limited to a subjective feeling of restlessnes. Threshold: Often (4-7 days/week) runs about climbs excessively. Problem has significant effect on functioning. (In addescents, may |
| Do you get into trouble for running down the hall in school? Does your mom often have to remind you to walk instead of run when you are out together? Do your parents or your teacher complain about you climbing things you shouldn't? What kinds of things? How often does this happen? Adolescents: Do you feel restless a lot? Feel like you have to move | 0 | () | () | Not Present. Subthreshdd: Occasionally runs about or climbs excessively. Problem has only minim effect on functioning. (In adolescents, may |

| Attention Deficit Hypera | activity | Disc | order | |
|---|---|---|---|---|
| | P | C | 5 | |
| 0. On the Go/Acts like Driven by Motor | () | () | () | 0 - No Information. |
| Do people tell you that your motor is always running? | () | () | () | 1 - Not Present. |
| Is it hard for you to slow down?<br>Can you stay in one place for long, or are you always on the go?<br>How long can you sit and watch TV or play a game? | () | () | () | <ol><li>Subthreshold: Occasionally, minimal effect on<br/>functioning.</li></ol> |
| Do people tell you to slow down a lot? | () | () | () | <ul> <li>Threshold: Often (4-7 days/week) acts as if<br/>"driven by a motor," Significant effect on<br/>functioning.</li> </ul> |
| | | | | PAST: P C S |
| | P | C | S | |
| 1. Difficulty Playing Quietly | () | () | () | 0 - No Information. |
| Do your parents or teachers often tell you to quiet down when you are | () | () | () | 1 - Not Present. |
| playing?<br>Do you have a hard time playing quietly? | () | () | () | <ul> <li>Subthreshold: Occasionally has difficulty<br/>playing quietly. Problem has only minimal effe<br/>on functioning.</li> </ul> |
| | () | () | () | <ul> <li>Threshold: Often (4-7 days/week) has difficulty<br/>playing quietly. Problem has significant effect<br/>on functioning.</li> </ul> |
| | | | | PAST: P C S |
| | <u>P</u> | C | <u>s</u> | |
| 2. Blurts Out Answers | () | () | () | 0 - No Information. |
| At school, do you sometimes call out the answers before you are called on? | () | () | () | 1 - Not Present. |
| Do you talk out of turn at home? Answer questions your parents ask your siblings? How often? | () | () | () | <ul> <li>2 - Subthreshold: Occasionally talks out of turn.</li> <li>Problem has only minimal effect on functionin</li> </ul> |
| | () | () | () | <ul> <li>Threshold: Often (4-7 days/week) talks out of<br/>turn. Problem has significant effect on<br/>functioning.</li> </ul> |
| | | | | PAST: |
| | P | C | <u>s</u> | |
| 3. Difficulty Waiting Turn | () | () | () | 0 - No Information. |
| Is it hard for you to wait your turn in games? | () | () | () | 1 - Not Present. |
| What about in line in the cafeteria or at the water fountain? | () | () | () | Subthreshold: Occasionally has difficulty<br>waiting his/her turn. Problem has only minima<br>effect on functioning. |
| | () | () | () | <ul> <li>Threshold: Often (4-7 days/week) has difficulty<br/>waiting his/her turn. Problem has significant<br/>effect on functioning.</li> </ul> |
| | | | | PAST: |

| | Attention [ | Deficit H | lype | ractivit | y Dis | order | _ | | page 5 | of 27 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | P | C | S | | | | |
| 4. Interrupts or Intrudes | | | | () | () | () | 0 - No | Information. | | |
| Do you get into trouble for talking out of turn a | | | | () | () | () | 1 - No | t Present. | | |
| Do your parents, teachers, or any of the kids you know complain<br>cut them off when they are talking?<br>Do kids complain that you break in on games? Does this happer | | | 1 | () | () | () | 2 - Su | bthreshold: C | ccasionally inte | rupts others. |
| | | | | () | () | () | 3 - Th | reshold: Offer | n (4-7 days/wee | k) interrunts |
| Rate based on data reported by informant observational data. | (parent/teacher) | or | | | | 0.7 | | hers. | ir ( r r days/irec | n, menapia |
| ovativational data. | | | | | | | PAST | | | |
| | | | | | _ | 2 | | P | c s | |
| | | | | P | C | <u>s</u> | | | | |
| 5. Talks Excessively | | | | () | () | () | | Information. | | |
| Do people say you talk too much? | | | | () | () | () | | t Present. | | |
| Do you get into trouble at school for talking wh<br>Do people in your family complain that you tall | too much? | upposed t | 07 | () | () | () | 2 - Su | bthreshold: C | ccasionally talk | s excessively. |
| What about humming or always making noise | | | | () | () | () | 3 - Th | reshold: Ofte | n talks excessiv | ely. |
| Do not rate vocal tics positively. | | | | | | | PAST | : 🖂 | | |
| Rate based on data reported by informant | (including pare | nt/teacher | r) or | | | | | | $\sqcup \sqcup$ | |
| observational data. | | | | | | | | Р | c s | |
| Codes for | Remaining Ite | ms: 0 | = No | | - | 1 = No | - | 2 = Yes | | |
| | Criteria | Pare | | Parer | | Chi | | Child<br>MSP | Summary | Summai |
| 3. Duration | 6 months<br>or more | 0 1 | 3.5 | 0 1 | 2 | 0 1 | 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| For how long have you had trouble (list symptoms that were positively endorsed)? | o, maio | | | L | | | 22.1. | | Jarrana | 1 |
| 7. Age of onset | Some | 0 1 | 2 | 0 1 | 2 | 0 1 | 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| low old were you when you started to have | symptoms | () () | () | ()() | () | () ( | () | ()()() | ()()() | ()()( |
| hese problems?<br>Did you have these problems in kindergarten? | present<br>before | | | | | | | | | |
| First Grade? Middle school? | age 12. | | | | | | | | | |
| ipecity. | | | | | | | | | | |
| 3. Impairment (Must be present in two settings) | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | 0 1 | 2 | 0 1 | 2 | 0 1 | 2 | 0 1 2 | 0 1 2 | 0 1 |
| A. Socially (with peers): | | ()() | () | ()() | () | ()( | () | ()()() | ()()() | ()()( |
| 7. Socially (Man poorey. | | | | | | | | | | |
| B. With family: | | 0 1 | 2 | 0 1 | 2 | 0 1 | 2 | 0 1 2 | 0 1 2 | 0 1 |
| | | () () | | () () | | () ( | | () () () | 000 | ()() |
| | | | | · | | | | | | |
| | | 0 1 | 2 | 0 1 | 2 | 0 1 | | 0 1 2 | 0 1 2 | 0 1 : |
| C. In school: | | ()() | 11 | ()() | 1.5 | () ( | 1.1 | ()()() | ()()() | ()()( |

Neurodevelopmental, Disruptive, and Conduct Disorders Supplement 2013 Attention Deficit Hyperactivity Disorder  Codes for Remaining Items: 0 = No Information Summary Summary CE MSP 19. DSM-5 Criteria; Evidence of ADHD 0 1 2 0 1 2 ()()() ()()() A. A persistent pattern of inattention and/or hyperactivity-impulsivity that interferes with functioning or development, as characterized by (1) and/or (2): I. Inattention: Six (or more) of the following symptoms have persisted for at least 6 months to a degree that is inconsistent with developmental level and that negatively impacts directly on social and academic/occupational activities a. Makes a lot of Careless Mistakes b. Difficulty Sustaining Attention on Tasks or Play Activities c. Doesn't Listen d. Difficulty Following Instructions e. Difficulty Organizing Tasks f. Dislikes/Avoids Tasks Requiring Attention g. Loses Things h. Easily Distracted Forgetful in Daily Activities 2. <u>Hyperactivity / Impulsivity</u>: <u>Six</u> or more of the following nine symptoms have persisted for at least <u>6 months</u>:

NOTE: For older adolescents and adults (age 17 and older), only <u>five</u> symptoms are required a. Fidgets b. Difficulty Remaining Seated c. Runs or Climbs Excessively d. Difficulty Playing Quietly e. On the Go/Acts as if Driven by a Motor f. Talks Excessively g. Blurts Out Answers h. Difficulty Waiting Turn i. Often Interrupts or Intrudes B. Some symptoms that caused impairment present before the age of 12; C. Several symptoms must be present in two or more situations (e.g. school and home); D. Clinically significant impairment; E. Symptoms do not occur exclusively during the course of psychotic disorder and not better accounted for by another mental disorder (e.g., mood disorder, anxiety disorder, dissociation, personality disorder). NOTE: Autism Spectrum Disorder is no longer a rule out for the diagnosis of ADHD. 0 1 2 0 1 2 20. Predominantly Inattentive Presentation ()()() ()()() Meets criterion A (I), but not criterion A (II) for past six months. 0 1 2 0 1 2 21. Predominantly Hyperactive-Impulsive Type ()()() ()()() Meets criterion A (II), but not criterion A (I) for past six months. Subject


| | Codes for Remaining Items: 0 = No Information 1 = No 2 = Yes | Summary | Summa |
|---|---|---|---|
| 2. Combined Ty Both criteria A (I | <u>pe</u><br>) and A (II) are met for past six months. | 0 1 2 | 0 1 |
| | d Attention Deficit Hyperactivity Disorder toms of inattention or hyperactivity-impulsivity that do not meet criteria for Attention Deficit sorder. | 0 1 2 | 0 1 2 |



| Oppositional Defi | ant Dis | orde | | |
|---|---|---|---|---|
| NOTE: A CHILD CANNOT MEET DSM-5 CRITERIA FOR ODD IF THEY DMDD. THIS SUPPLEMENT DOES NOT NEED TO BE COMPLETED, BU | | | | |
| When assessing for ODD, keep in mind that the essential feature of this disobedient, and hostile behavior toward authority figures that persists for a observed in individuals of comparable age and developmental level. If ODI | at least 6 | mont | hs and | occurs more frequently than is typically |
| parent-child relationshp diagnosis. | P | <u>c</u> | <u>s</u> | |
| 1. Easily Annoyed | () | () | () | 0 - No Information. |
| Do you have a short fuse? | () | () | () | 1 - Not Present. |
| Do people bug you and get on your nerves a lot? What kinds of things bug you or set you off? Do you get really annoyed when your parents tell you that you can't do | () | () | () | <ul> <li>Subthreshold: Easily annoyed or touchy on<br/>occasion, but less than once a week)</li> </ul> |
| something you want to do? Like what? What other things really get on your nerves? What do you do when you are feeling annoyed or bugged? How often would you say this happens? | () | () | () | Threshold: Easily annoyed or touchy. Annoyed more often than a typical child his/her age; at least one time per week. PAST: P C S |
| | <u>P</u> | c | <u>s</u> | |
| 2. Angry of Resentful | () | () | () | 0 - No Information. |
| | () | () | () | 1 - Not Present. |
| Do you get angry or cranky with your parents a lot? How about your teachers? brothers? sisters? friends? Do other people tell you that you get cranky a lot? Who? How often does it happen? | () | () | () | 2 - Subthreshold: Occasionally angry or resentful;<br>less than one time per week |
| Parent: is your child often resentful when you ask him/her to follow your rules or requests? | () | () | () | 3 - Threshold: Angry or resentful at least once per w<br>Angry more often than a typical child his/her a |
| | | | | PAST: P C S |
| A control (Section) | <u>P</u> | c | <u>s</u> | |
| 3. Spiteful and Vindictive | () | () | () | 0 - No Information. |
| When someone does something unfair to you, do you try or plan to try to get back at them? Do you go through with the plan? Give me some examples? | () | () | () | 1 - Not Present |
| What if your brother or a friend did something to get you into trouble or make you mad. Would you do something back to them? Has this happened before? How often? Are there times when people do something to you and you let it slide? Does this happen a lot? | () | () | () | <ul> <li>2 - Subthreshold; Sometimes lets things slide /<br/>occasionally gets back at people. (1-3<br/>times a week)</li> </ul> |
| Does this happen a lot? | () | () | () | <ol> <li>Threshold: Spiteful and/or vindictive once a<br/>week or more; Spiteful more often than a typical<br/>child his/her age.</li> </ol> |
| | | | | PAST: P C S |
| NOTE: DO NOT RATE ODD SYMPTOMS POSITIVELY IF SYMPTOMS EXCLUSIVELY WHEN USING ALCOHOL OR ELICIT SUBSTANCES. | OCCUR | EXC | LUSIV | ELY DURING A MOOD EPISODE,OR |
| Subject | | | | \$ E . |

| | Oppos | itional Defi | ant Diso | rder | | | page | 9 of 21 |
|---|---|---|---|---|---|---|---|---|
| | | | P | C | <u>s</u> | | | |
| . Annoys People on Purpose | | | () | () | () | 0 - No Information. | | |
| | | | () | () | () | 1 - Not Present. | | |
| Do you or do people say you do things on pu<br>Your parents? | rpose to annoy or | r bug them? | () | () | () | | | Contract to |
| Do you enjoy pushing your mom/dad's buttor<br>Peers? | ns? Teachers? S | Siblings? | | | | 2 - Subthreshold: Od<br>done things to a | | |
| How often do you like to do this? What kinds of things do they complain about! Are you a "pain in the neck"? | 2 Do you think tha | nt il's true? | () | () | () | <ul> <li>3 - Threshold: Often people. (at least</li> </ul> | | |
| Do not score teasing of a sibling. | | | | | | PAST: | | |
| | | | | | | P | c s | |
| | | | P | | • | | | |
| Plamas Others for Cum Mintalian | | | <u>P</u> | <u>c</u> | <u>s</u> | 2 5 8 2 22 | | |
| . Blames Others for Own Mistakes | | | () | () | () | 0 - No Information. | | |
| When you get into trouble, is it ever your faul | | AC 050 1904 | () | () | () | 1 - Not Present. | | |
| If you know that you did something wrong an<br>to it? Pretend that someone else did it? Blan<br>Is it usually your fault or someone else? | | | () | () | () | <ol> <li>Subthreshold: Or<br/>denies responsil</li> </ol> | | |
| Do you think most of your troubles are cause your own fault? | d by other people | e or are they | () | () | () | <ul> <li>3 - Threshold: Ofter responsibility for</li> </ul> | | |
| | | | | | | PAST: | c s | |
| Codes for | Remaining Ite | | | | <b>1</b> = No | P 2 = Yes | | |
| Codes for | Remaining Ite<br>Criteria | ms: 0 = No Parent CE | Information Parer MSP | ıt | 1 = No<br>Chi | P 2 = Yes | C S Summary CE | Summar<br> MSP |
| | Criteria | Parent | Parer | it | Chi | P 2 = Yes Id Child MSP | Summary | MSP |
| | - V. J. r | Parent<br>CE | Parer<br>MSP | 2 | Chi | P 2 = Yes Id Child MSP 2 0 1 2 | Summary<br>CE | 0 1 2 |
| Duration For how long have you had trouble (list | Criteria<br>6 months | Parent<br>CE<br>0 1 2 | Parer<br>MSP | 2<br>() | Chi<br>CE<br>0 1 | P 2 = Yes 1d Child MSP 2 0 1 2 0 () () () () | Summary<br>CE<br>0 1 2 | Summar<br>MSP<br>0 1 2<br>() () ( |
| Duration For how long have you had trouble (list symptoms that were positively endorsed)? | Criteria<br>6 months | Parent CE 0 1 2 () () () | Parer<br>MSP<br>0 1<br>() () | 2<br>() | Chi<br>CE<br>0 1 | P 2 = Yes Child MSP 2 0 1 2 () () () () | Summary CE 0 1 2 () () () () | 0 1 2<br>()()() |
| Duration For how long have you had trouble (list symptoms that were positively endorsed)? Impairment A. Socially (with peers): | Criteria<br>6 months | Parent CE 0 1 2 () () () () | Parer MSP 0 1 () () | 2 () | Chi CE 0 1 () () () | P 2 = Yes Id Child MSP 2 0 1 2 0 () () () () 2 0 1 2 0 () () () | Summary CE 0 1 2 () () () | 0 1 2<br>() () ( |
| Duration For how long have you had trouble (list symptoms that were positively endorsed)? Impairment | Criteria<br>6 months | Parent CE 0 1 2 () () () | Parer MSP 0 1 () () | 2<br>() | Chi CE 0 1 () () 0 1 () () | P 2 = Yes Id Child MSP 2 0 1 2 0 () () () () 2 0 1 2 () () () () | Summary CE 0 1 2 () () () | 0 1 2<br>() () () |
| Duration For how long have you had trouble (list symptoms that were positively endorsed)? Impairment A. Socially (with peers): B. With family: | Criteria<br>6 months | Parent CE 0 1 2 () () () () | Paret MSP 0 1 () () () | 2 () 2 () 2 () | Chi CE 0 1 () () 0 1 () () 0 1 () () | P 2 = Yes d | Summary CE 0 1 2 () () () () | MSP<br> 0 1 2<br> () () ( |
| Duration For how long have you had trouble (list symptoms that were positively endorsed)? Impairment A. Socially (with peers): | Criteria<br>6 months | Parent CE 0 1 2 () () () () 0 1 2 () () () () | Parer MSP 0 1 () () | 2 () 2 () 2 () 2 () | Chi CE (1) | P 2 = Yes d | Summary CE 0 1 2 () | 0 1 2 () |

| Codes for Remaining Items: | 0 = No Infor | mation 1 = | No 2 | = Yes | | |
|---|---|---|---|---|---|---|
| | Parent<br>CE | Parent<br>MSP | Child<br>CE | Child<br>MSP | Summary | Summar |
| Evidence of Precipitant (Specify): | 0 1 2 | 0 1 2<br>()()() | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| Are ODD symptoms present in the following environments: | 1.74 | | 4 4 | | | |
| A. With parents | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| With other adult family members (e.g. grandparents, aunts, uncles, etc.) | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| C. In school | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2<br>() () () | 0 1 2 | 0 1 2 |
| D. In community settings (e.g. coaches, police, heathcare provider, etc.) | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| E With peers | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 | 0 1 2 |
| DSM-5 Criteria: Evidence of Oppositional Defiant Disorder A. A pattern of angry/irritable mood, argumentative/defiant behavior, of as evidenced by four (or more) symptoms from any of the followin Angry/irritable Mood: 1. Often loses temper. 2. Often touchy or easily annoyed. 3. Often angry and resentful. | or vindictivenes:<br>g categories, ar | s lasting at leas | t 6 months,<br>h at least one i | individual who | 0 1 2<br>()()()()<br>Is not a sibling | 0 1 2 |
| Argumentative/Defiant Behaior: 4. Often argues with authority figures or, for children and adolesc 5. Often actively defies or refuses to comply with adults' requests 6. Often deliberately annoys others 7. Often blames others for his/her mistakes or behavior | | | roles | | | |
| Vindictiveness: | | | | | | |
| 8. Often spiteful or vindictive at least twice within the past 6 months | S | | | | | |
| B. The disturbance in behavior causes distress in the individual or of C. The behaviors do not occur exclusively during a Psychotic, Substi | | | | | | |
| NOTE: Conduct Disorder is no longer a rule out for the NOTE: CONSIDER CRITERION (A) MET ONLY IF THE BEHAVIOR INDIVIDUALS OF COMPARABLE AGE AND DEVELOPME | R OCCURS M | ORE FREQUE | NTLY THAN I | S TYPICALLY | Y OBSERVED | IN |
| Specify (current):Mild (one setting) Moderate (two settings) | | S | specify (past | | ild (one settin | |

Subject


| Oppositional Defiant Disorder Codes for Remaining Items: 0 = No Information 1 = No 2 = Yes | 1 | page | e 11 | of 2 | 7 | |
|---|---|---|---|---|---|---|
| Codes for Remaining Items. 0 - No Information 1 - No 2 - Fes. | Sui | mm | ary | Sur | nm | ar |
| *************************************** | 1 | CE | | \ \ \ | ISP | |
| 11. Evidence of Unsepcified Disruptive Behavior Disorder | 11 11/1 | 1 | | 100 | 1 | |
| If criteria is not met for CD or ODD, but symptoms are present. For example, there are multiple symptoms present, in addition to clinical impairment. | 10 | () | (.) | 1.1 | () | ( |
| 2. Evidence of Parent-Child Relational Problems | | 1 | 2 | 100 - | 1 | |
| 2. Evidence of Parent-Child Relational Problems | () | () | () | () | () | ( |
| | | | | _ | | |

Neurodevelopmental, Disruptive, and Conduct Disorders Supplement

| en prese<br>sorder,<br>r NOT g | ent du<br>MDE,<br>living | ADHI<br>both | n which the basic rights of others or major<br>ne past 12 months with at least one present i<br>D, psychosis, substance abuse.<br>diagnoses. However, in persistent |
|---|---|---|---|
| | | | diagnoses. However, in persistent |
| | ,,,,,, | migh | t consider giving both diagnoses. |
| P | C | s | |
| () | () | () | 0 - No Information |
| () | () | () | 1 - Not Present. |
| () | () | () | Subthreshold: Minor acts of deliberate destruction of other people's property on rare |
| | | | occasions (e.g., breaks another's toy on<br>purpose) OR one or two occasions of<br>significant destruction of property. |
| () | () | () | 3 - Threshold: Three or more instances of<br>moderate to severe vandalism/destruction of<br>property. |
| | | | P C S |
| | 3 | 4 | |
| _ | 100 | | 3 our ere |
| 1 | | | 0 - No Information |
| | | | 1 - Not Present. |
| 7.3 | () | () | 2 - Subthreshold: Has been with friends who bro<br>into a house, car, store, or building, but did n<br>actively participate. |
| () | () | () | <ul> <li>Threshold: Has broken into a house, car, stor<br/>or building 1 or more times.</li> </ul> |
| | | | PAST: P C S |
| Р | C | S | |
| 17 | | | 0 - No Information |
| () | () | () | 1 - Not Present. |
| () | () | () | <ul> <li>Subthreshold: Has been with friends who<br/>aggressively stole, but did not actively<br/>participate.</li> </ul> |
| () | () | () | Threshold: Mugging, purse-snatching, extorti-<br>armed robbery, etc. on 1 or more occasions. |
| | | | PAST: P C S |
| | 0<br>0<br>0<br>0<br>0 | P C O O O O O O O O O O O O O O O O O O | P C S 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 |

| Parameter | sorder | | | |
|---|---|---|---|---|
| Figure | Р | C | s | ,-3-1-2. |
| | () | () | () | 0 - No Information |
| Firesetting | () | () | () | 1 - Not Present |
| Have you set any fires? Why did you set the fire? Were you playing with matches and did you start the fire by accident, or did you start it on purpose? | () | () | () | <ul> <li>Subthreshold: Match/lighter play. No intent to<br/>cause damage, and fire(s) not started out of<br/>anger.</li> </ul> |
| Were you angry? Were you trying to cause a lot of damage or to get back at someone? What's the most damage you ever caused by starting a fire? | () | () | () | Threshold: Set 1 or more fires with the intent cause damage, or out of anger. |
| About how many fires have you set? | | | | PAST: C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| Often Stays out at Night | () | () | () | 0 - No Information. |
| What time are you supposed to come home at night? | () | () | () | 1 - Not Present. |
| Do you often stay out past your curiew? What is the latest you ever stayed out? Have you ever stayed out all night? | () | () | () | <ol> <li>Subthreshold: Stayed out all night, or several<br/>hours past curfew, on 1-2 isolated occasions<br/>(despite parent's prohibitions).</li> </ol> |
| How many times have you done that? NOTE: ONLY RATE POSITIVE INCIDENTS OF STAYING OUT IF IT BEGINS BEFORE THE AGE OF 13. | () | () | () | <ul> <li>Threshold: Stayed out all night, or several<br/>hours past curfew, on several occasions (3 o<br/>more times).</li> </ul> |
| | | | | PAST: P C S |
| | P | C | <u>s</u> | |
| | () | () | () | 0 - No Information. |
| Ran Away Overnight | | 91.5 | | |
| Ran Away Overnight | () | () | () | 1 - Not Present. |
| Have you ever run away? Why?<br>Was there something going on at home that you were trying to get away<br>from? | 3,7.3 | () | () | |
| Have you ever run away? Why?<br>Was there something going on at home that you were trying to get away | () | () | 100 | |

| Conduct Dis | order | | | |
|---|---|---|---|---|
| | Р | <u>c</u> | s | |
| . Use of a Weapon | () | () | () | 0 - No Information. |
| | () | () | () | 1 - Not Present |
| Have you ever used an object or item to hit/hurt someone? Have you ever carried a weapon? | () | () | () | 2 - Subthreshold: Has threatened use of a |
| Have you ever used or threatened to use:kitchen knife or pocket knife | 17 | 4.7 | 10 | weapon, but has never used one. |
| gunbrick, rocksbroken bottles | 0 | () | () | <ul> <li>Threshold: Used a weapon that can cause<br/>serious harm on 1 or more occasions (e.g.,<br/>knife, brick, broken bottle, gun).</li> </ul> |
| bat<br>brick | | | | PAST: |
| What about in self defense? | | | | P C S |
| | 2 | C | <u>s</u> | |
| . Physical Cruelty to Persons | () | () | () | 0 - No Information. |
| Have you ever beaten someone up for no reason? | () | () | () | 1 - Not Present |
| How bad? Was it just because the other person was different than you or because of the way they looked? | () | () | () | Subthreshold: Has been physical cruelty on one or two occasions. No significant injuries. |
| Did they get hurt? | () | () | () | 3 - Threshold: Has been physically cruel to an |
| NOTE: DO NOT COUNT TRIVIAL SIBLING RIVALRY, | | | | individual on 3 or more occasions, or on one occasion intentionally causing significant injury |
| | | | | PAST: P C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| Forced Sexual Activity | () | () | () | 0 - No Information. |
| Have you ever forced anyone to kiss you or touch you in your private parts? | () | () | () | 1 - Not Present. |
| Have you every forced another kid to touch you outside your clothes?<br>Has anyone ever said you forced another kid/person to go farther than they wanted? What did they say? | () | () | () | <ul> <li>Subthreshold: Forced or attempted to force<br/>someone to participate in mild sexual activity (e<br/>non-genital fondling) on one or more occasions</li> </ul> |
| | () | () | () | 3 - Threshold: Forced someone to participate in |
| | | | | severe sexual activity (e.g. genital fondling,<br>oral sex, vaginal intercourse and/or anal<br>intercourse) on one or more occasions. |
| | | | | PAST: P C S |
| Subject | | | | |

| | Con | duct | Dis | sore | ler | | | | | | | | | pag | ge : | 150 | f 27 | | - |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | P | C | | s | | | | | | | | | | | |
| 0. Cruelty to Animals | | | | | 0 | () | | ) | 0 | - No | Infor | mati | on | | | | | | |
| a sold and the sol | N. Oren error | | | | () | () | | ) | | - Nat | | | | | | | | | |
| Some kids like to hurt or torture animals. Have you h<br>animal on purpose? What did you do?<br>About how many times have you hurt an animal on p | | | | | () | () | | ) | | Sub | othre | sholo | | s repe | | | en m | ldly | сп |
| MOTE: DO NOT SCORE TRADITIONAL HUNTING CAREFUL ATTENTION TO THE COMMUNITY SET FARM, ETC.]. | | | | | () | () | ( | ). | | - Thr | esho | old: Fre oc | las ki | illed o | r tor | tured<br>peato<br>es to | lly ca | use | d |
| Codes for Remail | ning Items: | 0 = 1 | lo li | nfor | matic | in | 1.= | No | | 2 | = Ye | P | | С | | 5 | | | _ |
| | Criteria | P | are<br>CE | | | are<br>MSI | | ( | Chil | | | hile | | Sui | mm | ary | Su | mm | |
| 1. Impairment | | 1 | | | | | | 1000 | | 555 | 7.75 | 555 | | | | | | | 7 |
| A. Socially (with peers): | | () | 1 () | 2 | () | 1 | () | <b>0</b> () | 1 () | 2 | 0 | 1 () | 2 | () | 1 | 2 | () | () | ( |
| B. With family: | | 0 () | 1 () | 2 | 0 | 1 () | 2 | 0 () | 1 () | 2 | 0 () | 1 | 2 | 0 () | 1 | 2 | 0 () | 1 () | |
| C. In school: | ,,,,,,,,,, | 0 () | 1 () | 1 | 0 () | 1 () | 2 | 0 | -2 | 2 | 0 | 1 () | 2 | 0 () | 1 () | 2 | 0 () | 1 () | |
| 2. Duration For how long did you (list positively endorsed | 6 months or more | 0 | 1 () | | 0 | 1 | | 0 | 1 | 2 | 0 | 1 () | 2 | 0 | 1 | 2 | 0 | 1 () | |
| NOTE: PER THE DSM-5. "the Conduct Disorder or should be applied only when the behavior in quesymotomatic of an underlying dysfunction within individual and not simply a reaction to the immediant." | stion is | | | | | | | | | | | | | | | | | | |
| | | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 3 |
| Childhood Onset Type How old were you when you first started to (list positively endorsed items)? | Onset of at<br>least one<br>conduct | 11/30 | () | 7. | () | () | () | () | | () | 1.30 | () | | 1.7 | | () | () | () | - 1 |
| 4. Adolescent Onset Type | No conduct problems | 0 | 1 | | 0 () | 1 | 2 | 0 | | 2 | 0 | 1 | | 0 | 1 () | 2 | 0 | 1 | |

### CONFIDENTIAL Version 9.0


| | Con | duct Disorder | | | page 1 | 6 of 27 |
|---|---|---|---|---|---|---|
| <u>Codes for Ren</u> | naining Items: | 0 = No Information | <b>1</b> = No | 2 = Yes | Summary<br>CE | Summar<br>MSP |
| 5. Evidence of Conduct Disorder<br>DSM-5 Criteria | | | | | 0 1 2 | 0 1 2 |
| | to the fall than the blank | Company of the sale of the sale | | an Calman | (1111) | () () ( |
| A. A repetitive and persistent pattern of behavior<br>norms or rules are violoated, as manifested to<br>12 months, with at least one criterion present in<br>Aggression to People and Animals | y the presence of | three (or more) of the fo | | | | |
| 1) Often bullies, threatens or intimidates of | ners | | | | | |
| Often initiates physical fights Has used a weapon that can cause series. | | to others (e.g., a bat, b | rick, broken bot | tle, knife,gun). | | |
| 4) Has been physically cruel to people | | | | | | |
| <ul> <li>Has been physically cruel to animals</li> <li>Has stolen while confronting a victim (e.</li> <li>Has forced someone into sexual activity</li> </ul> | g., mugging, purse | snatching, extortion, as | med robbery) | | | |
| Destruction of Property 8) Has deliberately engaged in fire setting w 9) Has deliberately destroyed others' proper | | | e | | | |
| Deceitfulness or Theft 10) Has broken into someone else's house, 11) Often lies to obtain goods or favors or to a | | e "cons" others) | | | | |
| 12) Has stolen items of nontrivial value with | CONTRACTOR OF THE PROPERTY OF | And the state of t | ut without brea | king and entering | forgery) | |
| Serious Violation of Rules 13) Often stays out at night despite parenta | | | | ang and ontoning. | (orgory). | |
| <ol> <li>Has run away overnight at least twice v</li> <li>Is often truent from school, beginning be</li> </ol> | The state of the s | and the second s | e home (or once | e without returning | for a lengthy per | riod). |
| B. The disturbance in behavior causes clinically | significant impairm | nent in social, academic | or occupations | I functioning. | | |
| C. If the individual is age 18 years or older, criteria | are not met for An | ntisocial Personality Dison | der. | | | - |
| Specify (Current): With Limited Prosocial Emot | on | Spec | ify (Past): With | Limited Prosocial | Emotion | |
| Criteria: Displays at least two of the following chor guilt; 2) Callous, lack of empathy; 3) Unconce | | | | | | |
| Specify Severity (Current): Mild | Moderate | Severe | | | | |
| | /loderate | Severe | | | | |
| Criteria: Mild: Few problems in excess of those intermediate severity (e.g., stealing without concause considerable harm to others (e.g. forced | fronting a victim, v | andalism); Severe: Mar | y problems in e | xcess of those red | uired for the diagr | nosis, or prob |
| Subject | | | | | | E 1 |

| | Conduct Disorder | page 17 or | 27 |
|---|---|---|---|
| | Codes for Remaining Items: 0 = No Information 1 = No 2 = Yes | | |
| | | Summary<br>CE | Summar<br>MSP |
| 16 | Group Type | 0 1 2 | 0 1 2 |
| | Predominance of conduct problems occur as group activity with peers. | | |
| 17 | Solitary Aggressive Type | 0 1 2 | 0 1 2 |
| | Most conduct disorder activities initiated by the person (not as group activity). | () () () | ()()( |
| | | 1 | |
| 18 | . <u>Undifferentiated Type</u> Conduct symptoms cannot be classified as either group or solitary aggressive type. | ()()() | () () ( |
| | | | , |
| 10 | Callous and Unemotional | 0 1 2 | 0 1 2 |
| 10. | At least 2 of the following: 1. Lack of Remorse or Guilt2. Lack of Empathy3. Unconcerned about Performance | L | |
| 13. | 4. Shallow or Deficient Affect | | |
| | | 0 1 2 | 0 1 2 |
| 20 | | 0 1 2 | 0 1 2 |



Subject

Neurodevelopmental, Disruptive, and Conduct Disorders Supplement 2013 Simple and Complex Motor Disorders  Criteria for Items: 0 = No Information 1 = No 2 = Yes NOTE: FOR SYMPTOMS TO BE RATED POSITIVELY THEY MUST OCCUR MANY TIMES A DAY, OR HAVE OCCURRED INTER-MITTENTLY FOR ONE YEAR OR LONGER AND NOT BE BETTER ACOUNTED FOR BY ANOTHER NEUROLOGICAL DISORDER Child Child Parent Parent Summary Summary SIMPLE MOTOR CE MSP CE MSP CE MSP (Rate based on report and observation) 1. Eye Blinking 0 1 2 0 2 0 1 2 0 1 0 0 1 2 1 2 1 () () () () () 00 () Do your eyes blink a lot like this for no reason? (demonstrate) Other Facial Tics 1 2 0 1 2 0 1 2 0 1 2 0 1 2 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 Do other parts of your face sometimes move unexpectedly like this? (demonstrate facial grimaces, nose scrunching, and opening mouth as if to yawn) 3. Head Jerks 2 0 2 0 2 0 2 0 2 1 1 1 2 () ()()() 000000 00000000 Do you sometimes nod your head, shake your head, or turn your head to the side for no special reason? (demonstrate) 4. Shoulder Jerks 0 0 2 2 2 0 2 1 0 1 2 2 1 1 1 () 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 What about your shoulders, do your shoulders sometimes move unexpectedly like this (shrug shoulder or roll shoulder)? 5. Arm Movements 1 2 0 2 0 1 2 0 1 2 0 1 2 0 ()() () Do you sometimes flap your arms or throw your arms out as if to hit something that isn't there? (demonstrate) 1 2 0 6. Stomach Twitches 2 0 1 2 0 1 2 0 2 0 () () () () () () () 000000 Does your stomach sometimes move for no special reason? 2 0 2 0 1 2 0 1 2 0 1 2 0 7. Leg Movements () Do you ever stomp your feet or kick your legs out and you're not sure why you do it? Do you sometimes bang your legs up under your desk when you weren't planning on moving them?

Neurodevelopmental, Disruptive, and Conduct Disorders Supplement 2013 Simple and Complex Motor Disorders  Code for Remaining Items: 0 = No Information 2 = Yes Parent Parent Child Child Summary Summary MSP MSP CE CE MSP CE 8. Other 0 1 2 0 1 2 0 1 2 0 1 0 1 2 0 1 2 () Are there any other types of movements that you notice that I haven't asked you about? Specify: 9. Summation of all above 2 1 2 0 1 2 0 1 0 1 2 1 2 0 0 0 0 0 0 0 0 0 () () () 0000000 Simple motor tics occur many times a day or have occurred intermittently for 1 year or longer COMPLEX MOTOR 1. Touching/Tapping Things 2 1 2 0 1 2 0 2 0 2 () Do you ever touch your own body, your nose, your ear, or feel ike you have to touch other people, or other things...like having to touch the phone every time you walk by it, touch walls, or all the furniture in your room? Do you often tap your pencil or your fingers against your desk? 2. Hopping/Spinning 2 0 1 2 2 0 2 0 1 0 1 2 0 1 () When you are walking down the hall at school, do you sometimes find that you have to hop or spin rather than keep walking straight? 3. Echokinesis 2 0 1 2 0 1 2 0 2 0 2 0 2 1 1 1 1 () Do you ever find that you have to imitate other people's actions like pushing your hair back or rubbing your nose? Anything else? 4. Hurts Self 2 0 1 2 0 1 2 0 1 2 0 1 2 0 1 0 0 0 0 0 0 0 0 () () () 000000 Do you ever feel like you have to hit yourself in the face, pull your hair or bite your hand? 5. Other 1 2 0 1 2 0 1 2 0 1 2 0 1 2 0 1 2 () Are there any other types of movements that you notice that haven't asked you about? Specify. 6. Summation of all above 0 2 0 2 0 1 2 0 2 0 1 2 0 1 1 1 1 2 () Complex motor tics occur many times a day, or have occurred intermittently for 1 year or longer Subject

| Code for Remaining | g Iter | ns: | 0 = | No Ir | form | ation | 1 | = N | 0 | 2 = | Yes | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SIMPLE VOCAL PHONIC | F | Parer | nt | | arer<br>MSP | | | Chile | 1 | Child<br>MSP | | | Summary<br>CE | | | Summar<br>MSP | | |
| Sniffing/Coughing/Throat Clearing Do you ever sniff, cough, or clear your throat when | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 () | 1 () | 2 () | 0 () | 1 () | 2 | 0 | 1 () | 2 |
| you don't have a cold? Does this happen over and over again? | | | | | | | | | | | | | | | | | | |
| 2. Snorting/Grunting | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| Do you ever make noises through your nose or in your throat like this? (demonstrate) | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | ( |
| 3. Other | | | | | | | 12. | | | | | | | | | | | |
| Are there any other types of sounds that you make that I haven't asked you about? What about tongue clicking, lip smacking, or making | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | - |
| popping sounds? 4. Summation of all above | 0 | 1 | 2 | 0 | 4 | 2 | 0 | 4 | 2 | 0 | 4 | 2 | 0 | | 2 | 0 | 1 | |
| Simple vocal tics occur many times a day or intermittently for a year or longer. | 1000 | () | () | () | () | | () | () | Ö | 1 3 3 | () | | 100.0 | () | Ō | 150 | () | |
| COMPLEX VOCAL PHONIC | | | 4000 | | | | | | | | | | | | | | | |
| 1. Repeat Own Words/Sentences | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | - |
| Do you ever notice that you have to repeat<br>yourself, not because someone didn't hear you, but<br>because it didn't sound right, or maybe for no<br>special reason at all? | 17 | | | () | () | | Liz. | () | | () | () | () | 10 | () | () | () | () | |
| 2. Repeat Others Speech | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 |
| Do you find yourself sometimes repeating things other people have said for no special reason at all? | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | ( |
| 3. Coprolalia (Obscene Words) | | 4 | | | | | | | • | | | • | | | | • | | - |
| Do bad words ever pop out of your mouth in the middle of a sentence for no reason, or do you find yourself saying bad things under your breath and find you can't stop yourself? | () | () | () | () | () | () | () | 0 | () | () | O | () | () | Ò | () | Ö | () | |
| 4. Insults/Racial Slurs | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | - |
| Do you sometimes find yourself saying bad things<br>to people about how they look or something else<br>about them when you didn't really mean it? | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | - |
| Code for Remaining | na Iten | ns: | 0 = | No In | form | ation | 1 | = No | 0 | 2= | Yes | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 2200000 | | arer | | P | aren<br>MSP | t | | Child | - | ( | Child | | Sı | ımm<br>CE | ary | | mma<br>MSP |
| Other . | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 () |
| Are there any other things you sometimes find<br>yourself saying?<br>Are you afraid you might have one of these attacks? | | () | () | | () | | () | () | | () | () | | () | () | () | () | () |
| Summation of all above | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 |
| Vocal tics occur many times a day or intermittently for a year or longer. | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () |
| Impairment | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 |
| A. Socially (with peers): | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () | () |
| ~ | | | | | | | · | | , | | | | | | | | |
| B. With family: | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 |
| C. In school: | | | | | | • | | | | | | | | | | | |
| J. III 30/300/. | () | () | () | () | () | () | () | Ö | 2 () | () | () | () | () | () | () | () | () |
| | | | | | | | | | | .0000 | 0000 | 0006 | | | | و در | 00.00 |
| Criteria for Tourette's Disorder | | | | | | | | | | | | | 0 | 1 | 2 | 0 | 1 |
| DSM-5 Criteria A. Both multiple motor and one or more vocal tics have | | | | | | A | | | | | | | Line | 2222 | a a a l | 222 | 222 |
| necessarily concurrently. (A tic is a sudden, rapid, B. The tics may wax and wane in frequency, by have p C. Onset before age 18 years. D. The disturbance is not exclusively due to the direct p general medical condition (e.g., Huntington's disear | ersisted | for n | nore the | an 1 | year s | ince f | irst tic | onse | t. | | caliza | tion). | | | | | |
| gere ar medical corollion (e.g., nonlingiors diseas | se a po | Stvii a | CILC | prianti: | | | | | | | | | | | | | |

| Evidence of Persistent (Chronic DSM-5 Criteria A Single or multiple motor or vocal IB. The tics may wax and wane in free C. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T. Specify (Current): With motor tics of Specify (Past): With motor tics of D. Evidence of Provisional Tic Disturbance of Provisional Tic Disturbance is not exclusively B. The tics have been present for le C. Onset before age 18. D. The disturbance is not exclusive general medical condition (e.g. E. Criteria have never been met for | c) Motor or Voc<br>tics have been plequency, by have<br>ly due to the direct<br>Huntington's districted<br>Tourette's Disorder<br>only: | eal Tic Disord<br>resent during the<br>persisted for many the properties of the properties | the illness, but not both increthan 1 year since first effects of a substance (eal encephalitis). | motor and voca | | 0 | CE | 2 | 0 | mmma<br>MSP |
|---|---|---|---|---|---|---|---|---|---|---|
| DSM-5 Criteria A Single or multiple motor or vocal is. The tics may wax and wane in free. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T. Specify (Current): With motor tics of Specify (Past): With motor tics of Specify (Past): With motor tics of DSM-5 Criteria A. Single or multiple motor and/or v. B. The tics have been present for let C. Onset before age 18. D. The disturbance is not exclusively general medical condition (e.g. | tics have been pi<br>equency, by have<br>ly due to the direct<br>, Huntington's dis<br>Tourette's Disorde<br>only: | resent during the persisted for material physiological dease or postviral rice. With vocal tice | the illness, but not both increthan 1 year since first effects of a substance (eal encephalitis). | at tic onset. | | 0 | CE<br>1 | 2 | 0 | MSP<br>1 |
| DSM-5 Criteria A Single or multiple motor or vocal is. The tics may wax and wane in free. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T. Specify (Current): With motor tics of Specify (Past): With motor tics of Specify (Past): With motor tics of DSM-5 Criteria A. Single or multiple motor and/or v. B. The tics have been present for let C. Onset before age 18. D. The disturbance is not exclusively general medical condition (e.g. | tics have been pi<br>equency, by have<br>ly due to the direct<br>, Huntington's dis<br>Tourette's Disorde<br>only: | resent during the persisted for material physiological dease or postviral rice. With vocal tice | the illness, but not both increthan 1 year since first effects of a substance (eal encephalitis). | at tic onset. | | 15.00 | 1 | Wall. | 0 | 1 |
| DSM-5 Criteria A Single or multiple motor or vocal is. The tics may wax and wane in free. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T. Specify (Current): With motor tics of Specify (Past): With motor tics of Specify (Past): With motor tics of DSM-5 Criteria A. Single or multiple motor and/or v. B. The tics have been present for let C. Onset before age 18. D. The disturbance is not exclusively general medical condition (e.g. | tics have been pi<br>equency, by have<br>ly due to the direct<br>, Huntington's dis<br>Tourette's Disorde<br>only: | resent during the persisted for material physiological dease or postviral rice. With vocal tice | the illness, but not both increthan 1 year since first effects of a substance (eal encephalitis). | at tic onset. | | 15.00 | | Wall. | -52 | - 3-0 |
| A. Single or multiple motor or vocal IB. The tics may wax and wane in free C. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T. Specify (Current): With motor tics of Specify (Past): With motor tics of Specify (Past): With motor tics of DSM-5 Criteria A. Single or multiple motor and/or v. B. The tics have been present for is C. Onset before age 18. D. The disturbance is not exclusive general medical condition (e.g. | equency, by have fy due to the direct , Huntington's distrourette's Disorde only: | persisted for m<br>t physiological<br>ease or postvira<br>er. With vocal tic | effects of a substance (eal encephalitis). | at tic onset. | | () | () | () | () | () |
| B. The tics may wax and wane in fre C. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T Specify (Current): With motor tics of Specify (Past): With motor tics of D. Evidence of Provisional Tic Di DSM-5 Criteria A. Single or multiple motor and/or of B. The tics have been present for the C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g. | equency, by have fy due to the direct , Huntington's distrourette's Disorde only: | persisted for m<br>t physiological<br>ease or postvira<br>er. With vocal tic | effects of a substance (eal encephalitis). | at tic onset. | | | | | | |
| C. The onset is before age 18. D. The disturbance is not exclusively general medical condition (e.g., E. Criteria have never been met for T. Specify (Current): With motor tics of Specify (Past): With motor tics of D. Evidence of Provisional Tic Disturbance of Provisional Tic Di | iy due to the direct , Huntington's distributed in the content of | t physiological e<br>ease or postvira<br>er.<br>With vocal tic | effects of a substance (eal encephalitis). | | ora | | | | | |
| E. Criteria have never been met for T Specify (Current): With motor tics of Specify (Past): With motor tics of Specify ( | only: | With vocal tic | s only: | | | | | | | |
| D. Evidence of Provisional Tic Di DSM-5 Criteria A. Single or multiple motor and/or to B. The tics have been present for let. C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g. | only: | | | | | | | | | |
| D. Evidence of Provisional Tic Di DSM-5 Criteria A. Single or multiple motor and/or v B. The tics have been present for la C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g. | | With vocal fice | s only: | | | | | | | |
| DSM-5 Criteria A. Single or multiple motor and/or v B. The tics have been present for la C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g. | Disorder_ | | | | | | | | | |
| DSM-5 Criteria A. Single or multiple motor and/or v B. The tics have been present for la C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g. | Disorder | | | | | | | | | |
| A. Single or multiple motor and/or v B. The tics have been present for lace. C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g.) | | | >>> | | | 0 | 1 | 2 | 0 | 1 |
| B. The tics have been present for let C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g.) | | | | | | () | () | () | () | () |
| C. Onset before age 18 D. The disturbance is not exclusive general medical condition (e.g. | vocal tics. | | | | | | | | | |
| <ul> <li>D. The disturbance is not exclusive<br/>general medical condition (e.g.</li> </ul> | less than 1 year si | nce first tic ons | set, | | | | | | | |
| general medical condition (e.g. | all due to the dies | at physialagical | I officiate of a substance | o a stimulant | | | | | | |
| E Criteria have never been met for | | | | e.g., sumulano | s) Ot a | | | | | |
| | Tourette's Disord | der or Chronic N | Motor or Vocal Tic Disord | der. | | | | | | |
| Specify (Current): With motor tics of | only: | With vocal tics | s only: | | | | | | | |
| Specify (Past): With motor tics of | only: | With vocal tics | s only: | | | | | | | |
| Tic Disorder Not Otherwise Sp | pecified | | | | | 0 | 1 | 2 | 0 | 1 |
| DSM-5 Criteria | | | | | | O | () | () | () | () |
| This category is for disorders chara | acterized by tics the | hat do not meet | t criteria for a Specific Ti | c Disorder, Exa | mples | | | | | |
| include tics lasting less than 4 week | eks or tics with an | onset after age | 18 years. | | | | | | | |
| , | | | | | | | | | | |

| | Autism Spectrum | | | | |
|---|---|---|---|---|---|
| ote | : Assess symptoms with an onset in early childhood. | | | | |
| | | P | C | S | |
| | | () | () | () | 0 - No information. |
| 1. | Deficits in social-emotional reciprocity | () | () | () | 1 - Not present. |
| | Parent: s a young child, did your child show you toys and other things that<br>interested him or her, or did he or she play on his/her own with little or no<br>referencing to you | 0 | () | () | <ul> <li>2 - Subthreshold: Sometimes seeks to share; be<br/>not frequently or spontaneously.</li> </ul> |
| | If something good happens to your child now, like a good grade at school o<br>having some other success, will your child spontaneously share it with you?<br>Will she share the good news with friends? | () | () | () | 3 - Threshold: Does not spontaneously seek to<br>share enjoyment, interests or achievements |
| | Child: If something good happens to you, like you get a good grade at school or have some other success, do you keep it to yourself, or do you tell mom, dad, or someone else? | | | | with other people, or only shares when relat<br>to preoccupation. |
| | NOTE: DO NOT RATE POSITIVE IF IT IS ACCOUNTED FOR BY OTHER CONDITIONS SUCH AS ANXIETY, PSYCHOSIS, DEPRESSION, BEHAVIOR DISORDERS, OR NORMAL TEEN BEHAVIORS, | | | | P C S |
| | | <u>P</u> | <u>c</u> | <u>s</u> | |
| 2. | Deficits in developing and maintaining relationships, appropriate to developmental level | () | () | () | 0 - No information. |
| | developmentariever | () | () | () | 1 - Not present |
| | This may take different forms at different ages. Very young children may have<br>little or no interest in establishing friendships. Older children may have an<br>interest in friendship but lack understanding of the conventions of social<br>interaction. | () | () | () | <ol> <li>Subthreshold: Some personal relationships<br/>mostly in group situations or primarily in<br/>restricted interest areas.</li> </ol> |
| | Parent: Does your child have any good friends his/her age? Does your child get together with other children after school and on weekends? Does your child do better with younger kids or with adults than with kids | () | () | () | 3 - Threshold: Failure to develop peer relationsh<br>appropriate to developmental level. Unable<br>interpret peer reactions in social situations. |
| | his/her own age? Does s/he prefer to be by him or herself? Does your child wish to be social but fails to make relationships with peers? Does your child want to make friends, but says s/he does not know why other children do not want to be his/her friend? Is your child able to understand how other kids react in social situations? Or does s/he misinterpret or not "tune in" to peers' reactions in social situations? | | | | PAST: P C S |
| | Is he/she taken advantage of?<br>Can your child only be with other kids on his/her terms? | | | | |
| | Child: Do you like to be with other kids your age or would you rether be by<br>your self most of the time?<br>Do you have a best friend?<br>Do you get together after school or on the weekends? | | | | |
| | NOTE: BE CAREFUL TO WEIGH CHILD'S REPORT WITH COLLATERAL INFORMATION. DO NOT RATE THIS AS POSITIVE IF IT IS EXCLUSIVELY DUE TO OTHER CONDITIONS SUCH AS ADHD, SOCIAL ANXIETY, SCHIZOPHRENIA, OR SCHIZOID PERSONALITY. | | | | |

| Autism Spectrum | | | | |
|---|---|---|---|---|
| 11.00 | <u>P</u> | <u>c</u> | <u>s</u> | |
| Hyper-or hypo-reactivity to sensory input or unusual interest in<br>sensory aspects of environment | () | () | () | 0 - No information. |
| Is you child especially sensitive to sensory inputs? Is s/he sensitive to | () | () | () | 1 - Not present. |
| tags in clothes or the feel of different fabrics? Is you child very reactive to a change in lighting or sounds in the home? Alternatively, does you child seem oblivious to aspects of the | () | () | () | 2 - Subthreshold: Mild hyper- or hypo-reactivity to sensory inputs |
| environment around him/her? Does your child sometimes seem oblivious to pain or extreme chagnes in temperature? Are there any things your child likes to touch or smell? | () | 1) | () | - Threshold: Notable and impairing hyper- or<br>hypo-reactivity to sensory inputs |
| Child: Do you hate wearing certain clothing because the tags or fabric | | | | PAST: |
| really bother you? | | | | P C S |
| | <u>P</u> | <u>c</u> | <u>s</u> | |
| Motor deficits in performance of skilled movement not limited to social communication | () | () | () | 0 - No information |
| | () | () | () | 1 - Not present. |
| Parent: Is your child coordinated? Does s/he have trouble playing with<br>a ball or doing other sport-like activities? How is his/her manual<br>dexterity? Does s/he have trouble holding a pen or pencil? Using | () | () | () | 2 - Subthreshold: Mild motor deficits. |
| scissors? How is her/his balance? | () | () | () | 3 - Threshold: Moderate to severe motor defici |
| | | | | PAST: |
| | | | | PCS |
| NOTE: FOR ALL THE ABOVE QUESTIONS, NOTE WHETHER BEG., BEFORE PRESCHOOL), OR CURRENTLY. FOR AUTIS SHOULD HAVE STARTED WHEN THE CHILD WAS YOUNG. | M SPEC | TRU | M DIS | SORDERS, ALL THESE BEHAVIORS |
| OCD, SEVERE SOCIAL PHOBIA, MENTAL RETARDATION, A<br>THERE ARE CULTURAL ISSUES THAT CAN BETTER ACCOU | SEVER | E HIS | STOR | Y OF ABUSE OR NEGLECT, OR IF |

| | Au | tism | Spe | ctr | um | | | | | | | | 1 | page | 25 | of 27 | _ | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Codes for Remaining | Iten | ns: | 0 = | No I | nforn | natio | 1 1 | = N | 0 | 2: | Yes | 5 | | | | | | |
| | | Pare | | | arei<br>MSF | | | Child | ( | | Child<br>MSP | | Su | mm<br>CE | ary | | m m<br>MSP | - |
| 5. Communication and Social Deficits Common<br>Among Patients with Autism Spectrum Disorders | | | | | 107 | | | | | | 37.77 | | | | | | 7777 | |
| a. One Sided Verbosity | () | 1 | () | () | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | () | 0 | 1 | 2 |
| Does your child often go on and on talking<br>about one thing, almost like s/he is giving a<br>speech rather than having a conversation?<br>Have people ever said he seems like a "little<br>professor"? | Lee | | | 1 | | | | | | h-i | | | L | | | I | -99- | |
| b. Speech Pragmatic Deficits | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 | 1 | 2 | 0 | 1 | : |
| Does your child have trouble understanding the more subtle aspects of language, like how to take turns when having a conversation, or knowing what someone means when they use sarcasm or make analogies (e.g. "She's as heavy as a house")? | | 17 | 3.7 | 11/ | | | 17 | 17 | | 1.7 | 17 | <u> </u> | | | | 1.13 | 37 | |
| c. Abnormalities in Voice Modulation/Prosody | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 | 1 () | 2 | 0 | 1 () | 2 |
| Is there anything unusual about your child's<br>intonation? Is his/her voice monotone? Overly<br>sing-sangy? Does s/he have poor volume control<br>or unusual patterns of emphasis in speech? | Lii | | | 1 | | | le si si | | | | | rine- | | | | Jagan | | |
| d. Incessant and Insensitive Pursuit of Others | 0 | 1 | 2 | 0 | 1 | 2 | | 1 | 2 | 0 | 1 | 2 () | 0 | 1 | 2 | 0 () | 1 () | 2 |
| Does your child relentlessly pursue contact with others, even when they don't seem interested in talking or being with him/her? Does s/he have a hard time reading others' social cues? | L22. | | | 100. | -22 | . 2000 | 1555 | 2744 | -23- | Louis | -dd | | 1.32 | | -454 | 1,225 | | |
| NOTE: RATE BASED ON REPORT AND OBSERVA | TIO | <u>N.</u> | | | | | | | | | | | | | | | | |
| 6. Features of Patients with High Functioning Autism | | | | ç | -422 | | · · · | | | | | | | | | [ | | - |
| a. Social Isolation | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 1 |
| From the time your child was young, did your child<br>prefer to be alone? What about now, does she<br>seem uninterested in friends and other social<br>contacts? | Lein | -11 | | | -34 | | | | -442 | | | 21 | | | | 1.22 | | |
| b. Echolalic Speech | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 () | 2 | 0 | 1 | |
| Does your child repeat phrases she has heard<br>other's say, or nonsensical phrases over and<br>over? | bin n.a | | | | | | | | | | | | | | | | | |
| NOTE: RATE BASED ON REPORT AND OBSERVA | TIO | N. | | | | | | | | | | | | | | | | _ |

| CE | Summ<br>MSF<br>0 1<br>() () | (P |
|---|---|---|
| CE | MSF<br>0 1<br>() () | (P |
| a. Symptoms present in early childhood. O 1 2 0 1 2 | 0 1 | ) |
| b. Speech Pragmatic Deficits 0 | 0 1 | |
| Does your child have trouble understanding the more subtle aspects of language, like how to take turns when having a conversation, or knowing what someone means when they use sarcasm or make analogies (e.g. "She's as heavy as a house")? 8. Impairment A. Socially (with peers): () ( | - | |
| Does your child have trouble understanding the more subtle aspects of language, like how to take turns when having a conversation, or knowing what someone means when they use sarcasm or make analogies (e.g. "She's as heavy as a house")? 3. Impairment A. Socially (with peers): O 1 2 0 1 2 0 1 2 0 1 2 0 1 2 0 1 2 0 1 2 0 1 0 1 | () () | ) |
| A. Socially (with peers): () | | |
| A Socially (with peers): () | 0 1 | |
| | 0 0 | |
| b. vviii lainily. | 0 1 | |
| O. III SCHOOL | <b>0 1</b> () () | |

Neurodevelopmental, Disruptive, and Conduct Disorders Supplement 2013 **Autism Spectrum Disorder**  Codes for Remaining Items: 0 = No Information 2 = Yes Summary Summary Evidence of Autism Spectrum Disorders DSM-5 Criteria 0 1 2 0 1 2 () () () () () () A. Persistent deficits in social communication and social interaction across multiple contexts, as manifest by the following, currently or by history 1. Deficits in social-emotional reciprocity, ranging for example, from abnormal social approach or failure of back and forth conversation, to reduced sharing of interests, emotions, affect; to failure to initiate or respond to social interactions. 2. Deficits in nonverbal communicative behaviors used for social interaction, ranging from poorly integrated verbal and nonverbal communication, to abnormalities in eye contact and body-language, or deficits in understanding and use of gestures; to a total lack of facial expression and non-veral communication. 3. Deficits in developing, maintaining, and understanding relationships, ranging from difficulties adjusting behavior to suit different social contexts, to difficulties in sharing imaginative play and in making friend; to absence of interest in peers B. Restricted, repetitive patterns of behavior, interests, or activities as manifested by at least two of the following: 1. Stereotyped or repetitive speech, motor movements, or use of objects; (such as simple motor stereotypies, echolalia, repetitive use of objects, lining up of toys or flipping objects, or idiosyncratic phrases). 2. Insistence on sameness, inflexible adherence to routines, or ritualized patterns of verbal or nonverbal behavior (e.g. extreme distress at small changes, difficulties with transitions, need to take the same route or eat the same food every day). 3. Highly restricted, fixated interests that are abnormal in intensity or focus, (such as strong attachment to or preoccupation with unusual objects, excessively circumscribed or perseverative interests) 4. Hyper-or hypo-reactivity to sensory input or unusual interest in sensory aspects of environment; (such as apparent indifference to pain/heat/cold, adverse response to specific sounds or textures, excessive smelling or touching of objects, visual fascination with lights or movement. C. Syptoms must be present in early childhood (but may not become fully manifest until social demands exceed limited capacities, or may become masked by learned behavior or other mitigating measures). D. Symptoms cause clinically significant impairment in social, occupational, or other important areas of functioning. E. These disturbances are not better explained by intellectual disability or global developmental delay. Intellectual disability and autism spectrum disorder frequently co-occur; to make comorbid diagnoses of autism spectrum disorder and intellectual disability, social communication should be below that expected for general developmental level. Specify: With accompanying intellectual impairment Without accompanying intellectual impairment Without accompanying language impairment With accompanying language impairment Associated with a known medical or geneic condition or environental factor Associated with another neurodevelopmental, mental, or behavioral disorder Specify Severity: Level One - Requiring Support (e.g. decreased social interactions, to-and-fro conversations with others fail). Level Two - Requiring Substantial Support (e.g., speaks simple sentences, limited, narrow, special interests, odd non-veral communication). Level Three - Requiring Very Substantial Support (e.g., child with few intelligible words, rarely initiates interaction, makes unusual approaches). Subject

### SUMMARY DIAGNOSTIC CHECKLISTS TEMPLATES

| | | | | Date | e of A | ssessi | ment:/_ | |
|---|---|---|---|---|---|---|---|---|
| 0 = NO INFORMATIO<br>1 = NOT PRESENT<br>2 = PROBABLE | 4 = IN PA | ARTIAL REMIS | SION*<br>ng to the DSM-5) | 2. Meets<br>criteria r | crite<br>all bi<br>equire | ria for d<br>ut one,<br>ed for ti | ore symptoms o<br>or a minimum of<br>ne diagnosis<br>onal impairment | f 75% of the remainir |
| Ages:<br>Score in years | 1 1 | DIAGNOSIS<br>MOST SEVERE<br>PAST (MSP)<br>EPISODE | AGE OF<br>ONSET<br>MSP<br>EPISODE | | DIAGN<br>CURR<br>EPISC | ENT | AGE OF<br>ONSET<br>OF<br>CURRENT<br>EPISODE | |
| 1. Major Depressive Epis | sode | 0 1 2 3 | | 0 | 1 2 | 3 4 | | |
| 2. Dysthymia | | 0123 | | 0 | 1 2 | 3 4 | | |
| 3. Unspecified Depressi | ve Disorder | 0123 | | 0 | 1 2 | 3 4 | | |
| Adjustment Disorder Depressed Mood | W | 0123 | | 0 | 1 2 | 3 4 | | |
| 5. Mania | | 0123 | | 0 | 1 2 | 3 4 | | |
| 6. Hypmania | | 0123 | | 0 | 1 2 | 3 4 | Ħ | |
| 7. Cyclothymia | | 0123 | | | 1 2 | | Ħ | |
| 8. Bipolar Mixed Episo | de | 0123 | | | 1 2 | | | |
| (MDE & Mania) 9. Hypomania/Mixed Ep | oisode | 0123 | | | 1 2 | | | |
| 10. Unspecified Bipola | Disorder | 0123 | | | 1 2 | | | |
| 11. Unspecified Mood I | Disorder | 0123 | | | | | | |
| 12. Primary Mood Disord | ler w | 0123 | | | 1 2 | | | |
| Psychotic Features 13. Disruptive Mood | | 0123 | | | 1 2 | | | |
| Dysregulation Disord 14. Schlzoaffective Disor | | 0123 | | | 1 2 | | | |
| Schizophrenia | | | | | 1 2 | | | |
| | | 0123 | | 0 | 1 2 | 3 4 | | |
| 1. Schizophreniform Dis | | 0123 | | 0 | 1 2 | 3 4 | | |
| 17. Brief Reactive Psych | | 0123 | 1 1 | 0 | 1 2 | 3 4 | | |
| 1. Unspecified Psycho | otic DO | 0123 | . =1 | 0 | 1 2 | 3 4 | | |
| 896 | 2154 | YEA | R ID | 5-77 | - | | DATE | |

#### SUMMARY LIFETIME DIAGNOSES CHECKLIST DIAGNOSIS AGE OF AGE OF ONSET CURRENT MOST Ages: ONSET SEVERE PAST Score in years. DIAGNOSIS (MSP) MSP CURRENT EPISODE EPISODE EPISODE EPISODE 0 1 2 3 19. Panic Disorder 0 1 2 3 4 20. Agorophobia 0 1 2 3 0 1 2 3 4 21. Separation Aniety DO 0 1 2 3 0 1 2 3 4 22. Social Anxiety DO 0 1 2 3 4 0 1 2 3 23. Selective Mutism 0 1 2 3 4 0 1 2 3 24. Specific Phobia 0 1 2 3 0 1 2 3 4 0 1 2 3 25. Generalized Anxiety DO 0 1 2 3 4 26. Obsessive Compulsive DO 0 1 2 3 0 1 2 3 4 27. Posttaumatic Stress DO 0 1 2 3 0 1 2 3 4 28. Acute Stress Disorder 0 1 2 3 0 1 2 3 4 29. Unspecified Anxiety DO 0 1 2 3 0 1 2 3 4 30. Adjustment Disorder 0 1 2 3 0 1 2 3 4 w Anxious Mood 31. Enuresis 0 1 2 3 0 1 2 3 4 32. Encopresis 0 1 2 3 0 1 2 3 4 33. Anorexia Nervosa 0 1 2 3 0 1 2 3 4 34. Bulimia 0 1 2 3 0 1 2 3 4 0 1 2 3 35. Binge Eating DO 0 1 2 3 4



0 1 2 3

36. Eating DO NOS



0 1 2 3 4

| Ages:<br>Score in years | SEVERE PAST MI | E OF SET SP DIAGNOSIS CURRENT SODE EPISODE | AGE OF ONSET CURRENT EPISODE |
|---|---|---|---|
| 7. ADHD | 0 1 2 3 | 0 1 2 3 4 | |
| | Combined (1)<br>Inattentive (2)<br>Impulsive/Hyperad | Combined<br>O Inattentive<br>otive (3) Impulsive/I | (1)<br>(2)<br>Hyperactive (3) |
| 8. Unspecified ADHD | 0 1 2 3 | 0 1 2 3 4 | |
| 9. Conduct Disorder | 0 1 2 3 | 0 1 2 3 4 | |
| 10. Oppositional Defiant DO | 0 1 2 3 | 0 1 2 3 4 | |
| 11. Unspecified Disruptive Behav | 0 1 2 3 | 0 1 2 3 4 | |
| 42.Adj. Disorder w/Dist.<br>of Conduct | 0 1 2 3 | 01234 | 1 = 1 |
| 43. Adj. Disorder wMixed<br>Mood & Conduct | 0 1 2 3 | 0 1 2 3 4 | |
| 44. Tourettes | 0 1 2 3 | 0 1 2 3 4 | |
| 45. Chronic Motor or | 0 1 2 3 | 0 1 2 3 4 | |
| Vocal Tic Disorder<br>46. Transient Tic DO | 0 1 2 3 | 0 1 2 3 4 | |
| 47, Autism Spectrum DO | 0 1 2 3 | 0 1 2 3 4 | |
| 48. Alcohol Use Disorder | 0 1 2 3 | 01234 | |
| 49. Substance Use Disorder | 0 1 2 3 | 0 1 2 3 4 | |
| 50. Other Diagnoses (specify) | 0 1 2 3 | 0 1 2 3 4 | |
| 51. Other Diagnoses (specify) | 0 1 2 3 | 0 1 2 3 4 | |
| SUBSTANCE INDUCED MOOD A | ND ANXIETY | _ | |
| Substance Induced<br>Mood DO | 0 1 2 3 4 | 0 1 2 3 4 | |
| Specify M | OOD O Mania O Hypom | nania O Mixed O Depression C | Other/ Unknown |
| Substance Induced<br>Anxiety DO | 0 1 2 3 4 | 0 1 2 3 4 | |

| Outpatient Treatment | 0 | 1 | 2 | Psychiatric Hospitalization | 0 | 1 | 2 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Age of First Outpatient<br>Treatment (years) | | | | Age of First Psychiatric<br>Hospitalization (years) | Г | | | SUICIDAL | BE | НА | VIOR: |
| | _ | _ | | | | | _ | Ideation | 0 | 1 | 2 |
| Total Duration of Outpatient<br>Treatment (weeks) | | | | Number of Psychiatric<br>Hospitalizations | | | | Gesture: | 0 | 1 | 2 |
| | | | | Salar Salar Salar | | | | Attempt | 0 | 1 | 2 |
| | | | | Total Duration of Inpatient<br>Treatment (weeks) | | | | - | | | |



| Date of Last A | ssessment: | | | i i |
|---|---|---|---|---|
| 1 = NOT PRESENT 4 = IN<br>2 = PROBABLE | EFINITE<br>PARTIAL REMISS<br>applicable, accord | SION*<br>ing to the DSM-5) | | |
| Ages:<br>Score in years | DIAGNOSIS<br>MOST SEVERE<br>PAST (MSP)<br>EPISODE SINCE<br>LAST<br>INTERVIEW | AGE OF<br>ONSET<br>MSP<br>EPISODE<br>SINCE LAST<br>INTERVIEW | DIAGNOSIS<br>CURRENT<br>EPISODE | AGE OF<br>ONSET<br>OF<br>CURRENT<br>EPISODE |
| 1. Major Depressive Episode | 0 1 2 3 | | 0 1 2 3 4 | |
| 2. Dysthymia | 0123 | | 0 1 2 3 4 | |
| 3. Unspecified Depressive Disorder | 0123 | | 0 1 2 3 4 | |
| Adjustment Disorder w Depressed Mood | 0123 | | 0 1 2 3 4 | |
| 5. Mania | 0123 | - | 0 1 2 3 4 | |
| 6. Hypmania | 0123 | | 0 1 2 3 4 | |
| 7. Cyclothymia | 0123 | | 0 1 2 3 4 | |
| 8. Bipolar Mixed Episode<br>(MDE & Mania) | 0123 | | 0 1 2 3 4 | |
| 9. Hypomania/<br>Mixed Episode | 0 1 2 3 | | 0 1 2 3 4 | |
| 10. Unspecified Bipolar Disorder | 0123 | | 0 1 2 3 4 | |
| 11. Unspecified Mood Disorder | 0123 | | 0 1 2 3 4 | |
| 12. Primary Mood Disorder<br>w Psychotic Features | 0123 | | 0 1 2 3 4 | |
| 13. Disruptive Mood Dysregulation Disorder | 0 1 2 3 | | 0 1 2 3 4 | |
| 14. Schizoaffective Disorder | 0 1 2 3 | | 0 1 2 3 4 | |
| 15. Schizophrenia | 0123 | | 0 1 2 3 4 | |
| 16. Schizophreniform<br>Disorder | 0123 | | 0 1 2 3 4 | |
| 17 Brief Reactive Psychosis | 0123 | 7. 4 | 0 1 2 3 4 | |
| 18. Unspecified Psychotic DO | 0 1 2 3 | | 0 1 2 3 4 | |
| 8962154 | YEA | R ID | | DATE |

| | FOLLOW-UP SUMMARY DIA | AGNOSES CHECKLIST | | 52 |
|---|---|---|---|---|
| Ages:<br>Score in years | DIAGNOSIS AGE OF MOST ONSET SEVERE PAST MSP (MSP) EPISODE EPISODE SINCE SINCE LAST INTERVIEW INTERVIEW | DIAGNOSIS<br>CURRENT<br>EPISODE | AGE<br>OF<br>ONSET<br>CURRENT<br>EPISODE | |
| 19. Panic Disorder | 0 1 2 3 | 0 1 2 3 4 | | |
| 20. Agorophobia<br>Disorder | 0 1 2 3 | 0 1 2 3 4 | | |
| 21. Separation Aniety DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 22. Social Anxiety DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 23. Selective Mutism | 0 1 2 3 | 0 1 2 3 4 | | |
| 24. Specific Phobia | 0 1 2 3 | 0 1 2 3 4 | | |
| 25. Generalized Anxiety DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 26. Obsessive Compulsive DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 27. Posttaumatic Stress DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 28. Acute Stress Disorder | 0 1 2 3 | 0 1 2 3 4 | | |
| 29. Unspecified Anxiety DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 30. Adjustment Disorder w Anxious Mood | 0 1 2 3 | 0 1 2 3 4 | | |
| 31. Enuresis | 0 1 2 3 | 0 1 2 3 4 | | |
| 32. Encopresis | 0 1 2 3 | 0 1 2 3 4 | | |
| 33. Anorexia Nervosa | 0 1 2 3 | 0 1 2 3 4 | | |
| 34. Bulimia | 0 1 2 3 | 0 1 2 3 4 | | |
| 35. Binge Eating DO | 0 1 2 3 | 0 1 2 3 4 | | |
| 36. Eating DO NOS | 0 1 2 3 | 0 1 2 3 4 | | |





| | FOLLOW-U | P SUMMARY DI | AGNOSES CHECKLIS | эт | 53 |
|---|---|---|---|---|---|
| Actes:<br>Score in years | DIAGNOSIS<br>MOST<br>SEVERE PAST<br>(MSP)<br>EPISODE<br>SINCE LAST<br>INTERVIEW | AGE OF<br>ONSET<br>MSP<br>EPISODE<br>SINCE<br>LAST<br>INTERVIEW | DIAGNOSIS<br>CURRENT<br>EPISODE | AGE<br>OF<br>ONSET<br>CURRENT<br>EPISODE | |
| ADHD | 0 1 2 3 | | 0 1 2 3 4 | | |
| | O Combined (1)<br>O Inattentive (2)<br>O Impulsive/Hyp | peractive (3) | O Combined (<br>O Inattentive (<br>O Impulsive/H | 1)<br>2)<br>yperactive (3) | |
| Unspecified ADHD | 0 1 2 3 | | 0 1 2 3 4 | | |
| ). Conduct Disorder | 0 1 2 3 | | 0 1 2 3 4 | | |
| g. Oppositional Defiant DO | 0123 | | 0 1 2 3 4 | | |
| 1. Unspecified Disruptive Behav | 0 1 2 3 | | 0 1 2 3 4 | | |
| 42Adj. Disorder w/Dist.<br>of Conduct | 0 1 2 3 | | 0 1 2 3 4 | | |
| I3. Adj. Disorder w'Mixed<br>Mood & Conduct | 0 1 2 3 | | 0 1 2 3 4 | | |
| 4. Tourettes | 0 1 2 3 | | 0 1 2 3 4 | | |
| 45. Chronic Notor or<br>Vocal Tic Disorder | 0123 | | 0 1 2 3 4 | | |
| 46. Transient Tic DO | 0123 | | 0 1 2 3 4 | | |
| 47. Autism Spectrum DO | 0123 | | 0 1 2 3 4 | | |
| 48. Alcohol Use Disorder | 0123 | | 0 1 2 3 4 | | |
| 19. Substance Use Disorder | 0 1 2 3 | | 0 1 2 3 4 | | |
| 60. Other Diagnoses (specify) | 0 1 2 3 | | 0 1 2 3 4 | | |
| 51. Other Diagnoses (specify) | 0 1 2 3 | | 0 1 2 3 4 | | |
| UBSTANCE INDUCED MOOD A | | | | | |
| Substance Induced<br>Mood DO | 0 1 2 3 | | 0 1 2 3 4 | | |
| Specify Mo | OOD O Mania O H | ypomania O Mix | ed O Depression O | Other/ Unknown | |
| Substance Induced<br>Anxiety DO | 0 1 2 3 | | 0 1 2 3 4 | | |

| Outpatient Treatment | 0 | 1 | 2 | Psychiatric Hospitalization 0 1 2 | | | | |
|---|---|---|---|---|---|---|---|---|
| Age of First Outpatient<br>Treatment (years) | | | | Age of First Psychiatric<br>Hospitalization (years) | SUICIDAL | BE | НА | VIOR: |
| | | | | | Ideation | 0 | 1 | 2 |
| Total Duration of Outpatient Treatment (weeks) | | | | Number of Psychiatric Hospitalizations | Gesture: | 0 | 1 | 2 |
| | | | | Total Duration of Inpatient | Attempt | 0 | 1 | 2 |
| | | | | Treatment (weeks) | | | | |



## AMERICAN PSYCHIATRIC ASSOCIATION DSM-5 CROSS-CUTTING SYMPTOM MEASURES

http://www.psychiatry.org/practice/dsm/dsm5/online-assessment-measures#Level1

#### DSM-5 Parent/Guardian-Rated Level 1 Cross-Cutting Symptom Measure—Child Age 6-17

| Child's Name: | Age: | Sex: Male Female | Date: |
|---|---|---|---|
| Relationship with the child: | | | |
| Instructions (to the parent or guardian of child): The questic question, circle the number that best describes how much (past TWO (2) WEEKS. | | 이 마이지 이 프랑지 나 이번에 아르지 않는데 그렇게 그렇게 하지만데, 그렇게 아르지 않는 | The state of the s |

| | Dur | ing the past <b>TWO (2) WEEKS,</b> how much (or how often) has your child | None<br>Not at<br>all | Slight<br>Rare, less<br>than a day<br>or two | Mild<br>Several<br>days | Moderate<br>More than<br>half the<br>days | Severe<br>Nearly<br>every<br>day | Highest<br>Domain<br>Score<br>(clinician) |
|---|---|---|---|---|---|---|---|---|
| l. | 1. | Complained of stomachaches, headaches, or other aches and pains? | 0 | 1 | 2 | 3 | 4 | |
| | 2. | Said he/she was worried about his/her health or about getting sick? | 0 | 1 | 2 | 3 | 4 | |
| II | 3. | Had problems sleeping—that is, trouble falling asleep, staying asleep, or waking up too early? | 0 | 1 | 2 | 3 | 4 | |
| III. | 4. | Had problems paying attention when he/she was in class or doing his/her homework or reading a book or playing a game? | 0 | 1 | 2 | 3 | 4 | |
| IV. | 5. | Had less fun doing things than he/she used to? | 0 | 1 | 2 | 3 | -4 | |
| | 6. | Seemed sad or depressed for several hours? | 0 | 1 | 2 | 3 | 4 | |
| V. & | 7. | Seemed more irritated or easily annoyed than usual? | 0 | 1 | 2 | 3 | 4 | |
| VI. | 8. | Seemed angry or lost his/her temper? | 0 | 1 | 2 | 3. | 4 | |
| VII. | 9. | Started lots more projects than usual or did more risky things than usual? | 0 | 1 | 2 | 3 | 4 | |
| | 10. | Slept less than usual for him/her, but still had lots of energy? | 0 | 1 | 2 | 3 | 4 | |
| VIII. | 11. | Said he/she felt nervous, anxious, or scared? | 0 | 1 | 2 | 3 | 4 | |
| | 12. | Not been able to stop worrying? | 0 | 1 | 2 | 3 | 4 | |
| | 13. | Said he/she couldn't do things he/she wanted to or should have done, because they made him/her feel nervous? | 0 | 1. | 2 | 3 | 4 | |
| IX. | 14. | Said that he/she heard voices—when there was no one there—speaking about him/her or telling him/her what to do or saying bad things to him/her? | o | 1 | 2 | 3 | 4 | |
| | 15. | Said that he/she had a vision when he/she was completely awake—that is, saw something or someone that no one else could see? | 0 | 1 | 2 | 3 | 4 | |
| X. | 16. | Said that he/she had thoughts that kept coming into his/her mind that he/she would do something bad or that something bad would happen to him/her or to someone else? | 0 | 1 | 2 | 3 | 4 | |
| | 17. | Said he/she felt the need to check on certain things over and over again, like whether a door was locked or whether the stove was turned off? | o | 1 | 2 | 3 | 4 | |
| | 18. | Seemed to worry a lot about things he/she touched being dirty or having germs or being poisoned? | 0 | 1 | 2 | 3 | 4 | |
| | 19. | Said that he/she had to do things in a certain way, like counting or saying<br>special things out loud, in order to keep something bad from happening? | 0 | 1. | 2 | 3 | 4 | |
| | in th | ne past TWO (2) WEEKS, has your child | | | | | | |
| XI. | 20. | Had an alcoholic beverage (beer, wine, liquor, etc.)? | | Yes 🗆 | No | □ Don't | Know | |
| | 21. | Smoked a cigarette, a cigar, or pipe, or used snuff or chewing tobacco? | | Yes 🗆 | No | □ Don't | Know | |
| | 22. | Used drugs like marijuana, cocaine or crack, club drugs (like ecstasy), hallucinogens (like LSD), heroin, inhalants or solvents (like glue), or methamphetamine (like speed)? | | Yes 🗆 | No | □ Don't | Know | |
| | 23. | Used any medicine without a doctor's prescription (e.g., painkillers [like Vicodin], stimulants [like Ritalin or Adderall], sedatives or tranquilizers [like sleeping pills or Valium], or steroids)? | п | Yes 🗆 | No | □ Don't | Know | |
| XII. | 24. | In the past <b>TWO (2) WEEKS,</b> has he/she talked about wanting to kill himself/herself or about wanting to commit suicide? | 0 | Yes 🗆 | No | □ Don't | Know | |
| | 25. | Has he/she EVER tried to kill himself/herself? | | Yes 🗆 | No | ☐ Don't | Know | |

Copyright © 2013 American Psychiatric Association. All Rights Reserved. This material can be reproduced without permission by researchers and by clinicians for use with their patients.

#### Instructions to Clinicians

The DSM-5 Parent/Guardian-Rated Level 1 Cross-Cutting Symptom Measure—Child Age 6-17 assesses mental health domains that are important across psychiatric diagnoses. It is intended to help clinicians identify additional areas of inquiry that may have significant impact on the child's treatment and prognosis. The measure may also be used to track changes in the child's symptom presentation over time.

The measure consists of 25 questions that assess 12 psychiatric domains, including depression, anger, irritability, mania, anxiety, somatic symptoms, inattention, suicidal ideation/attempt, psychosis, sleep disturbance, repetitive thoughts and behaviors, and substance use. Each item asks the parent or guardian to rate how much (or how often) his or her child has been bothered by the specific symptom during the past 2 weeks. The measure was found to be clinically useful and had good test-retest reliability in the DSM-5 Field Trials in pediatric clinical samples across the United States.

#### Scoring and Interpretation

Nineteen of the 25 items on the measure are each rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3≕moderate or more than half the days; and 4=severe or nearly every day). The suicidal ideation, suicide attempt, and substance abuse items are each rated on a "Yes, No, or Don't Know" scale. The score on each item within a domain should be reviewed. Because additional inquiry is based on the highest score on any item within a domain, the clinician is asked to indicate that score in the "Highest Domain Score" column. Table 1 (below) outlines threshold scores that may be used to guide further inquiry for each domain. With the exception of inattention and psychosis, a rating of mild (i.e., 2) or greater on any item within a domain that is scored on the 5-point scale may serve as a guide for additional inquiry and follow-up to determine if a more detailed assessment for that domain is needed. A parent or guardian's rating of "Don't Know" on the suicidal ideation, suicide attempt, and any of the substance use items, especially for a child age 11-17, may be used as a guide for additional inquiry of the issues with the child. The DSM-5 Level 2 Cross-Cutting Symptom measures in Table 1 may be used as a resource to provide more detailed information on the symptoms associated with some of the Level 1 domains.

#### Frequency of Use

To track change in the child's symptom presentation over time, the measure may be completed at regular intervals as clinically indicated, depending on the stability of the child's symptoms and treatment status, and preferably by the same parent or guardian. Consistently high scores on a particular domain may indicate significant and problematic symptoms for the child that might warrant further assessment, treatment, and follow-up. Clinical judgment should guide decision making.

Table 1: DSM-5 Parent/Guardian-Rated Level 1 Cross-Cutting Symptom Measure—Child Age 6-17: domains, thresholds for further

| Domain | Domain Name | Threshold to guide<br>further inquiry | DSM-5 Level 2 Cross-Cutting Symptom Measure available online |
|---|---|---|---|
| l. | Somatic Symptoms | Mild or greater | LEVEL 2—Somatic Symptom—Parent/Guardian of Child Age 6–17 (Patient Health Questionnaire 15 Somatic Symptom Severity (PHQ-15) |
| III. | Sleep Problems | Mild or greater | LEVEL 2—Sleep Disturbance—Parent/ Guardian of Child Age 6–17 (PROMIS—<br>Sleep Disturbance—Short Form) <sup>1</sup> |
| III. | Inattention | Slight or greater | LEVEL 2—Inattention—Parent/Guardian of Child Age 6-17 (SNAP-IV) |
| IV. | Depression | Mild or greater | LEVEL 2—Depression—Parent/Guardian of Child Age 6–17 (PROMIS Emotional Distress—Depression—Parent Item Bank) |
| V. | Anger | Mild or greater | LEVEL 2—Anger—Parent/Guardian of Child Age 6–17 (PROMIS Emotional Distress—Calibrated Anger Measure—Parent) |
| VI. | Irritability | Mild or greater | LEVEL 2—Irritability—Parent/Guardian of Child Age 6–17 (Affective Reactivity Index) |
| VII. | Mania | Mild or greater | LEVEL 2—Mania—Parent/Guardian of Child Age 6–17 (adapted from the Altman Self-Rating Mania Scale) |
| VIII. | Anxiety | Mild or greater | LEVEL 2—Anxiety—Parent/Guardian of Child Age 6–17 (adapted from PROMIS<br>Emotional Distress—Anxiety—Parent Item Bank) |
| IX. | Psychosis | Slight or greater | None |
| Χ. | Repetitive Thoughts<br>and Behaviors | Mild or greater | None |
| XI. | Substance Use | Yes/<br>Don't Know | LEVEL 2—Substance Use—Parent/Guardian of Child Age 6–17 (adapted from the NIDA-modified ASSIST)/LEVEL 2—Substance Use—Child Age 11–17 (adapted from the NIDA-modified ASSIST) |
| XII. | Suicidal Ideation/<br>Suicide Attempts | Yes/<br>Don't Know | None |

Anot validated for children by the PROMIS group but found to have acceptable test-retest reliability with parent informants in the DSM-5 Field Trial.

Copyright © 2013 American Psychiatric Association. All Rights Reserved.

This material can be reproduced without permission by researchers and by clinicians for use with their patients.

#### DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure—Child Age 11-17

| Name: | Age: | Sex: Male Female | Date: |
|---|---|---|---|
| Instructions: The questions below ask about the describes how much (or how often) you have be | and the second s | | |

| | Dur | ing the past <b>TWO (2) WEEKS,</b> how much (or how often) have you | None<br>Not at all | Slight<br>Rare, less<br>than a day<br>or two | Mild<br>Several<br>days | Moderate<br>More than<br>half the<br>days | Severe<br>Nearly<br>every<br>day | Highest<br>Domain<br>Score<br>(clinician |
|---|---|---|---|---|---|---|---|---|
| ١. | 1. | Been bothered by stomachaches, headaches, or other aches and pains? | 0 | 1 | 2 | 3 | 4 | |
| | 2. | Worried about your health or about getting sick? | Ó | 1 | 2 | 3 | 4 | |
| II. | 3. | Been bothered by not being able to fall asleep or stay asleep, or by waking up too early? | 0 | 1 | 2 | 3 | 4 | |
| III | 4. | Been bothered by not being able to pay attention when you were in class or doing homework or reading a book or playing a game? | 0 | 1 | 2 | 3 | 4 | |
| IV. | 5. | Had less fun doing things than you used to? | 0 | 1 | 2 | 3 | 4 | |
| | 6. | Felt sad or depressed for several hours? | 0 | 1 | 2 | 3 | 4 | |
| v. & | 7. | Felt more irritated or easily annoyed than usual? | 0 | 1 | 2 | 3 | 4 | |
| VI. | 8. | Felt angry or lost your temper? | 0 | 1 | 2 | 3 | 4 | |
| VII. | 9. | Started lots more projects than usual or done more risky things than usual? | 0 | 1 | 2 | 3 | 4 | |
| | 10. | Slept less than usual but still had a lot of energy? | 0 | 1 | 2 | 3 | 4 | |
| VIII. | 11. | Felt nervous, anxious, or scared? | 0 | 1 | 2 | 3 | 4 | |
| | 12. | Not been able to stop worrying? | 0 | 1 | 2 | 3 | 4 | |
| | 13. | Not been able to do things you wanted to or should have done, because they made you feel nervous? | 0 | 1 | 2 | 3 | 4 | |
| IX. | 14. | Heard voices—when there was no one there—speaking about you or telling you what to do or saying bad things to you? | 0 | 1 | 2 | 3 | 4 | |
| | 15. | Had visions when you were completely awake—that is, seen something or someone that no one else could see? | 0 | 1 | 2 | 3 | 4 | |
| X. | 16. | Had thoughts that kept coming into your mind that you would do something bad or that something bad would happen to you or to someone else? | 0 | 1 | 2 | 3 | 4 | |
| | 17. | Felt the need to check on certain things over and over again, like whether a door was locked or whether the stove was turned off? | 0 | 1 | 2 | 3 | 4 | |
| | 18. | Worried a lot about things you touched being dirty or having germs or being poisoned? | 0 | 1 | 2 | 3 | 4 | |
| | 19. | Felt you had to do things in a certain way, like counting or saying special things, to keep something bad from happening? | 0 | 1 | 2 | 3 | 4 | |
| | in th | ne past TWO (2) WEEKS, have you | | | | | | |
| XI. | 20. | Had an alcoholic beverage (beer, wine, liquor, etc.)? | | ☐ Yes | | 0 1 | No | |
| | 21, | Smoked a cigarette, a cigar, or pipe, or used snuff or chewing tobacco? | - 01 | ☐ Yes | 9.1 | 0 1 | No | |
| | 22. | Used drugs like marijuana, cocaine or crack, club drugs (like Ecstasy), hallucinogens (like LSD), heroin, inhalants or solvents (like glue), or methamphetamine (like speed)? | | □ Yes | | <b>-</b> | No | |
| | 23. | Used any medicine without a doctor's prescription to get high or change the way you feel (e.g., painkillers [like Vicodin], stimulants [like Ritalin or Adderall], sedatives or tranquilizers [like sleeping pills or Valium], or steroids)? | 1 | □ Yes | 7 | 0 1 | No | |
| XII. | 24. | In the last 2 weeks, have you thought about killing yourself or committing suicide? | 1 | □ Yes | | | No | |
| | 25. | Have you EVER tried to kill yourself? | | ☐ Yes | | | No | |

 $Copyright @ 2013 \ American Psychiatric Association. All Rights Reserved. \\ This material can be reproduced without permission by researchers and by clinicians for use with their patients.$ 

#### Instructions to Clinicians

The DSM-5 Level 1 Cross-Cutting Symptom Measure is a self-rated measure that assesses mental health domains that are important across psychiatric diagnoses. It is intended to help clinicians identify additional areas of inquiry that may have significant impact on the child's treatment and prognosis. In addition, the measure may be used to track changes in the child's symptom presentation over time.

This child-rated version of the measure consists of 25 questions that assess 12 psychiatric domains, including depression, anger, irritability, mania, anxiety, somatic symptoms, inattention, suicidal ideation/attempt, psychosis, sleep disturbance, repetitive thoughts and behaviors, and substance use. Each item asks the child, age 11–17, to rate how much (or how often) he or she has been bothered by the specific symptom <u>during the past 2 weeks</u>. The measure was found to be clinically useful and had good test-retest reliability in the DSM-5 Field Trials conducted in pediatric clinical samples across the United States.

#### Scoring and Interpretation

Nineteen of the 25 items on the measure are each rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day). The suicidal ideation, suicide attempt, and substance abuse items are each rated on a "Yes or No" scale. The score on each item within a domain should be reviewed. Because additional inquiry is based on the highest score on any item within a domain, the clinician is asked to indicate that score in the "Highest Domain Score" column. Table 1 (below) outlines threshold scores that may be used to guide further inquiry for the domains. With the exception of inattention and psychosis, a rating of mild (i.e., 2) or greater on any item within a domain that is scored on the 5-point scale may serve as a guide for additional inquiry and follow-up to determine if a more detailed assessment for that domain is needed. The DSM-5 Level 2 Cross-Cutting Symptom measures listed in Table 1 may be used as a resource to provide more detailed information on the symptoms associated with some of the Level 1 domains.

#### Frequency of Use

To track change in the child's symptom presentation over time, it is recommended that the measure be completed at regular intervals as clinically indicated, depending on the stability of the child's symptoms and treatment status. Consistently high scores on a particular domain may indicate significant and problematic symptoms for the child that might warrant further assessment, treatment, and follow-up. Clinical judgment should guide decision making.

Table 1: DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure—Child Age 11–17: domains, thresholds for further inquiry, and associated Level 2 measures

| Domain | Domain Name | Threshold to guide<br>further inquiry | DSM-5 Level 2 Cross-Cutting Symptom Measure available online |
|---|---|---|---|
| ŀ | Somatic Symptoms | Mild or greater | LEVEL 2—Somatic Symptom—Child Age 11–17 (Patient Health Questionnaire Somatic Symptom Severity [PHQ-15]) |
| II. | Sleep Problems | Mild or greater | LEVEL 2—Sleep Disturbance—Child Age 11-17 (PROMIS—Sleep Disturbance—<br>Short Form) <sup>1</sup> |
| III. | Inattention | Slight or greater | None |
| IV. | Depression | Mild or greater | LEVEL 2—Depression—Child Age 11–17 (PROMIS Emotional Distress—<br>Depression—Pediatric Item Bank) |
| V. | Anger | Mild or greater | LEVEL 2—Anger—Child Age 11–17 (PROMIS Emotional Distress—Calibrated<br>Anger Measure—Pediatric) |
| VI. | Irritability | Mild or greater | LEVEL 2—Irritability—Child Age 11-17 (Affective Reactivity Index [ARI]) |
| VII. | Mania | Mild or greater | LEVEL 2-Mania-Child Age 11-17 (Altman Self-Rating Mania Scale [ASRM]) |
| VIII. | Anxiety | Mild or greater | LEVEL 2—Anxiety—Child Age 11–17 (PROMIS Emotional Distress—Anxiety—<br>Pediatric Item Bank) |
| IX. | Psychosis | Slight or greater | None |
| X. | Repetitive Thoughts<br>& Behaviors | Mild or greater | LEVEL 2—Repetitive Thoughts and Behaviors—Child 11–17 (adapted from the Children's Florida Obsessive-Compulsive Inventory [C-FOCI] Severity Scale) |
| XI: | Substance Use | Yes/<br>Don't Know | LEVEL 2—Substance Use—Child Age 11–17 (adapted from the NIDA-modified ASSIST) |
| XII. | Suicidal Ideation/<br>Suicide Attempts | Yes/<br>Don't Know | None |

Not validated for children by the PROMIS group but found to have acceptable test-retest reliability with child informants in the DSM-5 Field Trial.

Copyright © 2013 American Psychiatric Association. All Rights Reserved.

This material can be reproduced without permission by researchers and by clinicians for use with their patients.

#### 10.6 Columbia-Suicide Severity Rating Scales (C-SSRS)

## COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Lifetime Recent - Clinical

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in **The Columbia Suicide History Form**, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103 -130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

#### © 2008 The Research Foundation for Mental Hygiene, Inc.

| Ask questions 1 and 2. If both are negative, proceed to " | Cuicidal Relamine" section If the appropria | | | | | |
|---|---|---|---|---|---|---|
| question 2 is "yes", ask questions 3, 4 and 5. If the answer | | He/SI | ie: Time<br>he Felt<br>Suicidal | | st 1<br>nth | |
| "Intensity of Ideation" section below. 1. Wish to be Dead | | 111036 | , and the same | | - | |
| Subject endorses thoughts about a wish to be dead or not alive anymore<br>Have you wished you were dead or wished you could go to sleep and a | | Yes | No | Ves | No | |
| If yes, describe: | | 1 | | | | |
| <ol> <li>Non-Specific Active Suicidal Thoughts General non-specific thoughts of wanting to end one's life/commit suici of ways to kill oneself/associated methods, intent, or plan during the ass Have you actually had any thoughts of killing yourself?</li> </ol> | | Yes | No □ | Ves | No | |
| If yes, describe: | | | | | | Yes D |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) Subject endorses thoughts of suicide and has thought of at least one met specific plan with time, place or method details worked out (e.g., though who would say, "I thought about toking on overdose but I never made a it, and I would never go through with it." Have you been thinking about how you might do this? | hod during the assessment period. This is different than a-<br>nt of method to kill self but not a specific plan). Includes person | Yes | No | | No. | |
| If yes, describe: | | | | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, with Active suicidal thoughts of killing oneself and subject reports baying 80 thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on their | me intent to act on such thoughts, as opposed to "I have the | Yes | No. | 120 | No | |
| Il'yes, describe: | | | | | | |
| <ol> <li>Active Suicidal Ideation with Specific Plan and Intent<br/>Thoughts of killing oneself with details of plan fully or partially worked<br/>Have you started to work out or worked out the details of how to kill years.</li> <li>If yes, describe:</li> </ol> | | Yes | No. | 10000 | No | |
| INTENSITY OF IDEATION | was the state of t | _ | | | _ | |
| The following features should be rated with respect to the most:<br>the least severe and 5 being the most severe). Ask about time he | | | | | | |
| Lifetime - Most Severe Ideation: | Description of Idealian | | ost<br>vere | 100000 | | |
| Recent - Most Severe Ideation: | Description of Ideaton | 2 | 0.17 | 341 | 27 | |
| Frequency | trescription of mention | | | - | - | |
| How many times have you had these thoughts? | | | | | | |
| (1) Less than once a week (2) Once a week (3) 2-5 times in we<br>Duration | ek (4) Daily or almost daily (5) Many times each day | ~ | _ | - | - | |
| When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than I hour/some of the time (3) 1-4 hours/a lot of time | (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | - | | - | - | |
| Controllability | | | | | | |
| Could/can you stop thinking about killing yourself or want. (1) Easily able to central houghts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | 6 | | - | | |
| Deterrents | | | | | | |
| Are there things - anyone or anything (e.g., family, religion<br>die or acting on thoughts of committing suicide?<br>(1) Deterrents definitely stopped you from attempting suicide<br>(2) Deterrents probably stopped you<br>(3) Uncertain that deterrents stopped you | (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | 2 | - | _ | - | |
| Reasons for Ideation | | | | | | |
| What sort of reasons did you have for thinking about wants or stop the way you were feeling (in other words you could feeling) or was it to get attention, revenge or a reaction from (1) Completely to get attention, revenge or a reaction from others (2) Mostly to get attention, revenge or a reaction from others (3) Equally to get attention, revenge or a reaction from others and to end/stop the pain | t't go on living with this pain or how you were | - | | - | - | |

| SUICIDAL BEHAVIOR<br>(Check all that apply, so long as these are separate events; must ask about all types) | | Life | etime | | st 3 |
|---|---|---|---|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as oneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger we mouth but gun is broken so injury results, this is considered an attempt. Interring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstance highly tethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping fro high floor/story). Also, it someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. | an actual suicide<br>hile gun is in<br>as. For example, a<br>no window of a | | No | Yes | No 🖂 |
| Have you made a suicide attempt? Have you done anything to harm yourself? Have you done anything dangerous where you could have died? What did you do? Did you as a way to end your life? Did you want to die (even a little) when you ? Were you trying to end your life when you ? Or Did you think it was possible you could have died from ? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stres | s, feel better. | | al# of<br>empts | | al # of<br>empts |
| get sympathy, or get something else to happen)? (Self-lajurious Behavior without suicidal intent) If yes, describe: | | | 4.0 | | 1011 |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | Yes | No | Ves | No C |
| Interrupted Attempt: | | | | 100 | |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actualized accurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather that attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pull they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down Hunging: Person has noose around neek but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stop, you actually did anything? If yes, describe: | an an interrupted<br>ling trigger. Once<br>a from ledge | e Tota | No I al # of rupted | | No |
| n yes, describe. | | | _ | - | - |
| Aborted or Self-Interrupted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of bein something else. Has there been a time when you started to do something to try to end your life but you stopped yourself actually dld anything? If yes, describe: | g stopped by | abor | No al # of ted or cif- | abor | No II # of ted or alf-rupted |
| Bushnustom: Ante on Dahardan | | 10- | = | - | |
| Preparatory Acts or Behavior: Acts or preparation towards annumently making a suicide attempt. This can include anything beyond a verbalization or though assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things suicide note). | | Ves | No. | Yes | No |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collect getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | ing pills, | prepa | al # of<br>aratory<br>ects | prepa | al # of<br>anatory<br>ets |
| | Most Recent<br>Attempt<br>Date: | Most Lett<br>Attempt<br>Date: | | Initial/F<br>Attempt<br>Date: | |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding, sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns loss than 20% of body; extensive blood loss butcan recover, major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with instable vital signs; major damage to a vital area). 5. Death | Enter Code | Enler C | Code | Enter | Code |
| Detential Lethality: Only Answer if Actual Lethality=0 Likely tethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious tethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying, on train tracks with oncoming train but pulled away before run over). | Enier Code | Enter C | Tode | Enter | Code |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | _ | | | | |

© 2008 Research Foundation for Mental Hygiene, Inc.

C-5SR5—Lifetime Recent - Clinical (Version 1/14/09)

Page 2 of 2

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit - Clinical

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in **The Columbia Suicide History Form**, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience
of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY,
10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and
limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103
-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

| SUICIDAL IDEAT | ION | | | |
|---|---|---|---|---|
| | | | 1000 | e Las<br>isit |
| | | | Yes | No |
| If yes, describe: | | to be dead or not alive anymore, or wish to fall asteep and not wake up. It Thoughts Ing to end one's hielecommit suicide (e.g., "I've thought about killing anyault") without thoughts of ways to kill plan during the assessment period. If It Houghts Ing to end one's hielecommit suicide (e.g., "I've thought about killing anyault") without thoughts of ways to kill plan during the assessment period. If Alling yourself? In Any Methods (Not Plan) without Intent to Act Ind has thought of at least one motion seed in the assessment period. This is different than a specific plan with time, g., thought of nichaod to kill self but not a specific plan. Includes person who would any. "I thought about taking an for as to when, where or how I would actually do II. and I would never go through with II." In Some Intent to Act, without Specific Plan self and subject reports having some intent to act an aucht thoughts, as opposed to "I have the thoughts but I some intention of acting on them? In Specific Plan and Intent In Specific Plan and Intent In Open Intent to a plan and Intent In Specific Plan and Inte | | |
| | of wanting to end one's life/commit sui<br>tent, or plan during the assessment perio | | Ves | No. |
| If yes, describe: | | | - | |
| Subject endorses thoughts of seplace or method details worked | uicide and has thought of at least one mod<br>d out (e.g., thought of method to kill self<br>occific plan as to when, where or how I w | chod during the assessment period. This is different than a specific plan with time,<br>but not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| 4. Active Suicidal Ideati<br>Active suicidal thoughts of kill<br>definitely will not do anything | ling oneself and subject reports having so | ome intent to act on such thoughts, as opposed to "I have the thoughts but I | Yes | No |
| Thoughts of killing oneself wit | | d out and subject has some intent to carry it out. | Ves | No |
| INTENSITY OF IDEATION | | | | |
| The following features show<br>and 5 being the most severe | | severe type of ideation (i.e., I-5 from above, with I being the least severe | | ost |
| Most Severe Ideation: | Tona # (7.5) | Description of Ideation | Sev | vere |
| Frequency How many times have you (1) Less than once a weel | u had these thoughts? | X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X X | - | |
| Duration When you have the thoug (1) Fleeting - few second (2) Less than 1 hour/som (3) 1-4 hours/a lot of time | e of the time. | | - | |
| Controllability Could/can you stop think (1) Basily able to control (2) Can control thoughts (3) Can control thoughts | froughts with little difficulty | (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts | _ | |
| thoughts of committing so | uicide?<br>stopped you from attempting suicide<br>stopped you | (4) Deterrents most likely did not stop you<br>(5) Deterrents definitely did not stop you | | |
| Reasons for Ideation<br>What sort of reasons did<br>you were feeling (in other<br>revenge or a reaction fro<br>(1) Completely to get atten<br>(2) Mostly to get attention. | you have for thinking about warn<br>r words you couldn't go on thing<br>m others? Or both?<br>dion, revenge or a reaction from others<br>, revenge or a reaction from others<br>, revenge or a reaction from others | ting to die or killing yourself? Was it to end the pain or stop the way with this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) | | |

© 2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Since Last Visit - Clinical (Version 1/14/09)

Page I of 2

| SUICIDAL BEHAVIOR<br>(Check all that apply, so long as these are separate events; must ask about all types) | Since Last<br>Visit |
|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an actual societe attempt. There does not | Yes No |
| have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, this is considered an attempt. | 0 0 |
| Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies ment to die, but they thought that what they did could be lethal, intent may be inferred. | |
| Have you made a suicide attempt? | |
| Have you done anything to harm yourself?<br>Have you done anything dangerous where you could have died?<br>What did you do? | Total # of<br>Attempts |
| Did you as a way to end your life? | 1 |
| Did you want to die (even a little) when you ? | _ |
| Were you trying to end your life when you? Or did you think it was possible you could have died from? | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get | |
| sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) I yes, describe: | Ves No |
| | D D |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | 100 |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have necessarily before the person in the person in the person in the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have necessarily before the person in the person in the person in the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have necessarily before the person in the person in the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have necessarily before the person in the person in the person in the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have necessarily before the person in the perso | Yes No |
| Overdose, Person has pills in hand but is stopped from ingesting. Once they trigest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken many by someone else, or is somehow prevented from pullting trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around | |
| neck but has not yet started to hang - is stopped from doing so.<br>Has there been a time when you started to do something to end your life but someone or something stopped you before you | Total # of |
| next ally did anything? | interrupted |
| fyes, describe. | _ |
| Aborted or Self-Inferrupted Attempt; When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. | Yes No |
| Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you includely did anything? If yes, describe: | Total # of<br>aborted or<br>self- |
| | interrupted |
| Preparatory Acts or Behavior:<br>Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a | Yes No |
| specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide altempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? | Total # of |
| If yes, describe: | preparatory<br>acts |
| Suicide: | Yes No |
| Death by snicide occurred smee last assessment. | |
| | Most Lethal<br>Attempt<br>Date: |
| Actual Lethality/Medical Damage: 1. No physical damage or very minor physical damage (e.g., surface scratches). | Enter Code |
| Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree burns lass than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; | |
| extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying ontrain tracks with oncoming train but pulled away before run over). | Enter Code |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result indeath despite available medical care | |
| © 2008 Research Foundation for Montal Physicine, Inc. C-SSRS—Since Last Visit - Clinical (Version 1/14/09) | Page 2 of 2 |

#### 10.7 Swanson, Nolan and Pelham Rating Scale-Revised (SNAP IV)

| For each item, check the column which best describes this child | Not At | Just A<br>Little | Pretty<br>Much | Yery<br>Much |
|---|---|---|---|---|
| . Fails to give close attention to details or makes careless mistakes in schoolwork or tasks | | | | |
| 2 Has difficulty sustaining attention in tasks or play activities | 200 | | | |
| 3. Does not seem to listen when spoken to directly | - | | | |
| Does not follow through on instructions and fails to finish schoolwork, chores, or duties | | | | |
| 5. Has difficulty organizing tasks and activities | | | | |
| 8. Avoids, dislikes, or reluctantly engages in tasks requiring sustained mental effort | | | | |
| Loses things necessary for activities (e.g., toys, school assignments, pencils, or books) | | 1 - 3 | | 1 |
| 3. Is distracted by extraneous stimuli | 1 | | | |
| ). Is forgetful in daily activities | | | | |
| 0. Fidgets with hands or feet or squirms in seat | | | 1- 3 | |
| 1. Leaves seat in classroom or in other situations in which remaining seated is expected | | | | |
| 2. Runs about or climbs excessively in situations in which it is inappropriate | | | | |
| 3. Has difficulty playing or engaging in leisure activities quietly | | | | |
| 4. Is "on the go" or often acts as if "driven by a motor" | | | | |
| 5. Talks excessively | 1 | | | |
| 6. Blurts out answers before questions have been completed | | | | |
| 7. Has difficulty awaiting turn | | | | |
| 8. Interrupts or intrudes on others (e.g., butts into conversations / games) | | | - | |
| 9. Loses temper | | | | |
| 0. Argues with adults | | | | |
| 1. Actively defies or refuses adult requests or rules | | - | | |
| 2. Deliberately does things that annoy other people | | | | |
| 3. Blames others for his or her mistakes or misbehavior | | | | |
| 4. Is touchy or easily annoyed by others | | | | |
| 5. Is angry and resentful | | | | 1 |
| 6 le spiteful or vindictive | | | - | |

Rater Initials: \_\_\_\_\_

#### 10.8 Simpson-Angus Rating Scale

#### 1. GAIT

The patient is examined as he walks into the examining room, his gait, the swing of his arms, his general posture, all form the basis for an overall score for this item. This is rated as follows:

- 0 = Normal
- 1 = Diminution in swing while the patient is walking
- 2 = Marked diminution in swing with obvious rigidity in the arm
- 3 = Stiff gait with arms held rigidly before the abdomen
- 4 = Stopped shuffling gait with propulsion and retropulsion

#### 2. ARM DROPPING:

The patient and the examiner both raise their arms to shoulder height and let them fall to their sides. In a normal subject, a stout slap is heard as the arms hit the sides. In the patient with extreme Parkinson's syndrome, the arms fall very slowly:

- 0 = Normal, free fall with loud slap and rebound
- 1 = Fall slowed slightly with less audible contact and little rebound
- 2 = Fall slowed, no rebound
- 3 = Marked slowing, no slap at all
- 4 = Arms fall as though against resistance; as though through glue

#### 3. SHOULDER SHAKING:

The subject's arms are bent at a right angle at the elbow and are taken one at a time by the examiner who grasps one hand and also clasps the other around the patient's elbow. The subject's upper arm is pushed to and fro and the humerus is externally rotated. The degree of resistance from normal to extreme rigidity is scored as follows.

- 0 = Normal
- 1 = Slight stiffness and resistance
- 2 = Moderate stiffness and resistance

- 3 = Marked rigidity with difficulty in passive movement
- 4 = Extreme stiffness and rigidity with almost a frozen shoulder

#### 4. ELBOW RIGIDITY:

The elbow joints are separately bent at right angles and passively extended and flexed, with the subject's biceps observed and simultaneously palpated. The resistance to this procedure is rated. (The presence of cogwheel rigidity is noted separately.)

- 0 = Normal
- 1 = Slight stiffness and resistance
- 2 = Moderate stiffness and resistance
- 3 = Marked rigidity with difficulty in passive movement
- 4 = Extreme stiffness and rigidity with almost a frozen shoulder

#### 5. WRIST RIGIDITY or Fixation of position:

The wrist is held in one hand and the fingers held by the examiner's other hand, with the wrist n1oved to extension, flexion and ulner and radial deviation:

- 0 = Normal
- 1 = Slight stiffness and resistance
- 2 = Moderate stiffness and resistance
- 3 = Marked rigidity with difficulty in passive movement
- 4 = Extreme stiffness and rigidity with almost a frozen shoulder

#### 6. LEG PENDULOUSNESS:

The patient sits on a table with his legs hanging down and swinging free. The ankle is grasped by the examiner and raised until the knee is partially extended. It is then allowed to fall. The resistance to falling and the Jack of swinging form the basis for the score on this item:

- 0 = The legs swing freely
- 1 = Slight diminution in the swing of the legs

- 2 = Moderate resistance to swing
- 3 = Marked resistance and damping of swing
- 4 = Complete absence of swing

#### 7. HEAD DROPPING:

The patient lies on a well-padded examining table and his head is raised by the examiner's hand. The hand is then withdrawn and the head allowed to drop. In the normal subject the head will fall upon the table. The movement is delayed in extrapyramidal system disorder and in extreme parkinsonism it is absent. The neck muscles are rigid and the head docs not reach the examining table. Scoring is as follows:

- 0 = The head falls completely with a good thump as it hits the table
- 1 = Slight slowing in fall, mainly noted by lack of slap as head meets the table
- 2 = Moderate slowing in the fall quite noticeable to the eye
- 3 = Head falls stiffly and slowly
- 4 = Head does not reach the examining table

#### 8. GLABELLA TAP:

Subject is told to open eyes wide and not to blink. The glabella region is tapped at a steady, rapid speed. The number of times patient blinks in succession is noted:

- 0 = 0 5 blinks
- 1 = 6 10 blinks
- 2 = 11 15 blinks
- 3 = 16 20 blinks
- 4 = 21 and more blinks

#### 9. TREMOR:

Patient is observed walking into examining room and is then reexamined for this item:

0 = Normal

- 1 = Mild finger tremor, obvious to sight and touch
- 2 = Tremor of hand or arm occurring spasmodically
- 3 = Persistent tremor of one or more limbs
- 4 = Whole body tremor
- 10. SALIVATION:

Patient is observed while talking and then asked to open his mouth and elevate his tongue. The following ratings are given:

- 0 = Normal
- 1 = Excess salivation to the extent that pooling takes place if the mouth is open and the tongue raised.
- 2 = When excess salivation is present and might occasionally result in difficulty in speaking
- 3 = Speaking with difficulty because of excess salivation
- 4 = Frank drooling

#### 10.9 Barnes Akathisia Rating Scale (BARS)

| Name: | Park. |
|-------|-------|
| name: | Date: |

#### Barnes Akathisia Rating Scale (BARS)

**Instructions:** Patient should be observed while they are seated, and then standing while engaged in neutral conversation (for a minimum of two minutes in each position). Symptoms observed in other situations, for example while engaged in activity on the ward, may also be rated. Subsequently, the subjective phenomena should be elicited by direct questioning.

#### Objective

- Normal, occasional fidgety movements of the limbs
- Presence of characteristic restless movements: shuffling or tramping movements of the legs/feet, or swinging of one leg while sitting, and/or rocking from foot to foot or "walking on the spot" when standing, but movements present for less than half the time observed
- Observed phenomena, as described in (1) above, which are present for at least half the observation period
- Patient is constantly engaged in characteristic restless movements, and/or has the inability to remain sealed or standing without walking or pacing, during the time observed

#### Subjective

#### Awareness of restlessness

- 0 Absence of inner restlessness
- 1 Non-specific sense of inner restlessness
- The patient is aware of an inability to keep the legs still, or a desire to move the legs, and/or complains of inner restlessness aggravated specifically by being required to stand still
- 3 Awareness of intense compulsion to move most of the time and/or reports strong desire to walk or pace most of the time

#### Distress related to restlessness

- No distress
- 1 Mild
- 2 Moderate
- 3 Severe

#### Global Clinical Assessment of Akathisia

- Absent. No evidence of awareness of restlessness. Observation of characteristic movements of akathisia in the absence of a subjective report of inner restlessness or compulsive desire to move the legs should be classified as pseudoakathisla
- Questionable. Non-specific inner tension and fidgety movements
- 2 Mild akathisia. Awareness of restlessness in the legs and/or inner restlessness worse when required to stand still. Fidgety movements present, but characteristic restless movements of akathisia not necessarily observed. Condition causes little or no distress.
- 3 Moderate akathisia. Awareness of restlessness as described for mild akathisia above, combined with characteristic restless movements such as rocking from foot to foot when standing. Patient finds the condition distressing
- 4 Marked akathisia. Subjective experience of restlessness includes a compulsive desire to walk or pace. However, the patient is able to remain seated for at least five minutes. The condition is obviously distressing.
- 5 Severe akathisia. The patient reports a strong compulsion to pace up and down most of the time. Unable to sit or lie down for more than a few minutes. Constant restlessness which is associated with intense distress and insomnia.

#### Scoring the Barnes Akathisia Rating Scale (BARS)

The Barnes Akathisia Rating Scale is scored as follows:

Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness are rated on a 4-point scale from 0-3 and are summed yielding a total score ranging from 0 to 9.

The Global Clinical Assessment of Akathisia uses a 5-point scale ranging from 0-4.

Citation: Barnes TR: A Rating Scale for Drug-Induced Akathisia. British Journal of Psychiatry 154:672-676, 1989.

#### 10.10 Abnormal Involuntary Movement Scale (AIMS)

Abnormal Involuntary Movement Scale (AIMS)

### Abnormal Involuntary Movement Scale (AIMS)

www.cnsforum.com

Abnormal Involuntary Movement Scale (AIMS)

#### **Examination Procedure**

Either before or after completing the examination procedure, observe the patient unobtrusively at rest (e.g., in the waiting room).

The chair to be used in this examination should be a hard, firm one without arms.

- Ask the patient whether there is anything in his or her mouth (such as gum or candy) and,
  if so, to remove it.
- Ask about the \*current\* condition of the patient's teeth. Ask if he or she wears dentures.
   Ask whether teeth or dentures bother the patient \*now\*.
- 3. Ask whether the patient notices any movements in his or her mouth, face, hands, or feet. If yes, ask the patient to describe them and to indicate to what extent they \*currently\* bother the patient or interfere with activities.
- 4. Have the patient sit in chair with hands on knees, legs slightly apart, and feet flat on floor. (Look at the entire body for movements while the patient is in this position.)
- Ask the patient to sit with hands hanging unsupported if male, between his legs, if female and wearing a dress, hanging over her knees. (Observe hands and other body areas).
- Ask the patient to open his or her mouth. (Observe the tongue at rest within the mouth.)Do this twice.
- Ask the patient to protrude his or her tongue. (Observe abnormalities of tongue movement.) Do this twice.
- Ask the patient to tap his or her thumb with each finger as rapidly as possible for 10 to 15 seconds, first with right hand, then with left hand. (Observe facial and leg movements.)
- Flex and extend the patient's left and right arms, one at a time.
- Ask the patient to stand up. (Observe the patient in profile, Observe all body areas again, hips included.)
- Ask the patient to extend both arms out in front, palms down. (Observe trunk, legs, and mouth.)
- Have the patient walk a few paces, turn, and walk back to the chair. (Observe hands and gait.) Do this twice.

| Patient Information | | | | | | | |
|---------------------|------|-----|------|------|------|------|-----|
| Patient | Date | Day | Mth. | Year | Time | Hour | Mir |
| Personal notes | | | | | | | |

#### **Scoring Procedure**

Complete the examination procedure before making ratings. For the movement ratings (the first three categories below), rate the highest severity observed. 0 = none, 1 = minimal (may be extreme normal), 2 = mild, 3 = moderate, 4 = severe. According to the <u>original</u> AIMS instructions, one point is subtracted if movements are seen **only on activation**, but not all investigators follow that convention.

| Facial and Oral Movements | |
|---|---|
| Muscles of facial expression, e.g., movements of forehead, eyebrows, periorbital area, cheeks. Include frowning, blinking, grimacing of upper face. | 0 1 2 2 3 4 |
| Lips and perioral area, e.g., puckering, pouting, smacking. | 0 1 1 2 3 3 4 |
| 3. Jaw, e.g., biting, clenching, chewing, mouth opening, lateral movement. | 0 0 1 2 2 3 4 |
| 4. Tongue. Rate only increase in movement both in and out of mouth, not inability to sustain movement. | 0<br>1<br>2<br>3<br>4 |

www.cnsforum.com

| Extremity Movements | |
|---|---|
| v | T |
| 5. Upper (arms, wrists, hands, fingers). Include movements that are choreic (rapid, objectively purposeless, irregular, spontaneous) or athetoid (slow, irregular, complex, serpentine). Do not include tremor (repetitive, regular, rhythmic movements). | 0<br>1<br>2<br>3<br>4 |
| 6. Lower (legs, knees, ankles, toes), e.g., lateral knee movement, foot tapping, heel dropping, foot squirming, inversion and eversion of foot. | 0 1 1 2 3 4 |
| Trunk Movements | |
| 7. Neck, shoulders, hips, e.g., rocking, twisting, squirming, pelvic gyrations. Include diaphragmatic movements. | 0 1 2 3 4 |
| Global Judgements | |
| 8. Severity of abnormal movements. Based on the highest single score on the above items. | □ 0<br>□ 1<br>□ 2<br>□ 3<br>□ 4 |
| 9. Incapacitation due to abnormal movements. | none, normal minimal mild moderate severe |
| 10. Patient's awareness of abnormal movements. | no awareness aware, no distress aware, mild distress aware, moderate distress aware, severe distress |

www.cnsforum.com

4

| Dental status | |
|--------------------------------------------------|----------|
| 11. Current problems with teeth and/or dentures. | ☐ no yes |
| 2. Does patient usually wear dentures? | □ no |

www.cnsforum.com

5

#### 10.11 Child Health Questionnaire Parent Form 28-item (CHQ-PF28)

| П | | | | | $\Box$ | | ODAY'S D | ATE |
|---|---|---|---|---|---|---|---|---|
| ID NU | MBER | | | M | ONTH | DAY | Y | EAR |
| - | | | | | | | | |
| are no | right or wrong r | responses. If you are | ir child's health and we<br>unsure how to respond | | | | | |
| that yo | ou fill in each qu | estion. Please use blu | ue or black ink. | | | | | |
| Corre | ct Marks: | X M = | | | | | | |
| | | | | | 2 | ППГ | | |
| 050 | TION 4. VOUD | CHILDING CO DEAL IN | TATE TO THE PARTY OF THE PARTY | | 11 | | | |
| SEC | FION 1: YOUR | CHILD'S GLOBAL H | Exce | lent Very good | G | ood | Fair | Po |
| 1.1. | In general, wo | ould you say your child | s's health is: | | | | | |
| | 1 1 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | | | | | |
| | | CHILD'S PHYSICAL | | | | | | |
| | | | ACTIVITIES al activities your child r | night do during a day | <b>V</b> | | | |
| | following questi<br>During the pa | ions ask about physica<br>st 4 weeks, has your | al activities your child r<br>child been limited in an | | Yes, | Yes, | Yes, | |
| The | following questi<br>During the pa | ions ask about physica | al activities your child r<br>child been limited in an | | Yes,<br>limited | limited | limited | 100 |
| The | following questi During the pa the following a a. Doing thing | ions ask about physica<br>st 4 weeks, has your of<br>activities due to health<br>gs that take a lot of en | al activities your child r<br>child been limited in an | y of | Yes, | | and the second second | limite |
| The | following questi<br>During the pa<br>the following a<br>a. Doing thing<br>or running | ions ask about physical<br>ist 4 weeks, has your of<br>activities due to health<br>gs that take a lot of er<br>? | al activities your child r<br>child been limited in an<br>n problems?<br>nergy, such as playing | y of soccer, | Yes,<br>limited<br>a lot | limited<br>some | limited<br>a little | limite |
| The | During the pa<br>the following a<br>a. Doing thing<br>or running<br>b. Doing thing | ions ask about physical st 4 weeks, has your of activities due to health gs that take a lot of eregs that take some energy. | al activities your child r<br>child been limited in an<br>n problems? | y of soccer, | Yes, limited a lot | limited some | limited a little | limite |
| The | During the pa<br>the following a<br>a. Doing thing<br>or running<br>b. Doing thing | ions ask about physical<br>ist 4 weeks, has your of<br>activities due to health<br>gs that take a lot of er<br>? | al activities your child r<br>child been limited in an<br>n problems?<br>nergy, such as playing | y of soccer, | Yes,<br>limited<br>a lot | limited<br>some | limited<br>a little | No, no limite |
| The 2.1. | During the pa<br>the following:<br>a. Doing thin<br>or running<br>b. Doing thin<br>c. Bending, li | ions ask about physical st 4 weeks, has your cactivities due to health gs that take a lot of er? gs that take some eneithing or stooping? | al activities your child r<br>child been limited in an<br>n problems?<br>nergy, such as playing<br>ergy such as riding a bi | y of soccer, | Yes, limited a lot | limited some | limited a little | limite |
| The 2.1. | During the pa<br>the following:<br>a. Doing thin<br>or running<br>b. Doing thin<br>c. Bending, li | ions ask about physical st 4 weeks, has your of activities due to health gs that take a lot of eregs that take some energy. | al activities your child r<br>child been limited in an<br>n problems?<br>nergy, such as playing<br>ergy such as riding a bi | y of soccer, | Yes, limited a lot | limited some | limited a little | limite |
| The 2.1. | During the pathe following: a. Doing thing or running: b. Doing thing: c. Bending, li CTION 3: YOUR During the pa | ions ask about physical st 4 weeks, has your of activities due to health gs that take a lot of errors that take some energy gs that take some energifting or stooping? CHILD'S EVERYDAY at 4 weeks, has your of the street of the | al activities your child r child been limited in an n problems? nergy, such as playing ergy such as riding a bi Y ACTIVITIES child been limited in the | y of soccer, ke or skating? | Yes, limited a lot | limited some | limited a little | |
| The 2.1. | During the pathe following: a. Doing thing or running: b. Doing thing: c. Bending, li CTION 3: YOUR During the pa | ions ask about physical st 4 weeks, has your of activities due to health gs that take a lot of errors that take some energy gs that take some energifting or stooping? CHILD'S EVERYDAY at 4 weeks, has your of the street of the | al activities your child r child been limited in an n problems? mergy, such as playing ergy such as riding a bi Y ACTIVITIES child been limited in the IONAL difficulties or pro- | y of soccer, ke or skating? | Yes, limited a lot | limited some | limited a little | |
| The 2.1. | During the pathe following: a. Doing thing or running: b. Doing thing: c. Bending, li CTION 3: YOUR During the pa | ions ask about physical st 4 weeks, has your of activities due to health gs that take a lot of errors. The state of the st | al activities your child rechild been limited in an approblems? Therefore, such as playing argy such as riding a bit of ACTIVITIES child been limited in the IONAL difficulties or progress, limited some | soccer, ke or skating? e AMOUNT of time he oblems with his/her E | Yes, limited a lot | limited some | limited a little | |
| The 2.1. | During the pathe following: a. Doing thing or running: b. Doing thing: c. Bending, li CTION 3: YOUR During the pa | ions ask about physical st 4 weeks, has your cactivities due to health gs that take a lot of er? gs that take some energifting or stooping? CHILD'S EVERYDAY st 4 weeks, has your of friends due to EMOTI | al activities your child r child been limited in an n problems? mergy, such as playing ergy such as riding a bi Y ACTIVITIES child been limited in the IONAL difficulties or pro- | soccer,<br>ke or skating?<br>e AMOUNT of time he<br>oblems with his/her E | Yes, limited a lot | limited some | limited a little | limite |
| SEC 3.1. | During the pa<br>the following: a. Doing thing<br>or running: b. Doing thing c. Bending, li CTION 3: YOUR During the pa<br>activities with | ions ask about physical st 4 weeks, has your activities due to health gs that take a lot of ergos that take a lot of ergos that take some eneighting or stooping? CHILD'S EVERYDAY at 4 weeks, has your of friends due to EMOTI Yes, limited a lot | al activities your child rechild been limited in an approblems? Therefore, such as playing argy such as riding a bit of the control of the c | y of soccer, ke or skating? e AMOUNT of time he oblems with his/her E Yes, limited a little | Yes, limited a lot | d spend on the control of the contro | limited a little | limite |
| The 2.1. | During the pathe following: a. Doing thing or running: b. Doing thing: c. Bending, li CTION 3: YOUR During the pathe | ions ask about physical st 4 weeks, has your activities due to health gs that take a lot of ergos that take a lot of ergos that take some eneighting or stooping? CHILD'S EVERYDAY at 4 weeks, has your of friends due to EMOTI Yes, limited a lot | al activities your child rechild been limited in an approblems? mergy, such as playing ergy such as riding a bit of the control of the contr | y of soccer, ke or skating? e AMOUNT of time he oblems with his/her E Yes, limited a little | Yes, limited a lot | d spend on the control of the contro | limited a little | limite |
| SEC 3.1. | During the pathe following: a. Doing thing or running: b. Doing thing: c. Bending, li CTION 3: YOUR During the pathe | ions ask about physical st 4 weeks, has your activities due to health gs that take a lot of er? gs that take some energifting or stooping? CHILD'S EVERYDAY st 4 weeks, has your of friends due to EMOTI Yes, limited a lot | al activities your child rechild been limited in an approblems? mergy, such as playing ergy such as riding a bit of the control of the contr | y of soccer, ke or skating? e AMOUNT of time he oblems with his/her E Yes, limited a little | Yes, limited a lot | d spend on the control of the contro | limited a little | limite |

| SECTION 4: PAIN 4.1. During the past 4 weeks, how often has your child had bodily pain or discomfort? None of the time Once or twice A few times Fairly often Very often every day \[ \begin{array}{cccccccccccccccccccccccccccccccccccc | |
|---|---|
| None of the time Once or twice A few times Fairly often Very often every day | |
| None of the time Once or twice A few times Fairly often Very often every day | |
| None of the time Once or twice A few times Fairly often Very often every day | |
| | , |
| SECTION 5: BEHAVIOR Below is a list of items that describe children's behavior or problems they sometimes have. 5.1. How often during the past 4 weeks did each of the following | |
| statements describe your child? | Urios / |
| diffen offen tithes ne | never Nev |
| a. Argued a lot? | |
| a. Argued a lot? b. Had difficulty concentrating or paying attention? | |
| a. Argued a lot? b. Had difficulty concentrating or paying attention? c. Lied or cheated? | |
| a. Argued a lot b. Had difficulty concentrating or paying attention c. Lied or cheated? 5.2. Compared to other children your child's age, in general would you say his/her behavior is: | |
| a. Argued a lot b. Had difficulty concentrating or paying attention c. Lied or cheated 5.2. Compared to other children your child's age, in general would you say his/her behavior is: Excellent Very good Good Fair Poor | |
| a. Argued a lot b. Had difficulty concentrating or paying attention c. Lied or cheated 5.2. Compared to other children your child's age, in general would you say his/her behavior is: Excellent Very good Good Fair Poor | |
| a. Argued a lot b. Had difficulty concentrating or paying attentions c. Lied or cheated 5.2. Compared to other children your child's age, in general would you say his/her behavior is: Excellent Very good Good Fair Poor | |



| The f | TION 7: SELF-ESTEEM following ask about your child's satisfactic<br>keep in mind how other children your child | | | helpful if | | |
|---|---|---|---|---|---|---|
| 7.1. | During the past 4 weeks, how satisfied your child has felt about: | do you think<br>Very<br>satisfied | Somewhat satisfied | Neither<br>satisfied<br>nor<br>dissatisfied | Somewhat dissatisfied | Very<br>dissatisfie |
| | a. His/her school ability? | | | | | |
| | b. His/her friendships? | | | | | |
| | c. His/her life overall? | | | | | |
| The f | TION 8: YOUR CHILD'S HEALTH following statements are about health in g How true or false is the statement for your a. My child seems to be less healthy the | ur child? C | true t | ostly Por | | Definite<br>false |
| | b. My child has never been seriously ill. | | | 0 0 | | |
| | c. I worry more about my child's health worry about their children's health. | than other people | | 0 0 | | |



| SEC | TION 9: YOU AND YOUR FAMILY | | | | | | |
|---|---|---|---|---|---|---|---|
| 9.1. | During the past 4 weeks, how MUCH concern did each of the following cau | | None<br>at all | A little | Some | Quite<br>a bit | A lot |
| | a. Your child's physical health | | | | | | |
| | b. Your child's emotional well-being | or behavior | | | | | |
| 9.2. | During the past 4 weeks, were you L! of time YOU had for your own needs | | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>some | Yes,<br>limited<br>a little | No, no |
| | a. Your child's physical health | | | | | | |
| 9.3. | b. Your child's emotional well-being of During the past 4 weeks, how often health or behavior: | as your child's | Vely<br>often | Fairly | Sometimes | Almost<br>never | Never |
| | a. limited the types of activities you o | ould do as a family? | | | П | П | |
| | <ul> <li>b. interrupted various everyday famil<br/>(eating meals, watching tv)?</li> </ul> | y activities | | | | | |



#### 10.12 Parenting Stress Index-Short Form (PSI-4-SF)



#### Record/Profile Form

Richard R. Abidin, EdD

#### Instructions:

On the inside of this form, write your name, gender, date of birth, ethnic group, and marital status; today's date; and your child's name, gender, and date of birth. This questionnaire contains 36 statements.

Read each statement carefully. For each statement, please focus on the child you are most concerned about and circle the response that best represents your opinion. Answer all questions about the same child.

Circle SA if you strongly agree with the statement.

Circle A if you agree with the statement.

Circle NS if you are not sure.

Circle D if you c sage or with the statement.

For example, if you sometimes enjoy going to the movies, you would circle A in response to the following statement:

I enjoy going to the movies.

SA (A) NS D SD

While you may not find a response that exactly states your feelings, please circle the response that comes closest to describing how you feel. Your first reaction to each question should be your answer.

Circle only one response for each statement, and respond to all statements. Do not erase! If you need to change an answer, mark an "X" through the incorrect answer and circle the correct response. For example:

I enjoy going to the movies.

SA A NS 🕅 🚱

• 16204 N. Florida Ave. • Lutz, FL 33549 • 1.800.331.8378 • www.parinc.com

Copyright @ 1990, 1995, 2012 by PAR. All rights reserved. May not be reproduced in whole or in part in any form or by any means without written permission of PAR. This form is printed in green and orange ink on carbonless paper. Any other version is unauthorized

Reorder #RO-10271

WARNING! PHOTOCOPYING OR DUPLICATION OF THIS FORM WITHOUT PERMISSION IS A VIOLATION OF COPYRIGHT LAWS.

| PSI-4 | Answer | Sł |
|-----------|-------------|----|
| HORT FORM | T5-2710 UK. | |

| ame | Gender | Date of | birth | | 114 | 1 | |
|---|---|---|---|---|---|---|---|
| hnic group | Marital status | Today's | date | | / | 1 | |
| nild's name | Child's gender | Child's | date of bir | th_ | -1 | _ / | / |
| A Transpired | | | | | Disease | <u> </u> | _ |
| SA = Strongly Agree A = Agree | THE R. P. LEWIS CO., LANSING, MICH. | 201,011,000 | D = Stro | ngıy | Disag | ree | 4 |
| <ol> <li>I often have the feeling that I cannot ha</li> <li>I find myself giving up more of my life</li> </ol> | to meet my children's ne | eeds than I ever | (ent | A | NS | D | SE |
| expected | | | SA | A | NS | D | SI |
| 3. I feel trapped by my responsibilities as | | | | A | NS | D | SI |
| <ol><li>Since having this child, I have been una</li></ol> | | | | A | NS | D | SE |
| 5. Since having a child, I feel that I am alm | | And I say the second the said of the said | | A | NS | D | SI |
| <ol><li>I am unhappy with the last purchase of</li></ol> | | | | A | NS | D | SI |
| 7. There are quite a few things that bother | | | | Α | NS | D | SE |
| 8. Having a child has caused more proble | ms than I expected in m | y relationship with | SA | Α | NS | D | SI |
| my spouse/parenting partner 9. I feel alone and without friends | | | | A | NS | D | SI |
| <ol><li>I feel alone and without friends</li><li>When I go to a par v, Lusually expect n</li></ol> | | | | A | NS | D | SI |
| 1. I am not as interested in people is tus. | the state of the s | | A CONTRACTOR OF THE PARTY OF TH | A | NS | D | SI |
| 2. I don't enjoy things as I used to | | | SA | A | NS | D | St |
| 3. My child rarely does things for me that | make me feel good | | SA | Α | NS | D | SI |
| 4. When I do things for my child, I get the | | | | Α | NS | D | SI |
| very much. | | | | A | NS | D | SI |
| <ol> <li>My child smiles at me much less than I</li> <li>Sometimes I feel my child doesn't like i</li> </ol> | | | | A | NS | D | SI |
| | | | | A | NS | D | SE |
| | | | | A | NS | D | SI |
| | | | | A | NS | D | SI |
| 22 2327 24 4 4 4 | | | | A | NS | D | SI |
| <ol> <li>My child is not able to do as much as I'</li> <li>It takes a long time and it is very hard I</li> </ol> | | | | A | NS | D | SI |
| 2. I feel that I am: (Choose a response from | n the choices below.) | | 1 | 2 | 3 | 4 | 5 |
| a very good parent a better-than-avera | t. | | | | | | |
| 3. an average parent. | | | | | | | |
| 4. a person who has s<br>5. not very good at b | some trouble being a par | ent. | | | | | |
| 3. I expected to have closer and warmer for | | | 1 | | | 3 | 20 |
| | ******** | | SA | A | NS | D | SI |
| 4. Sometimes my child does things that b | other me just to be mean | | SA | A | NS | D | SI |

| | SA = Strongly Agree A = Agree NS = Not Sure D = Disagree SD = | = Stro | ngly | Disag | jree | |
|---|---|---|---|---|---|---|
| 25. | My child seems to cry or fuss more often than most children. | SA | Α | NS | D | SE |
| 26. | My child generally wakes up in a bad mood | SA | A | NS | D | SE |
| 27. | I feel that my child is very moody and easily upset. | SA | A | NS | D | SE |
| 28. | Compared to the average child, my child has a great deal of difficulty in getting | | | | | |
| | used to changes in schedules or changes around the house | SA | A | NS | D | SE |
| 29. | My child reacts very strongly when something happens that my child doesn't like. $\ \ .$ . | SA | A | NS | D | SE |
| 30. | When playing, my child doesn't often giggle or laugh. | SA | A | NS | D | SE |
| 31. | My child's sleeping or eating schedule was much harder to establish than I expected. | SA | A | NS | D | SE |
| 32. | I have found that getting my child to do something or stop doing something is: (Choose a response from the choices below.) | 1 | 2 | 3 | 4 | 5 |
| 33. | 5. much easier than I expected. Think carefully and count the number of things which your child does that bothers yo For example, dawdles, refuses to listen, overactive, cries, interrupts, fights, whines, etc. (Choose a response from the choices below.). | | 2 | 3 | 4 | 5 |
| | 1. 1-3<br>2. 4-5<br>3. 6-7<br>4. 8-Do not duplica | + | 2 | | | |
| | "DU HULUUPIICA | 1 | ~ | | | |
| 34. | There are some things my child does that really bother me a lot. | SA | A | NS | D | SD |
| 34. | | SA | A | NS<br>NS | D<br>D | SE |

## Please do not write in this area.